# The Botswana Combination Prevention Project (BCPP) Evaluation Protocol (Protocol #1)

# **Research Design and Impact Evaluation**

Version 7.0

January 16, 2019

# **Collaborating Institutions:**

Botswana–Harvard AIDS Institute Partnership (BHP)
Botswana Ministry of Health (MOH)
Harvard T.H. Chan School of Public Health
U.S. Centers for Disease Control and Prevention (CDC)

**Funded by**: The United States President's Emergency Plan for AIDS Relief (PEPFAR) through the Centers for Disease Control and Prevention (CDC)

#### i. PRINCIPAL INVESTIGATORS

Myron Essex, DVM, PhD Lasker Professor of Health Sciences Harvard T.H. Chan School of Public Health FXB 402, 651 Huntington Avenue Boston, MA 02115-6017

Email: messex@hsph.harvard.edu

Phone: +1-617-432-0975 +1-617-739-8348 Fax:

Joseph Makhema, MBChB, FRCP Chief Executive Officer **Botswana Harvard AIDS Institute** Private Bag BO320 Gaborone, Botswana

Email: jmakhema@bhp.org.bw

**Phone:** +267-390-2671 Fax: +267-390-1284

Shahin Lockman, MD, MS

Associate Professor of Medicine; Associate Professor in the Department of Immunology and Infectious Diseases

Harvard T.H. Chan School of Public Health

FXB 406a, 651 Huntington Avenue

Boston, MA 02115

Email: shahin.lockman@gmail.com

**Phone:** +1-617-771-8780 Fax: +1-617-739-8348

Eric Tchetgen Tchetgen, PhD

Professor of Biostatistics and Epidemiologic Methods

Departments of Biostatistics and Epidemiology

Kresge, Room 822 677 Huntington Avenue

Boston, MA 02115

Email: etchetge@hsph.harvard.edu

**Phone:** 617-432-5970 Fax: 617-432-1884

Molly Pretorius Holme, MS Senior Research Manager Department of Immunology and Infectious Diseases Harvard T.H. Chan School of Public Health

FXB 406a, 651 Huntington Avenue

Boston, MA 02115

Email: mpretori@hsph.harvard.edu

**Phone:** +1-617-432-4377 **Fax:** +1-617-739-8348

#### ii. ROLES OF INSTITUTIONS AND PRINCIPAL INVESTIGATORS

 Institutions: Close coordination between MOH, Harvard Chan School, CDC, and BHP is needed to ensure seamless implementation of research and program activities. However, MOH and CDC will lead, and ultimately be responsible for, program implementation and monitoring and evaluation, while Harvard Chan School/BHP will lead, and ultimately be responsible for, the evaluation of HIV incidence and viral genetic linkage analyses.

#### • Principal Investigators:

**Myron Essex:** Harvard Principal Investigator (PI) responsible for preparation of the study protocol, design and evaluation of research, monitoring of research progress, creation and monitoring of research budgets, and preparation of research progress reports; responsible for design of initial proposal, including virological analyses, and supervision of Harvard and BHP investigators.

**Joseph Makhema:** BHP Co-Principal Investigator (Co-PI) responsible for preparation of study protocol, preparation of progress reports, and overseeing field research staff in Botswana.

**Shahin Lockman:** Harvard Co-Principal Investigator (Co-PI) responsible for preparation of the study protocol, and monitoring of research progress / revisions of research protocol and procedures as needed; and assisting with monitoring/revision of research budgets and preparation and review of research progress reports.

**Eric Tchetgen Tchetgen:** Harvard Co-Principal Investigator (Co-PI) responsible for monitoring of research progress, facilitation of internal and external study monitoring, and preparation of research progress reports; responsible for overseeing statistical design and analyses as well as their interpretation.

**Molly Pretorius Holme:** Harvard Co-Principal Investigator (Co-PI) responsible for preparation of the study protocol, and monitoring of research progress / revisions of research protocol and procedures as needed; and assisting with monitoring/revision of research budgets and preparation and review of research progress reports.

# iii. INVESTIGATOR LISTS BY INSTITUTION

# Botswana Ministry of Health (MOH), Gaborone, Botswana (Alphabetical Order)

| Name | Role | Contact Email |
|------------------------------|----------------------|---------------------|
| Marina Anderson, MD, MPH | Surveillance | manderson@gov.bw |
| Shenaaz El-Halabi (DPS), MPH | In-country oversight | sel-halabi@gov.bw |
| Ernest B. Fetogang, PhD | M&E | efetogang@gov.bw |
| Refeletswe Lebelonyane, MD | In-country oversight | rlebelonyane@gov.bw |
| Madisa Mine, PhD | Laboratory | mmine@bhp.org.bw |

# Harvard T.H. Chan School of Public Health, Boston, MA, USA (Alphabetical Order)

| Name | Role | Contact Email |
|---|---|---|
| Ingrid Bassett, MD | Cost-effectiveness | ibassett@partners.org |
| Kara Bennett, MS | Statistical Consultant | karabennett@earthlink.net |
| Victor DeGruttola, DSc | Senior Statistical Scientist | degrut@hsph.harvard.edu |
| Scott Dryden-Peterson, MD | Treatment and PMTCT | scott_peterson@post.harvard.edu |
| Kenneth Freedberg, MD | Cost-effectiveness | kfreedberg@partners.org |
| Vladimir Novitsky, MD, PhD | Lab | vnovi@hsph.harvard.edu |
| Kathleen Powis, MD, MPH | Research Operations, Treatment and PMTCT | kpowis@partners.org |
| Roger Shapiro, MD, MPH | Treatment and PMTCT | rshapiro999@gmail.com |
| Rochelle Walensky, MD | Cost-effectiveness | rwalensky@partners.org |
| Rui Wang, PhD | Statistics | rwang8@partners.org |
| Kathleen Wirth, ScD | Statistics | kwirth@hsph.harvard.edu |

# Botswana-Harvard AIDS Institute Partnership (BHP), Gaborone, Botswana (Alphabetical Order)

| Name | Role | Contact Email |
|---|---|---|
| Tendani Gaolathe, MD | Treatment and PMTCT, Field research operations | tgaolathe@bhp.org.bw |
| Simani Gaseitsiwe, PhD | Lab | gaseitsiwe@bhp.org.bw |
| Poloko Kebaabetswe, PhD, MPH | Qualitative research consultant | polokokebaabetswe@yahoo.com |
| Mompati Mmalane, MD, FRCS-Ed, MSc | BHP oversight and research operations | mmmalane@bhp.org.bw |
| Mosepele Mosepele, MBBS, MSc | Clinical outcomes | mmosepele@bhp.org.bw |
| Sikhulile Moyo, MSc, MPH, PhD | Lab | smoyo@bhp.org.bw |
| Rosemary Musonda, MSc, PhD | Lab | rmusonda@bhp.org. bw |
| Erik van Widenfelt, BA | Research data systems | ewidenfelt@bhp.org.bw |

# <u>Centers for Disease Control and Prevention (CDC), Atlanta, GA, USA, and Gaborone, Botswana (Alphabetical Order)</u>

| Name | Role | Contact Email |
|-------------------------|--------------------------|-----------------|
| Pam Bachanas, PhD, MS | НТС | dtt6@cdc.gov |
| Ebi Bile, BSc, MA | In-country lab oversight | efb6@bw.cdc.gov |
| Arielle Lasry, PhD | HTC Costing | ftn9@cdc.gov |
| Tafireyi Marukutira, MD | Clinical | xwt5@cdc.gov |
| Lisa A. Mills, MD | Co-Investigator | lmills1@cdc.gov |
| Janet Moore, PhD | Co-investigator | jym3@cdc.gov |
| Sherri Pals, PhD | Statistics | sfv3@cdc.gov |
| Elliot Raizes, MD | Clinical Consultant | gwq0@cdc.gov |
| Chunfu Yang, PhD | Laboratory | cxy0@cdc.gov |

# iv. TABLE OF CONTENTS

| I. | PF | RINCIPAL INVESTIGATORS | 2 |
|---|---|---|---|
| II. | RC | ROLES OF INSTITUTIONS AND PRINCIPAL INVESTIGATORS | |
| Ш | . IN | INVESTIGATOR LISTS BY INSTITUTION | |
| IV | '. TA | TABLE OF CONTENTS | |
| ٧. | LIS | ST OF TABLES AND FIGURES | 9 |
| VI | | CRONYMS AND ABBREVIATIONS | |
| | | OTSWANA COMBINATION PREVENTION PROJECT SCHEMA | |
| VI | II. EV | /ALUATION PROTOCOL SYNOPSIS | 20 |
| 1. | IN | ITRODUCTION AND BACKGROUND | 22 |
| | 1.1. | EPIDEMIC IN BOTSWANA | 22 |
| | 1.2. | COMBINATION PREVENTION | 22 |
| | 1.3. | THE PROPOSED COMBINATION PREVENTION (CP) PACKAGE | 23 |
| 2. | ST | TUDY OBJECTIVES | 24 |
| | 2.1. | Primary Study Hypothesis | 24 |
| | 2.2. | Primary Objectives | 24 |
| | 2.3. | EVALUATING THE IMPACT OF COMBINATION PREVENTION: DESIGN AND RATIONALE TO ADDRESS PRIMARY OBJECTIVES | |
| | 2.4. | SECONDARY OBJECTIVES | |
| | 2.5. | DESIGN AND RATIONALE TO ADDRESS SECONDARY OBJECTIVES | 28 |
| 3. | 0 | VERVIEW OF STUDY METHODS | 31 |
| 4. | ST | TUDY POPULATIONS | 32 |
| | 4.1. | SELECTION OF STUDY COMMUNITIES | 32 |
| | 4.2. | Matching of Study Communities | 33 |
| | 4.3. | DEFINITION OF A STUDY COMMUNITY RESIDENT | 34 |
| | 4.4. | STUDY INCLUSION AND EXCLUSION CRITERIA | 35 |
| | 4.5. | RATIONALE FOR ELIGIBILITY CRITERIA | 38 |
| 5. | SA | AMPLE SIZE AND SAMPLE SELECTION METHODS | 41 |
| | 5.1. | SAMPLE SIZE CALCULATIONS RELATED TO PRIMARY OBJECTIVE #1 | 41 |
| | 5.2. | SAMPLE SIZE CALCULATIONS RELATED TO PRIMARY OBJECTIVE #2 | 50 |
| | 5.3. | EXPECTED NUMBERS OF STUDY PARTICIPANTS | 58 |
| | 5.4. | Planned Interim Analysis of Data | 60 |
| 6. | ST | TUDY PROCEDURES | 61 |
| | 6.1. | Baseline Household Survey (BHS) | 61 |
| | 6.2 | HIV INCIDENCE COHORT (HIC) | 69 |

| 6.3. | FOCUS GROUP DISCUSSIONS AND INDIVIDUAL IN-DEPTH INTERVIEWS RELATED TO BARRIERS TO AND FACILITATORS ( | OF |
|---|---|---|
| LINKAG | E TO CARE AND ART INITIATION AMONG A SUBSET OF BHS PARTICIPANTS | |
| 6.4. | RESEARCH BLOOD DRAW PROCEDURES IN COMBINATION PREVENTION COMMUNITIES, OUTSIDE OF THE BHS | 76 |
| 6.5. | THE END OF STUDY SURVEY (ESS) AND FINAL T2 STUDY VISIT FOR PREVIOUSLY ENROLLED 20% HOUSEHOLDS | 77 |
| 7. CO | ST EFFECTIVENESS ANALYSIS | 80 |
| 7.1 | CEPAC Model Structure | 81 |
| 7.2 | Data Inputs | 82 |
| 7.3 | MODEL VALIDATION AND APPROACH TO UNCERTAINTY | 85 |
| 7.4 | COST-EFFECTIVENESS ANALYSIS PLAN | 86 |
| 8. LAE | SORATORY METHODS | 87 |
| 8.1. | OVERVIEW OF LABORATORY METHODS | 87 |
| 8.2. | TRAINING OF LABORATORY PERSONNEL | 88 |
| 8.3. | SPECIMEN COLLECTION, TRANSPORT, AND PROCESSING | 88 |
| 8.4. | LABORATORY TESTING FOR BHS, HIC, AND ESS (RETURNED TO PARTICIPANT AND/OR PARTICIPANT FILE) | 89 |
| 8.5. | RESEARCH LABORATORY TESTING (RESULTS NOT RETURNED TO PARTICIPANT) | 90 |
| 8.6. | QUALITY ASSURANCE | 94 |
| 8.7. | BIOSAFETY AND WASTE MANAGEMENT | 94 |
| 8.8. | SPECIMEN STORAGE AND SHIPMENT | 94 |
| 9. DA | TA COLLECTION AND MANAGEMENT | 95 |
| 9.1. | Data Management team | 95 |
| 9.2. | DATA FLOW | 95 |
| 9.3. | DATA FLOW FROM BHS, HIC, ESS, AND RESEARCH BLOOD DRAWS | 95 |
| 9.4. | THE BCPP RESEARCH DATA MANAGEMENT CENTER (DMC) | 97 |
| 9.5. | REPORTING STUDY PROGRESS | 97 |
| 10. AN | ALYSIS PLANS | 97 |
| 10.1. | Analysis Plan to Meet Primary Objectives | 97 |
| 10.2. | Analysis Plan to Meet Key Secondary Objectives | 99 |
| 11. ETH | IICAL CONSIDERATIONS | 103 |
| 11.1. | ETHICAL REVIEW | 103 |
| 11.2. | Informed Consent | 103 |
| 11.3. | Risks | 108 |
| 11.4. | Benefits of Research Participation | 108 |
| 11.5. | CONFIDENTIALITY | 108 |
| 11.6. | COMPENSATION AND INCENTIVES | |
| 11.7. | PROTOCOL COMPLIANCE AND COMPLIANCE WITH UN CONVENTION ON THE RIGHTS OF THE CHILD | 109 |
| 11.8. | FUTURE USE OF STORED SAMPLES | 109 |
| 12. STU | JDY SAFETY AND MONITORING PLAN | 110 |
| 12.1. | REPORTING ADVERSE EVENTS | 110 |
| 12.2. | DSMB | 111 |
| 12.3. | Protocol Violations | 111 |
| 12.4. | STUDY MONITORING PLAN | 111 |

| 13. | ADN | MINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION | 111 |
|-----|------|-------------------------------------------------------|-----|
| 1 | 3.1. | STUDY RECORDS AND DOCUMENT RETENTION | 111 |
| 1 | 3.2. | Information Dissemination and Publication Plan | 111 |
| 14. | REF | ERENCES | 112 |
| 15. | APP | ENDICES | |

| Cross-<br>Protocol<br>Appendix | |
|---|---|
| Number | Title |
| C2 | Table A: Study Communities and Matching Criteria for Community Pairs |
| | Table B: Back-up Communities if Selected 30 Communities Decline, are Unavailable or Deemed Unsuitable for Study Inclusion Figure A: Map of Study Communities in Three Regions Figure B: Map of Study Communities in the Southern Region Figure C: Map of Study Communities in the Central Region Figure D: Map of Study Communities in the Northern Region |
| С3 | Table of Study Population Sizes |
| C4 | Data Safety Monitoring Plan |

| Protocol 1<br>Appendix | Title |
|---|---|
| LOA#1 | Letter of Amendment #1 (December 13, 2013) to Protocol 1 v1.0 dated September 24, |
| | 2013 |
| 1-1 | Summary of Protocol Changes |

# v. **LIST OF TABLES AND FIGURES**

| Table 1A | Original Model Input Parameters for the Primary Model to Estimate Impact of Combination Prevention (CP) Package Scale-Up in CP Communities Versus Enhanced Care (EC) Communities over 4 Years |
|---|---|
| Table 1B | Model Input Parameters for the Updated Primary Model to Estimate Impact of Combination Prevention (CP) Package Scale-Up in CP Communities Versus Enhanced Care (EC) Communities over 4 Years |
| Table 2A | Projected Cumulative HIV Incidence in Enhanced Care (EC) versus Combination Prevention (CP) Communities over 4 Years of Study Follow-Up Using Original Parameters and with ART for Individuals with CD4≤350 cells/µL or Viral Load ≥10,000 copies/ml in the CP Arm |
| Table 2B | Projected Cumulative HIV Incidence and Study Power with Universal Test and Treat in the Combination Prevention (CP) Arm and Different Scenarios of Botswana National Guidelines Changes in the Enhanced Care (EC) Arm |
| Table 3 | Cluster Size versus Cluster Number Needed to Achieve >85% Power to Detect Anticipated Effect Size by the End of the 3rd Year of Follow-up across a Range of Coefficients of Variation (k), Assuming ART is Offered to HIV-Infected Individuals with CD4≤350 or Viral Load≥10,000 copies/ml in the Combination Prevention Arm based on the original set of parameters |
| Table 4 | Estimated Precision of 95% Confidence Interval Surrounding HTC, ART (including VL suppression), and MC Coverage Proportions at Baseline and Study End |
| Table 5 | Inputs for Calculating CI Widths Surrounding HTC, ART (including VL suppression), and MC Coverage Proportions at Baseline and Study End |
| Table 6 | Estimated Power of Detecting Differences in Coverages in HTC, ART, VL suppression, and MC between Enhanced Care (EC) and Combination Prevention (CP) Arms in the ESS |
| Table 7 | Expected Numbers of Participants in Study Components |
| Table 8 | Resource Utilization and Cost Data Needs |
| Table 9 | Individual Healthcare Utilization, Cost, and Quality of Life Assessments |
| Table 10 | Prevention Strategies and Outcomes of Interest |
| Table 11 | BCPP Evaluation Protocol Laboratory Testing Responsibilities |
| Table 12 | Summary of Approach to Consent, Various Components of the Study |
| FIGURE S1 | Overview of Surveys and HIV Incidence Cohort in the Evaluation Protocol |
| Figure 1 | Number of Clusters Versus Cluster Size Needed to Ensure >85% Power to Detect Anticipated Differences in Cumulative HIV Incidence Between Enhanced Care and Combination Prevention Arms |
| Figure 2A | Power to Detect Various Potential Reductions in Observed HIV Incidence In CP Communities when EC Communities have a Cumulative Incidence of $4.1\%$ |
| Figure 2B | Power to Detect Various Potential Reductions in Observed HIV Incidence In CP Versus EC Communities under different Annual EC Incidence Rates |

| Figure 3 | Flow of participants from 20% Household Survey to BHS and HIC |
|---|---|
| Figure 4A | BHS Procedures for Individuals with no Documentation of HIV-Positive Status |
| Figure 4B | BHS Study Procedures for Individuals with Documentation of HIV-Positive Status |
| Figure 4C | Follow-up Procedures for HIC Enrollees During T1 |
| Figure 4D | Procedures for Individuals in 20% Households who are Newly Identified During T1 and who have No Documentation of HIV-Positive Status |
| Figure 4E | Procedures for Individuals in 20%Households who are Newly Identified During T1 and who HAVE Documentation of HIV-Positive Status |
| Figure 5A | Procedures for the End of Study Survey in 80% Households in 6 Communities |
| Figure 5B | Procedures for the Final Survey Visit at T2 in 20% BHS/HIC Households |
| Figure 6 | A simulated patient trace from South Africa |
| Figure 7 | CD4 Trajectory in the CEPAC-I model as compared to the HPTN-052 trial |

#### vi. ACRONYMS AND ABBREVIATIONS

AE adverse event

AHS annual household surveys (follow-up visits of the BHS and HIC)

ANC antenatal clinic (or care)

ART antiretroviral treatment (or therapy)

ARV antiretroviral

BCPP Botswana Combination Prevention Project
BHHRL Botswana—Harvard HIV Reference Laboratory
BHP Botswana—Harvard AIDS Institute Partnership

BHS baseline household survey CCC closed clinical cohort

CDC Centers for Disease Control and Prevention

CEPAC Cost-Effectiveness of Preventing AIDS Complications

CI confidence interval
CP combination prevention
CRT community-randomized trial
DMC Data Management Center

EDC electronic data capture (system used by BHP)

EC enhanced care

ELISA enzyme-linked immunosorbent assay

ESS end-of-study survey

ETC expanded treatment cohort

FDE full disk encryption FGD focus group discussion

FRR false recent rate FTE full-time equivalent

GCLP Good Clinical and Laboratory Practice
HIV-1 RNA HIV-1 RNA load in plasma, viral load

HIC HIV Incidence Cohort

HPLC high performance liquid chromatography

HSPH Harvard School of Public Health
HTC HIV testing and counseling
IAS International AIDS Society
IDI individual in-depth interviews
IDR immunodominant region
IRB institutional review board

IPMS integrated patient management system

ISPOR International Society for Pharmacoeconomics and Outcomes Research

LTC linkage to care

LTCM Linkage-to-care Manager LTFU loss/lost to follow-up

MC male circumcision

M&E monitoring and evaluation
MoH Botswana Ministry of Health

MTCT mother-to-child (HIV) transmission

NNRTI non-nucleoside reverse transcriptase inhibitor

OHRP Office for Human Research Protections

OI opportunistic infection

Option B+ indefinite continuation of ART for women who start ART for PMTCT

PEPFAR President's Emergency Plan for AIDS Relief

PI protease inhibitor

PII personally identifiable information

PIMS Patient Information Management System

PMTCT prevention of mother-to-child (HIV) transmission

POB pregnancy/breastfeeding

POC point-of-care

PSA probabilistic sensitivity analysis
QA/QC quality assurance/quality control

QALY quality adjusted life-year

QOL quality of life

RDS respondent driven sampling
SAE serious adverse event
SD standard deviation

SMC Safe Male Circumcision (Botswana government initiative)

SOC standard of care

SOP standard operating procedures SRH sexual and reproductive health

study arm a group of 15 communities that is randomized to receive either enhanced

care or combination prevention

TB tuberculosis

TDR transmitted drug resistance

UNAIDS Joint United Nations Programme on HIV/AIDS

UTT universal test and treat VPN virtual private network

VDC Village Development Committee WHO World Health Organization

YLS Year of Life Saved

#### vii. BOTSWANA COMBINATION PREVENTION PROJECT SCHEMA

#### INTRODUCTION

#### **Background on Combination Prevention**

In recent years, several new HIV prevention interventions have proven to be highly effective at reducing transmission of HIV and have offered hope for containing and possibly reversing epidemics in sub-Saharan Africa. Despite considerable success in scaling up these interventions in many sub-Saharan African countries, adult HIV incidence remains high in many regions in Southern Africa. This may in part be attributed to the insufficient scale and quality of HIV prevention interventions. Modeling studies suggest that investment in rapid, coordinated scale-up of a combination of evidence-based HIV prevention interventions, including HIV testing and counseling (HTC), male circumcision (MC), antiretroviral therapy (ART) and prevention of mother-to-child transmission (PMTCT), can significantly reduce population-level HIV incidence and may be cost-effective or even cost-saving in the long term. Rigorous evidence-based outcomes to support these projections of population-level impact are needed if national and international bodies are to justify further investment in combination prevention strategies.

# **Study Hypothesis**

The BCPP study was designed to test the hypothesis that implementing a combination prevention package (described below) will impact the HIV/AIDS epidemic by significantly reducing population-level, cumulative HIV incidence in a defined geographic area over a period of 3 years and will be cost-effective. With the changes introduced in version 5.0 of this protocol, HIV incidence will be measured over a shorter period, approximately 2.5 years.

# **Proposed Combination Prevention Package**

The proposed combination prevention package for the BCPP includes:

- Rapid scale-up of HTC services, with a target of ensuring >90% of HIV-infected adults aged 16-64 have documentation of their HIV-infected status.
- Rapid scale-up of universal ART for all HIV-infected adults, with a target of ensuring that >93% of adults diagnosed with HIV infection are receiving ART.
- Rapid scale-up of retention in care and adherence interventions, with a target of ensuring that >95% of HIV-infected adults receiving ART are virally suppressed with HIV-1 RNA <400 copies/ml.
- Rapid scale-up of linkage to male circumcision services, with a target of ensuring >60% of HIV-negative men (aged 16–49) are circumcised.
- Rapid strengthening of PMTCT services, with a target of ensuring >90% of women initiated on indefinite ART (Option B+) during pregnancy remain in care and on treatment at 12 months postdelivery.

# **Study Arms**

Thirty communities (described in *Appendix C2*) in three geographic areas considered representative of Botswana have been proposed for inclusion in the community randomized trial (CRT): (1) around Gaborone in the south east, (2) around Francistown in the north east, and (3) in the region around Mahalapye, Serowe, and Palapye in the central eastern region. Communities will be randomized to either the Combination Prevention arm or the Enhanced Care arm. Combination Prevention

communities will receive the proposed combination prevention package described above. Enhanced Care Communities will receive guidance and technical support for quality management and data systems at all laboratories and local clinics at which individuals receive HIV care and treatment (and participants in the survey occurring in ~20% of households in the Enhanced Care communities may benefit from study provision of home-based HIV counseling and testing and, for HIV-infected residents, point of care CD4 count and HIV-1 RNA testing).

# High Viral Load Treatment and Universal Test and Treat as Combination Prevention Package Components

Data show that higher levels of HIV-1 RNA (viral load) are independently associated with both higher rates of HIV transmission and more rapid HIV clinical disease progression and CD4 decline. This study therefore originally included the use of a modified "treatment as prevention" approach that targeted not only those adults who need ART for their own health, but also those adults who are most likely to perpetuate HIV transmission within the community (those with viral load  $\geq$ 10,000 copies/mI). At the time of designing the BCPP in 2012 there was strong experimental evidence supporting initiation of ART at CD4 $\leq$ 350 cells/ $\mu$ L, or WHO Stage III/IV, but conclusive experimental evidence supporting patient benefit of ART initiation at higher CD4 counts, especially CD4 >500 cells/ $\mu$ L was lacking.

The 2013 WHO guidelines recommended initiation of ART in all HIV-infected adults with CD4 $\leq$ 500 cells/ $\mu$ L regardless of clinical stage. In an attempt to provide programmatic data for an anticipated change in CD4 threshold for ART initiation in the future in Botswana and to enhance the power of the study to answer its primary objective, the threshold for ART initiation in the Combination Prevention arm was modified in early 2015 (from CD4 $\leq$ 350 to CD4 $\leq$ 500 regardless of viral load, in addition to offering expanded ART to persons with CD4>500 and viral load  $\geq$ 10,000).

Shortly thereafter, in July 2015, the WHO announced that it would revise ART guidelines to recommend universal treatment (regardless of CD4 count or HIV disease severity). The WHO's plans were informed by results from two clinical ART trials. One, the START trial, reported that early drug treatment of people with HIV cut their risk of serious illness or death by 57% (Lundgren, Babiker et al. 2015). Another, the TEMPRANO study, released findings that early ART significantly decreased morbidity overall and when restricted to patients with baseline CD4>500 cells/µL (Danel, Moh et al. 2015). WHO published an early release guideline on when to start ART and on pre-exposure prophylaxis for HIV in September 2015 (World Health Organization 2015). The BCPP study team, with the support of the DSMB and funder, revised the intervention treatment initiation criteria to take these results and WHO guidelines into account. Universal test and treat (UTT) is therefore included in the combination prevention package starting with version 4.0 of the protocols as of June 2016.

Also as of June 2016, with the launch of its "Treat All" campaign, Botswana treatment guidelines allow initiation of ART for all HIV-infected citizens regardless of CD4 count or WHO stage. Enhanced Care community residents are eligible to receive ART according to these updated Botswana national guidelines. Residents in the Combination Prevention communities are continuing to receive additional expanded treatment as prevention.

Through additional modeling, the study team adjusted effect size and power calculations to reflect a move to universal ART in both the Combination Prevention and Enhanced Care arms, using a range of roll-out timelines. This revised modeling also used estimates of coverage (by HTC, linkage to care, ART,

and MC) that are consistent with what had been observed in BCPP thus far, rather than using the higher coverage "targets". Model-based estimates suggest that the impact of a change in treatment policy on the power to detect a difference in cumulative incidence (the primary objective of BCPP) may still yield at least 60% power, but the impact depends on the exact nature and timing of the actual implementation of changes in policy as well as other prevailing conditions. The retention of this level of power even with Enhanced Care communities moving to expanded access to ART is at least in part attributable to the fact that BCPP is implementing multiple HIV prevention interventions (including higher HTC coverage, linkage to HIV care/treatment, adherence support, etc.). With version 5.0 of the protocol, we are dropping the third annual household survey and instead performing the second annual household survey approximately 6 months later than originally planned. This will result in a total average follow-up of the BHS/HIC participants of approximately 30 months rather than 36 months. This change is being made for budgetary reasons, and also because the randomized arms are becoming more similar over time with regard to HIV treatment (particularly with the move to UTT in both arms in June 2016). Shortening the follow-up period from the originally planned 36 months to an average of 30 months with version 5.0 of the protocol reduces estimated power for the first primary objective to approximately 63%.

# Indefinite ART following PMTCT (Option B+)

Women completing ART for PMTCT will be offered indefinite ART continuation (regardless of pretreatment CD4, viral load or clinical stage). Option B+ was part of the original combination prevention package at the launch of this study in 2013. Upon the Botswana government's adoption of Option B+ as national policy (April 2015), Option B+ is offered to qualifying women in Enhanced Care communities as well as Combination Prevention communities per national guidelines.

# **Relationship of BCPP Study Protocols**

The Botswana Combination Prevention Project and related procedures were initially described in three separate, but inter-related, protocols: an *Evaluation Protocol (#1), Closed Clinical Cohort Protocol (#2),* and *Intervention Protocol (#3)*.

In 2015, the *Closed Clinical Cohort Protocol* (#2) was terminated due to concerns about low study power, evolving ART guidelines, and feasibility.

#### **BCPP STUDY OBJECTIVES**

Primary objectives covered by the BCPP study protocols include:

- 1. To determine whether implementation of a combination prevention (CP) package can significantly reduce population-level, cumulative HIV incidence in 16-64 year old residents in Botswana over a period of approximately 30 months. This evaluation is a primary objective of the *Evaluation Protocol*. Implementation of the combination prevention package is described in detail in the *Intervention Protocol*.
- 2. To estimate population-level uptake of HIV testing, ART, VL suppression, male circumcision, and PMTCT services and compare service uptake between Enhanced Care communities and Combination Prevention communities at baseline and at study end. This is a primary objective of the *Evaluation Protocol*.
- 3. To estimate the cost per additional infection averted in Combination Prevention communities compared with Enhanced Care communities. This is a primary objective of the *Evaluation Protocol*.

4. To implement the combination prevention intervention package in Combination Prevention communities and describe uptake of these interventions in Combination Prevention communities (expanded HIV Testing and Counseling, strengthened Male Circumcision, expanded HIV Care and Treatment, and strengthened PMTCT services). This is the primary objective of the *Intervention Protocol*.

#### **STUDY DESIGN**

The over-arching design is a pair-matched CRT that will be completed over the course of approximately 5 years. A randomized design is selected to provide experimental evidence of combination prevention package impact, and because population-level HIV incidence is the outcome of interest, we propose a community (rather than individual) randomized trial. A detailed description of the combination prevention package and how these interventions go beyond standard of care (SOC) are described in detail in the *Intervention Protocol*. In brief, the interventions consist of the following four components:

- 1) Expand HTC and strengthen linkage-to-care services
- 2) Strengthened and expanded HIV care and treatment services
- 3) Expand male circumcision (MC) services
- **4)** Strengthened PMTCT services, specifically identification, linkage, and treatment of HIV-positive pregnant women

#### **STUDY METHODS**

The study communities will be matched into pairs based on community characteristics thought to be associated with the outcome of interest (adult HIV incidence). Pair-matching is done to improve balance between study arms and statistical efficiency.

The study methods are divided into five components that are described in detail in the BCPP protocols and summarized here.

1) Baseline Household Survey (BHS) followed by Annual Household Survey (AHS)\* Visits Following matching, within each community, a baseline household survey (BHS) of approximately 20% of randomly selected households will be implemented to (1) establish an HIV incidence cohort (HIC) consisting of all eligible consenting HIV-negative household members aged 16-64 years, and (2) estimate baseline and annual coverage of the combination prevention package. The BHS and subsequent annual household survey (AHS) visits are described in the *Evaluation Protocol*. Individuals who enroll in BHS will be followed with AHS visits, regardless of whether they are assigned to the HIC (see below) to assess uptake in both study arms of HTC, ART including viral suppression, MC and PMTCT services and describe major outcomes.

\*Revisions in Version 5.0 of the protocol extended the interval between the first annual household follow-up visit at T1 and the second/final household visit at T2 to approximately 18 months, rather than 12. "AHS" will still be used to refer to follow-up visits to the 20% households.

#### 2) HIV Incidence cohort (HIC)

The HIC, enrolled during the BHS, will be followed to assess cumulative HIV incidence over approximately 30 months, which is the primary study outcome of interest. HIV genotypes of incident infections will be analyzed to allow description of which incident infections in the HIC are linked to HIV-

infected persons residing in the same study arm. Comparison of linked HIV incidence rates between arms may inform analysis of intervention effectiveness. The HIC is described in the *Evaluation Protocol*.

ART, Strengthened PMTCT and MC Services)

Matched community pairs will be randomized 1:1 to Enhanced Care or Combination Prevention arms (15 communities per arm). Combination Prevention communities will receive the combination prevention intervention package, which includes strengthened HIV testing and counseling, universal ART, and strengthened male circumcision services. To reach high coverage levels of HTC, campaigns will be implemented after BHS and continue with ongoing services in the Combination Prevention arm. Universal ART with linkage to care and adherence support will be offered to eligible HIV-infected persons referred through the study from BHS/AHS or HTC services and routine testing, as well as to existing patients already enrolled in care at the Combination Prevention community clinics. Services for pregnant women will be strengthened for third trimester retesting of women with a previous HIV-negative test; linkage to HIV treatment for all HIV-infected pregnant and post-partum women; and retention on ART post-delivery. To reach high coverage levels of male circumcision in HIV-uninfected adult men, MC campaigns with strengthened linkage to MC services will be conducted in Combination Prevention communities. Programmatic intervention activities are described in the *Intervention Protocol*.

# 4) End of study survey (ESS)

An end of study survey (ESS) targeting 100% of households in three community pairs (3 Combination Prevention communities and 3 Enhanced Care communities) will be used to estimate and compare Combination Prevention package uptake between arms. The ESS is described in the *Evaluation Protocol*.

5) Laboratory Research Activities (Viral Genotype Analysis and Point-of-Care Viral Load Validation) Laboratory research activities will be used to map genotypes from HIV-infected individuals identified during the BHS, HTC, and ESS and from seroconverted individuals in the HIC. All HIV-infected adults will be asked for consent to allow viral genotype analysis. Genotyping will help to inform viral genotype maps of Enhanced Care community and Combination Prevention community arms. These viral genotype analyses will be used to assess whether the proportion of new infections that are linked to circulating HIV-1 variants in the same arm, declines over time in the Combination Prevention arm. Procedures related to this genotyping are described in the *Evaluation Protocol*. The accuracy and feasibility of point-of-care viral load testing will also be assessed in comparison to standard viral load platforms.

FIGURE S1: Overview of Surveys and HIV Incidence Cohort in the Evaluation Protocol



# **Equipoise**

In individually randomized trials involving human participants, equipoise is the ethical requirement that, at the start of a trial, there be a state of honest, professional disagreement in the community of expert practitioners as to the preferred treatment. Beneficence, the moral obligation not to harm needlessly, and when possible, to promote the welfare of research subjects, is a key ethical principle underpinning the concept of equipoise.

In this study, investigators believe there is equipoise, since impact of combination HIV prevention programs on population-level adult HIV incidence has not yet been rigorously demonstrated, and professional disagreement about the effectiveness of combination prevention and the need for a thorough evaluation of its impact has been published in the scientific literature. Therefore, based on current scientific evidence for and against the combination prevention package, randomizing a community to either Enhanced Care or Combination Prevention arms does not breach the trust relationship between the state and the community.

Combination prevention will be compared to an enhanced standard of care in the Enhanced Care communities. The Enhanced Care communities will benefit in several ways from participation in the project. First, residents in the 20% households participating in the BHS and related activities (outlined in the Evaluation Protocol) will be offered the following procedures, which may confer direct health benefits: home-based HIV counseling and testing; point-of-care CD4 testing for HIV-infected, treatment-naive residents; HIV-1 RNA testing for HIV-infected residents (HIV-1 RNA sample drawn in the household); and referral to local HIV care and treatment clinics for HIV-infected residents who are not on treatment and/or not actively engaged in care. Second, the BCPP will also provide guidance and technical support for quality management and data systems at all laboratories and local clinics at which individuals receive HIV care and treatment, including those in the Enhanced Care communities. The MOH will receive technical assistance to support improved implementation and utilization of

clinical data systems (primarily PIMS2 and IPMS) in all 30 study communities. It is likely that resulting improvements in medical data systems and in quality management will help improve the general quality of care and treatment of all community residents attending these clinics.

To maintain the trust relationship between the study team and the community during study conduct, analyses are proposed for interim DSMB review to ensure that the DSMB can recommend early stopping of the trial if efficacy is demonstrated early. If efficacy is demonstrated, scale-up of the combination prevention package in Enhanced Care communities would be encouraged by investigators, although implementation would be based on funding availability and guidelines from the MOH.

#### **BCPP STUDY COORDINATION AND GOVERNANCE**

Implementation of the BCPP protocols will be coordinated using BCPP standard operating procedures and manuals, integrated across protocols where possible. Roles and responsibilities for program implementers and study investigators are defined in each of the protocols and will be described in detail in the BCPP Study Manual. While some overlap exists due to the design of the different protocols, Harvard Chan School/BHP will have primary responsibility for the *Evaluation Protocol* and CDC/MOH will have primary responsibility for the *Intervention Protocol*. During its abbreviated implementation the CDC/MOH had primary responsibility for the *CCC Protocol*. Due to the interlocking nature of the BCPP protocols, a joint project data management team, chaired by representatives from MOH, Harvard Chan School, BHP, and CDC, will be formed to build and manage the research data collection systems/overall research database for the BCPP.

#### viii. **EVALUATION PROTOCOL SYNOPSIS**

The *Evaluation Protocol* of the BCPP describes the rationale for and procedures related to evaluation of the primary endpoint (HIV incidence), as well as some key related secondary endpoints. This protocol therefore focuses on the Baseline Household Survey; the HIV Incidence Cohort; research-related blood sample collection; and an End of Study Survey.

# **Primary Objectives of the Evaluation Protocol:**

- 1. To determine whether implementation of a combination prevention (CP) package can significantly reduce population-level, cumulative HIV incidence in 16-64 year old residents in Botswana over a period of approximately 30 months.
- 2. To estimate population-level uptake of HIV testing, ART, VL suppression, male circumcision, and PMTCT services and compare service uptake between Enhanced Care and Combination Prevention communities at baseline and at study end.
- 3. To estimate the cost per additional HIV infection averted in combination prevention compared with Enhanced Care communities.

# **Study Design:**

The study is a pair-matched community-randomized trial.

# **Study Population:**

Thirty community clusters will be selected from three geographic regions in Botswana. Prior to randomization, community pairs will be matched on community characteristics thought to be associated with the outcome of interest (HIV incidence). The average total population size of each of the targeted communities is 6,027, giving a total population across all 30 communities of about 180,800, of whom about 105,000 are adults aged 16-64.

#### **Study Procedures:**

Matched community pairs will be randomized 1:1 to Enhanced Care or Combination Prevention arms (15 communities per arm). Randomization will occur prior to initiation of study activities (including the BHS).

Within each community, a baseline household survey (BHS) of approximately 20% of randomly selected households will be implemented to (1) establish an HIV incidence cohort (HIC) consisting of eligible consenting HIV-negative household members aged 16-64 years, and (2) estimate baseline coverage of the CP package.

Combination Prevention communities will receive the Combination Prevention intervention package immediately after completion of the BHS. All study communities, including Enhanced Care communities will receive guidance and technical support for quality management and data systems at all laboratories and local clinics at which individuals receive HIV care and treatment.

The HIC will be followed during AHS visits to assess cumulative HIV incidence over approximately 30 months, which is the primary study outcome of interest. Study participants who are not eligible for the

HIC will also be followed in the AHS, to assess, in both study arms, uptake of HTC, ART, MC and PMTCT in each arm and to describe major health outcomes (such as death).

To meet the second primary objective, an end-of-study survey (ESS) targeting 100% of households in selected pairs of communities will be used to estimate and compare CP package uptake between arms.

To understand HIV transmission patterns in Combination Prevention and Enhanced Care communities, HIV-1 genotyping will be performed. Because sexual mixing outside of a study arm will likely be an important source of contamination, circulating HIV-1 variants in Combination Prevention and Enhanced Care communities will be genotyped, and genotyping data will be translated into HIV transmission network(s). The genotyping data will be used to estimate the spatial location (community) of HIV infection for identified newly infected individuals. Specifically, the HIV genotyping data will estimate a potential link for each incident case in the study, and distinguish between linked (new incident infections between members of the same study arm), and unlinked (new incident infections transmitted from outside the study arm). The HIV-1 genotyping in Enhanced Care and Combination Prevention arms will be performed through sample collection from consenting HIV-infected adults in the BHS and newly infected individuals in the 20% households taking part in the household surveys throughout the study; from HIV-infected adults newly-identified through the HTC campaigns in the Combination Prevention communities; from all HIV-infected adults accessing HIV care and treatment at local clinics in the Combination Prevention communities; and from participants in the ESS in both the Enhanced Care and Combination Prevention arms. The HIV genotyping data will also be used to assess whether the proportion of new infections that are linked to circulating HIV-1 variants in the same arm declines over time at a different rate from those infections that are not linked to circulating variants from the same arm, in the Combination Prevention communities.

#### **Duration:**

Study activities will occur over a period of approximately 50 months. The BHS will be completed in approximately 24 months. Each incidence cohort will be followed for an average of approximately 30 months.

#### Sample Size:

With approximately 300 HIV-negative individuals enrolled in the HIC in each of 30 communities, the estimated size of the HIC will be 4,500 per study arm or 9,000 in total. Original model simulations estimate that over a 3-year study follow-up period of the HIC, rapid scale-up of interventions will result in cumulative adult HIV incidence of 0.024 in the Combination Prevention arm compared with 0.041 in the Enhanced Care arm (40% reduction). Assuming a coefficient of variation (k) of 0.26, and alpha of 0.05, an average community HIC size of 300, with 15 communities per arm, in a pair-matched design, should allow 86% power to detect the estimated difference in cumulative adult HIV incidence between study arms, by the end of three years of HIC follow-up. Sample size was determined based on these original power estimates. To update estimates of study power, a simulation study was undertaken using a range of updated input parameters. These were based on observed BCPP data from the first several community pairs and on speculation regarding roll-out of UTT. As expected, these demonstrate some reduction in power compared to that described in the previous versions of the protocol, but power exceeded 60% in the tables displayed in Section 5.1.1.

# 1. INTRODUCTION AND BACKGROUND

# 1.1. Epidemic in Botswana

Thirty years into the global HIV pandemic, HIV prevalence and incidence remain high in sub-Saharan Africa. Although this region represents only 12% of the world's population, it accounts for approximately 67% of the world's 34 million HIV-infected persons, and annually, about 70% of the world's 2.7 million new infections occur in this region (UNAIDS 2010). Despite Botswana's substantial progress in providing HIV treatment and prevention of mother-to-child transmission services (PMTCT) to its citizens, an estimated 25% of its adult residents are HIV-infected, the second highest adult HIV prevalence in the world; and about 14,000 persons in Botswana are newly infected with HIV annually, the third highest national HIV incidence rate globally (UNAIDS 2010).

#### 1.2. Combination Prevention

In recent years, several new HIV prevention interventions have proven to be highly effective at reducing transmission of HIV and have offered hope for containing and possibly reversing epidemics in sub-Saharan Africa. For HIV-negative men, male circumcision has been shown to significantly reduce HIV acquisition from HIV-infected female partners. Three randomized controlled trials of circumcision, involving more than 10,000 men in sub-Saharan Africa, demonstrated a 60% reduction in HIV acquisition risk (Auvert, Taljaard et al. 2005; Bailey, Moses et al. 2007; Gray, Kigozi et al. 2007). Additionally, antiretroviral treatment (ART) of HIV-infected persons has been shown to reduce viral load and consequently the risk of HIV transmission to uninfected partners in sero-discordant couples by as much as 96% (Cohen, Chen et al. 2011). Similarly, the use of antiretrovirals to prevent transmission of HIV from infected mothers to their infants during pregnancy, birth, and breastfeeding can reduce transmission to about 1% (Shapiro, Hughes et al. 2010).

Despite considerable success in scaling up these interventions in many sub-Saharan African countries, especially those supported by the U.S. President's Emergency Plan for AIDS Relief (PEPFAR), adult HIV incidence has remained high (>1%) in many regions in Southern Africa (Botswana, Swaziland, Lesotho, Kwa-Zulu Natal in South Africa, and Southern Mozambique). Multiple factors may account for high HIV incidence in this part of the world. Firstly, viral characteristics of HIV-1 subtype C, endemic in Southern Africa, may make it more infectious than other viral subtypes (Novitsky, Wang et al. 2010; Novitsky, Ndung'u et al. 2011). For example, recent evidence suggests that about one third of persons infected with HIV-1 subtype C, maintain very high viral loads (VL>50,000 copies/ml) for more than 6 months after sero-conversion.

Secondly, the scale and quality of the HIV prevention interventions (HTC, ART, MC and PMTCT) may have been insufficient to reduce HIV incidence among adults in Southern Africa to levels observed in other parts of the world. For example, the main mechanism by which scale-up of HTC and ART reduces HIV transmission risk in the community, is by reducing viral load in resident HIV-infected persons, ideally to undetectable levels (VL<400 copies/ml). Studies have suggested that every 0.5 log reduction in an individual's HIV-1 viral load is equivalent to a 40% reduction in individual HIV transmission risk (Modjarrad, Chamot et al. 2008), and once the viral load is fully suppressed (VL <400 copies/ml) individual HIV transmission risk is virtually zero (Attia, Egger et al. 2009). Despite considerable scale-up

of access to HTC and ART, poor retention of HIV-infected persons in the HIV care and treatment cascade from diagnosis to ART follow-up (Rosen and Fox 2011), has certainly mitigated the ability of HTC and HIV care and treatment programs in Southern Africa to reduce the prevalence of HIV-infected persons with detectable viral loads (VL>400 copies/ml). In a meta-analysis of pre-ART retention in Africa, Rosen et al. reported that only 59% of newly diagnosed adults are successfully linked to HIV care and treatment services, only 46% are retained from initial registration and staging at the facility to ART-eligibility, and only 68% are retained from ART eligibility to ART initiation (Rosen and Fox 2011). Of those adults who initiate ART, ~30% are no longer on therapy by 3 years of follow-up, with most of those no longer in care considered lost to follow-up (Fox and Rosen 2010). Therefore, even if 50% of HIV-infected adults in Botswana know their HIV status (Central Statistics Office 2009), a considerably lower proportion are expected to have a suppressed viral load (Gardner, McLees et al. 2011). The remaining HIV-infected adults with unsuppressed viral load are still infectious and spreading virus in the community. Additionally, achieving high coverage of male circumcision among HIV-negative males has also been challenging with most countries, including Botswana, unable to meet ambitious 80% coverage targets to date (Curran, Njeuhmeli et al. 2011).

In summary, despite having the tools to end the HIV epidemic (Fauci and Folkers 2012), insufficient scale, quality, and coordination of prevention interventions has significantly limited southern Africa's ability to sufficiently curb the HIV epidemic. This has led public health experts to call for a "combination prevention" strategy that involves implementing multiple prevention interventions with known efficacy in a geographic area at a scale, quality, and intensity to impact the epidemic (Merson, Padian et al. 2008). Although most experts agree that synchronized implementation of a combination of prevention interventions is needed, there remains considerable debate about what components should be included in the essential combination prevention package (Merson, Padian et al. 2008; Halperin 2009). However, four evidence-based interventions including HTC, ART, MC and PMTCT followed by indefinite ART are recommended for scale-up by almost all prevention experts and will form the cornerstone of the combination prevention package proposed as part of this project (see Section 1.3 below).

#### 1.3. The Proposed Combination Prevention (CP) Package

Based on experimental evidence for prevention interventions discussed above, the proposed combination prevention (CP) package to be delivered as part of the BCPP *Intervention Protocol* will include accelerated scale-up and expansion of HTC, active linkage to HIV care and treatment according to local eligibility criteria, expanded ART among all HIV-infected residents regardless of WHO Stage or CD4 count; strengthened support for retention in care and ART adherence, and strengthened active linkage to expanded MC and PMTCT services. Under versions 1.0 and 2.0 of this protocol, the combination prevention package included expanded ART for individuals with CD4>350 cells/μL plus HIV-1 RNA ≥10,000 copies/mL, or pregnancy/breastfeeding (Option B+). Under version 3.0 of this protocol, the combination package included expanded ART for individuals with WHO Stage I/II and CD4 counts 351–500 cells/μL or with WHO Stage I/II and CD4 counts >500 cells/μL and high HIV-1 RNA levels (≥10,000 copies/mL). Option B+ was offered beginning with version 3.0 in both Combination Prevention and Enhanced Care communities with the adoption of this policy by the Botswana government in April 2015. Beginning with version 4.0 of this protocol, universal test and treat was offered in the Combination Prevention arm. Enhanced Care communities have received the Botswana standard of care in effect as it changes over time (see the Schema and Section 5.1.1 for discussion of

the standard of care and services in Enhanced Care communities). Version 5.0 of the Evaluation Protocol takes into account that universal ART is available to residents of both Enhanced Care and Combination Prevention Communities following the Botswana government's adoption of "Treat All" in June 2016.

In 2014, the Joint United Nations Programme on HIV/AIDS (UNAIDS) proposed new targets directed at ending the AIDS epidemic (UNAIDS 2014). Namely, that by 2020, 90% of all people living with HIV will know their HIV status; 90% of all people with diagnosed HIV infection will receive sustained combination antiretroviral therapy (ART); and 90% of all people receiving ART will have viral suppression The targets of the study combination prevention package meet, and in some cases exceed, those for the UNAIDS 90-90-90.

To reach stated scale-up targets (see BCPP Schema) several service uptake initiatives will need to be implemented, including (1) community mobilization to encourage HTC and MC uptake, (2) strengthening linkage to ART and/or PMTCT services for newly diagnosed HIV-infected adults, (3) strengthening of linkage to MC services for HIV negative males identified at HTC services, (4) expansion of HTC, ART, PMTCT and MC services through recruitment of additional health care personnel, and where necessary, creation of new infrastructure (e.g. new male circumcision surgical units), and (5) monitoring and evaluation of prevention programs to ensure stated targets are reached.

Adults aged 16-64 will be targeted for service uptake because recent, nationally representative surveys of HIV prevalence and incidence (Central Statistics Office 2009) suggest that HIV incidence remains high (>1%) throughout this age group. Modeling exercises (presented in Section 5) suggest that meeting scale-up targets by the end of two years of program implementation, and maintaining treatment coverage thereafter, could result in community HIV incidence reductions of approximately 40% by the end of 2.5 years of implementation.

The *Intervention Protocol* describes the details of implementing the CP package in the study communities.

# 2. STUDY OBJECTIVES

#### 2.1. Primary Study Hypothesis

Implementing the CP package will impact the HIV/AIDS epidemic by reducing the incidence of HIV infection in a defined geographic area within approximately 2.5 years and will be cost-effective.

# 2.2. Primary Objectives

1) To determine whether implementation of a combination prevention (CP) package can significantly reduce population-level, cumulative HIV incidence in 16-64 year old residents in Botswana over a period of approximately 30 months.

- 2) To estimate population-level uptake of HIV testing, ART, VL suppression, male circumcision, and PMTCT services and compare service uptake between Enhanced Care and Combination Prevention communities at baseline and at study end. The service uptake indicators will include:
  - The proportion of 16-64 year-old community residents who report knowing that they are HIV-infected, or report testing HIV-negative in the preceding 12 months.
  - The proportion of 16-49 year-old HIV-negative men, resident in the study communities who are circumcised.
  - The proportion of HIV-infected 16-64 year-old adult community residents who know they are HIV-positive and are receiving ART.
  - The proportion of HIV-infected 16-64 year-old community residents who know they are HIV-positive, are receiving ART, and have HIV-1 RNA ≤400 copies/mL.
  - The proportion of eligible, HIV-infected pregnant women, resident in study communities, who remained in care and on treatment 12 months post-delivery after initiating ART for Option B+.
- 3) To estimate the cost per additional HIV infection averted in Combination Prevention compared with Enhanced Care communities.

# 2.3. Evaluating the Impact of Combination Prevention: Design and Rationale to Address Primary Objectives

Although modeling studies suggest that implementation of the stated CP Package can significantly reduce HIV incidence and may be cost-effective, rigorous evidence to support these projections of population-level impact is needed if national and international bodies are to justify further investment in combination prevention strategies (Lancet 2010; Padian, McCoy et al. 2011). For funders to be confident in the effectiveness of the proposed CP package, this evaluation would need to: (1) demonstrate a measureable reduction in adult HIV incidence and (2) be able to attribute any observed incidence reduction to scale-up of the CP package. The first two primary study objectives for the BCPP Evaluation Protocol are designed to meet these needs.

Current global economic realities have resulted in level or declining availability of funding for HIV/AIDS programs (Stover, Korenromp et al. 2011). Therefore, the proposed third primary objective is to evaluate the cost-effectiveness of CP package implementation in Botswana.

A randomized design is proposed to provide experimental evidence of CP package impact, and because population-level HIV incidence is the outcome of interest, we propose a community (rather than individual) randomized trial (CRT).

In summary, 30 study communities, considered representative of the rural and peri-urban populations of Botswana, will be selected and matched into pairs based on community characteristics thought to be associated with HIV incidence, which is the outcome of interest (see section 4.2 and Appendix C2 for matching criteria). Pair-matching is done to improve balance between study arms and statistical efficiency (Hayes and Moulton 2009). Communities within pairs will be randomized to Combination Prevention or Enhanced Care arms. Following community matching and randomization, a baseline 20% household survey (BHS) will be implemented to recruit an HIV incidence cohort (HIC) of eligible, consenting, HIV-negative adults aged 16-64. Through activities described in the BCPP *Intervention Protocol*, the CP package will be scaled up to target levels within two years post-randomization in

Combination Prevention communities with treatment coverage levels maintained thereafter. The HIC will be followed at approximately 12 months (T1) and 30 months (T2) after enrollment to measure cumulative HIV incidence. A small number of communities may receive a third follow-up at 36 months (T3) as stipulated by protocol versions 1.0-4.0, depending upon the timing of approval and roll-out of version 5.0 of the *Evaluation Protocol*. In addition, a small number of communities will have had their second follow-up visit at T2 according to the original study design and schedule. All data collected from these study visits under previous versions of the protocol and the former study schedule will contribute to the final analyses. Cumulative HIV incidence will be compared between Enhanced Care and Combination Prevention arms to assess CP package impact. Households that participated in the BHS will be visited (as part of the HIC follow-up activities). Residents of these households who are not participating in the HIC will also be asked to complete a survey at each follow-up visit to help provide CP package coverage estimates during the course of the study. The overall evaluation study design is illustrated in Figure S1 in the BCPP Schema (section vii), and the rationale for the sample sizes is provided in Section 5.

We propose a parallel group CRT design rather than a step-wedge design primarily because a step-wedge design is considered infeasible. A step-wedge design would entail enrollment of multiple HIV incidence cohorts sampled, recruited and followed within the short time period of any one "step" and this would be expensive and beyond the realm of feasibility. In addition, a parallel group CRT is generally regarded as providing stronger experimental evidence of impact compared with a step-wedge design because any pre-existing trends in HIV incidence will be controlled for at the design stage, rather than modeled in an adjusted analysis as would need to occur in a step-wedge trial (Hussey and Hughes 2007; Hayes and Moulton 2009).

A pre- versus post-study design would not generate evidence of similar strength to that of a parallel group CRT (Habicht, Victora et al. 1999; Hayes and Moulton 2009). Previous pair-matched CRTs to assess impact of complex program interventions on adult HIV incidence have been successfully implemented in Africa, and this lends support to the feasibility of our proposed design (Hayes, Mosha et al. 1995).

We propose directly measured HIV incidence as the primary outcome of interest, because fewer assumptions are required for direct HIV incidence measures, and this is still regarded as the gold standard technique for estimating incidence (Kim, Hallett et al. 2011).

We propose that the HIV incidence cohort (HIC) remain open such that HIV-negative adults aged 16-64 who migrate into HIC households, or adolescents who age into eligibility during study conduct, or other participants who become eligible during study conduct, be offered the opportunity to enroll in the HIC at T1. An open, rather than a closed cohort, has been selected because (1) this should help to keep the incidence cohorts representative of their respective communities, (2) this has some sample size advantages, and (3) analysis techniques to manage open rather than closed HIV incidence measures are available and not inferior. The advantages of an open, rather than a closed, cohort should outweigh the disadvantages, which includes possible intervention contamination of Enhanced Care communities (see Section 2.5.1).

To meet the second primary objective, CP package coverage in the community will be estimated at baseline and annually in the 20% households, and through an end of study survey (ESS) that targets all

households in 6 of the 30 study communities. Targeting 100% of households in 6 communities in the ESS allows for obtaining more precise estimates of CP package coverage (see Section 5 for precision estimates), and permits comparison of estimated coverage in the 20% households with that in the rest of the community.

To meet the third primary objective, costing data will be collected prospectively, and used in combination with impact estimates derived from the CRT. The cost-effectiveness analysis and methods for collecting costing data are described in Section 7.

# 2.4. Secondary Objectives

- 1) To estimate the extent to which incident HIV infections in Combination Prevention and in Enhanced Care communities arise from HIV strains circulating within communities randomized to the same study arm as the incident case or from strains circulating outside those communities (sexual network mixing) by: (1) genotyping the circulating HIV-1 variants in Enhanced Care and Combination Prevention arms, and (2) estimating the proportions of new HIV infections that can and cannot be phylogenetically linked to HIV-infected persons in the same study arm.
- 2) To estimate the efficacy of the Combination Prevention package on reducing the rate of new infections with HIV strains circulating within communities in the same study arm.
- 3) In the intervention arm only, to estimate over time, the proportion of incident HIV-1-infections that can be linked to HIV-infected adults of the same study arm.
- 4) During the end of study survey (ESS) to compare Combination Prevention (CP) package uptake within 20% households to CP package uptake in the broader communities they represent.
- 5) To obtain secondary cross-sectional estimates of community HIV incidence at baseline and study end in Enhanced Care and Combination Prevention communities through use of HIV-incidence assays.
- 6) At baseline, during study conduct, and at study end, to estimate the proportion of recent HIV infections in Combination Prevention and Enhanced Care communities with evidence of transmitted HIV drug resistance.
- 7) To estimate the proportion of HIV-infected adults with undetectable viral load (VL<400 copies/ml) and to estimate the community viral load at baseline, during study conduct, and study end in Combination Prevention and Enhanced Care communities.
- 8) To estimate the association between HIV-1 viral load and HIV transmissions using viral linkage data.
- 9) To project HIV infections and deaths (attributable to AIDS) averted in the combination prevention and Enhanced Care communities beyond the time frame of the trial.
- 10) To estimate the cost of provision of intervention services.

- 11) To estimate the cost-effectiveness of combination prevention (taking into account both infections averted and clinical costs) using the two arms from the trial as well as an additional model-based strategy.
- 12) To compare CD4 and viral load trajectories over time, among HIV-infected ART-naive persons who reside in Combination Prevention vs. Enhanced Care communities.
- 13) To assess the accuracy and feasibility of point-of-care viral load testing in comparison to standard viral load platforms.
- 14) To understand (through qualitative interviews) barriers to and facilitators of linkage to care and ART initiation among BHS participants.
- 15) To use BCPP data in analyses of the rates of and risk factors for major AIDS and non-AIDS illnesses/injuries/mortality among persons living with and without HIV in Botswana.

# 2.5. Design and Rationale to Address Secondary Objectives

#### 2.5.1. Contamination

There are several sources of potential contamination in the proposed trial. This contamination can affect interpretation of results concerning the efficacy of the ART-related interventions in reducing HIV transmission in this trial, and is hence addressed in secondary objectives #1-2 (sexual network contamination) and secondary objective #4 (intervention contamination).

**Sexual network contamination** will almost certainly occur; available evidence from a recently conducted community survey in Mochudi (a district in southern Botswana) showed at least 30% of surveyed adults reported sexual partnerships with adults outside the community (unpublished data). Therefore, during trial conduct, sexual network contamination may occur in four ways:

- o Enhanced Care HIC members may become HIV-infected through relationships with: (1) non-study community members, or (2) Combination Prevention community members
- o Combination Prevention HIC members may become HIV-infected through relationships with: (1) non-study community members, or (2) Enhanced Care community members

Because Botswana's population is congregated largely in the eastern part, which constitutes a relatively small geographic area, and because the population is widely mobile anyway (Central Statistics Office 2009), attempting to separate study communities by large "buffer zones" or geographic boundaries (e.g. mountainous regions) is not considered a feasible option for trying to reduce sexual network contamination. Instead, investigators propose HIV-1 genotyping to enumerate circulating HIV-1 variants in Combination Prevention and Enhanced Care communities. Clustering of HIV-1 sequences implies that hosts are connected by a chain of viral transmission. Clustered HIV-1 sequences represent viral variants that circulate and spread in the communities where the analyzed blood specimens originate. The planned genotyping will help assess which new incident infections in the HICs were transmitted from members of the same study arm (phylogenetically linked infections), and which were transmitted from outside the study arm (unlinked infections). Similar methodology

has been successfully used in HIV prevention trials involving sero-discordant couples (Cohen, Chen et al. 2011). More details related to the proposed analyses are described in Sections 8 and 10.

A high density of sampling is necessary to increase the accuracy of viral linkage analysis. To assess patterns of HIV-1 transmission, blood samples for HIV-1 genotyping will be collected from:

- All consenting HIV-infected individuals identified in the BHS upon enrollment, and at AHS visits and during the ESS in participating Combination Prevention and Enhanced Care communities.
- All consenting newly identified HIV-infected adults identified in the HIC in both Combination Prevention and Enhanced Care communities, at T1 and T2.
- All consenting HIV-infected adults who present to HIV care/treatment clinics after being identified in the first HTC campaigns in Combination Prevention communities.
- All consenting HIV-infected adults receiving HIV care and/or treatment at local clinics in the Combination Prevention communities (including those already in care/on ART at the start of the study).
- All consenting newly diagnosed HIV-infected adults in the second HTC campaign (HTC2) and thereafter in the Combination Prevention communities who present to HIV care/treatment clinics.

The importance of genotyping in assessing and possibly controlling for sexual network contamination is captured in the first two secondary objectives. To meet the first secondary objective, we will assess the proportions of *linked* vs. *unlinked* incident cases in the Combination Prevention and Enhanced Care communities that are identified within the 20% of households participating in surveys, over the course of the study. This will allow us to estimate the extent of sexual network contamination of the HIV incidence cohorts.

To meet secondary objective #2, we will evaluate genotypes from the same groups as in secondary objective #1 (i.e., HIV-infected residents of the 20% of households participating in surveys over the course of the study, in both arms). This analysis, however, will include only phylogenetically *linked* incident cases. This analysis will therefore control for sexual network contamination by including only linked incident cases in the analysis of CP package impact.

The additional purpose of HIV-1 genotyping is captured in the 3<sup>rd</sup> secondary objective, which targets all HIV-infected residents in Combination Prevention communities. In secondary objective #3, we will estimate how the proportion of linked incident cases (in Combination Prevention communities only) changes over time. If the CP package is effective in reducing population-level HIV incidence, there should be a reduction in the proportion of recent infections that can be phylogenetically linked to HIV-infected persons in Combination Prevention communities.

**Intervention contamination** will occur mainly in three ways: (1) through Enhanced Care community members accessing interventions in Combination Prevention communities, (2) through Combination Prevention community members accessing Enhanced Care outside the Combination Prevention communities, and (3) through study procedures (such as HIV counseling and testing) related to the BHS and HIC (which may affect the Enhanced Care communities, in particular).

Several approaches (detailed in the *Intervention Protocol*) will be undertaken in an attempt to decrease intervention contamination between Enhanced Care and Combination Prevention communities. However, to assess the extent and nature of the intervention contamination that will inevitably occur, CP package uptake will be compared between Enhanced Care and Combination Prevention communities during the end of study survey (ESS), as described in primary objective #2.

With regard to contamination related to the BHS and HIC, BHS and HIC study procedures include: (1) HTC and point-of-care CD4 and referral of HIV-infected persons to HIV care and treatment services, and (2) encouragement of annual HTC and risk reduction measures for HIV-negative adults, combined with counseling about MC benefits for HIV-negative males. These procedures could introduce an unintentional intervention in the Enhanced Care communities (in the BHS and HIC participants). These procedures could also make the HIC less representative of the broader community of residents, even in the Combination Prevention communities. Unfortunately, this type of contamination is unavoidable as the study cannot be conducted without implementing these study procedures in all communities. To assess possible intervention contamination introduced by study procedures in the BHS and HIC, investigators propose the 4<sup>th</sup> secondary objective.

Another aspect of study design may result in HIV incidence measured in the HIC not being representative of broader study communities (in addition to the intervention contamination described above): despite being an open cohort, observed incidence in the HIC may be different than incidence in the communities that it represents, because behavior of HIC enrollees may change simply because they are part of a study (the Hawthorne effect). Laboratory-based methods for estimation of HIV incidence are important tools for monitoring of HIV/AIDS epidemics and are attractive due to their simplicity, ease of use, low cost and application to single cross-sectional specimens collected during routine surveys. For accuracy of testing and reliable scale-up, cross-sectional HIV incidence estimates need to be compared with the longitudinal HIV incidence data and properly validated. Use of incidence assays will categorize HIV infections observed at baseline (during the BHS and first HTC campaign), and newly diagnosed and incident HIV-infections during study conduct (during HTC activities thereafter), during follow-up of the 20% households including the HIC, and at study end (during the ESS) as either prevalent or recent (new infection in the preceding 3-12 months depending on the algorithm of incidence testing). For cross-sectional estimates of HIV incidence, the cross-sectional assay-based data will be compared and validated by the longitudinal data on HIV incidence. In sum, the 5<sup>th</sup> secondary objective will assess whether cumulative HIV incidence observed in the HIC is representative of community incidence.

# 2.5.2. Transmission Dynamics

Surveillance of transmitted HIV drug resistance (TDR) among recently infected individuals can inform treatment guidelines and provide feedback on the success of HIV-1 treatment and prevention programs. Increasing prevalence of transmitted drug-resistance mutations in the population may adversely impact the use of HIV treatment regimens. Therefore, surveillance of transmitted HIV drug resistance will address whether a rapid scale-up of ART in Combination Prevention communities is associated with the increasing prevalence of transmitted drug resistance (as compared with Enhanced Care communities). Secondary objective #6 addresses this concern.

As described earlier, the mechanism by which expanded access to ART should achieve a prevention effect is through lowering the proportion of HIV-infected adults in the intervention community with detectable viral loads (VL>400 copies/ml) (Montaner, Lima et al. 2010). To explore whether the treatment strategy in Combination Prevention communities achieved this aim, investigators propose to estimate the proportion of HIV-infected adults participating in the BHS, HIC and ESS with undetectable HIV-1 viral loads. This is captured in the 7<sup>th</sup> secondary objective.

Assessing the prevention efficacy of any single prevention intervention on its own will not be possible as part of this CRT as multiple prevention interventions will be implemented simultaneously. However, among linked recent HIV infections that are identified at baseline, during 20% household follow-up, during HTC in Combination Prevention communities, and ESS, assessing the proportion that are associated with HIV transmission from adults with high viral load (e.g. VL ≥10,000 copies/ml and other thresholds) could improve understanding of the proportion of incident infections in study communities that might be averted by the initially proposed treatment-as-prevention strategy and/or UTT. This is captured in the 8th secondary objective.

# 2.5.3. Cost and Cost-effectiveness

Assessing cost-effectiveness of the proposed CP package is crucial if potential funders and national governing bodies are to continue investment in the CP package after study completion.

The Cost-Effectiveness of Preventing AIDS Complications International (CEPAC-I) model will be used to assess expected outcomes from the proposed combination prevention programs in Botswana. The cost effectiveness analysis will evaluate three combination HIV prevention strategies: the two arms from the trial and an additional model-based strategy, the "optimized package". The "optimized package" provides a model-based scenario based on the intervention arm, but will assess the case where linkage to routine HIV care, ART, and HIV screening are further optimized, pre-exposure prophylaxis is administered, and may incorporate additional prevention strategies.

Model-based cost-effectiveness analysis is critical to understanding the value of clinically effective prevention and therapeutic strategies. Model-based analyses have a number of attractive features, such as allowing one to: a) organize and synthesize trial data; b) handle uncertainty and forecast beyond a single trial via sensitivity and "what-if" analysis and c) extrapolate to longer time horizons, new geographic settings, and alternative target populations. With regard to HIV/AIDS, models have been used in multiple settings to evaluate the epidemiologic and policy implications of preventive interventions, to study the cost effectiveness of different treatments, to evaluate screening programs, to determine future resource needs, and to inform the design of clinical trials.

Secondary objectives (#9-11) pertain to cost and cost-effectiveness analyses. These will provide critical information to policy makers, following completion of the trial.

# 3. OVERVIEW OF STUDY METHODS

As described in the BCPP Schema (section vii), the over-arching design is a pair-matched community randomized trial (CRT) that will be completed over the course of approximately 5 years. To facilitate

description in this protocol the study methods are divided into six components. Harvard/BHP will have responsibility for 1, 2, 4, and 5 and CDC/MOH will have responsibility for 3.

- 1) The baseline household survey (BHS) (with subsequent annual household surveys, AHS)
- 2) Follow-up of the HIV incidence cohort (HIC) and BHS participants
- 3) Programmatic interventions in Combination Prevention communities
- 4) The End of Study Survey (ESS)
- 5) Laboratory Research Activities (Viral Genotype Analyses)

This protocol describes the BHS/AHS, HIC, and ESS, and the viral genotype analyses of the BCPP impact evaluation including the following: study population eligibility criteria (Section 4.4), sample size estimates and sampling methods (Section 5), study procedures for the BHS/AHS, HIC and ESS and Research Blood Draws (Section 6), cost effectiveness analysis (Section 7), laboratory procedures (Section 8), data management issues (Section 9), approaches to analysis (Section 10) and issues related to ethical interaction with human subjects (Section 11). Section 12 provides a suggested study safety and clinical monitoring plan, and Section 13 a description of study logistics and responsibilities, including a data dissemination plan.

# 4. STUDY POPULATIONS

# 4.1. Selection of Study Communities

Thirty communities (Appendix C2) in three geographic areas in Botswana: (1) around Gaborone in the south east, (2) around Francistown in the north east, and (3) in the region around Mahalapye, Serowe, and Palapye in the central eastern region, are proposed for inclusion in the CRT. The rationale for selecting 30 communities is provided in Section 5 (sample size calculations). The communities in Appendix C2 are purposively selected and proposed based on (1) desired size, and (2) feasibility.

# Community size

Communities need to be large enough to meet sample size requirements yet not be so large that achieving ambitious CP package coverage targets is infeasible. Results of sample size calculations show that an average cluster size of about 300 HIV incidence cohort (HIC) enrollees per community is needed. To achieve this sample size, we are aiming to enroll approximately 500 potential HIC enrollees per community (300/0.85/0.70=500). The proportion of potential enrollees incorporates the expected impact of missing, refusal, capping the size of larger communities, and using back-up households.

Because investigators wish to minimize intervention contamination that may be introduced by repeat HIV testing and counseling of the HIC in Enhanced Care communities, we propose to keep the community HIC size at no more than 20% of the entire study community. Therefore, the ideal average community size proposed by investigators is about 5,750 persons [500/(0.58\*0.75\*0.2) = 5,747] [Note: 0.58 is the proportion of the community considered age-eligible (Appendix C2), 0.75 is the proportion of adults HIV-negative, and 0.2 is the desired sampling proportion for the HIC]. Investigators therefore searched for communities of size 2,500—15,000, aiming for an average size of 5,750. Slightly less than 20% of households from the 30 study communities will take part in the BHS and HIC. Note that although this sample will likely be somewhat less than 20% of households,

we will refer to these as the "20% households" from this point forward, for ease of reference (please see Sections 5.1.3 and 5.1.4 for details regarding selection of the 20% households).

# Feasibility

This project represents a significant logistical operation over the course of 5 years. To maintain feasibility, investigators propose that all communities need to:

- Have a health center, from which HIV care and treatment, PMTCT, and HTC or MC services can be provided.
- Be reachable by road, via a ≤8 hour drive from Gaborone or Francistown. (CDC and MOH have permanent, well-staffed offices in Gaborone and Francistown, while Harvard has a permanent office in Gaborone. This makes the study easier to implement and monitor for quality control purposes).
- Have a clear geographic boundary such that it is reasonably easy to identify a household as either being part of, or outside of, the study community.

These feasibility inclusion criteria resulted in the exclusion of urban areas from the study, and the inclusion of rural and peri-urban areas.

The 30 study communities proposed meet the criteria described above. The average total population size of each of the targeted communities is 6,027. Therefore, we estimate a total population in study communities of about 180,800 people, with 58% (104,864) aged 16-64 (Appendix C3). HIV prevalence among residents aged 16-64 is estimated at 25%, resulting in an estimated 26,216 HIV-infected residents aged 16-64, or 13,108 per study arm.

# 4.2. Matching of Study Communities

Due to the small number of communities that can be enrolled in community randomized trials for cost and feasibility reasons, there exists a chance of imbalance of potential confounders between study arms. Therefore, in this study we considered restricted randomization, matching, and stratification as strategies to ensure balance between arms. We chose a pair-matched design because:

- This approach is more likely than stratification to achieve balance between study arms;
- Matching has the added advantage of improving statistical efficiency compared with restricted randomization, and;
- Chosen matching covariates (see below) are quite closely correlated with the outcome of interest (adult HIV incidence), making a matched design of similar or increased statistical efficiency compared with a stratified design, even though a matched design entails greater loss of degrees of freedom.

Possible disadvantages of a pair-matched design include:

- Loss of both communities in a pair if one community drops out.
- It is not possible to assess whether the intervention effect varies between matched pairs, whereas, in a stratified design, opportunity to assess effect modification across strata would be possible.

The following community matching criteria were chosen:

- Community size: Although community size in Botswana may not be associated with the outcome of interest (HIV incidence), achieving sample size balance between arms improves statistical efficiency. Appendix C2 provides a comparison of communities within proposed matched pairs. Overall, proposed community HIC sizes range from 230 to 1,105; however, following matching, the median difference between community HIC size within matched pairs is 61, and ranges from 1-313.
- Baseline Access to Health Services including ART: Access to ART is associated with a decrease in new HIV diagnoses (Montaner, Lima et al. 2010; Tanser, Bärnighausen et al. 2013). Although some communities within matched pairs have access to primary care clinics, and others have access to primary care hospitals, investigators believe that in the context of Botswana, this does not represent a significantly different level of access to health services.
- Age structure: Adult HIV prevalence and incidence are correlated with adult age (Central Statistics Office 2009). Age structures are very similar within the study community pairs. If we use the proportion of adults (16-64) who are at highest risk for HIV infection (25-34) as an indicator of age structure, the median difference in this proportion is 2% (range 0-7%). Note that residents up to age 64 are included in the study, due to relatively high HIV prevalence (15-25%) in persons aged 50-64 years in Botswana, as well as a spike in HIV incidence (5.5%) in 60-64-year old men, both noted in the 2008 Botswana AIDS Indicator Survey, or BAIS. [Note: we do not have age structure data for Mandunyane or Mmadinare, but based on the age structure of the other 28 selected communities, do not expect any significant differences in age structure within the matched pairs].
- Geographic location as measured by proximity to major urban centers (Hayes, Mosha et al. 1995).
  Geographic locations of communities within pairs, as estimated by average distance to the nearest
  large urban centers, are quite similar. For example, across 30 communities, the range of average
  distances to nearby urban centers ranges from 18-380 kilometers. However, following matching,
  the median difference in distance to an urban center between communities in a matched pair is 20
  kilometers (range 3-150).

We do not have access to community-specific measures of HIV prevalence [e.g. HIV prevalence measured from antenatal care (ANC) clinics]. Previous successful pair-matched CRTs (Hayes, Mosha et al. 1995), where HIV incidence was the outcome of interest, have also addressed the problem of absent baseline HIV prevalence estimates by using geographic location and other proxies of HIV prevalence as matching criteria.

# 4.3. Definition of a Study Community Resident

The following definitions of study community residents will be used in the protocol:

• **Permanent study community resident:** An individual who reports spending on average ≥14 nights each month in that community over the preceding 12 months or an individual who recently moved into the community and reports spending on average ≥14 nights each month since arriving.

- Part-time study community resident: An individual who reports spending on average 3–13 nights each month in that community over the preceding 12 months or an individual who recently moved into the community and reports spending on average 3-13 nights each month since arriving.
- **Non-study community resident:** An individual who reports spending on average <3 nights each month in that community over the preceding 12 months.
- **Household member:** an individual who reports spending more nights (on average) in the household being sampled than in any other household in the same community over the preceding 12 months.
- Botswana Citizen: A Botswana citizen is anyone who can produce proof of Botswana citizenship.
  Usually this is the Omang number, which can be found on national ID cards, drivers licenses,
  Botswana passports, or an Omang application receipt. The Omang number is needed in Botswana
  to access routine government services. It is anticipated, based on a community survey in Mochudi,
  and the 2011 census (Central Statistics Office 2009), that less than 3% of residents will be noncitizens.
- **Spouse of Botswana Citizen:** A spouse of a Botswana citizen is a person who can produce evidence of being married to a Botswana citizen, usually a marriage certificate, and is therefore eligible to receive free medical services in Botswana.
- **Non-citizen:** A non-citizen is anyone who declares himself or herself as a non-citizen and/or cannot produce proof of Botswana citizenship.

# 4.4. Study Inclusion and Exclusion Criteria

# 4.4.1. Baseline 20% Household Survey (BHS)

The BHS will be conducted in the 20% households that are sampled from the participating study communities that have a total population of ≤6,000 residents; and approximately 273 households from the participating study communities that have a population over 6,000 residents (the latter is approximately 20% of residential and habitable plots for 6,000 residents). Eligible adults residing within these households will be asked to take part in the BHS. Eligible residents of the participating 20% households who did not take part in the BHS at T0--e.g. due to absence, etc.--and who are present during the subsequent AHS visits (prior to the final visit) will also be asked to complete the same procedures that are offered in the BHS. Following, we define inclusion/exclusion criteria (with regard to the BHS) for: (1) households, and (2) adults living within selected households.

# • **Household** Eligibility Criteria for BHS: Inclusion criteria

 The household should be located within the study community enumeration area map established for the 2011 national population census (Central Statistics Office 2009) or within established community boundaries where these maps are not available.

# • Household Representative Eligibility Criteria for BHS:

#### Inclusion criteria:

- Aged 18 years or older
- Household member
- o Willing to provide household information following administration of verbal consent script

# • Household Member Eligibility Criteria for BHS:

# **Inclusion criteria:**

- Aged 16-64 years
- o Permanent or part-time study community resident in any of the 30 study communities
- Household member
- O Botswana citizen or spouse of a Botswana citizen
- O Able to provide informed consent if  $\geq$ 18 years old, or able to provide assent to complement a guardian's permission, if a minor (aged 16 or 17)

# 4.4.2. HIV Incidence Cohort (HIC)

The HIV Incidence Cohort (HIC) will be enrolled from the 20% households participating in the BHS. The HIC will largely be enrolled during the BHS at T0; however, eligible residents of the participating 20% households who are present during AHS visits (prior to the final visit) and who were not previously enrolled to the HIC (e.g. due to absence, 15 years of age, etc.) will also be asked to enroll in the HIC (i.e., the HIC is an open cohort). Therefore, the **household** inclusion criteria described above for the BHS will apply to the HIC. Eligibility criteria for **HIV Incidence Cohort members** are as follows:

#### Inclusion criteria:

- Documented to be HIV-uninfected according to the rapid HIV test algorithm
- Aged 16-64 years
- Permanent study community resident in any of the 30 study communities
- Household member
- Does not intend to move out of the study community in the next 12 months
- Botswana citizen or spouse of Botswana citizen
- Agrees to annual home visits, as well as other study procedures
- Provision of contact details (such as telephone numbers, physical and/or alternate addresses)
   that would allow the study team to trace him/her
- Able to provide informed consent if ≥18 years old, or able to provide assent to complement a guardian's consent, if a minor (aged 16 or 17)

**Note:** The above HIC eligibility criteria apply during the BHS (T0) and AHS visits prior to the final visit (i.e. the HIC is an open cohort).

#### 4.4.3. Individuals Eligible for Research Blood Draw in Combination Prevention Communities
For HIV-infected residents of Combination Prevention communities who did not take part in the research blood draw through the BHS, the following eligibility criteria will apply for the blood draw for HIV-1 RNA and genotyping/incidence assay/TDR/storage:

#### **Inclusion Criteria:**

- Any individual with documented HIV infection, including newly-diagnosed individuals and HIV-infected persons already receiving care and/or antiretroviral treatment at the clinic. (note: blood draws for HIV-1 RNA, genotyping, incidence assay, TDR and storage will be obtained once from HIV-infected clinic patients throughout the study.)
- Adult aged 16-64 years
- Permanent or part-time resident of combination prevention communities
- Botswana citizen or spouse of Botswana citizen
- Able to provide informed consent for study enrollment if ≥18 years old, or able to provide assent to complement a guardian's permission, if a minor (aged 16 or 17)

#### 4.4.4. End of Study Survey (ESS)

The ESS will be conducted at the end of the study in 3 pairs of communities (6 communities) selected out of the 30 participating communities. It will be conducted in the  $^{80}$ % of the population that is not taking part in the 20% household surveys. At T2, residents of the 20% households will also contribute data toward the ESS analyses.

#### Inclusion criteria:

- Aged 16-64 years
- Permanent or part-time study community resident in any of the selected 3 pairs of study communities (for ~80% households to be newly enrolled at ESS), or any of the 30 communities (for ~20% BHS/HIC households having final evaluation at T2/ESS)
- Able to provide informed consent for study enrollment if ≥18 years old, or able to provide assent to complement a guardian's permission, if a minor (aged 16 or 17)

#### 4.4.5. Economic Assessment

Participants in the 20% household surveys will be asked to answer questions to estimate healthcare costs and quality of life; these questions are included as supplemental sections in the annual resident survey that participants will complete. The eligibility criteria for this group of participants in the economic assessments are therefore the same as for the BHS.

There will be additional sampling of individuals with opportunistic illnesses or low CD4 cell count. The eligibility criteria for these assessments are as follows:

#### Inclusion criteria for Supplemental Economic Assessment:

- Permanent or part-time study community resident in any of the study communities
- Aged 18-64 years
- Documented to be HIV-infected.

- Measured CD4<200 cells/μL or WHO stage 3 or 4 illness</li>
- Botswana citizen or spouse of Botswana citizen
- Able to provide informed consent for study enrollment

Records for a small subset of community residents (up to 80 residents) who die during the course of the study will be abstracted to evaluate for healthcare costs at the end of life. These individuals need not necessarily be part of one of the study cohorts. This aspect of the research does not involve human subjects per the definition at 45CFR46.102(f) that a human subject is a *living* individual. The eligibility criteria for the record review is as follows:

#### Inclusion criteria for Record Abstraction:

- Resident in any of study communities (defined by at-home death in a study community and/or recorded as a resident in the medical record)
- Aged 18-64 years at the time of death
- Botswana citizen or spouse of Botswana citizen
- Died during the years of the course of the study
- Records available for review

# 4.4.6. Barriers to and Facilitators of Linkage-to-Care (LTC) and ART Initiation

A small subset of participants in the 20% household surveys will be invited to participate in a focus group discussion (FGD) or individual in-depth interview (IDI) to provide information on barriers to and facilitators of linkage-to-care (LTC) and ART initiation. Staff from the BHS (Research Assistants) and MOH (Nurse Prescribers) will be invited to participate in separate FGDs to provide insight into the dynamics surrounding linkage to care and initiation of ART.

#### Inclusion Criteria for BHS Participants in FGDs or IDIs

- BHS participant (enrolled in the 20% household survey prior to the FGD)
- Resident of study community in the Combination Prevention arm
- Aged 18-64 years
- Documented to be HIV-infected
- Eligible for ART initiation (to be used for purposive selection for focus group discussion and indepth interviews)
- Able to provide informed consent for FGD or IDI participation

#### <u>Inclusion Criteria for Staff Participants in FGDs</u>

- BHS staff member or Nurse Prescriber in any of the Combination Prevention communities
- At least 18 years of age
- Able to provide informed consent for FGD participation

#### 4.5. Rationale for Eligibility Criteria

#### Rationale Surrounding Need for Botswana Citizenship for BHS/HIC:

Although the Botswana Government provides free HTC services to non-citizens, free access to health services, including ART, MC and PMTCT is restricted to a) persons who can produce valid

documentation of Botswana citizenship or b) spouses of Botswana citizens. The BCPP package of intervention services will therefore not be available to non-citizens of Botswana unless married to a citizen, per regulations of the MOH (Presidential Directive Cab. 5 (b)/2004).

As the households are followed longitudinally under the auspices of the study team but non-citizens cannot access free public health services unless married to a citizen, the eligibility criterion of Botswana citizenship (or being married to a Botswana citizen) is included for BHS/HIC participants, but not for ESS participants who are not followed longitudinally.

Rationale for Including Non-Citizens in ESS: The intervention package implemented in Combination Prevention communities includes the following for non-citizens: expanded HTC services, including a referral to the health clinic in their community of residence to connect them with available fee-based services including treatment; and enhanced linkage to MC services, including for men who decline HIV testing or have indeterminate results. A major goal of the ESS is to evaluate and compare coverage of the intervention package components between arms, particularly HTC coverage which cannot be evaluated in the 20% BHS cohort. Comprehensively surveying all potential recipients of services in the study communities is an important aspect of achieving the goal of the ESS. Other key objectives of the ESS are to improve mapping of viral genetic linkage, and to accurately estimate how viral burden and viral suppression are distributed across HIV-infected residents of the study communities. Obtaining a sample from as many HIVinfected residents of the study communities as possible at ESS is critical for these objectives. Finally, the lack of access to free ART for non-citizens residing in Botswana represents a potentially significant gap in achieving the 90-90-90 goal for viral suppression that will be important to understand and quantify if Botswana is to consider expanding its treatment program, and for potentially further reducing HIV incidence in Botswana. Non-citizens will be included in the crosssectional survey at ESS only, and will be offered anonymous participation to protect their identity. Non-citizens living in Botswana without legal documentation and others in the same household may face the risk of penalty (see Section 11). Participation in ESS may help non-citizens by providing free HIV testing and counseling with referral to services that they would be able to access.

#### Rationale for Age Limits:

Persons <16 years of age will be excluded from study participation because our intervention is targeting individuals age 16−64, and we hope to measure relevant study outcomes among this population. In Botswana, all persons aged ≥16 can access medical services, including HTC, without needing guardian permission. Although individuals aged 16-17 can access medical services without guardian permission, participation in research still requires guardian permission, because the age of consent for research in Botswana is 18. Therefore, eligible 16-17 year-olds will be asked for assent to participate in research activities if/after permission is provided by the guardian.

#### Rationale for Number of Nights Spent per Month in the Community:

For the BHS, we propose that adults who report spending ≥3 nights each month in the community over the past year, on average, be included, because these adults will be eligible for interventions if the community is randomized to the intervention arm (please see the *Intervention Protocol* for details on rationale for use of this definition of community residence vis a vis eligibility for

interventions). We need to estimate baseline and subsequent service uptake among a similar (representative) group of adults enrolled in the BHS (and subsequent household surveys), to allow assessment of baseline use of and uptake of interventions over time, and comparison between study arms.

For the HIC, we propose that adults who report spending on average  $\geq$ 14 nights each month in the community over the past 12 months, and who do not intend to move out of the community over the next 12 months be included, because we believe that these adults are more likely to:

- 1) have sexual relationships with individuals residing inside versus outside the study community (hopefully reducing sexual network contamination),
- 2) access available health services in the community versus outside the study community (hopefully reducing intervention contamination of the HIC cohorts), and,
- 3) be easier to retain in the study (hopefully avoiding possible selection bias introduced by excessive loss to follow-up).

For research blood draws in all HIV-infected adults in the Combination Prevention arm, investigators propose that adults who report spending on average  $\geq$ 3 nights per month in the community over the past year be included in blood draws for viral phylogenetic linkage.

For the ESS, investigators propose that adults who report spending ≥3 nights per month in the community over the past year be eligible because: (1) we need to measure coverage of the CP package within this group of adults, and (2) consenting HIV-infected adults identified during the ESS will contribute blood samples to improve completeness of the HIV-1 genotype map in Enhanced Care and Combination Prevention communities (important for secondary objectives 1-3).

# • Rationale for Number of Nights Spent per Month in the Household:

It is important to determine that participants in household-based procedures (BHS and HIC) are indeed at least part-time residents of the approximately 20% of households that are sampled (rather than casual visitors). The definition of household membership used (spending more nights on average in the household being sampled than in any other household in the same community over the preceding 12 months) is relatively straightforward to implement, and also helps decrease the chance of a given individual being asked to take part in household procedures in more than one household per community (although this criterion will not affect the chance of a participant enrolling in more than one community).

Note: we intend to avoid enrolling the same individual more than once in the same component of the study (the BHS or the HIC). We will try to achieve this through the following means:

- Inclusion of the household membership eligibility criterion.
- Avoid enrollment of residents in the study if they state that they already took part in the study, with confirmation through other means.
- Using the unique citizen Omang number to reduce the number of instances in which a resident is enrolled twice.

# 5. SAMPLE SIZE AND SAMPLE SELECTION METHODS

# 5.1. Sample Size Calculations Related to Primary Objective #1

To estimate the required sample size to detect predicted differences in cumulative HIV incidence between combination prevention and enhanced care incidence cohorts, we: (1) modeled the potential impact of the originally proposed intervention package on adult HIV incidence, and (2) used impact estimates in standard formulae for pair-matched CRTs to estimate the number of community clusters, size of incidence cohorts, and duration of incidence cohort follow-up, required to detect the originally estimated impact with sufficient power (≥85% power).

# 5.1.1. Estimating Impact of Combination Prevention on Adult HIV Incidence

We used two epidemic models to estimate the potential impact on adult HIV incidence of scale-up of the CP package to high population-level coverage levels.

- Primary model: The primary model is an agent-based network epidemic simulation model. Using models for generating degree distribution for sexual network described by Jones and Handcock (Jones and Handcock 2003) and implemented as an R package (Handcock, Hunter et al. 2003), we constructed stochastic degree distributions based on data from Likoma Island (Helleringer and Kohler 2007). Methods in Blitzstein and Diaconis (Blitzstein and Diaconis 2006) allow for the uniform sampling of networks with the prescribed degree sequence. For the sampled networks we select only those networks that match the prescribed level of mixing between communities. Using techniques similar to Eaton et al. (Eaton, Hallett et al. 2011), the model allows investigators to take into account community characteristics, including varying coverage levels for different prevention modalities, and population sizes, as well as individual characteristics including transmission risk, disease progression, condom use, linkage to care, and circumcision status.
- <u>Secondary model</u>: We also used the published Goals model available at (<a href="http://futuresinstitute.org/Default.aspx">http://futuresinstitute.org/Default.aspx</a>.) which is part of the Spectrum suite of models (Stover, Bollinger et al. 2011), to estimate CP impact on population-level HIV incidence. The Goals model is widely used by national governments, including Botswana (Stover, Fidzani et al. 2008), to plan HIV prevention programs and also estimate impact on HIV incidence and other indicators (e.g. number of AIDS deaths). We used the Goals model primarily to assess whether Goals impact estimates were similar to impact estimates from the primary model. The Goals model produced comparable results when using the same set of input parameters.

Table 1A lists input parameters used in the original primary model where we assumed the expanded ART intervention would be offered to HIV-infected individuals with CD4≤350 cells/μL or viral load ≥10,000 copies/ml in the Combination Prevention arm throughout the study, and that the Botswana national guidelines for ART initiation would not change during the study period. Original estimates of model input parameters were obtained from Botswana Government data and from the population-based Mochudi Prevention Project that was conducted from May 2010 to May 2013 (see below for a detailed explanation of input parameters). Timely linkage to care and treatment was assumed to be

80% in Enhanced Care and 90% in Combination Prevention communities during the study period. We assume that sexual mixing between communities is on average 20% with a 95% confidence interval of 15% to 25%.

Table 1A: Original Model Input Parameters for the Primary Model to Estimate Impact of Combination Prevention (CP) Package Scale-Up in CP Communities Versus Enhanced Care (EC) Communities over 4 Years

| | EC Arm | CP Arm | | |
|---|---|---|---|---|
| | Anticipated True Coverage of | of Services in the EC | CP Scale-up with ART at CD4≤350 or VL≥10K in | |
| | Communit | ty | CP Arm | |
| Time | HTC outside of study cohort | Male Circumcision | HTC* | Male Circumcision* |
| Baseline | | | | |
| Survey | 37% | 12.7% | 37% | 12.7% |
| End Y1 | 41% | 31.4% | 90%** | 46.4% |
| End Y2 | 45% | 50.0% | 90% | 80% |
| End Y3 | 49% | 60.0% | 80% | 80% |
| End Y4 | 53% | 70.0% | 70% | 80% |

<sup>\*</sup>Intervention Community scale-up targets

For version 5.0 of the protocol, we conducted new simulations using updated baseline parameters based upon observed data in the first several community pairs. Treatment initiation is assumed to be 80% in the Enhanced Care communities and 90% in the Combination Prevention communities during the study period. Table 1B lists input parameters used in the updated primary model. Note that the updated model was undertaken to assess power under more realistic assumptions related to baseline parameters and coverage by interventions and under different scenarios for expanded ART.

Table 1B: Model Input Parameters for the Updated Primary Model to Estimate Impact of Combination Prevention (CP) Package Scale-Up in CP Communities Versus Enhanced Care (EC) Communities over 4 Years

| | EC A | rm | | CP Arm |
|---|---|---|---|---|
| Time | Anticipated True Coverage of Services in the EC Community | | CP Scale-up with Universal Test and Treat in CP Arm | |
| | HTC outside of study | | | |
| | cohort | Male Circumcision | HTC | Male Circumcision |
| Baseline | | | | |
| Survey | | 35% | | 35% |
| End Y1 | 27% | 40% | 79% | 50% |
| End Y2 | 31% | 45% | 85% | 55% |
| End Y3 | 35% | 50% | 80% | 60% |

#### Explanation of input parameters:

#### • HTC Service Uptake

HTC coverage is defined as the probability of a person of unknown status being tested for HIV anytime in the previous 12 months. We assumed 79% and 85% HTC coverage for the CP arm in

<sup>\*\*</sup>Allowing 4 months of scale-up period

the updated model, more conservative than the 90% target, in years one and two, respectively. HTC uptake will likely increase in Enhanced Care communities during the study period as well. We assumed that HTC coverage in Enhanced Care communities would increase 4% per year during the study period.

#### Male Circumcision Service Uptake

A 2010–2011 survey of the Mochudi district in Botswana suggests MC coverage is 12.7% (the MOH Spectrum estimate is 11%). Linkage to male circumcision services in Enhanced Care communities will be ongoing. The original model parameters assumed that MOH, and the original *Intervention Protocol* targets for MC would be met in the EC, and CP arm, respectively by the end of Year 4 post-randomization. According to BAIS reports, the prevalence of circumcision among males in Botswana aged 16–64 was approximately 13% in 2008 and 28% in 2013, an increase of only 15% in 5 years. In addition, version 4.0 of the *Intervention Protocol* includes a lower MC target of 60% in Year 3. In the updated model, we therefore set the baseline MC prevalence at 35%, revised the coverage in the EC arm to increase by 5% per year, and assumed the revised MC coverage target of 60% would be achieved by the end of Year 3 in the CP arm.

# • ART Service Uptake

In the primary model using either the original or updated parameters, ART coverage is an intermediate outcome of HTC coverage and linkage to care. In the updated model we assumed baseline ART coverage of 88.7%.

# • PMTCT service uptake

We have not listed PMTCT coverage input parameters because in both models, PMTCT coverage increases have no direct impact on adult HIV incidence. However, in real program settings, with an estimated 10% of adult women becoming pregnant each year, we expect ANC clinics to be an important avenue for adult HTC and entry into HIV care and treatment. The primary PMTCT coverage goal of the CP package is to increase the proportion of HIV-infected post-partum women who are enrolled in care clinics (linked) and are retained in care and on ART (Option B+).

# Sexual Mixing between Study Communities

One of the main reasons for building the primary model was to allow for potential sexual network contamination of HIV incidence cohorts in intervention and Enhanced Care communities. Therefore, the primary model assumed that an average of 21% (SE: 2.6%) of sexual relationships occurred between persons in opposite study arms. Data from a survey of Mochudi district in Southern Botswana showed that 30% of the relationships were from outside of Mochudi, with 25% of the out-of-community relationships in Gaborone, the capital of Botswana. We decided to assume, on average, 21% sexual mixing for two primary reasons: (1) many of the study communities are more rural than Mochudi; and (2) some of the out-of-community relationships in Enhanced Care communities will not be with Combination Prevention community residents.

Table 2A below provides model estimates of differences in cumulative HIV incidence between Enhanced Care and Combination Prevention communities. Table 2A reflects modeling conducted with the original expanded ART design offered in CPCs at the time of launching the study in 2013. The input parameters are based on the Mochudi survey, Botswana government data before the study launched, and the HTC and MC coverage levels as listed in Table 1A.

Table 2A: Projected Cumulative HIV Incidence in Enhanced Care (EC) versus Combination Prevention (CP) Communities over 4 Years of Study Follow-Up Using Original Parameters and with ART for Individuals with CD4≤350 cells/μL or Viral Load ≥10,000 copies/ml in the CP Arm

| | EC Arm | CP Arm CP Scale-up with ART at CD4≤350 or VL≥10K in CP Arm | |
|---|---|---|---|
| Time | | Cumulative Incidence | (% Reduction vs. EC) |
| End of Y1 | 1.79% | 1.40% | (22% ↓) |
| End of Y2 | 3.05% | 2.01% | (34% ↓) |
| End of Y3 | 4.05% | 2.44% | (40% ↓) |

Table 2B reflects modeling conducted with change in CD4 threshold from 350 to 500 in 2015, and move to UTT in Combination Prevention communities (implemented with version 4.0 of this protocol) and Botswana's "Treat All" policy in place starting June 2016. The input parameters for the projections in Table 2B are based on observed data in the first several community pairs and HTC and MC coverage levels listed in Table 1B. In the updated models, we assumed 80% ART initiation in the EC arm and 90% in the CP arm.

The Botswana MoH adoptetd universal ART as national policy effective June 2016. Therefore, we simulated this scenario of treatment eligibility in the Enhanced Care arm compared to UTT in the Combination Prevention arm: CD4≤350 followed by universal ART in 2016. Guidelines changes are assumed to become policy in June 2016, and ramp up to full scale over the following 12 months. The CP arm was simulated as follows: launching with the original design (CD4≤350 or VL>10,000), followed by CD4≤500 or VL≥10,000 in the third quarter of 2015, followed by UTT in June 2016. These simulations were done with the updated input parameters shown in Table 1B above.

Table 2B: Projected Cumulative HIV Incidence and Study Power with Universal Test and Treat in the Combination Prevention (CP) Arm and "Treat All" in the Enhanced Care (EC) Arm

| Treatment Eligibility | | Length of<br>Follow-up | Cumulative Incidence Rate (CIR) (%) | | Reduction<br>in CIR (%) | Power (%) |
|---|---|---|---|---|---|---|
| ECC | СРС | rollow-up | ECC | CPC | III CIK (%) | |
| CD4≤350 → CD4≤350 or VL≥10k at study launch → CD4≤500 or VL≥10k in | 2 Years | 1.45 | 0.93 | 36 | 47 | |
| | 2.5 Years | 1.70 | 1.00 | 41 | 63 | |
| 2016 | 2015 → UTT in 2016 | 3 Years | 1.84 | 1.06 | 42 | 70 |

Since the exact timing of UTT roll-out is unknown in Enhanced Care communities under Botswana's "Treat All" program, we made a simple assumption that each Enhanced Care community will have the same (reflecting the average) amount of time of follow-up before and after UTT. This assumption was also made for the Combination Prevention communities, but these communities will receive UTT earlier. While the reality will undoubtedly depart from these assumptions, the models are useful in providing a first-order approximation of power.

# 5.1.2. Estimating Needed Number of Community Clusters and Size of Incidence Cohorts to Detect Estimated HIV Incidence Differences

We examined the number of communities and incidence cohort size needed to detect a 40% difference in cumulative HIV incidence (originally 4.05% in the Enhanced Care arm vs. 2.44% in the Combination Prevention arm), which we hoped would be achieved by the end of the third year of follow-up if Botswana national guidelines remain at ART initiation for individuals with CD4≤350 throughout the entire study. Required sample size was determined based on the original combination prevention package design prior to the launch of the study (see version 1.0 of the Evaluation Protocol). See Sections 5.1.1, 5.2.1, and 5.2.2 for updated study power estimates based on the current design and assumptions.

We aimed to have  $\geq$ 85% power to detect the anticipated effect size with alpha set at 0.05.

We used the formula from Hayes and Moulton, appropriate for a pair-matched CRT (Hayes and Moulton 2009).

$$c=2+\left(z_{1-\frac{\alpha}{2}}+z_{1-\beta}\right)^2\frac{\pi_0(1-\pi_0)/m+\pi_1(1-\pi_1)/m+k_m^2(\pi_0^2+\pi_1^2)}{(\pi_0-\pi_1)^2}\text{, where,}$$

c is the number of clusters (community clusters) per arm,

 $Z_{1-\alpha/2}$  is the standard normal deviate corresponding to the upper tail probability of  $\alpha/2$  where  $\alpha$  is the probability of a type I error.

 $Z_{1-\beta}$  is the standard normal deviate corresponding to the upper tail probability of  $\beta$  where  $\beta$  is the probability of a type II error,

 $\pi_0$  is the cumulative HIV incidence in the control arm,

 $\pi_1$  is the cumulative HIV incidence in the intervention arm,

m is the cluster size in each community cluster (examined a range – see below)

 $k_m$  is the matched pair, between-cluster coefficient of variation of the true proportions in both the control and intervention arms (based on primary model simulations, the estimate of  $k_m$  is 0.24. To be conservative, we used 0.26, but we examined a range of  $k_m$  from 0.2 - 0.35).

The table and graph below illustrate the community and cluster sizes needed to ensure  $\geq$ 85% power to detect the anticipated effect size by the end of the third year of follow-up.

Table 3: Cluster Size versus Cluster Number Needed to Achieve >85% Power to Detect Anticipated Effect Size by the End of the 3<sup>rd</sup> Year of Follow-up across a Range of Coefficients of Variation (k), Assuming ART is Offered to HIV-Infected Individuals with CD4≤350 or Viral

Load≥10,000 copies/ml in the Combination Prevention Arm based on the original set of parameters

| | Number of clusters required, depending on the size of k | | | | |
|---|---|---|---|---|---|
| Cluster size (m) | k=0.2 | k=0.24 | k=0.26 | k=0.3 | k=0.35 |
| 1000 | 7 | 9 | 9 | 11 | 14 |
| 900 | 7 | 9 | 10 | 11 | 14 |
| 800 | 8 | 9 | 10 | 12 | 14 |
| 700 | 8 | 10 | 10 | 12 | 15 |
| 600 | 9 | 10 | 11 | 13 | 15 |
| 500 | 9 | 11 | 12 | 13 | 16 |
| 400 | 10 | 12 | 13 | 14 | 17 |
| 300 | 12 | 14 | 14 | 16 | 19 |
| 200 | 16 | 17 | 18 | 20 | 22 |
| 100 | 27 | 28 | 29 | 31 | 33 |



<sup>\*</sup>Assumes ART is offered to HIV-infected individuals with CD4≤350 or viral load≥10,000 copies/ml in the Combination Prevention arm based on the original set of parameters

With 15 clusters per arm and on average 300 HIV-negative HIC participants per community (i.e., 4,500 HIC participants per arm or 9,000 HIC participants total), we have 86% power to detect the anticipated difference in cumulative HIV incidence between Enhanced Care and Combination Prevention communities (4.05% vs. 2.44%) by the end of the third year of follow-up, if Botswana national guidelines remain at ART initiation for individuals with CD4≤350 throughout the entire study, assuming the coefficient of variation (k) is 0.26. Under the Combination Prevention package introduced with version 4.0 of this protocol (ART for all HIV-infected individuals), the estimated

power based on more conservative assumptions (Table 1B) is >72% if national guidelines change to also offer universal ART in 2016.

Investigators note that power calculations are based on differences in proportions of the population infected over the 3-year period for each pair of communities, and do not take into account all of the variability that could arise from the interval-censoring that allows for making use of partial information for dropouts, irregular schedules of visits, and delayed entry into the cohort. However, we believe that the power calculations will be reasonable because the available information should not be sharply reduced by these factors. While some information will be lost because of dropout, the open nature of the HIC, use of the results from multiple tests throughout the study period, and the interval-censored data, which reflects the actual time of infection, would add information.

Assuming cumulative HIV incidence in the Enhanced Care arm is 4.1% at 3 years, we examined the range of effect sizes that might be detected if 30 communities are enrolled with 300 HIV-negative adults per incidence cohort (see Figures 2A and 2B below).





The above power estimates suggest that, for 15 matched pairs, with average HIC size 300 per community, if cumulative incidence in the Combination Prevention arm is  $\geq$ 38% lower than in the Enhanced Care arm (4.1%), we should have >80% power to detect the difference by the end of the third year of follow-up, assuming k is 0.26 (Figure 2A). If the annual incidence rate in the Enhanced Care arm turns out to be as low as 1.0%, we will still have >80% power if we can achieve a reduction of at least 41% in cumulative incidence in the Combination Prevention arm (Figure 2B).

#### 5.1.3. Study Community Selection

Our rationale for selection of the 30 study communities is provided in Section 4.1. Here we describe in more detail how selected study communities facilitate enrollment of HIV incidence cohorts of sufficient average size (averaging 300 persons per HIC).

The total estimated population in the 30 targeted communities is 180,800, on average 6,027 individuals per community, ranging from 2,409 (Ranaka) to 12,086 (Mmadinare). The age-eligible (16-64 year olds) subset is estimated at 58% or 3,495 per community including 2,622 HIV-negative and 874 (25%) HIV-positive individuals. Assuming 20% of household members are absent, and 85% of present members consent to participate in the study, sampling 20% of households from communities of population ≤6,000 and approximately 333 households from communities of population >6,000, should facilitate identification of on average 300 HIV-negative persons per community, sufficient to meet sample size requirements for the CRT. Assuming 4.2 persons per household (Central Statistics Office 2009), 2.4 of whom are adults, and 1.8 of whom are HIV-negative adults, this would suggest we need to visit at baseline and annually on average 240 households per community.

#### 5.1.4. Incidence Cohort Selection – the Baseline 20% Household Survey

The primary purpose of the baseline 20% household survey is to identify and recruit HIV negative individuals for the HIV incidence cohort. To reach a 20% household sample size (on average 240 households per community), a 25% sample of households (possibly ranging from 115 to 576, and averaging 360 households per community) will initially be randomly selected. The initial unit of selection will be a plot using google area maps (and potentially population census and other publicly available sources); in some instances there may be more than one household on a plot and all houses on a selected plot will be asked to take part. The specifics of the household selection process are described in the BHS/HIC manual. In villages with population under 6,000, the required 20% households will be randomly selected from the 25% sample and approached first for participation in the study. In villages with population over 6,000, 333 households will be randomly selected from the 25% sample and approached first for participation in the study.

The remaining households in the 25% sample will be ordered randomly (e.g. from 1-49). If some of those households in the primary 20% sample in smaller villages (population ≤6,000) or the 333 households in larger villages (population >6,000) do not participate (e.g. refuse consent), the additional households in the full 25% sample will be approached sequentially, in the order specified by the random sampling scheme. In villages with population under 6,000, the enrollment will stop when either a 20% sample of the entire community has been achieved or the full 25% household sample list is exhausted. In villages with population over 6,000, after at least 273 households have been enrolled, the enrollment will continue until 20% of the households in the village have enrolled, or 23 working days have been reached, whichever comes first.

Based on previous survey experience in Mochudi and northern Botswana, we anticipate that we will be able to enroll 20% of households from the baseline 25% household sample. Our reason for not wishing to approach more than 25% of households is to avoid excessive intervention contamination of the Enhanced Care arm.

Figure 3 depicts the numbers and flow of participants from the 20% household sample.

Figure 3: Flow of participants from 20% Household Survey to BHS and HIC



# 5.2. Sample Size Calculations Related to Primary Objective #2

# 5.2.1. Estimating Precision Surrounding HTC, ART, VL Suppression, MC, and PMTCT Coverage Proportions

The rationale for the size of the baseline 20% household sample is provided above.

The end of study survey (ESS) will provide the primary estimates of intervention coverage. It should be noted that the model inputs related to intervention coverage used to estimate power for Primary Objective #1 (Tables 1B and 2B) differ from the intervention coverage values used to estimate power for Primary Objective #2. Modeling for Primary Objective #1 used a combination of observed coverage (from the first several communities) and targets (for MC). For Primary Objective #2, actual coverage of the intervention package will generally be assessed in distinct populations according to the service uptake indicators outlined in Section 2.2 and the targets of the Intervention Protocol (Table 4).

At the ESS we will compare coverage of HTC, ART, VL Suppression, and MC between the two study arms. We will have limited power (<60%) to detect a difference in PMTCT coverage proportions between study arms due to small sample size; the number of HIV-positive, pregnant women at ESS is estimated to be 270 per study arm. However, HIV-positive pregnant women will be included in measurement of coverage of the ART and VL suppression targets.

The ESS will be conducted in 3 pairs of communities (6 communities in total, 3 in each arm) selected out of the 30 participating communities. The ESS will attempt to survey the ~80% of the population that is not taking part in the BHS/HIC, in these 6 communities (in addition, the 20% households in these communities will participate in T2 surveys (or T3 surveys, in a small number of communities completing T3 visits prior to the roll-out of version 5.0), leading to the target of 100% community assessment in these 6 communities at the end of the study). The final surveys among residents in the 20% households in the remaining 24 communities will also provide data.

The rationale for seeking a 100% community census in three Enhanced Care and three Combination Prevention communities is as follows: (1) to measure HTC coverage in both study arms and more accurately measure study-end MC and ART coverage, (2) to improve mapping of viral genetic linkage, (3) to accurately estimate how the viral burden and viral suppression are distributed across HIV-infected people in Enhanced Care and Combination Prevention communities, (4) to compare CP package uptake within 20% households to CP package uptake in the broader communities they represent, and (5) to improve precision of cross-sectional assay-derived HIV-incidence estimates in Enhanced Care communities. The ESS was restricted to 6 (rather than 30) communities as it provides sufficient data for these analyses and requires significantly fewer resources.

The average total population size of the study communities is 6,027. Therefore, we estimate a total population in the six ESS communities of 36,162 people, with 58% (20,974) aged 16-64. Approximately 20% of these residents will be visited at T2 (or T3 in communities having this visit prior to version 5.0) as part of the BHS/HIC follow-up visits. Residents of the remaining approximately 80% will be invited to participate in the ESS as a one-time household survey. Assuming 80% of residents are present at the time of an ESS/T2 visit, and 85% consent to participate, there will be on average 2,377 participants per community, and approximately 14,262 in total, including residents of the previously enrolled 20% households and new enrollees from the remaining 80% of households.

In the table below we estimate precision of confidence intervals surrounding coverage proportions of the HIV prevention interventions to be compared (HTC, ART including VL suppression, and MC) in all study communities at baseline and, separately in Enhanced Care and Combination Prevention communities at study end.

Table 4: Estimated Precision of 95% Confidence Interval Surrounding HTC, ART (including VL suppression) and MC Coverage Proportions at Baseline and Study End

| | y and the coverage i roportions at baseline and | Baseline | | |
|---|---|---|---|---|
| | | Household | | |
| | | Survey (BHS) | End of Study | Survey (ESS) |
| | | All Study | | |
| | | Communities | EC Arm | CP Arm |
| | Denominator (n=residents aged 16–64 years) | 12,000 | 5,931 | 5,931 |
| | Numerator (n=residents aged 16–64 years who know | | | |
| HTC | they are HIV-positive or have tested HIV-negative within | 4,440 | 2,847 | 5,338 |
| Coverage | the past 12 months) | | | |
| | HTC coverage proportion | 37% | 48% | 90% |
| | Width of 95% CI (+-) | ±1.6% | ±4.9% | ±8.9% |
| | Denominator (n=HIV-positive people aged 16–64 years) | 3,000 | 2,971 | 2,971 |
| | Numerator (n=HIV-positive people aged 16–64 years | | | |
| ART | who know they are HIV-positive and are currently | 2,190 | 2,405 | 2,763 |
| Coverage | receiving ART) | | | |
| | ART coverage proportion | 73% | 79.5% | 93% |
| | Width of 95% CI (+-) | ±3.0% | ±4.3% | ±4.8% |
| | Denominator (n=HIV-positive people aged 16–64 years) | 3,000 | 2,971 | 2,971 |
| | Numerator (n= HIV-positive people aged 16–64 years | | | |
| VL | who know they are HIV-positive, are currently receiving | 2,100 | 2,264 | 2,822 |
| Suppression | ART and with HIV viral load ≤400 copies/mL) | | | |
| | VL suppression coverage proportion | 70% | 76.2% | 95% |
| | Width of 95% CI (+-) | ±3.0% | ±4.1% | ±4.9% |
| | Denominator (n=HIV-negative men aged 16-64 years) | 4,320 | 4,278 | 4,278 |
| 146 | Numerator (n=HIV-negative men aged 16-64 years who | 4.542 | 2.420 | 2.567 |
| MC | are circumcised) | 1,512 | 2,139 | 2,567 |
| Coverage | MC coverage proportion | 35% | 50% | 60% |
| | Width of 95% CI (+-) | ±1.9% | ±2.9% | ±3.4% |

A detailed explanation of the contents of Table 4 is provided below. Total populations sizes may be found in Appendix C3.

# HTC coverage numerators and denominators:

- The BHS denominator is calculated as (average number of BHS enrollees per community)\*number of communities = 400\*30 = 12,000.
- The **BHS numerator** is calculated as 12,000 (BHS enrollees)\*(expected proportion of residents who either know they are HIV-positive or have tested HIV-negative within the past 12 months) = 12,000\*0.37 = **4,440** (note that the definition of HTC coverage used here differs slightly from the definition used in section 5.1, due to requirements related to model structure).
- The ESS denominator includes all residents aged 16-64 years outside of the BHS 20% sample in the 3 pairs of selected communities. The BHS 20% sample cannot be used to assess HTC coverage because all BHS participants are tested at enrollment per study design. The same proportions expected to be present and consent to BHS at T0 were assumed for the ESS at T2.

Therefore the **ESS denominator per arm** is calculated as [ (average population size per community)\*(proportion expected to be age-eligible)\*(proportion expected to be present)\*(proportion expected to consent) – (average number of BHS enrollees per community) ]\*(# communities per arm) = [ (6,027\*0.58\*0.80\*0.85) – (400) ]\*3 = (2,377–400)\*3 =**5,931**.

- We assumed that HTC coverage in EC communities would increase 7% in the first year and 4% per year thereafter during the study period (note that the definition of HTC coverage used here differs slightly from the definition used in section 5.1, due to requirements related to model structure). Therefore the ESS numerator in the EC arm is calculated as 5,931\*(expected proportion who know they are HIV-positive or have tested HIV-negative within the past 12 months at T2) = 5,931\*(0.48) = 2,847
- The **ESS numerator for the CP arm** is calculated as 5,931\*(target outlined in Protocol 3) = <math>5,931\*0.90 = 5,338.

#### ART coverage numerators and denominators:

- The BHS denominator includes HIV-positive persons aged 16-64 years in the BHS 20% sample and is calculated as (the total number of BHS enrollees)\*(proportion HIV-positive) = 12,000\*0.25 = 3,000.
- The **BHS numerator** is calculated as 3,000\*(proportion HIV-positive persons expected to know their status and currently on ART based on preliminary BHS data) = 3,000\*0.73 = **2,190**.
- The ESS denominator includes HIV-positive adults from the BHS 20% sample in the 24 communities not selected for participation in the ESS and all HIV-positive adults (100% sample) in the 6 ESS communities. Based on preliminary follow-up data at T1, we expect 90% of participants enrolled at T0 to be present at T2. In addition, we expect additional household members will be added to the cohort at T1. Based on preliminary data from T1, we assume an increase in enrollment of 10% at T1.

The number of HIV-positive adults from the BHS 20% sample from the 24 non-ESS communities and 6 ESS communities is calculated as (average number of BHS enrollees per community)\*(proportion expected to be present at T2)\*(additional proportion newly enrolling at T1)\*(proportion HIV-positive)\*(number of communities) = 400\*0.90\*1.10\*0.25\*30 = 2,970.

The number of HIV-positive adults in the 6 ESS communities outside the BHS 20% samples is calculated as [ (average population size per community)\*(proportion expected to be age-eligible)\*(proportion expected to be present)\*(proportion expected to consent)\*(proportion HIV-positive)—(average number of HIV-positive BHS enrollees per community at T2) ]\*(number of ESS communities) = [ (6.027\*0.58\*0.8\*0.85\*0.25) - (2.970/30) ]\*6 = 2,972.

Therefore the **ESS denominator per arm** is 2,970 + 2,972 = 6,050/2 =**2,971**.

Based on preliminary BHS data, we found that 87% of HIV-positive participants who knew their status were on ART representing 73% of all HIV-positive persons (irrespective of prior knowledge of status). Assuming that HIV diagnosis among HIV-positives will increase by 3% over 2 years in the EC arm and that 87% of these new diagnoses will initiate ART, we expect an additional 2.6% of all HIV positive-persons will be on ART by T2. Additionally, we expect that by T2 UTT will have been scaled up and available in EC communities for approximately 6 months. Therefore, all ART-naïve individuals will be eligible for ART including those with CD4≤350 at

baseline. Based on preliminary BHS data, 7.8% of HIV-positive, ART-naïve persons have a CD4>350 cells/mm<sup>3</sup>. Since UTT will only have been in place for approximately 6 months by T2, we assume that 50% of these ART-naïve individuals with a CD4>350 cell/mm<sup>3</sup> will be on ART by T2 or 7.8%\*0.5 = 3.9%.

Thus, the **ESS numerator for the EC arm** is calculated as 2,971\*[ (proportion of HIV-positive persons expected to know their status and currently on ART at T0) + (additional proportion of HIV-positive, ART-naïve at T0 expected to be on ART by T2 due to increased diagnosis and under UTT) ] = 2,971\*(0.73+0.026+0.039) = 2,971\*0.795 = 2,405

• The **ESS numerator for the CP arm** is calculated as 2,971\* (target outlined in Protocol 3) = 3,516\*0.93 = 2,763.

# • VL suppression numerators and denominators:

- The BHS denominator includes HIV-positive persons aged 16-64 years in the 20% BHS sample and is calculated as described above for the BHS denominator for ART coverage = 3,000.
- The BHS numerator is calculated as 3,000 \* (proportion HIV-positive persons expected to know their status, be on ART and have a VL ≤400 copies/mL based on preliminary BHS data) = 3,000\*0.70 = 2,100.
- The ESS denominator by arm includes all HIV-positive adults from the BHS 20% sample in the 24 communities not selected for participation in the ESS and all HIV-positive adults in the 6 ESS communities as described above for the ESS denominator for ART coverage = 2,971.
- Based on preliminary BHS data, we found that 96% of HIV-positive participants who knew their status and were on ART were virologically suppressed representing 70% of all HIV-positive persons (irrespective of prior knowledge of status and ART status). Therefore, the additional 3% increase in diagnosis among HIV-positive persons by T2 in the EC arm contributes to an increase in VL suppression coverage of 3%\*87%\*96% = 2.5%. As described above, due to UTT, there will be an increase in VL suppression coverage among previously ART-naïve individuals with a CD4>350 cells/mm³ of 3.9%\*96% = 3.7%.

Therefore, the **ESS numerator for the EC arm** is calculated as 3,516\*[(proportion of HIV-positive persons expected to know their status who are on ART and virologically suppressed) + (additional proportion on ART and virologically suppressed due to increased diagnosis and UTT)] =**2,971\***<math>(0.70+0.025+0.037) =**2,971\***(0.762 =**2,264**.

The ESS numerator for the CP arm is calculated as 2,971\*(target outlined in Protocol 3) = 2,971\*0.95 = 2,822.

#### MC coverage numerators and denominators:

- The BHS denominator includes HIV-negative men in the BHS 20% sample and is calculated as average number of BHS enrollees per community)\*(proportion who are male)\*(proportion HIV-negative)\*(number of communities) = 400\*0.45\*0.8\*30 = 4,320.
- The **BHS numerator** is calculated as 4,320\*(proportion of HIV-negative men circumcised based on preliminary BHS data) = 4,320\*0.35 = **1,512**.
- The ESS denominator includes HIV-negative men from the BHS 20% sample in the 24 communities not selected for participation in the ESS and all HIV-negative men (100% sample)

in the 6 ESS communities. The assumptions regarding additional enrollment at T1 are described in detail above for ART coverage.

The number of HIV-negative men from the BHS 20% sample in the 24 non-ESS communities and 6 ESS communities is calculated as (average number of BHS enrollees per community)\*(proportion expected to be present at T2)\*(additional proportion newly enrolling at T1)\*(proportion male)\*(proportion HIV-negative)\*(number of communities) = 400\*0.90\*1.10\*0.45\*0.8\*30 = 4,277.

The number of HIV-negative men in the 6 ESS communities outside the BHS 20% sample is calculated as [ (average population size per community)\*(proportion expected to be age-eligible)\*(proportion expected to be present)\*(proportion expected to consent)\*(proportion male)\*(proportion HIV-negative) – (average number of HIV-negative BHS male enrollees per community at T2) ]\*(number of ESS communities) = [ (6.027\*0.58\*0.8\*0.85\*0.45\*0.8) - (4.277/30) ]\*6 = 4.279.

Therefore the ESS denominator per arm is 4,277 (HIV-negative from the BHS 20% sample in 30 communities) + 4,279 (HIV-negative men from the 80% sampled in 6 ESS communities) = 8,556/2 = 4,278.

- The **ESS numerator for the EC arm** is calculated as **4,278**\* (proportion of HIV-negative men expected to be circumcised) = **4,278**\*0.5 = **2,139**.
- The ESS numerator for the CP arm is calculated as 4,278\*(target outlined in Protocol 3) = 4,278\*0.6 = 2,567.

#### Widths of the 95% confidence intervals:

 Based on the variance formula from Hayes and Moulton (2009), the 95% CI widths are calculated as follows:

$$precision = 1.96 \sqrt{\frac{p(1-p)DEFF}{n}}$$
 
$$DEFF = 1 + (m-1)k^{2} \frac{p}{(1-p)}$$
 
$$m = \frac{n}{c}$$

precision is the width of the 95% CI
p is the proportion for which the 95% CI is calculated
DEFF is the design effect
n is the total sample size from which p is calculated (i.e., denominator)
k is the between-cluster coefficient of variation of the true proportion
c is the number of clusters (i.e., number of communities)

Table 5 summarizes the inputs for calculating the widths of the 95% CIs shown in Table 4.

Table 5: Inputs for Calculating CI Widths Surrounding HTC, ART (including VL suppression), and MC Coverage Proportions at Baseline and Study End

| | | Baseline Household | | |
|---|---|---|---|---|
| | | Survey (BHS) | End of Study Surv | urvey (ESS) |
| | Input | All Study Communities | EC Arm | CP Arm |
| | р | 0.37 | 0.48 | 0.90 |
| HTC | n | 12,000 | 5,931 | 5,931 |
| Coverage | С | 30 | 4 | 4 |
| | k | 0.1 | 0.1 | 0.1 |
| | р | 0.73 | 0.795 | 0.93 |
| ART | n | 3,000 | 2,971 | 2,971 |
| Coverage | С | 30 | 15 | 15 |
| | k | 0.1 | 0.1 | 0.1 |
| | р | 0.70 | 0.762 | 0.95 |
| VL | n | 3,000 | 2,971 | 2,971 |
| Suppression | С | 30 | 15 | 15 |
| | k | 0.1 | 0.1 | 0.1 |
| | р | 0.35 | 0.50 | 0.60 |
| MC | n | 4,320 | 4,278 | 4,278 |
| Coverage | С | 30 | 15 | 15 |
| | k | 0.1 | 0.1 | 0.1 |

# 5.2.2. Power to detect difference in coverages of HTC, ART, VL suppression, and MC at the end of study

The coverage of ART, VL suppression, and MC will be assessed in eligible participants in 100% of 3 pairs of randomly selected communities and 20% of the remaining 12 pairs of communities. The coverages of ART, VL suppression, and MC in the 12 pairs of communities will be adjusted based on the difference in coverage observed between the 20% cohort and the remaining 80%. HTC coverage over the past 12 months and 24 months will be assessed in eligible participants in 80% of the 3 pairs of communities, outside of the 20% cohort. This is because the 20% cohort in both arms is expected to receive 100% HTC coverage by study design.

The projected coverage of HTC, ART, VL suppression, and MC at the end of year 3 is 52%, 80%, 76% and 50%, respectively, in the Enhanced Care arm, and 90%, 93%, 95% and 60%, respectively, in the Combination Prevention arm (see Table 4 above). Assuming a coefficient of variation of 0.1 for HTC, ART, VL suppression, and MC coverage, the power in detecting the aforementioned differences in coverage in the ESS is 99%, 96%, 99% and 98% for HTC, ART, VL suppression, and MC, respectively (see Table 6).

Table 6. Estimated Power of Detecting Differences in Coverages in HTC, ART, VL Suppression, and MC between Enhanced Care (EC) and Combination Prevention (CP) Arms in the ESS

| | | HTC | ART | VL | MC |
|--------------------------|----|-----|-----|-----|-----|
| Projected | EC | 48% | 80% | 76% | 50% |
| Coverage at ESS | СР | 90% | 93% | 95% | 60% |
| Coefficient of Variation | | 0.1 | 0.1 | 0.1 | 0.1 |
| Power | | 99% | 96% | 99% | 98% |

# 5.2.3. Sampling Strategy for End of Study Survey (ESS)

To ensure on-time completion of the ESS, which will be conducted by one team in each arm, ESS communities must be selected with consideration given to the sequence of the rollout of BHS, population size and region. To select 3 feasible pairs of ESS communities, we considered the anticipated rollout sequence and selected one pair of communities from each of the three regions represented in the study. This resulted in the inclusion of the 5<sup>th</sup>, 7<sup>th</sup> and 13<sup>th</sup> pairs as the initial list of ESS communities. No further adjustment of selection is expected to be necessary, but in the event of unanticipated changes in logistical or operational activities, the selection procedure described above may be repeated prior to any outreach for the ESS.

To sample 100% of households in 3 pairs of Combination Prevention and Enhanced Care communities at the end of the study, all households in the selected Combination Prevention and Enhanced Care communities will be approached for: (1) GPS mapping, (2) enumeration of number and demographics of persons living in households, and (3) offering of HTC services. The ESS will therefore include residents of the 80% of households not participating in the BHS/HIC in the 3 selected pairs of communities, and ESS data will be complemented by data from the residents of the 20% of households participating in the BHS/HIC in all 30 communities at T2.

Note that it is likely we will reach all 20% of households with BHS/HIC enrollees during the ESS, because HIC households will have previously agreed to study procedures. However, it is less certain what proportion of the remaining 80% of households will agree to the survey.

Possible reasons for not reaching non-HIC households in Enhanced Care and Combination Prevention communities at study end include:

- **Refusal**: We expect rates of refusal for participation in the ESS to be <15%, based on experience from northern Botswana and Mochudi district.
- Not at home during the household visit: This may apply particularly to men. If the survey team determines that certain household members are best reached for the survey after hours during the week or on weekends, arrangements will be made to visit the households during these convenient times.

Investigators will need to assess whether participation rates in the household survey introduces any potential selection bias.

# **5.3.** Expected Numbers of Study Participants

Study participants will be recruited to participate in and provide data for different aspects of the study per the Table below.

**Table 7. Expected Numbers of Participants in Study Components** 

| Study component | Targeted subjects | Expected # of Participants | Data Collection |
|---|---|---|---|
| Household<br>structure | Household representative in 20% households | 7,244 | <ul> <li>Household Composition Form (updated at each visit)</li> <li>Baseline Household Survey at TO</li> </ul> |
| BHS/HIC | Age-eligible members of 20% households, a subset of whom will be enrolled into the HIC (HIV-negative and meeting additional HIC eligibility critieria) | 12,000 total (9,000 in HIC) | <ul> <li>Baseline Resident Survey at first visit</li> <li>Annual Resident Survey at subsequent visits</li> </ul> |
| Qualitative Research on Barriers to and facilitators of LTC and ART initiation among BHS participants | HIV-infected BHS participants BHS Research Assistants and Nurse Prescribers | 60 BHS participants in FGDs 40 BHS participants in IDIs 20 Research Assistants and Nurse Prescribers inFGDs | <ul> <li>Focus Group Discussions</li> <li>In-depth semi-structured interview guide</li> </ul> |
| Blood draw for research purposes | HIV-infected individuals (or seroconverters in BHS/HIC | 3,270 (part of 12,000 above) | Same as for BHS |
| | HIV-infected BHS residents who decline survey participation but are willing to give a blood sample | 150 | Research blood draw form |
| | All HIV-infected persons in CP community clinics | 11,934 | Research blood draw form |
| End of study<br>survey | All eligible residents in 3 pairs of selected communities | 14,262 total: ~2,400 from the 20% households at T2 and ~11,862 from the remaining 80% of households. | End of Study Resident Survey (for participants enrolling for the first time at ESS) Final Resident Survey (modified annual follow-up survey) for previous enrollees from 20% households) |
| Supplemental<br>Economic<br>Assessment | Individuals experiencing OIs seeking out- or inpatient care | Up to 150 (depending on how many respondents from 20% households meet this criteria) | Economic Assessment |
| | Individuals with low CD4 without OIs seeking out- or inpatient care | Up to 300 (depending on how many respondents from 20% households meet this criteria) | Economic Assessment |
| Point-of-care Viral<br>Load Pilot Study | ART-naïve HIV-infected individuals in BHS | Up to 400 | |

#### 5.4. Planned Interim Analysis of Data

The BCPP is divided into three interlocking protocols (two active protocols, after Protocol 2 was terminated in 2015), and the investigators expect that DSMB review will require information regarding interim study results and study conduct from all three. The combination prevention package under study includes provision of ART for all HIV-infected adults regardless of WHO Stage or CD4 count. Hence, the reports will provide information needed to evaluate the adverse and favorable effects of this intervention on individually treated patients as well as on the villages in which they reside. The study will require at least 5 reviews, DSMB 1-5, proposed to take place at baseline and at the end of years 1, 2, 3, and 4. DSMB 3 will evaluate intervention rollout and safety. To demonstrate that the study has reasonable power to answer the study questions given information up to the time of each review, investigators will provide the DSMB with assessments of the adequacy of coverage of proposed interventions; estimated conditional power given available incidence information will be provided at DSMB 4. Investigators (other than statisticians preparing DSMB reports) will remain blinded to HIV incidence data collected from the HIC, during the conduct of the study. Details of the DSMB review plan for each protocol are provided in that protocol, and the full detailed plan is provided in Appendix C4.

#### 5.4.1. Proposed Schedule of DSMB Reviews

The incidence cohorts (HIC) will be enrolled in all 30 communities over a period of approximately two years. The enrollment of incidence cohorts for one matched pair (2 study communities) will begin simultaneously. The number of working days required to complete each community in the pair will vary depending on the sizes of the communities. The BHS/HIC households will be revisited approximately 12 months, and 30 months after they were enrolled. Figure A in Appendix C4 illustrates the planned schedule of enrollment and follow-up.

As demonstrated in Figure A in Appendix C4, there are 5 proposed DSMB reviews. The proposed components of each DSMB review are summarized in Table A in Appendix C4. Harvard investigators will provide at least 5 DSMB reports related to activities covered in this *Evaluation Protocol*: one for protocol review before enrollment, one each at DSMB 2 and 3 with reports of baseline parameters; one at DSMB 4 (after the end of calendar year 3) with assessment of conditional power based on available incidence information and relevant coverage information in intervention implementation, and one at study end at DSMB 5. At DSMB 5, we will provide reports on all data collected during the BHS, HIC follow-up, and ESS.

# 6. STUDY PROCEDURES

In this section we describe detailed study procedures for each of the following study segments: (1) the Baseline Household Survey (BHS), (2) the HIV Incidence Cohort (HIC), (3) Research Blood Draws, and (4) the End of Study Survey (ESS).

### 6.1. Baseline Household Survey (BHS)

Overview: During the BHS conducted in the 20% households, voluntary HIV testing and counseling (HTC) will be conducted, and the HIC will be identified and enrolled (note: the HIC is an open cohort, so additional eligible residents of the same 20% households may enroll in the HIC in subsequent years). HIV-positive participants will be referred to the local clinic for evaluation and if eligible, related interventions in Combination Prevention communities. All eligible consenting residents of the 20% households will be asked to take part in a survey (and, if HIV-infected, a research blood draw). All of these participating residents will be asked to respond to the same core survey (Resident Survey, Baseline).

Data collected under previous versions of the protocol with the original follow-up schedule will still be used, i.e. data and samples from participants whose communities had a T2 and/or T3 visit under the former follow-up schedule will be included in analyses. This protocol outlines the visit schedule and procedures to be implemented following the roll-out of version 5.0 but does not invalidate approved protocol procedures conducted prior to the roll-out of version 5.0.

Starting with version 5.0 of the protocol, during the subsequent visit to the household at T1, newly-identified eligible residents will be asked to enroll in the BHS/AHS, including the HIC (or, if HIV-infected, for a research blood draw); and all eligible residents will be asked to complete a survey focused on assessing uptake of key components of the combination prevention package (and changes in risk behavior), regardless of whether or not they are participating in the HIC or are referred for interventions.

#### 6.1.1. Selection and Recruitment of Households for the BHS

• Random Selection: As described in Section 5, for each study community, a complete list of households will be obtained from google area maps (and potentially complemented by data from other sources). From this sample frame, 25% of households will be selected using simple random sampling. In villages with population under 6,000, the required 20% households will be randomly selected from the 25% sample and approached first for participation in the study. In villages with population over 6,000, 333 households will be randomly selected from the 25% sample and approached first for participation in the study. The remaining 5% of selected households will be considered back-up households in case some of the households in the primary 20% sample refuse to participate. Households in the back-up list will be ordered (e.g. 1-49) to indicate the order in which they should be approached to meet sample size requirements.

**Recruitment:** Trained community liaison officers (CLOs) may do reconnaissance visits in advance of the survey team, for example, to identify households in the sample that are not actually inhabited or are not residential dwellings. These staff may also try to find out the ideal time for the survey team to visit, and the approximate size of the household so that the survey team may plan to accommodate potential participants. Research staff may perform these functions in the absence of CLOs. Each of the households in the 20% primary sample will be approached by the survey team for participation in the study. If some of these selected 20% households elect not to participate (e.g., all residents are repeatedly absent or refuse consent), the additional households in the full 25% sample will be approached, in the order specified, until either the pre-specified sample (described above) has been achieved or this 25% sample list is exhausted. All eligible residents will be asked to take part in activities related to the BHS (using the BHS/HIC Consent). Those who are confirmed HIV-uninfected and meet additional HIC eligibility criteria will be enrolled in the HIC (see Section 6.2). ART-naive HIV-infected residents will be referred to local clinics for WHO staging and in CP communities immediate ART initiation (see Intervention Protocol). See Figure 3.

**Training:** Prior to approaching the community, survey staff will have been trained in study procedures, including the informed consent process, HTC counseling, questionnaires and sample collection/processing/transport methods. Training will occur following structured procedures, to ensure that all study staff are trained in the same procedures. Survey staff will be arranged into teams of sufficient size and number, such that the study schedule can be met.

#### 6.1.2. Household Visit Procedures for the BHS

Interview of Household Representative: Trained study staff will approach the household representative of a selected household, which will preferably be the household head when available, but may be any other eligible household representative. Verbal consent will be requested using an IRB-approved script (Household Script). If consent is granted, general household information will be obtained from the household representative using the Household Composition Form. Information to be recorded includes:

- Household GPS
- Household address
- Household Size
- Household Composition. For each household member:
  - o Age
  - First name or initials
  - Gender
  - o Presence at the time of the household visit
  - Estimated number of nights spent per month outside the community over the past 12 months (which will be confirmed by individual household members)
  - Relationship to the head of the household or representative
- Common household socioeconomic indicators (Household Survey, Baseline)

#### Classification of Households that Cannot be Enumerated

All visited households selected for BHS need a final disposition status so that a decision can be made about whether any household is eligible for replacement. In cases where the residency status of a plot remains uncertain after a total of three visits, a research staff member will approach either a neighbor or a representative at the Village Development Committee (VDC) for assistance. This representative, who must be 18 years of age or older, will be asked whether a plot/household is regularly occupied by potentially eligible residents (Household Residency Status Assessment) to assist in making a final determination of the plots/households' residency status.

# Interview with Age-Eligible Household Members (16-64):

HIV counseling and testing (also, see HIV Testing Procedures below): to avoid creating an impediment to HIV testing that would not exist for residents accessing routine health services (by requiring written informed consent for, and participation in, study procedures), HTC (and POC CD4 as needed) will be offered to household members who decline participation in the research survey. Whereas only BHS study team members in Enhanced Care communities will offer HTC testing, HTC may be offered either by the BHS study team or by the HTC campaign team in Combination Prevention communities; the BHS study team will also refer individuals who decline testing to local clinics where HIV testing is available. Note: HIV and CD4 results (and accompanying information that is routinely collected as part of public HTC programs) will be collected on the HTC Intake form (see Intervention Protocol) in Combination Prevention communities and made available to the linkage to care manager for monitoring and evaluation of the intervention package (and as will be done as part of the HTC campaigns in the Combination Prevention communities). The linkage to care manager and HTC campaign team will be aware of the location of households selected for BHS/HIC in Combination Prevention communities, and will be informed of numbers of those who were not reached during the household survey due to refusal or absence. Residents declining HIV testing can still take part in the BHS, if they agree.

Written informed consent for participation in the BHS and annual follow-up visits will be obtained from each willing individual aged ≥18 who meets BHS eligibility criteria (BHS/HIC Consent). For residents aged 16 or 17 who meet BHS eligibility criteria, parental permission followed by minor assent will be obtained. Up to two revisits will be scheduled for absent individuals. The BHS consent will request permission for the study questionnaire, blood draws for research purposes for persons testing HIV-positive (including blood draw for HIV genotype, HIV incidence assay, and viral load) at the current visit or in cases of future seroconversion to HIV-positive status, optional storage of leftover blood for future testing, CD4 and viral load testing at T1 and/or T2 for HIV-positive individuals who are ART-naïve at enrollment or who seroconvert and are ART-naive after enrolling, and annual household questionnaire completion (at T1, T2--and T3 [for any communities completing T3 prior to the roll-out of version 5.0]) by all participants. With the elimination of the T3 visit in version 5.0 of this protocol, a Dear Participant letter will be used to inform enrolled participants that T2 will be their final visit. HIVinfected participants who decline participation in the BHS survey can still provide informed consent to donate blood for HIV VL and genotyping/incidence assay, using a separate consent form (Research Blood Draw Consent).

#### Questionnaire:

Each consenting eligible household member will be interviewed/complete a questionnaire in a private environment within the household or at an agreed upon space. A questionnaire will be completed at the BHS enrollment visit (Resident Survey, Baseline); in addition, a shorter followup questionnaire (Resident Survey, Annual) will be administered to BHS participants, including HIC members, at subsequent visits. During the final T2 visit, a Final Resident Survey will be administered to BHS/HIC participants. The first questionnaire (Resident Survey, Baseline) will include questions on basic demographic variables, current health status, medical history, prior coverage of HTC, current coverage of MC, prior or current pregnancies, sexual risk behavior, basic screening for active tuberculosis by symptoms-questions, and (among HIV-infected persons), prior/current use of antiretrovirals for treatment or PMTCT. All residents will complete a core questionnaire. When possible, residents may be randomly assigned to complete different short supplemental questionnaires in order to keep the duration of the interview as short as possible while still collecting key variables. Skip patterns will ensure that appropriate questions are asked depending on the self-reported HIV status, gender, and prior participation of the consenting adult. Subsequent questionnaires will include variables related to CP package intervention uptake, general health (e.g. history of serious illnesses, and in a sample of willing respondents, blood pressure and hip/waist circumference), and sexual risk behavior. Data will be collected on a mobile electronic device (e.g. notebook); these devices will use authentication/password protection and encryption to render information electronically unusable, unreadable, or indecipherable to unauthorized individuals. Mobile devices and the staff operating them will not be equipped with the encryption keys to decrypt select sensitive data fields. Secure and lockable rooms will be used to store mobile devices when not in use.

#### HIV testing procedures, BHS:

HIV testing will be offered to all adults who do not have documentation of HIV-positive status. Documentation of HIV-positive status is participant self-report of positive HIV status, in combination with: (1) an official MOH HIV test result card indicating HIV-positive status, (2) documentation of prior ART or PMTCT ARV prescription, or (3) documentation of pre-ART care including either a CD4 count, a WHO Stage, or some specific mention of medical care for the HIV-infected patient by a clinical care provider. When in doubt, HIV status will be considered "undocumented".

## a) Adults with no Documentation of HIV-Positive Status, BHS:

These individuals include those reporting being HIV-negative at their last test, individuals reporting never having HIV tested, or individuals reporting being HIV-infected but not having documentation of HIV-positive status as described above.

- Pre- and post-test counseling will be provided by trained staff, as per Botswana Government guidelines and standards.
- ➤ Capillary blood samples will be collected by fingerprick using a sterile disposable lancet. Blood will be aliquoted into a microtube. This blood will be used for both the rapid HIV test and subsequently (among HIV-positive individuals), for point-of-care CD4 cell count (POC CD4). If a capillary blood sample cannot be obtained a venous blood sample (4-5 ml) may be drawn instead for the rapid HIV test and subsequently (among those testing HIV-positive), used for POC CD4.

- The capillary (or venous) blood sample will first be tested using parallel HIV rapid testing algorithms (see Section 8.4). HIV rapid test results will be released to the participant at the time of the visit.
- ➤ Discordant HIV test results will be resolved by collection of a venous blood sample (~ 4-5 ml) that will be sent to the laboratory for HIV enzyme immune-assay (EIA) testing as per the National Algorithm. Contact details of individuals with sero-discordant results will be obtained and when HIV EIA results are available, the study personnel make arrangements provide the results (either in the person's home or in the clinic, depending on the participant's preference) and perform the appropriate post-test counseling and remaining study procedures.
- > Subsequent management of the individual will depend on the HIV test result:
  - HIV Negative Participants: HIV negative household members meeting eligibility criteria for the HIV Incidence Cohort (HIC) will be enrolled in the HIC (see Sections 4.4 and 6.2). HIV-negative participants meeting criteria for the BHS but not the HIC will participate only in the BHS and subsequent surveys.
  - HIV-Positive Participants: Residual blood remaining after HIV testing will be used to perform a POC CD4 test using the PIMA CD4 machine at the household. If insufficient blood remains from the sample taken for the HIV rapid test, venous blood should be drawn (4-5 ml) along with the tubes for VL and genotyping/incidence assay (see below) to avoid a separate prick. POC CD4 results will be provided to the participant immediately following testing. Participants will have venous blood drawn for viral load/HIV incidence assay/genotyping/storage. The blood for viral load, HIV genotyping, and HIV incidence assay testing will be collected in 2 tubes: 4-5 ml for viral load and up to 10 ml for HIV genotype/incidence assay/storage. The viral load results will be returned to HIV care clinics. The pre-ART viral load is not standard of care and is not required to determine ART eligibility in Botswana. Therefore, while it will be shared with clinics, it will be of limited clinical use. The incidence assay and viral phylogenetic tests are being performed primarily for research purposes, and will not be run in real time; therefore results will not be returned to the patient. Efforts will be made to avail results indicating transmitted drug resistance to participants. However, this testing will be done retrospectively and therefore may be of limited clinical utility.

All HIV-infected persons who are not yet in HIV care and/or on ART will be referred for immediate HIV care and treatment at the study community clinic according to national guidelines in all Enhanced Care and Combination Prevention communities. If the patient is treatment-naive, the patient will also be referred to the study community clinic in Combination Prevention communities for immediate ART initiation. Access to universal ART is described in the separate *Intervention Protocol* that is part of the BCPP.

Verbal Consent Script for Household Representative Household Structure Survey Approach Eligible HH Members for Survey Participation Questionnaire No Documentation of Documentation of HIV-**HIV Status** HIV-positive status positive status Finger capillary blood sampling HIV RT + sample for POC CD4 See Figure 4B Below HIV POS^ 10ml EDTA **HIV IND HIV NEG** -Genotype -Incidence **Run POC** 4-5ml EDTA **INCIDENCE COHORT\*** 4-5ml EDTA CD4 EIA/WB/PCR 4-5ml EDTA only In CPCs, refer to clinic Results to if needed: stored for ART initiation. In **Participant** ECCs. refer for WHO staging and national ART program

Figure 4A: BHS Procedures for Individuals with no Documentation of HIV-Positive Status

Abbreviations: CPC, Combination Prevention Community; ECC, Enhanced Care Community; HH, Household; HTC, HIV Testing and Counseling; RT, Rapid Test; POC, Point-of-Care; C, consent procedures; IND, indeterminate; VL, viral load; EIA, enzyme immuno-assay; WB, Western Blot. \*Eligible persons only (See section 4.4).

^Leftover sample from either the fingerprick or 4-5mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

#### b) Adults who Have Documentation of HIV-Positive Status, BHS:

These individuals include residents who report being HIV-positive and have documentation supporting this (MOH HIV test card, documentation of prior ART, CD4, WHO staging, or specific mention of HIV-related clinical care). Subsequent management of the participant will depend on whether the participant reports taking ART:

- All BHS participants documented to be HIV-infected (regardless of ART status): A venous blood draw for a 4-5ml EDTA tube for HIV viral load, and a 10ml EDTA tube for genotyping/HIV incidence assay will be requested.
- Residents documented to be HIV-infected but ART-naive: these residents will have a POC CD4 test run (and will be provided with the result). Generally, the sample for this POC CD4 in ART-naive residents documented to be HIV-infected will be drawn along with the venous blood for VL and genotyping/incidence assay, to avoid a separate prick. For residents declining the research blood draw, sample for POC CD4 can be obtained by finger stick for capillary blood. All HIV-infected persons who are not yet in HIV care and/or on ART will be referred for immediate HIV care and treatment at the study community clinic according to national guidelines in all Enhanced Care and Combination Prevention communities. Patients will also be

referred to the study community clinic in Combination Prevention communities, for universal ART, which is described in the separate *Intervention Protocol* that is part of the BCPP.

Verbal Consent Script for Household Representative Household Structure Survey Approach Eligible HH Members for Survey Participation Questionnaire **No** Documentation of Documentation of HIV-**HIV Status HIV-positive Status** positive status See Figure 4A Above Reports prior/current ART Reports No Prior/current ART^ 10ml EDTA -Genotype 4-5ml EDTA or finger capillary -Incidence 10ml EDTA blood sampling for POC CD4 4-5ml EDTA -Genotype -Incidence -VL 4-5ml EDTA In CPCs, refer to clinic for ART initiation. In -VL ECCs, refer for WHO staging and national ART program

Figure 4B: BHS Study Procedures for Individuals with Documentation of HIV-Positive Status

Abbreviations: CPC, Combination Prevention Community; ECC, Enhanced Care Community; HH, Household; HTC, HIV Testing and Counseling; POC CD4, Point-of-Care CD4; C, consent procedures; VL, viral load.

Note about Test Results During BHS: Individuals participating in HTC will be offered the result of their rapid HIV test with post-test counseling. During the BHS, POC CD4 results will be given to the participants in all communities. The viral load results will be returned to HIV care clinics. The pre-ART viral load is not standard of care and is not required to determine ART eligibility in Botswana. Therefore, while it will be shared with clinics, it will be of limited clinical use. The incidence assay and viral phylogenetic tests are being performed primarily for research purposes; therefore results will not be returned to the patient. Genotyping will not be run in real time and therefore will be of limited utility for patient care. However, if results indicate transmitted drug resistance, efforts will be made to avail this information to the participant upon completion of testing.

#### • Compensation:

BHS participants will receive 20 pula in cell phone airtime as compensation for their time to participate in the survey.

<sup>\*</sup>Consent administered to eligible household members only (see section 4.4).

<sup>^</sup>Leftover sample from either the fingerprick or 4-5mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

#### 6.1.3. Household Visit Procedures for Non-HIC Members at T1:

These procedures pertain to consenting residents (both HIV-uninfected and HIV-infected) in 20% households who are not participating in the HIC. This group will include residents who took part in the original BHS, as well as residents newly-identified at T1 who are not enrolled in the HIC.

For residents who already consented to and took part in the BHS (and are not in the HIC), a short survey will be administered at T1, primarily to assess combination prevention intervention uptake (and to assess risk behavior/risk compensation and general health). HTC will be offered to those without documentation of HIV-positive status. Point-of-care CD4 and viral load testing will be offered at T1 to HIV-positive individuals who were ART-naïve upon enrollment into BHS, or who seroconvert and are ART-naïve after enrolling in BHS. POC CD4 results from T1 will be shared with participants in both arms, and viral load results will be shared with clinics (or with patients, if a validated point-of-care viral load test is introduced). A research blood draw (for HIV genotype/incidence assay testing/optional storage) will be obtained from anyone newly identified with HIV infection. Procedures for the final visit to BHS/HIC households at T2 are described with those for the end of study survey (ESS). See Figure 5B.

For residents who did not take part in the BHS at TO (and are not in the HIC), the same procedures as outlined for the BHS will be offered at T1.

# 6.1.4. Data Collection and Handling:

- Questionnaires: For consenting BHS participants, all questionnaire data, HIV test results, POC CD4 test results, and information regarding collection of sample for genotyping/incidence assay/storage will be collected electronically using notebook computers. These devices will use authentication/password protection and encryption to render information electronically unusable, unreadable, or indecipherable to unauthorized individuals. Mobile devices and the staff operating them will not be equipped with the encryption keys to decrypt select sensitive data fields. Secure and lockable rooms will be used to store mobile devices when not in use.
- Consent Forms: Investigators will document consent procedures on the notebook application.
   One copy of the signed consent form will be kept by investigators while a second copy will be kept by the participant.
- Blood samples will be labeled with barcoded stickers and transported to the study clinic or lab, as appropriate.

#### 6.1.5. Criteria for Study Discontinuation

Participants will be discontinued from longitudinal follow-up in the BHS (or HIC) if the participant (or guardian if < age 18) requests to withdraw.

# 6.1.6. Data Collection on Cause-of-Death for Deceased Study Participants

If study staff learn that an enrolled study participant has died during the course of the study, basic information related to the cause of death will be recorded. A deceased study participant is no longer a human subject per the definition at 45CFR46.102(f); a human subject is a *living* individual. Data for the Cause-of-Death Form may be collected from official sources, such as medical records, a death certificate, or from health care providers.

# 6.2. HIV Incidence Cohort (HIC)

Methods for household selection and identification of eligible persons for HIC enrollment are described above (Section 6.1).

### 6.2.1. Enrollment Procedures, HIC

- Consent: As described in Figure 4A above, residents of the 20% households will be asked for consent for survey participation (BHS/HIC Consent). This consent will request permission for the baseline study questionnaire, subsequent HIV testing and questionnaire at follow-up visits, future blood draw for research purposes if seroconversion to HIV-positive status occurs (blood for HIV viral load/genotype/incidence assay/optional storage), POC CD4 and viral load at T1 and/or T2 (among a subset, as described above) if seroconversion occurs, and storage of blood remaining from the HIV rapid test microtube finger prick draw. The latter will be used for confirmation of negative HIV status at enrollment, if future HIV seroconversion occurs. Consenting residents who are determined to meet HIC eligibility criteria will be enrolled in the HIC.
- Venous blood draw: In the event that insufficient blood remains from the sample drawn for the
  HIV rapid test, HIC enrollees will have a venous blood sample drawn for storage at the research
  lab. If the participant sero-converts during HIC follow-up the baseline sample will be available
  to confirm that the participant was truly HIV-negative at enrollment. The storage of this
  baseline blood sample is indicated for this protocol and covered in the main body of the
  BHS/HIC consent form. This blood draw will also mitigate the potential for inadvertent HIV
  status disclosure that could occur if venous blood draws only pertain to HIV-infected
  individuals.
- Questionnaire and Forms: All consenting residents will be administered an enrollment questionnaire (Resident Survey, Baseline), and contact information (mobile phone numbers, alternate addresses, and addresses of a friend/family member) will be obtained to facilitate tracing (Locator Form). At T1, a shorter questionnaire (Resident Survey, Annual) including questions related to CP package intervention uptake, general health, and sexual risk behavior will be administered. Those who decline enrollment in the HIC will be asked to take part in the BHS only. Residents declining both the HIC and BHS will be thanked for their time and asked, via an IRB-approved verbal consent script (Refusal Script) to provide basic information about their reason for declining via the Refusal Survey Form. This will assist in characterizing the impact of refusal on study outcomes.

#### 6.2.2. HIC Follow-up

- HIC Follow-up Schedule: Subsequent household surveys of the HIC will be conducted at approximately 12 and 30 months after enrollment (T1 and T2, respectively). Procedures for the final visit at T2 visit are described with those for the end of study survey (ESS). Therefore, in this section, we restrict description of procedures to those that apply to T1. HIC activities conducted during the T1 follow-up household visits include: (1) updating the household structure to assess who might be newly eligible for BHS/HIC enrollment, (2) repeat HIV testing and questionnaire administration to HIC enrollees, and (3) screening non-HIC enrollees for HIC eligibility. These three activities are described in detail below. Wherever possible, via telephone or other communication channels, study teams will arrange a suitable time and venue to meet, and perform study procedures, for HIC household members. When necessary, study interviews may be conducted by phone.
- Activity #1, HIC Follow-up: Update Household Structure: Study staff will approach the household head or representative of the selected household. A previously enrolled household member can serve as the household representative, where appropriate. Updated household information will be obtained. Information to be recorded includes:
  - Household GPS (confirmed not re-measured)
  - Household address updated if there have been changes
  - Household Composition (updated)

# Activity #2, HIC Follow-up: Questionnaire, Repeat HIV Testing, and Other Lab Draws in Existing HIC Enrollees (Figure 4C):

HIC participants will have previously consented to the questionnaires and blood draws described here (as part of the BHS/HIC consent process). Previous enrollees of the HIC will be engaged in a follow-up questionnaire (Resident Survey, Annual), administered using devices such as notebook computers; these devices will use authentication/password protection and encryption. In addition, HIC enrollees will be re-tested for HIV using point of care rapid tests (two different rapid tests in parallel) performed on blood collected from a fingerstick in a microtube. Even if the HIC enrollee indicates that he/she has tested HIV-positive and enrolled in care since the earlier negative HIV test, repeat HTC will be offered to existing HIC enrollees to confirm HIV positive status one time.

If the existing HIC enrollee tests HIV-negative, the enrollee will be offered routine post-test counseling, and, in Combination Prevention communities only, those services for HIV-negative adults that constitute part of the CP package (TB screening and referral of uncircumcised HIV-negative males for MC).

If the participant tests HIV-positive, (or if the participant reports knowing HIV-positive status and refuses repeat HTC), a venous blood draw will be performed for HIV viral load (10mL EDTA tube) and for genotyping/incidence assay/optional storage (10mL EDTA tube) among HIC participants in both the Enhanced Care and Combination Prevention communities.

Procedures will differ slightly for HIC members in the Enhanced Care vs. Combination Prevention communities with regard to linkage-to-care services:

### • Procedures For HIC Members Testing Positive for HIV During Follow-up:

- Participants Reporting no Previous ART: a POC CD4 test will be run on residual sample from the HIV test, and the CD4 result shared with the participant. If the residual sample is insufficient a venous blood draw (4-5 ml) may be performed. Linkage-to-care services will be provided in Combination Prevention Communities. Participants in Enhanced Care communities will receive the Enhanced Care referral to care and treatment services described in the BCPP Intervention Protocol.
- Participants Reporting Prior ART Initiation: Management will be the same as for pre-ART participants, except no POC CD4 will be run.
- HIC Members who test positive for HIV at T1: These participants will still have a follow-up visit at T2. Participants who seroconvert between T0 and T1, and report no previous ART at T1 will have point-of-care CD4 and viral load testing again at T2. See Figure 5B.

\*Note about Test Results During Follow-up: Individuals participating in HTC during T1 and T2 will be offered the result of their rapid HIV test with post-test counseling. During follow-up, POC CD4 results will be given to the participant during the study visit. Viral load results will be returned to HIV care clinics. The pre-ART viral load is not standard of care and is not required to determine ART eligibility in Botswana. The incidence assay and viral phylogenetic tests are being performed primarily for research purposes; therefore results will not be returned to the patient. Genotyping will not be run in real time and therefore will be of limited utility for patient care. However, if results indicate transmitted drug resistance, efforts will be made to avail this information to the participant upon completion of testing.



Figure 4C: Follow-up Procedures for HIC Enrollees During T1

Abbreviations: CP, Combination Prevention; EC, Enhanced Care; HH, Household; RT, Rapid Test; POC CD4, Point-of-Care CD4; IND, indeterminate; VL, viral load; EIA, enzyme immuno-assay; WB, Western Blot. #Verbal consent script need not be re-administered if the respondent is the same person at follow-up visits, or an enrolled survey participant.

^Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5). \*\*At T1, previous HIC enrollees who have seroconverted since T0 will have POC CD4 run if they are ART-naïve. At T2, these HIC enrollees who had POC CD4 at T1, i.e. those who were ART-naïve at T1, will have another POC CD4 at T2, even if they have started ART between the T1 and T2 visits (see Figure 5B).

- Activity #3, HIC Follow-up: Screening of non-HIC Members for HIC Eligibility: Adults identified as possibly being newly eligible for the HIC, based on the interview with the household head/representative, will be approached at T1. For example, residents in the 20% of households originally selected who were too young to enroll in the HIC during the BHS may turn 16 years of age during follow-up, and now be eligible for the HIC, or a new resident may be present. These adults will be invited to participate in the research, asked to sign the BHS/HIC Consent, respond to the questionnaire, and then be offered HTC services, similar to procedures conducted during the BHS. Similar to the BHS, adults in the HIC household will either have documentation of HIV status, or not. Subsequent management depends on whether the adult already has documentation of HIV-positive status or not:
  - No documentation of HIV-positive Status: These procedures are summarized in Figure 4D below. Potential new participants will be asked consent to join the research study. Eligible HIV-negative adults will be offered the opportunity to enroll in the HIC (refusers and those who are not eligible for the HIC will be asked to participate in the same procedures summarized in the BHS (see Section 6.1). If consent is granted, the same questionnaire administered during the BHS (Resident Survey, Baseline) will be administered to these newly identified individuals. HTC will be offered. HIV-infected adults will be asked for research blood draws, and further managed according to whether the patient is in a Combination Prevention or Enhanced Care community (Figure 4D).
Figure 4D: Procedures for Individuals in 20% Households who are Newly Identified During T1 and who have No Documentation of HIV-Positive Status



Abbreviations: HH, Household; HTC, HIV Testing and Counseling; RT, Rapid Test; POC CD4, Point-of-Care CD4; C, consent procedures; IND, indeterminate; VL, viral load; EIA, enzyme immuno-assay; WB, Western Blot.

#Verbal consent script need not be re-administered if the respondent is the same person at follow-up visits, or an enrolled survey participant.

**Documented HIV-Positive Status:** Newly identified household members with a documented HIV-positive status will be interviewed and asked for research blood draws and further managed according to whether the individual is in an Combination Prevention or Enhanced Care community (Figure 4E). These participants will still have a follow-up visit at T2. HIV-positive participants who enroll at T1, and report no previous ART will have point-of-care CD4 and viral load testing again at T2 (see section 6.1.3 and Figure 5B).

<sup>\*</sup>Eligible persons only (See section 4.4).

<sup>^</sup>Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

<sup>\*\*</sup>HIV-positive pre-ART participants enrolled at T1 will have POC CD4 and viral load tests at T1 (as shown above) and again at T2 (see section 6.1.3 for follow-up procedures of non-HIC enrollees).

Figure 4E: Procedures for Individuals in 20% Households who are Newly Identified During
T1 and who HAVE Documentation of HIV-Positive Status



Abbreviations: HH, Household; HTC, HIV Testing and Counseling; POC CD4, Point-of-Care CD4; C, consent procedures; VL, viral load.

#Verbal consent script need not be re-administered if the respondent is the same person at follow-up visits, or an enrolled survey participant.

- HIV Incidence Cohort Retention Procedures: Three attempts to make appointments for follow-up visits are made by phone for each study participant before the survey team returns to enrolled households. Once the survey resumes in the community, three attempts, either household visits or calls, will be performed in an effort to reach each enrolled member and complete follow-up study procedures.
- <u>Data Collection</u>: Questionnaires to be administed to HIC enrollees will be approved by IRBs prior to use in the field. All data will be collected electronically on devices such as notebook computers that are encrypted and password protected. Investigators will store signed paper consent forms and will also indicate electronically whether participant consent has been obtained. Paper copies of informed consent forms will be provided to the HIC enrollees. Blood samples may have bar codes linked to study IDs that are applied at the point of sample collection.

<sup>\*</sup>Consent administered to eligible household members only (see section 4.4).

<sup>^</sup>Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

<sup>\*\*</sup>HIV-positive pre-ART participants enrolled at T1 will have POC CD4 and viral load tests at T1 (as shown above) and again at T2 (see section 6.1.3 for follow-up procedures of non-HIC enrollees and Figure 5B).

- <u>Compensation</u>: Each HIC participant will receive 20 Pula (about \$3) worth of air time as compensation for time dedicated to the study at each scheduled follow-up study home visit.
- 6.3. Focus Group Discussions and Individual In-Depth Interviews related to barriers to and facilitators of linkage to care and ART initiation among a subset of BHS participants

  In order to understand locally-relevant barriers to and facilitators of linkage to care and ART initiation, including initiation of "expanded" ART outside of local guidelines, we will conduct focus group discussions (FGDs) and individual in-depth interviews (IDIs) with a subset of HIV-infected BHS participants. The goal is to improve/optimize approaches to linkage to care and ART initiation in the context of the overall trial and ultimately in Botswana.

#### 1) Recruitment

Recruitment will occur at or after T1, because at that time we will be assessing whether HIV-infected persons referred for care and ART at T0 actually linked/started ART.

We will invite HIV-infected BHS participants 18 years of age or older who, within their own community: 1) have not linked to care since initiation of the BHS, 2) have linked to care and were found to be eligible for treatment but did not start ART, or 3) linked to care, started and continued ART. We will convene up to two focus groups for each one of the three categories to learn about barriers to linkage and ART initiation as well as attitudes and approaches that can facilitate linkage to care and ART adherence. We aim to include in the FGDs a subset of individuals who were eligible to start ART by current local guidelines and a subset who were eligible by expanded ART guidelines. These FGDs will be semi-structured and done using an FGD guide. We will also conduct semi-structured IDIs focusing on the three groups described above.

We will convene up to 6 FGDs among BHS participants from CPCs that will each include between 8 and 10 participants. Participants will be purposefully selected to participate in one of the three categories of focus groups based on demographic and laboratory values (data collected in BHS). The BHS/HIC consent form states that participants may be invited to participate in additional aspects of the research. Using the BHS database and the eligibility criteria (see section 4.4.6) a Research Assistant will contact potential participants and ask to schedule a dedicated home visit to discuss participation in the FGD or IDI. Potential participants will be given a consent form and, if selected for a FGD, a confidentiality agreement to review. If a participant agrees to participate in a FGD, he/she will be informed of the date and time of the scheduled event. IDIs will be scheduled with participants based on their and staff member availability. Written informed consent will be obtained at the time the participant arrives for the scheduled FGD or IDI, and before any study procedures take place.

The BHS field team and the MOH nurse prescribers may have vital insight into the dynamics surrounding linkage to care and initiation of ART. Therefore, we will invite up to 20 members of these two groups to participate in separate FGDs. These FGDs will be semi-structured and done using an FGD guide. Findings from these FGDs will be used to finalize the FGD guides for HIV-infected BHS participants.

In general, different individuals will participate in FGDs and IDIs. We will continue to invite participants for IDIs until thematic saturation is achieved. We plan to conduct up to 40 IDIs. As

above, we will aim to include participants who met the eligibility criteria for expanded treatment (to investigate their understanding of expanded treatment, and motivators/barriers to starting ART) as well as those who were eligible by current local guidelines. Findings from the FGDs will be used to finalize the IDI guides.

#### 2) Consent

All individuals taking part in the qualitative research will sign a separate written consent form (ART Start Focus Group Consent for BHS, ART Start Focus Group Consent for Staff, or ART Start Interview Consent). Those participating in FGDs will also sign a confidentiality agreement.

# 3) Data Collection and Handling

FGDs and IDIs will be conducted in a private setting by a trained research assistant in the local language (usually Setswana). Focus group discussions and interviews will be audio recorded, transcribed and translated; all study records will be collected using study identification numbers (without personal identifiers), and will be kept locked and accessible only to relevant study staff. Overall results (without identifiers) will be shared with the study team and implementing partners, in an effort to enhance linkage to care and ART initiation.

# 4) Compensation

Participants in FGDs or IDIs will receive 30 Pula to compensate them for their time and up to 30 pula in transport reimbursement to attend the FGD or IDI.

# 6.4. Research Blood Draw Procedures in Combination Prevention Communities, Outside of the BHS

Procedures for the HTC campaigns are detailed in the *Intervention Protocol* and described in brief below. Under that protocol, community residents identified as HIV-infected in Combination Prevention communities will be referred by counselors and linked by Linkage-to-Care Managers (LTCMs) to HIV care and treatment clinics. These patients will be asked to consent to research participation including a blood draw for viral load/HIV genotype/incidence assay testing/optional storage. In addition, all other HIV-infected residents of Combination Prevention communities (including those already in HIV care; those eligible for ART by Government guidelines; and those already on ART) will be invited at the clinic to participate in the research blood draw.

# 1) Recruitment

- Research blood draw eligibility: All HIV-infected adult residents of Combination Prevention communities are eligible for the research blood draw. All eligible adults presenting to the HIV care and treatment clinics will be offered the opportunity to participate in the research, including those already in care (even those on ART). During the study (prior to the ESS), HIV-infected Combination Prevention community residents will be asked/consented to give a sample for genotyping/phylogenetics/transmitted drug resistance. Each consenting participant will be asked a few basic questions (e.g. age, gender, ART status) that will permit interpretation of results even if the participant did not take part in other surveys/questionnaires.
- Sample size: Based on the average population size of the study communities and 25% HIV prevalence, 11,608 HIV-infected individuals are estimated to reside in the 15 Combination

Prevention communities at the time the study starts. These individuals will be invited at local clinics to participate in the research blood draw. The expected number of additional participants in the clinic-based research blood draws following the first year is based on incident cases and therefore expected to be much lower (approximately 326).

• Consent: Eligible research participants will be consented for a venous blood draw at the time of their visit to the clinic that will include a 10mL tube for HIV viral load and a 10ml EDTA tube for HIV genotyping/incidence assay/storage (Research Blood Draw Consent). The participant may elect to receive the program blood draws (for viral loads only) without the research blood draw (blood draw for HIV genotyping/incidence assay/storage), if he/she chooses.

**Blood draw:** Trained staff will draw the relevant blood samples from consenting patients. Patients will receive their viral load result. Results of phylogenetic analysis and other research assays will not be returned to participants or their providers. Genotyping will not be run in real time and therefore will be of limited utility for patient care. However, if results indicate transmitted drug resistance, efforts will be made to avail this information to the participant upon completion of testing.

2) <u>Follow-up and Retention:</u> Program follow-up and retention of HIV-infected patients is described in the *Intervention Protocol*.

# 3) Data Collection and Handling

All research data will be collected electronically on devices such as notebook computers that are encrypted and password protected. Investigators will: (1) securely store original written signed consent pages, (2) record participant granting of consent electronically, and (3) ensure paper copies of informed consent forms are provided to the research participants. Blood samples may have barcodes linked to study IDs applied at the point of sample collection.

#### 4) <u>Compensation</u>

There will be no compensation for participating in the HTC campaign nor for participating in blood/data collection for this research component of the study.

# 6.5. The End of Study Survey (ESS) and Final T2 Study Visit for Previously Enrolled 20% Households

#### 1) ESS Recruitment

- **ESS Community Selection:** 3 pairs of communities (6 communities in total) will be selected to take part in the ESS. Section 5.2.3 details the process for selecting the ESS communities. As noted previously, residents of the 20% households in all 30 communities will undergo final follow-up evaluations at this T2 time as well.
- ESS Household Selection: 100% of households in the 3 pairs of Enhanced Care and Combination Prevention communities (6 total communities) will be targeted for the ESS--the 20% households already participating in the repeat surveys (T2 survey), and the 80% of households not yet approached for participation in the evaluation research. Google maps (and other publicly available sources) will be used to identify eligible households.

 Recruitment: Each of the study community households will be approached for participation in the study. If the heads of eligible households, or a suitable household representative, are not available at the time of the first home visit, up to two re-visits to the household will be scheduled.

**Schedule**: The ESS will be scheduled to coincide with the T2 visit to 20% households.

- 2) The remaining ESS study activities (training; household visit procedures; data collection and handling) will be very similar to those in the BHS, with a few exceptions:
  - Participants will be consenting to a one-time questionnaire and blood draw, and not longitudinal follow-up in any cohort.
  - Participants will be referred to local treatment facilities for HIV care and treatment (if HIV-infected) and male circumcision (if HIV-uninfected), and no linkage to care interventions will be implemented.
  - Non-citizens will be eligible to participate anonymously in this one-time survey.

In sum, the ESS will consist of HTC (if not documented to be HIV-infected); informed consent of eligible residents of the 80% households in the participating 6 communities (or newly-eligible residents of the 20% households in the participating 6 communities), followed by completion of a questionnaire that focuses on combination prevention intervention uptake; and (among consenting HIV-infected residents) collection of a sample for HIV viral load/genotyping/incidence assay/optional storage (see Figure 5A).

Verbal Consent Script for Household Representative Household Structure Survey Approach Eligible HH Members Questionnaire No Documentation of Documentation of HIV-**HIV Status** HIV-positive Status Positive status Finger capillary blood sampling **HIV RT** 10ml EDTA -Genotype -Incidence **HIV POS** HIV IND **HIV NEG** 10ml EDTA Routine post-- VL test counseling 4-5ml EDTA + encourage EIA/WB/PCR If reports No Prior/current ART^ MC uptake among men Run POC CD4 # Results to Participant Referred to HIV Care and **Treatment Clinic** 

Figure 5A. Procedures for the End of Study Survey in 80% Households in 6 Communities

Abbreviations: HH, Household; C, consent procedures; RT, rapid test; VL, viral load; MC male circumcision; IND, indeterminate; EIA, enzyme immuno-assay; WB, Western Blot.

3) T2 visit: procedures during the T2 visit among 20% household residents will be very similar to those in the ESS participants (with the exception that participants who previously consented to taking part in the BHS or HIC will not need to provide additional consent for study procedures). Note that eligible consenting residents of 20% households in the 30 communities who did not previously participate in the BHS/AHS will complete the ESS consent and survey/procedures.



Figure 5B. Procedures for the Final Survey Visit at T2 in 20% BHS/HIC Households

Abbreviations: HH, Household; C, consent procedures; RT, rapid test; VL, viral load; MC male circumcision; IND, indeterminate; EIA, enzyme immuno-assay; WB, Western Blot.

#Verbal consent script need not be re-administered if the respondent is the same person at follow-up visits, or an enrolled survey participant.

<sup>\*</sup>Consent administered to eligible household members only (see section 4.4).

<sup>^</sup>Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5). # Sample for the POC CD4 in previously documented HIV-positive participants may be drawn along with the venous blood for VL, to avoid a separate finger prick. Otherwise, capillary blood sample leftover from rapid HIV test may be used.

<sup>\*</sup>Consent required from newly identified residents who did not enroll and consent previously at BHS or T1. Consent administered to eligible household members only (see section 4.4.4).

<sup>^</sup>Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

<sup>\*\*</sup>HIV-positive participants who were ART-naïve upon enrollment at a prior visit will have POC CD4 repeated at T2, even if they have started ART since enrollment. Generally, the sample for the POC CD4 at T2 in previously documented HIV-positive participants will be drawn along with the venous blood for VL, to avoid a separate finger prick.

# Newly identified HIV-positive participants (i.e. no prior study documentation of HIV-positive status) who are ART-naïve will have POC CD4 run on leftover capillary blood. If a capillary blood sample cannot be obtained, a venous blood sample (4-5 ml) may be drawn instead.



Figure 5C. Procedures for the End of Study Survey for Non-Citizen/Spouse of Citizen Respondents

Abbreviations: HH, Household; C, consent procedures; RT, rapid test; VL, viral load; MC male circumcision; IND, indeterminate; EIA, enzyme immuno-assay; WB, Western Blot.

# Sample for the POC CD4 in previously documented HIV-positive participants may be drawn along with the venous blood for VL, to avoid a separate finger prick. Otherwise, capillary blood sample leftover from rapid HIV test may be used.

\*\*Sample will be collected for confirmatory testing and study staff will arrange for participant to obtain confirmed result. Real-time result will be made available to participant at mobile lab/clinic. Research Blood Draw and Viral Load will be collected simultaneously in the event the confirmed result is positive. Similar to other study participants, anonymous non-citizen participants may obtain their viral load results. Non-citizen participants will be provided with a receipt matching their coded specimen. They may present the receipt to the mobile lab/clinic to obtain their result.

# 7. COST EFFECTIVENESS ANALYSIS

In this section we describe the Cost-Effectiveness of Preventing AIDS Complications International (CEPAC-I) model, the novel data collection, and the analysis plan to determine the cost per HIV infection averted under the intervention and related secondary objectives of estimating cost per quality adjusted life year (QALY) saved under the observed and ideal conditions.

<sup>\*</sup>Waiver of requirement for written documentation of informed consent. Administer Consent Script/Written Statement (see section 11.2).

<sup>^</sup>Leftover sample from either the fingerprick or 10mL sample will be run in a small subset of HIV+ participants not currently on ART to validate POC VL (run in parallel with standard VL) (see Section 8.5).

#### 7.1 CEPAC Model Structure

The CEPAC model is comprised of a CEPAC-I state-transition model of HIV disease progression linked to a dynamic CEPAC model of HIV transmissions.

### 1) CEPAC-I state transition model

CEPAC-I, as a *state-transition* model characterizes disease progression as a sequence of monthly transitions from one "health state" to another as depicted in the following diagram: chronic, acute, and death (Kreke, Schaefer et al. 2004; Walensky, Wood et al. 2008).



Health states are defined by current and setpoint HIV RNA, current and nadir CD4 count, and history of opportunistic infections (OIs). OIs are divided into groups based on country-specific data and are classified as severe or mild. From each health state in each month, individuals face competing mortality risks from non-HIV causes. The efficacy of sequential ART regimens is characterized by their impact on HIV RNA and CD4 count (Cole, Hernan et al. 2003; Losina, Yazdanpanah et al. 2007). A random number generator and set of estimated probabilities determine the clinical pathway that a patient follows until death. The entry characteristics of simulated patients (age, sex, CD4 count, HIV RNA) are randomly drawn from a distribution based on data from the setting of interest. A tally of clinical events, time spent in each health state, and cost associated with each health state is maintained. Upon the patient's death, summary statistics for that person are recorded. Results from large numbers of individual simulations are averaged to develop stable population estimates. Simulation sizes of 1 million patients are typically sufficient for treatment strategies.

### 2) CEPAC HIV dynamic model

We have completed a pilot transmission model incorporated into CEPAC-I (Walensky, Ross et al. 2012) and are developing a full agent-based, dynamic transmission model of the HIV epidemic linked to the CEPAC-I Model. This transmission model will be incorporated into this analysis to estimate the additional potential population-wide impact of HIV treatment interventions on incidence. While several dynamic transmission models have been published (Alam, Meyer et al. 2009; Leclerc, Matthews et al. 2009; Bendavid, Brandeau et al. 2010; Enns and Brandeau 2011; Gray, Ghaus et al. 2011; Hallett, Baeten et al. 2011; Phillips, Pillay et al. 2011; Prabhu, Farnham et al. 2011; Schneider, Puthanakit et al. 2011; Bershteyn, Klein et al. 2012; Ventelou, Arrighi et al. 2012), the CEPAC Dynamic Model combines behavioral, demographic, and biological parameters to project HIV transmission from and to individuals on a population level and links to the clinical detail of CEPAC-I (natural history, treatment outcomes, and costs of care). Outcomes include incidence and prevalence over user-defined time periods. Using a fitting procedure based on Bayesian melding methods (Poole and Raftery 2000; Alkema, Raftery et al. 2008; Johnson, Alkema et al. 2010), we have fit the model to HIV prevalence in South Africa

from 1990-2002 prior to the introduction of ART, and are currently fitting it to 2003-2012 in the presence of ART (Joint United Nations Programme on HIV/AIDS (UNAIDS) 2010).

# 7.2 Data Inputs

#### 1) Natural History

We have derived CD4-stratified model input parameters from Côte d'Ivoire and South Africa to describe the natural history of HIV in sub-Saharan Africa (Holmes, Wood et al. 2006; Losina, Anglaret et al. 2006; Wang, Kumarasamy et al. 2006). Natural history data from South Africa are primarily from the Cape Town AIDS Cohort (CTAC), a cohort of 2,088 patients followed by Wood et al. (Holmes, Wood et al. 2006). These model parameters will be compared with observed CD4 trajectories and clinical outcomes in the Baseline Household Survey to confirm that the model accurately describes the experience of the Botswana population.

# 2) ART Efficacy

Efficacy data for 1<sup>st</sup>-line NNRTI- or PI-based regimens (66-88% viral suppression at 48 weeks) are from both clinical trials and observational cohorts in Africa with similar efficacy for 2<sup>nd</sup>-line regimens (Coetzee, Hildebrand et al. 2004; Nachega, Stein et al. 2004; DART Virology Group and Trial Team 2006; Charalambous, Innes et al. 2007; Barth, van der Meer et al. 2008; Boulle, Van Cutsem et al. 2008; Delfraissy, Flandre et al. 2008; Hammond and Harry 2008; Losina, Chang et al. 2008; Wouters, Van Damme et al. 2008; Bierman, van Agtmael et al. 2009; Gandhi, Moll et al. 2009; Fox, Ive et al. 2010). CD4 increase on 1<sup>st</sup>-line ART averages 113-236 cells/μl at 48 weeks, with the sharpest increase occuring in the first two months, followed by a more gradual increase (Charalambous, Innes et al. 2007; Seyler, Adje-Toure et al. 2007; Barth, van der Meer et al. 2008; Hammond and Harry 2008; Pujades-Rodriguez, O'Brien et al. 2008; Wouters, Van Damme et al. 2008; Gandhi, Moll et al. 2009; Fox, Ive et al. 2010). While data from clinical trials are more complete in terms of virologic and CD4 response, as well as loss to follow up (LTFU) and toxicity, they generally provide higher estimates of suppression than data from large community cohorts (DART Virology Group and Trial Team 2006; Delfraissy, Flandre et al. 2008; Hammond and Harry 2008). We will therefore use data from trials to represent primarily bestcase scenarios in terms of efficacy and LTFU (Cohen, Chen et al. 2011; Anglaret and Eholié 2012; Grinsztejn and Mugyenyi 2012) and cohorts (Cornell, Schomaker et al. 2012; Wandeler, Keiser et al. 2012) for more likely generalizable programmatic outcomes. Efficacy and effectiveness data will be updated as studies emerge with data from newer regimens (1<sup>st</sup>-, 2<sup>nd</sup>-, and 3<sup>rd</sup>- line) as treatment provision, regimens, and experience matures (Pujades-Rodriguez, O'Brien et al. 2008; Fox, Ive et al. 2010; Saravanan, Madhavan et al. 2012). We will assess both trial- and cohort-reported efficacies to assess how differences may change policy conclusions.

# 3) <u>Costs</u>

We will fully update the cost parameters for direct medical care in the CEPAC-I model. We will carry out a facility-based costing study in Botswana using an 'ingredients-based' methodology (UNAIDS 2011) that leverages longitudinal utilization records over a retrospective two-year period in several of the community clinics. This will allow us to quantify utilization of services for routine care, OI treatment, treatment of HIV-related co-morbidities, and end-of-life care (see Table 8).

We will use facility-based staffing records, inventories, procurement and accounting records, and other site-specific data to generate a unit cost per outpatient visit, per inpatient day, per procedure, per laboratory test, and per monthly medication cost. To determine the total unit cost for each service we will define each facility's service centers and measure their output, for example an inpatient day. We will then define and measure the input required by the service center in terms of capital resources (buildings, equipment and other one-off costs such as consultant fees) and recurrent resources (staff salaries, consumables and monthly costs such as electricity bills). Once we have determined the total input we will calculate the monetary value of each item to establish the current financial price and to calculate the unit cost of each service center output. Through this UNAIDS-recommended (UNAIDS 2011) costing methodology we will reflect the most current utilization patterns and unit costs, and will tailor HIV care recommendations to Botswana cost structures. All costs will be updated to constant year dollars and discounted at 3%/year (Gold, Siegel et al. 1996).

**Table 8. Resource Utilization and Cost Data Needs** 

| Parameter | Stratified by |
|---|---|
| Start-up costs | Intervention, Site, Monthly for first 3 months |
| Scale-up costs | Incremental cost of increasing coverage levels by 10% increments; Quarterly |
| Personnel costs | FTEs for all hired staff per implemented intervention* Salaries for each staff member |
| Medications | 1 <sup>st</sup> and 2 <sup>nd</sup> line ART<br>Cotrimoxazole<br>OI treatment |
| Patient visits to healthcare setting | Average frequency on ART Average frequency by CD4 stratum (off ART) Urgent care visits (by ART status) Hospitalizations and length of stay (by ART status and with diagnosis) Death costs Costs by visit type † |
| Laboratory‡ | HIV test, Confirmatory HIV test, CD4 monitoring, HIV-1 RNA, Screening chemistries, Screening CBCs |

<sup>\*</sup> Including but not limited to: home visits, nurses, care and treatment, doctors for ART, surgical sMC

The measurements of healthcare utilization and personal health care costs are included in the questionnaire to be used at T1 (Resident Survey, Annual) and during the ESS (Resident Survey, ESS). These supplementary items will be requested from at least 1,500 participants drawn from both Enhanced Care and Combination Prevention communities at T1 and T2.

In order to more accurately estimate changes in health resource utilization during periods of illness and during periods with low CD4 cell count (CD4200 cells/ $\mu$ L), supplementary sampling of individuals in clinics and hospitals serving study communities will be conducted. Up to 150

<sup>†</sup> Urgent care, per diem hospital stay, routine visit

<sup>‡</sup> Includes anticipated frequencies and associated costs

consenting participants experiencing opportunistic illnesses and 300 without opportunistic illness but with low CD4 counts will be recruited from outpatient and inpatient settings.

Possible participants will be approached in three settings. First, individuals participating in the 20% household surveys with low CD4 count or current opportunistic illness will be identified and selected for completion of these supplemental items. Second, qualifying individuals receiving care in the Combination Prevention community clinics will be identified and referred for possible participation in these questionnaires. Finally, if these settings are inadequate to achieve the target sample size, other patients seeking care in clinics or inpatient facilities serving study communities will be identified through review of care logs and conversations with clinical staff. Participants recruited from the clinics, and those not previously part of a study cohort, will be required to provide written informed consent prior to completion of these questionnaires (Economic Consent). Consenting participants will be interviewed for health resource utilization and quality of life (Economic Assessment).

Health care costs frequently are concentrated at the end of life and these costs may be missed during community surveys and during a focused clinical survey described above. Consequently, we will abstract health resource utilization during the 30 days before death from existing medical records in up to 80 residents of study communities (40 HIV-infected, 40 HIV-uninfected) who die during the course of the study (Death Economic Abstraction). Of these, 20 non-accidental deaths that occur outside of the hospital will be targeted as costs associated with these deaths are anticipated to be different. Study teams will learn of deaths of community residents from the community clinic staff, and from review of inpatient care logs for facilities providing care for study communities. Family members or contacts of the decedent will not be interviewed. No identifiable information will be recorded during record abstraction. This aspect of the research does not involve human subjects per the definition at 45CFR46.102(f) that a human subject is a *living* individual.

Table 9. Individual Healthcare Utilization, Cost, and Quality of Life Assessments

| Instruments | Sample Size | Timing | Recruitment |
|---|---|---|---|
| Annual Resident Survey and End of | At least 3,000 (at least 1,500 at | T1 and T2 | Participants in BHS/AHS |
| Study Survey. These instruments | each time point) | | |
| include EQ5D5L, resource utilization | | | |
| (including HIV-related costs for HIV- | | | |
| infected), lost economic activity | | | |
| Economic Assessment: EQ5D5L, | 150 with opportunistic illness | Throughout study | 1) Participants in |
| resource utilization (including HIV- | | | BHS/ESS |
| related costs for HIV-infected), lost | 300 with low CD4 ≤200 cells/μL | | 2) Participants in IDCC |
| economic activity | without opportunistic | | 3) Other patients |
| | illnesses | | treated in facilities |
| CEA Enrollment checklist for | | | caring for residents |
| participants outside BHS/ESS | | | of study |
| | | | communities |
| Death Economic Abstraction: Resource | 80 | Throughout study | Clinics and hospitals |
| utilization | | | caring for residents |
| | | | of study |
| | | | communities |

# 4) Quality of Life

Quality of life implications of HIV treatment in resource-limited settings are becoming more important in the evaluation of innovations that incrementally improve clinical management of HIV than a decade ago, when survival gains were appropriately the overriding concern. To enable the CEPAC-I model to estimate QALYs as an outcome, we will synthesize existing evidence on preference-based measures of QOL (EuroQol Group 1990; World Health Organization Division of Mental Health and Prevention of Substance Abuse 1997; Brazier, Usherwood et al. 1998; Brazier, Roberts et al. 2002; Sullivan, Lawrence et al. 2005) for HIV health states from the literature (Jelsma, Maclean et al. 2005; Louwagie, Bachmann et al. 2007; Zimpel and Fleck 2007; Lara, Wakholi et al. 2008; Robberstad and Olsen 2010; Rajeev, Yuvaraj et al. 2012; Tran, Ohinmaa et al. 2012). The largest study to date of QALY-weights in HIV used the EQ5D instrument in a trial involving 21,000 US patients and has been used in model-based analyses (Simpson, Luo et al. 2004; Pitter, Kahn et al. 2007; Meyer-Rath and Over 2012). To produce estimates that can be adapted to the CEPAC-I model structure, we will adjust the QALY-weights as needed by collecting EQ5D data at T1 and T2 and use new methods for synthesizing evidence on QALYs (Tengs and Lin 2002; Isogai, Rueda et al. 2012) and predicting health-related QOL among HIV-infected persons (Isogai, Rueda et al. 2012).

The EQ5D is included in the questionnaire instrument used at T1 (Resident Survey, Annual) and at T2 to estimate QOL in the study communities. Supplementary sampling of individuals with opportunistic infections and low CD4 will be conducted. The EQ5D will be administered to up to 150 consenting individuals with opportunistic illnesses and 300 individuals with CD4<200 cells/ $\mu$ L receiving care in inpatient and outpatient facilities serving study communities (Economic Assessment), as described above for medical cost estimation.

# 7.3 Model validation and approach to uncertainty

Medical decisions and guidelines for care are nearly always formulated without perfect information. This is particularly true with rapid advances in knowledge and, thus, justifies both the use of model-based approaches and an inclusive attitude toward the data used in modeling studies. Because hypotheses cannot be tested using traditional measures of statistical significance in microsimulation modeling, we have a particular responsibility to both validate models and to investigate the impact of uncertainty with care and transparency. Here we describe approaches to model validation and sensitivity analysis.

# 1) Validation

We ascertain internal consistency in the model in several steps: First, we examine the face validity of randomly selected, individual patient "traces" (Figure 5). These detailed views of a patient's month-to-month experience offer a check on the reasonableness of the output and a mechanism for debugging. Second, we check "internal validity," verifying that model output accurately approximates the data used to derive input parameters. This is an area of increasing importance in disease policy modeling. Figure 6 illustrates the validation of model runs using HPTN 052 trial data inputs with trial outcomes (Losina, Yazdanpanah et al. 2007; Walensky, Ross et al. 2012).





Figure 5: A simulated patient trace from South Africa

Figure 6: CD4 Trajectory in the CEPAC-I model as compared to the HPTN-052 trial

#### 2) Deterministic sensitivity analysis

The US Panel on Cost-Effectiveness in Health and Medicine and the International Society for Pharmacoeconomics and Outcomes Research (ISPOR) Task Force on Good Modeling Practice both recommend deterministic sensitivity analysis to provide insight about uncertainty where small changes in model input data produce large changes in model results (Weinstein, Siegel et al. 1996; Paltiel 2001; Drummond, Brown et al. 2003; Weinstein, O'Brien et al. 2003; Ades, Claxton et al. 2006; Briggs, Weinstein et al. 2012). We will use deterministic methods (one-way, multi-way, best-case, worst-case, and threshold approaches) to assess how uncertainty in current data or lack of data about treatments still in development may affect policy conclusions, or when application of data from alternative regions or countries yields different results (Gold, Siegel et al. 1996; Paltiel 2001; Uhler, Kumarasamy et al. 2010).

<u>Probabilistic approaches.</u> In contrast to deterministic sensitivity analyses, probabilistic sensitivity analysis (PSA) generates values for multiple inputs simultaneously based on predefined probability distributions for each input. PSA is recommended under guidelines elaborated by the ISPOR-Medical Decision Making Task Force (Society for Medical Decision Making and International Society for Pharmacoeconomics and Outcomes Research; Briggs, Weinstein et al. 2012). We have developed the capacity to conduct PSA on output from the CEPAC-I model. Parameters of interest will be chosen based on importance to the results (as identified by deterministic sensitivity analyses described above) and also on whether data are available to specify distributions (Ades, Claxton et al. 2006). We will use these analyses to calculate the expected cost-effectiveness of each prevention strategy, the uncertainty surrounding that result, and the number of times each strategy is optimal.

#### 7.4 Cost-Effectiveness Analysis Plan

The CEPAC International model will be used to assess expected outcomes from the proposed combination prevention programs. Table 10 shows the prevention strategies and outcomes of interest that will be examined; the main outcome of interest will be the comparison of the three strategies to each other. An additional "no regular screen, no ART" strategy will be modeled for historical comparison only. In addition to life expectancy, cost, and cost-effectiveness of alternative HIV combination prevention strategies, the impact of these strategies on secondary transmission and HIV incidence will also be examined by estimating the number of secondary cases per infected individual in

each combination prevention scenario. Results will be stratified showing life expectancy for the entire population, life expectancy for only the HIV-infected residents, and the number of new HIV infections averted. Table 8 shows resource utilization and cost data needs.

**Table 10. Prevention Strategies and Outcomes of Interest** 

| Prevention strategy | Outcomes of interest |
|---|---|
| Enhanced Care communities (Current Standard of Care) | |
| Combination Prevention communities (expanded HTC, MC, PMTCT, and universal testing and treatment) | Total population QALYs Mortality at 2 years Number of new HIV infections at 2 years Reduction in HIV incidence |
| "Optimized Package" (model-based scenario based on the Combination Prevention arm, but will assess the case where linkage to routine HIV care is ideal, ART is optimized, HIV screening is more frequent, and pre-exposure prophylaxis is administered) | Per person total direct costs Cost-effectiveness (\$/HIV infection averted) Cost-effectiveness (\$/YLS*, \$/QALY) |

<sup>\*</sup>year of life saved: YLS

Incremental cost-effectiveness ratios – both dollars per year of life saved (\$/YLS or \$/QALY), and dollars per HIV infection averted (\$/infection averted) – will be used to assess the comparative value of these alternative combination HIV prevention strategies. The incremental cost-effectiveness ratios will be determined by ranking strategies in order of increasing cost. Incremental cost-effectiveness is defined as  $\Delta C/\Delta E$ , where  $\Delta C$  is the difference in costs between two rank-ordered strategies, and  $\Delta E$  is the difference in effectiveness, as defined either by life expectancy (when calculating \$/YLS or \$/QALY) or number of new HIV infections (when calculating \$/infection averted). Before assessing the incremental costs and benefits of increasingly expensive strategies, we will eliminate strategies that are less effective and more costly. Analyses will be conducted from the modified societal perspective (not including time and productivity costs), and discounted at 3% per annum. Additional analyses will be done to include time and productivity costs, with data derived from external sources and consistent with other combination prevention trials.

# 8. LABORATORY METHODS

Detailed laboratory procedures, including procedural guides during actual specimen and data collection and study-specific SOPs are described in the BCPP Manual and outlined in brief below.

# 8.1. Overview of Laboratory Methods

An overview of the types of laboratory tests, sample types, and the location of the testing is provided below. The study will use the following laboratories and locations:

- 1. BHHRL: Botswana Harvard HIV Reference Laboratory (Gaborone)
- 2. NHHRL: MOH regional HIV Reference Lab (Francistown)
- 3. MOH Local Program Labs (Botswana, multi-sites)

- 4. Field sites: Households and community venues conducting surveys and HTC campaigns
- 5. Harvard Chan: Harvard T.H. Chan School of Public Health (Boston)
- 6. CDC: International Laboratory Branch at Centers for Disease Control and Prevention (Atlanta)

**Table 11: BCPP Evaluation Protocol Laboratory Testing Responsibilities:** 

| Test | Location of Testing* |
|---|---|
| HIV Rapid Tests | Field Sites |
| CD4 | MOH Local Program Lab and Field Sites (POC) |
| HIV-1 RNA Viral Load | BHHRL/NHHRL |
| Laboratory-based incidence assays | BHHRL |
| Viral linkage | Harvard Chan/BHHRL or collaborators |
| Minor drug-resistant variant genotyping | Harvard Chan/BHHRL or collaborators |
| QA/QC Procedures | BHHRL and NHHRL |
| Tandem mass spectrometry/HPLC | Harvard Chan/BHHRL or collaborators |
| Point of care viral load | Field sites |

<sup>\*</sup>Collaborating institutions may participate in testing activities if requested by the responsible institution listed above.

# 8.2. Training of Laboratory Personnel

All laboratory personnel will participate in study-specific training prior to study initiation. Training will include an overview of the BCPP study design and study-specific laboratory methodologies in addition to Research Ethics, GCLP (Good Clinical and Laboratory Practice), QA/QC (quality assurance/quality control), and laboratory record keeping procedures. Study staff responsible for providing HIV testing and counseling will complete the required training curriculum recognized by the MOH. Staff will also be trained on the use and completion of all study forms related to these services. Study staff members who will collect blood samples or conduct laboratory analyses will receive training in universal precautions, sample collection, and testing of study samples. Additional refresher trainings will be scheduled during the study to ensure consistency and address training needs as they arise.

#### 8.3. Specimen Collection, Transport, and Processing

Specimens will be collected from participants at study field sites and samples transported to designated laboratories for processing, testing and storage. Testing may also occur at study field sites.

#### Sample types:

a) <u>Capillary blood samples</u>: Finger prick samples will be collected in a microtube using a sterile disposable lancet, by trained staff at study field sites according to the appropriate blood collection SOP and used for the HIV rapid test, POC CD4 test, and (in a subset), POC viral load test.

- b) <u>Venous blood samples</u>: Samples will be collected by trained phlebotomists according to policies and procedures described in a SOP for blood collection. The number and types of samples will vary by the study group as described in Section 6. Tube sizes have been standardized to streamline collection of specimen in the field and integration into existing laboratory testing sites. Samples will be labeled with participant ID/barcodes and transported using coolers or portable refrigerators to the designated research laboratory, processed within 24 hours, and aliquots at -70°C. In brief, the following specimen sizes will be used:
  - 4-5 ml EDTA tube or 10ml EDTA tube: Viral Load
  - 10 ml EDTA tube: Genotyping, TDR, incidence assays

In cases in which sample for POC CD4 is obtained from venous blood (rather than lancet fingerstick)--e.g. among ART-naive patients with documented HIV infection in whom a rapid test is not being performed—an additional 4-5 ml EDTA tube will be collected.

Note: consenting pre-ART participants may also have blood drawn for baseline safety labs as part of the "research blood draw" in Combination Prevention communities, to avoid multiple sticks and to help expedite time to treatment initiation. More detailed procedures related to this phlebotomy are described in the *Intervention Protocol*.

c) <u>Plasma and buffy coats:</u> Plasma and buffy coats will be collected from whole blood specimens (EDTA tube) by centrifugation (1,500 x g or ~3,000 rpm for 10 min), then aspirate plasma into 1 ml aliquots, followed by aspirate of buffy coat into 1 ml aliquots. Both plasma and buffy coats will be stored frozen (-70°C).

#### 8.4. Laboratory testing for BHS, HIC, and ESS (returned to participant and/or participant file)

a) <u>HIV Diagnostic Testing:</u> HIV diagnostic testing will be conducted by the study sites as per National HIV Testing guidelines using Botswana-government—approved parallel rapid tests. The current algorithm includes KHB and Unigold™ HIV rapid test in parallel. If results are discordant, a 4-5 ml blood specimen will be taken at the visit and sent to a reference laboratory for further testing using ELISA or Nucleic Acid testing per BHHRL HIV testing algorithm (e.g. Murex HIV 1.2.0 test, Genetic Systems Biorad HIV-1/2) and/or Western blot and/or DNA/RNA PCR. The results of EIA and/or Western Blot and/or DNA/RNA PCR at the BHHRL lab will supersede the discordant and/or indeterminate results obtained in the field. All HIV tests will be conducted according to the manufacturer's guidelines.

If results of anonymous HIV diagnostic testing in the household are discordant, the confirmatory HIV testing will be performed at the mobile lab in real-time. The Cepheid Xpert POC HIV-1 Qual will be used according to the manufacturer's instruction. Xpert HIV-1 Qual provides a total nucleic acid based test for viral RNA and proviral DNA in one integrated cartridge by using 100 ul of whole blood. If the result of Xpert HIV-1 Qual test is negative, the person is considered to be HIV-negative. If result of Xpert HIV-1 Qual test is positive, the person is considered to be HIV-positive.

- b) <u>POC CD4</u>: Capillary blood samples (obtained from the lancet fingerprick blood draw also used for the HIV rapid test) will be tested using the Pima™ CD4 with the Pima analyzer (Alere, Inc.) described previously (Mtapuri-Zinyowera, Chideme et al. 2010; Jani, Sitoe et al. 2011) to obtain an absolute count of CD4 cells.
- c) <u>HIV-1 Viral Load:</u> Testing will be conducted by NHHRL at Francistown and BHHRL at Gaborone using licensed assays. HIV-1 RNA VL in plasma will be performed by Roche TaqMan Assay using the Roche COBAS AmpliPrep/COBAS TaqMan version 2 HIV-1 Test or Abbott m2000sp/m2000rt. The BioMeriuex platforms are also available in the reference or national laboratories and may be used for viral load testing. All results will be made available to be keyed or electronically transfered to the protocol database after appropriate user validation.

Several POC VL devices are currently undergoing field performance characteristic evaluations [ALERE HIV NAT POC system (Alere, Inc.), Cepheid Xpert POC VL]. The potential future use of the POC VL tests through an amendment to the BCPP *Evaluation Protocol* may be considered depending on successful evaluation of the POC VL device. POC VL using best available devices will be conducted on a subset of treatment-naïve individuals and may also be conducted on individuals receiving ART.

d) <u>Transmitted Drug Resistance:</u> Efforts will be made to return results indicating transmitted drug resistance to participants upon completion of testing. Note that these results will only be available retrospectively (e.g. about 1 year or later after sampling), and may therefore be of limited clinical utility.

# 8.5. Research laboratory testing (results not returned to participant)

# a) Viral Genotyping

Plasma and buffy coats will be the primary sample source for viral genotyping. The algorithm of viral genotyping based on the V1C5 region of HIV-1 *env* gp120 and HIV-1 *gag* are in place in the Harvard Chan lab (Novitsky, Lagakos et al. 2009; Novitsky, Wang et al. 2009; Novitsky, Wang et al. 2010; Novitsky, Wang et al. 2011). A newly developed technique of long-range HIV genotyping (Novitsky, Zahralban-Steele et al. 2015) will be also applied, as it provides better resolution of HIV transmission clusters (Novitsky, Moyo et al. 2015).

- Details of sample processing, amplification, sequencing and troubleshooting are summarized in (Novitsky, Zahralban-Steele et al. 2015).
- The "gray zone" samples will be resolved by applying more sensitive methods such as Single Genome Amplification and Sequencing and 454-based next generation "deep sequencing."

The viral linkage analysis includes all generated viral sequences. QA/QC procedures will be applied routinely.

Cluster analysis using generated viral sequences from each participating community will be performed as described recently (Novitsky, Bussmann et al. 2013; Novitsky, Moyo et al. 2014; Novitsky, Kuhnert et al. 2015). Potential links and clustering will be analyzed for all available

prevalent and incident HIV infections. The optimal evolutionary model will be identified for the aligned set of query sequences using jModelTest (Posada 2008).

HIV clusters will be identified by a combination of bootstrapped ML (Felsenstein 1985; Nei and Kumar 2000; Felsenstein 2004) and internode certainty (Salichos and Rokas 2013; Salichos, Stamatakis et al. 2014). The ML phylogeny will be inferred in RAxML (Stamatakis 2006; Stamatakis 2014) under the GAMMA model of rate heterogeneity. To account for phylogenetic uncertainty, from 100 to 1,000 bootstrap trees will be inferred using the rapid bootstrap in RAxML (Stamatakis 2006). The bootstrap threshold will be set to 0.80, and we will perform the sensitivity analysis at 0.70 and 0.90. We will use 0.70 as the internode certainty threshold (Salichos and Rokas 2013; Salichos, Stamatakis et al. 2014).

To estimate effective reproductive number R, HIV transmission rate  $\lambda$ , and the rate of becoming non-infectious  $\delta$  for the identified HIV lineages, we will use the BDSKY model in BEAST2 (Bouckaert, Heled et al. 2014; Novitsky, Kuhnert et al. 2015). The chain length of Markov Chain Monte Carlo runs will be set to  $2x10^8-3x10^8$  with the first 25% of states of each run burned-in. The generated trees will be sampled to estimate effective reproductive number, R, HIV transmission rate,  $\lambda$ , rate of becoming non-infectious,  $\delta$ , effective population size,  $N_e$ , and the tMRCA. Convergence will be evaluated by Tracer v1.5 (http://beast.bio.ed.ac.uk/Tracer) and effective sample sizes of >200.

Transmitted drug resistance will be analyzed using samples from new incident cases and samples identified as recent HIV infections using laboratory-based incidence assays (see below). Up to 200 samples will be analyzed annually. Identified incident cases will be prioritized for inclusion into TDR analysis.

Viral mutations associated with HIV drug-resistance will be analyzed in bulk using plasma and buffy coat specimens (Novitsky, Zahralban-Steele et al. 2015). Analysis of viral mutations associated with HIV drug-resistance will be performed at the BHHRL lab using the IAS recommendations for ART-experienced patients (Johnson, Calvez et al. 2011) and WHO-recommendations (Bennett, Camacho et al. 2009). Drug resistance testing at BHHRL will use the validated resistance testing assay developed at International Laboratory Branch, CDC, USA (Zhou, Wagar et al. 2011), or an alternative assay (Wallis, Papathanasopoulos et al. 2010). In addition, more sensitive methods such as next-generation sequencing and allele-specific PCR will be used for analysis of HIV-1 drug-resistant mutations at low frequency in a subset of samples at investigators discretion and this testing will be conducted at a Harvard Chan School lab.

# b) Laboratory-based tests for HIV Incidence

Results of cross-sectional HIV incidence testing obtained at the BHHRL will be compared with the longitudinal HIV incidence data. The study may also compare HIV incidence estimates derived from multi-assay algorithms including available laboratory and clinical data. HIV incidence tests and algorithms will be validated for accuracy and scale-up.

HIV seropositive specimens will be tested using the LAg-Avidity assay in combination with additional information on antiretroviral treatment exposure (ART status) and HIV-1 RNA viral load for incidence estimate as described below. Contemporary methods for estimating incidence may be used as well, or instead, as these methods evolve.

LAq-Avidity EIA: The LAg-Avidity EIA is a CDC-developed new incidence assay (Duong, Qiu et al. 2012; Duong, Kassanjee et al. 2015) now commercially available from Sedia BioSciences (Portland, OR). The LAg-Avidity assay uses a multi-subtype recombinant protein that covers the immunodominant region (IDR) of gp41 of HIV-1, group M, rIDR-M. Briefly, microwell plates are coated with limiting concentration of rIDR-M antigen. Limiting the antigen allows binding of only high-avidity antibodies which are further dissociated by a pH 3.0 buffer step. ODn values are calculated for each specimen using a pre-defined calibrator specimen (CAL) tested on the same plate as follows: ODn = specimen OD/Median CAL OD. Specimens with an ODn value less than or equal to 2.0 during initial testing are confirmed by further testing of the sample in triplicate, where the median value of the three results is considered the final ODn for the specimen. All specimens with ODn values greater than 1.5 are classified as long-term infections. The HIV-1 sero-positive status of specimens with ODn values of <0.4 is confirmed with EIA, as any HIV-negative samples would incorrectly score as recent in the assay. Any HIV seronegative specimens identified at this step are excluded from the total HIV positives and incorporated into the total number of negative specimens (N) for the incidence estimation. Recent (ODn<1.5) infections are likely to have seroconverted within a mean duration of recency of 130 days (Rehle, Johnson et al. 2015).

ART status is collected routinely during the household surveys. Individuals who can provide evidence of being on ART during the household survey are considered long-term, not recent, cases of HIV infection for the purposes of cross-sectional estimates of HIV incidence. To rule out false recent infections, specimens with ODn in LAg-Avidity assay below 1.5 may be tested for the presence of ARV drugs, including but not limited to Tenofovir, Emtricitabine, Zidovudine, Nevirapine, Efavirenz, Lopinavir, Atazanavir and Darunavir by High Performance Liquid Chromatography (HPLC) coupled to Tandem Mass Spectrometry (Rehle, Johnson et al. 2015). Specimens with detectable traces of ARV drugs are considered long-term cases. Testing for the presence of ARVs is an evolving field and other methods will be considered and possibly used as they become available locally and regionally.

HIV-1-positive specimens from ART-naïve individuals with an ODn value less than or equal to 1.5 will be subjected to HIV-1 viral load (VL) analysis as an indirect indicator of ART usage or a natural ability to control HIV infection (elite controllers). Specimens with a LAg ODn ≤1.5 from ART-naïve individuals and a VL ≥400 copies/mL will be classified as recent infections. Results from the LAg-Avidity testing, including ART status and VL testing, will be maintained in a computer-based data management file. Therefore, a separate false recent rate (FRR) correction is not relevant or necessary, and will be set to zero (Rehle, Johnson et al. 2015). The use of multi-assay algorithms (see below) continues to provide evidence that use of additional data or assays improves accuracy of HIV recency testing.

#### • Multi-assay algorithms:

Other algorithms for cross-sectional estimation of HIV incidence may include a combination of BED-capture EIA, Avidity assay (AxSYM or BioRad), (Braunstein, Nash et al. 2011; Laeyendecker, Brookmeyer et al. 2012) and/or multi-assay algorithms that include a combination of BED and Avidity assays and accompanied by CD4 and VL data. These algorithms will be used in a subset of samples for validation and comparison with the data generated previously in the country and/or with other studies.

Incidence calculations are assay- and algorithm-specific. Methods for calculating estimated incidence are described in section 10.

# c ) POC viral load assay

A pilot study of POC viral load testing will be performed to permit assessment of accuracy of POC viral load vs. standard viral load assays as well as assessment of operating characteristics of POC viral load assay(s). The first component will include POC viral load testing in the mobile lab settings by XPERT HIV-1 Viral Load from Cepheid. The second component will include POC viral load testing in households. Both components of POC viral load testing will be accompanied by HIV-1 RNA testing in the Botswana-Harvard HIV Reference Lab (BHHRL) using standard protocol. Currently, we are awaiting a viable potential candidate to be used in the pilot study in the second component. Each component of POC viral load testing will use only one POC viral load platform (and it is possible that both components will use the same POC viral load platform).

Mobile lab POC viral load testing procedures: The same blood sample that is already drawn for standard viral load testing by phlebotomy in households (and processed in the mobile lab placed in each participating community) will be used for POC viral load testing. Approximately 200 POC viral load tests will be performed in mobile labs in real-time (the same day) using whole blood and plasma from this blood draw. Results of POC viral load testing from this pilot study will not be returned to participants, as the platform will not yet have been validated; results of the standard viral load assay will be returned to the local clinic. The same plasma sample tested in the mobile lab will also be tested at BHHRL in Gaborone using standard procedures. The targeted population for this portion of the pilot will be approximately 200 (but up to 400) ART-naïve HIV-infected individuals. The range in sample size is necessary because investigators do not know the precise viral load distribution of participants and we need to ensure that 1/3 of the participants have a viral load below the threshold of 10,000 copies/ml to allow for assessment of the performance of POC viral load tests at lower viral loads.

POC viral load testing in households procedures: Blood for POC viral load testing will be collected according to the manufacturer's instructions in households. Approximately 200 POC viral load tests will be performed in households in real-time using these blood samples. Results of POC viral load testing from this pilot study will not be returned to participants, as the platform will not yet have been validated; results of the standard viral load assay will be returned to the local clinic. A parallel sample drawn in the household will be tested in BHHRL in Gaborone using standard procedures. The targeted population for this portion of the pilot will be approximately 200 (but up to 400) ART-naïve HIV-infected individuals. The range in sample size is necessary because investigators do not know the precise viral load distribution of participants and we need to ensure that 1/3 of the participants have a viral load below the threshold of 10,000 copies/ml to allow for assessment of the performance of POC viral load tests at lower viral loads.

If high concordance is observed between POC viral load assays and standard viral load assays, POC viral load may be used in lieu of standard viral load assays, among pre-ART BHS participants, as noted previously in Section 8.4c). If this is done, then viral load results will be shared with clinics.

Operational characteristics will be evaluated in both components. We will record the time it takes to obtain viral load result in each test, reported ease of use by field operators, and stability under different conditions.

# 8.6. Quality Assurance

A quality management plan with monitoring and evaluation of key indicators will be implemented at the BHHRL and NHHRL. Standard operating procedures (SOPs) will be used for all tests as well as QA/QC procedures. Laboratory staff conducting testing will participate in proficiency testing and 5% of all tests will be subjected to internal QC processes. The QA/QC plan will include periodic monthly reviews of EQA performance and corrective actions implemented. Procedures will be in place for performing and documenting the quality of a specimen, including storage and transport conditions, monitoring of equipment and temperatures, and function indicators. The QA/QC plan will include routine collaboration with the CDC laboratories, enrollment in appropriate EQA schemes, and interlaboratory comparisons. Field sites will participate in EQA and proficiency testing for all POC assays used.

Certification status for laboratory tests will be maintained including: HIV ELISA, POC HIV Rapid EIA, POC CD4 count, and HIV-1 RNA load. Laboratories will be monitored throughout the study by the study team and external monitors as requested by the study sponsor.

# 8.7. Biosafety and Waste Management

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate blood and secretion precautions will be employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the CDC. All infectious specimens will be transported in accordance with the IATA (International Air Transport Association) guidelines using designated courier services.

#### 8.8. Specimen Storage and Shipment

Specimens will be stored until all protocol-related and quality assurance testing have been completed. In addition, study participants will be asked to provide written informed consent for long term storage and potential future testing of their specimens. Specimens without consent for long-term storage and additional testing will be discarded at the end of the study and destruction documented in the study files. Future human subjects research on stored specimens will require submission and approval of a separate study protocol to all engaged IRBs and appropriate study team committee.

The study site will coordinate shipment of specimens as required. Samples (buffy coats, plasma, and/or isolated nucleic acid) for research components of viral genotyping will be shipped to a Harvard Chan School lab in Boston, MA. Selected samples may be transferred to the CDC Laboratories and HPTN Central Laboratory for cross-studies analyses. Other specimens will be stored at BHHRL.

#### 9. DATA COLLECTION AND MANAGEMENT

# 9.1. Data Management team

A project data management team, chaired by representatives from MOH, BHP, Harvard Chan School, and CDC, will be formed to build the research data collection systems. The data management team will:

- (1) Design the data collection and management systems required for BCPP;
- (2) Coordinate data usage for project progress reports to funders;
- (3) Coordinate data usage by the DSMB (as described in Section 5.4), and,
- (4) Coordinate data usage for analysis of primary and secondary study objectives.

This section outlines data collection and management guidelines; detailed methodologies for data collection and management will be developed and placed into SOPs or described in the manual.

# 9.2. Data Flow

Research data will be collected on mobile electronic devices during household surveys. Research data that are not collected during household surveys include routine clinical monitoring data collected in the electronic medical record system (PIMS2 or IPMS) for Combination Prevention community clinic patients (described in the *Intervention Protocol*); data from participants who consent to research-related blood draws (see section 6.3); and data on health resource utilization and quality of life from a subset of participants experiencing opportunistic illnesses (see Section 7).

#### 9.3. Data Flow From BHS, HIC, ESS, and Research Blood Draws

**Data entry**: Field teams will be trained in the use of appropriate mobile devices (e.g. notebooks) for data entry during the BHS, HIC, ESS, and research blood draws. Skip patterns, legal ranges, and consistency checks will help to ensure high quality data are collected.

From the point of entry, BHS study data will be synchronized from the field devices into the community server at the end of each shift. Data from the community server will be synchronized over encrypted virtual private network (VPN) channels to the central server at the BHP Data Management Center (DMC) in Gaborone nightly. Backups of the community server are transferred to the BHP DMC nightly and then included in the DMC's general backup routine. Database backups will be encrypted and stored on encrypted drives before transfer to removable media. Secure and lockable rooms will be used to house all workstations and servers and to store mobile devices when not in use.

All information will be collected and transmitted electronically except consent forms and laboratory labels. A paper copy of the informed consent/assent forms will be offered to the participants. The consent forms with participants' signatures and Omang numbers will be collected and, at the end of the day, secured in locked file cabinets at the base sites. Laboratory labels with bar code will be used for sample tracking. The sample labels will contain a computer-generated Subject Identifier, sample date, date of birth, and coded HIV status, and the type of sample. No personal identifying information can be derived from the labels.

Management of Personally Identifying Information (PII): The national identity card, Omang, required by the MoH for access to health care services including ART, is also needed to: (1) help identify study participants during research follow-up, and (2) link study data to HIV care and treatment data collected in routine HIV care and treatment systems.

However, once entered into the data system, observations with unique Omang numbers will be allocated, and referred to thereafter, by a unique computer-generated Subject Identifier. PII (such as first and last name, and omang number) may be viewed in the context of the BHP Electronic Data Capture (EDC) system by authorized EDC users. PII will only be used outside of the EDC in sending results to healthcare staff providing care who are required to reliably identify a patient. When EDC data are transferred to partners for operational purposes, the data will be transmitted through an encrypted VPN network between servers deployed with full disk encryption (FDE). When EDC data are transferred to partners for analytical purposes, PII values are not decrypted, if included, and the data will be transmitted through an encrypted VPN between servers deployed with FDE.

Protection of Electronically Stored Subject Data: Security of electronic records and data is a significant concern. All components of the distributed data systems will use authentication and encryption to render electronically stored subject identity and personal health information unusable, unreadable, or indecipherable to unauthorized individuals for "data in use" (e.g. data being analyzed by BCPP investigators), "data in motion" [e.g. data being transferred between data entry points and the Data Management Center (DMC) in Gaborone] and "data at rest" (e.g. data in storage at DMC in Gaborone).

Full Drive Encryption will be implemented at the hardware layer of all devices storing protected health information. A three-factor scheme will be used to authenticate users through the hardware layer to the application layer where personal health information is available. The applications will have user profiles to control access to certain data and reports. The application and database layers will use a combination of hashing and encryption for sensitive and personal data. Mobile devices and the staff operating them will not be equipped with the encryption keys to decrypt select sensitive data fields.

#### Special EDC/Data Considerations for Anonymous Participation of Non-citizens

In the ESS, enumerated subjects who are non-citizens not married to a citizen of Botswana are eligible to participate anonymously. The EDC will be used to collect survey data for these subjects without collecting any PII should they choose to participate. Following enumeration, each subject will be asked about their citizenship status prior to completing the Eligibility Checklist. If the subject is willing to participate anonymously given their non-citizen status, the EDC will redirect the RA to the Anonymous Eligibility Checklist. If the non-citizen subject is eligible for the survey and accepting of verbal consent, the EDC will do the following to protect the anonymity of the participant and maintain data integrity and completeness across anonymous and identified participants: 1) de-link the participant's enumeration record from the household; 2) generate an electronic consent record filling all PII variables with computer-generated ones; 3) allocate a Subject Identifier; 4) redirect the RA to the survey tool for completion with the participant. In this way there is no requirement for the RA to have proof of identification in order to proceed with data collection, electronically captured data will not be associated with a location in the community and PII will not be collected into the EDC nor in any manual manner.

# 9.4. The BCPP Research Data Management Center (DMC)

All research data collected from the BHS, AHS, HIC, and ESS will be housed centrally at the BCPP Research Data Management Centre (DMC), a secure facility within the Botswana Harvard HIV Reference Laboratory (BHHRL) that is co-owned by the MOH and BHP. Designated representatives from Harvard, MOH, and CDC will manage these data, and keep record of data management progress and access.

Sharing of program clinical data, that are stored in the MOH M&E unit, and which reflect routine care of consenting research participants with BCPP investigators, will be described in a data sharing agreement.

#### 9.5. Reporting Study Progress

On a monthly basis, a data manager at the Harvard Chan School will be responsible for providing indicators of project progress to project investigators and directors.

#### 10. ANALYSIS PLANS

#### 10.1. Analysis Plan to Meet Primary Objectives

# • 1<sup>st</sup> Primary Objective

To estimate the impact of the CP package on cumulative HIV incidence, we will perform pairwise comparisons within matched pairs of communities using a method that estimates the incidence ratio between the two communities and allows for interval censored time to event data (Finkelstein 1986). Interval censored time to HIV infection will arise from the fact that only the time interval in which subjects have become infected will be known and that some subjects will enter the incidence cohort after the start of the study, miss a follow-up survey, or drop-out. A permutation test will be used to test the null hypothesis of no intervention effect on incidence ratio. The test statistic will be an inverse-variance weighted average of the incidence ratio of every pair. The null distribution of the test statistic will be obtained by calculating the test statistic with the treatment assignment permuted within each pair (resulting in a sign change of the log of the incidence ratio estimate for each pair). The permutation test is valid even if the variances for the incidence ratio estimates are not accurately estimated; however, efficiency increases as the variance estimates get closer to the truth. Assuming independence of the incidence ratio among different pairs, the variance of the overall estimate of the incidence ratio can be estimated as a weighted sum of the variance of incidence ratio for each pair, where the weights are the inverse of the variance squared.

Secondary analyses will be performed to investigate the potential impact of informative censoring, which would arise if the probability of being tested was associated with risk of infection. Doubly robust methods based on weighting by the inverse of the probability of a subject receiving a test will be used for each pairwise comparison, and the method above will be employed for inference. To compare our results with those from other approaches, a secondary analysis will be performed

based on the method of Zhang and Sun (Zhang, Sun et al. 2007) for interval-censored community-level data. Missing data will be handled using approaches described in Tsiatis (Tsiatis 2006) and Little and Rubin (Little and Rubin 2002). Sensitivity analysis will be performed to assess the robustness of inference to various assumptions.

**Covariate-Adjusted Analyses**: Pair-matching in this CRT controls for certain factors associated with the outcome of interest, at the design stage. Nonetheless, there could be imbalance between arms for a number of other baseline community covariates (e.g., despite best attempts at matching there may be baseline imbalances in HIV prevalence between arms). By adjusting for these covariates, precision and power of the trial can be improved.

Covariate adjustment through a two-stage procedure has been proposed by Gail et al. (Gail, Byar et al. 1992). First, a proportional hazard model for interval-censored data will be fit, including the covariates of interest, as well as terms for the matched pairs, but excluding the intervention effect. The expected incidence rate of each community will be estimated based on the fitted model. We will then perform a permutation test on the difference between the expected and observed incidence rate to test the null hypothesis of no intervention effect while adjusting for imbalances in these covariates.

# • 2<sup>nd</sup> Primary Objective

To estimate coverage of HTC, ART (including viral suppression), and MC at baseline and study end in Enhanced Care and Combination Prevention communities, the following proportions will be estimated with 95% confidence intervals:

- The proportion of 16-64 year-old community residents who report knowing that they are HIV-infected, or report testing HIV-negative in the preceding 12 months.
- The proportion of 16-49 year-old HIV-negative men resident in the study communities who are circumcised.
- The proportion of HIV-infected 16-64 year-old community residents who know they are HIV-positive and are receiving ART.
- The proportion of HIV-infected 16-64 year-old community residents who know they are HIV-positive, are receiving ART, and have HIV-1 RNA ≤400 copies/mL.

To compare proportions between arms at the end of study, we will use cluster-level analysis. The main outcome measure will be the proportion of eligible persons successfully covered by the intervention. Cluster-specific proportions will first be calculated for each cluster within a pair. Then within-pair coverage rate ratios  $\binom{r_{1j}}{r_{0j}}$ , coverage rate differences  $\binom{r_{1j}-r_{0j}}{r_{0j}}$ , and their

standard errors will be estimated (where " $r_1$ " and " $r_0$ " are the coverage proportions for Combination Prevention and Enhanced Care clusters respectively, and "j" represents the jth cluster pair). The change in coverage between ESS and baseline will also be compared.

To estimate the overall coverage proportion, we calculate coverage proportion among all eligible survey participants within each arm at baseline and ESS. The ratio and difference of coverage proportions between Enhanced Care and Combination Prevention communities at baseline and ESS are then calculated. We will additionally consider inclusion of data collected from non-citizens in

analyses of the second primary objective. To this end, we will conduct both stratified and pooled analyses.

Baseline characteristics of the two treatment arms will be examined to characterize the population and to identify any imbalance between the arms. Where a large difference in baseline characteristics is observed between treatment groups the relevant covariate may be included in an adjusted analysis.

# • 3<sup>rd</sup> Primary Objective

The estimated cost per additional HIV infection averted will be estimated using the CEPAC-I model.

# 10.2. Analysis Plan to Meet Key Secondary Objectives

 1<sup>st</sup> Secondary Objective: To estimate the extent to which incident HIV-infections in Combination Prevention and in Enhanced Care communities arise from HIV strains circulating within communities randomized to the same study arm as the incident case or from strains circulating outside those communities (sexual network mixing).

Statistical concepts applicable to assessing genetic linkage of incident infections within the HIC are described in section 8. Using these analysis techniques, incident infections observed in the HIC will be classified as either phylogenetically linked to HIV-1 variants in the same study arm, or unlinked. The proportion of incident infections that are unlinked will be provided with 95% confidence intervals.

 2<sup>nd</sup> Secondary Objective: To estimate the efficacy of the Combination Prevention package on reducing the rate of new infections with HIV strains circulating within communities in the same study arm.

Maps of circulating HIV-1 genotypes will be generated in Enhanced Care and Combination Prevention communities through sample collection during the BHS, HIC and ESS. In addition, HIV genotyping will be done through blood sample collection among all HIV-infected persons attending clinics in Combination Prevention communities. However, to avoid biased comparisons between Combination Prevention and Enhanced Care arms, only HIV-1 genotype maps generated from the BHS, HIC, and ESS in both Combination Prevention and Enhanced Care arms will be used to categorize incident infections as either linked or unlinked for analysis of this secondary objective. To meet this secondary objective, pairwise comparison of HIV incidence between Enhanced Care and Combination Prevention arms (as described in section 10.1 above), limited only to linked infections in each arm, will be performed.

 3<sup>rd</sup> Secondary Objective: In the Combination Prevention arm only, to estimate over time, the proportion of recent HIV-1-infections that can be linked to HIV-infected adults of the same study arm.

In Combination Prevention communities, we will carry out phylogenetic clustering using data collected at baseline and all subsequent timepoints. By comparing all newly diagnosed cases each

year and at ESS against clusters established at baseline, we will be able to assess the trend in newly diagnosed cases linking to existing cases or with each other.

 4<sup>th</sup> Secondary Objective: During the ESS, to compare Combination Prevention (CP) package uptake within 20% HIC households to CP package uptake in the broader communities they represent.

Coverage of ART, MC, and PMTCT at the ESS will be estimated separately for participants within the 20% households in all 30 communities, and in the remaining 80% of households in each of the 6 communities selected for the ESS. The proportions for the coverage are as defined in 2<sup>nd</sup> primary objective. We will do pair-wise comparisons of the proportions between the study cohort and those in the same community outside of the cohort using cluster-level analysis stratified by treatment status. The within-community coverage ratio and difference and their standard errors will be calculated for ART, MC, and PMTCT, in Enhanced Care and Combination Prevention arms separately.

• 5<sup>th</sup> Secondary Objective: To obtain secondary cross-sectional estimates of community HIV incidence at baseline and study end in Enhanced Care and Combination Prevention communities through use of HIV-incidence assays.

Assay-based HIV incidence is calculated as the number of recent infections divided by the population at risk (those testing HIV-negative plus those recently seroconverting), then annualized by multiplying by 365 divided by the accepted mean seroconversion duration for the assay.

To calculate the incidence as an annual instantaneous rate ( $I_r$ ) the following formula, or a contemporary equivalent, may be used:

$$I_r = \frac{R - \varepsilon P}{(1 - \varepsilon)\omega N}$$

Where the survey counts (N, P, R) are as follows:

N = number of HIV negative individuals in the survey

P = number of HIV positive individuals in the survey

R = number of individuals classified incidence assay positive

The calibration parameters are as follows:

 $\omega$  = mean incidence assay duration specified in units of years

 $\varepsilon$  = false recent rate (FRR) of the incidence assay. In the presence of more data such as viral load, documented ART status and documented testing history, FRR adjustments may not be neccessary as per the WHO guideline on recent infection testing algorithm (World Health Organization 2011; UNAIDS 2013; Rehle, Johnson et al. 2015).

Confidence intervals are computed using a delta method approximation which may include the error, assumed to be normally distributed, associated with calibration parameters. The coefficient of variation ( $C_v$ ,  $C_v$ ) is computed as follows:

$$C_{v} = \sqrt{\frac{1}{P} \left( \frac{N+P}{N} + \frac{(P-R)R[1+\varepsilon/(1-\varepsilon)]^{2}}{[R-\varepsilon/(1-\varepsilon)(P-R)]^{2}} \right) + \frac{\sigma_{\omega}^{2}}{\omega^{2}} + \frac{\sigma_{\varepsilon}^{2}(P-R)^{2}}{(1-\varepsilon)^{4}[R-\varepsilon/(1-\varepsilon)(P-R)]^{2}}},$$

where

 $\sigma_{\omega}$  is the standard deviation of the mean RITA duration (assumed normally distributed)

 $\sigma_{arepsilon}$  is the standard deviation of the FRR (assumed normally distributed).

The 95% confidence interval (CI) for  $I_r$  is then computed as:

$$I_r \pm 1.96 \times I_r C_v$$

Sampling weights will be applied accordingly in the national adult incidence estimate calculation (15-59 years and 15-49 years), and survey design effects will be computed to estimate the variance for calculating the 95% CI around the estimates. Overall incidence estimates and sub-group incidence estimates (15-59 years and 15-49 years), where possible, will be calculated to highlight peak incidences that can be targeted by HIV prevention programs. Bi- and multivariate analysis using STATA and or SAS software will examine associations between demographic, behavioral or other characteristics and HIV recency status.

6<sup>th</sup> Secondary Objective: At baseline, during study conduct, and at study end, to estimate the
proportion of recent HIV infections in combination prevention and enhanced care communities
with evidence of transmitted HIV drug resistance.

The proportion of patients with evidence of transmitted HIV drug resistance will be calculated as the proportion of patients identified with drug resistance through drug resistance assays among patients with new or recent HIV infections identified through assay-based testing. Testing for TDR will be performed on samples from HIV-infected persons residing in the 20% BHS/HIC households and from ESS participants in both arms; and from consenting HIV-infected persons identified through the HTC campaigns in Combination Prevention communities. The proportion and its standard error will be calculated for each arm at baseline, annually, and at study end.

• 7<sup>th</sup> Secondary Objective: To estimate the proportion of HIV-infected adults with undetectable viral load (VL<400 copies/ml) at baseline, during study conduct, and study end in Combination Prevention and Enhanced Care communities.

This analysis will be performed using measurements of HIV-1 RNA throughout the study. The threshold of 400 copies/ml will be used for enumeration of HIV-infected individuals either above or below the threshold. Testing for HIV-1 RNA will be performed on samples from HIV-infected persons residing in the 20% BHS/HIC households and from ESS participants in both arms; and from consenting HIV-infected persons identified throughout the study in Combination Prevention

communities. The proportion and the 95% confidence intervals with transmitted drug resistance will be estimated and compared between Combination Prevention and Enhanced Care communities at baseline, annually, at the study end.

 8<sup>th</sup> Secondary Objective: To estimate the association between HIV-1 viral load and HIV transmissions using viral linkage data.

The hypothesis to be tested is that individuals with high HIV-1 RNA load are responsible for the majority of new HIV transmissions. To estimate HIV-1 RNA load within clusters we will use two sets of data, results of phylogenetic clustering and measurements of HIV-1 RNA load in HIV-positive individuals participating in the study. Specifically, HIV-infected individuals will be grouped based on clustering patterns of their viral sequences, and cluster-specific (within each cluster) HIV-1 RNA load will be estimated. We will compare HIV-1 RNA load between two groups of clusters, clusters with and without incident cases identified over the study. The assumption is that HIV-1 RNA is higher within clusters with incident cases.

Analysis plans for **Secondary Objectives 9-11** are covered in Section 7 (concerning cost-effectiveness).

• 12<sup>th</sup> Secondary objective: To compare CD4 and viral load trajectories over time, among HIV-infected ART-naive persons who reside in Combination Prevention vs. Enhanced Care communities.

We will compare CD4 count and viral load over time between randomized arms, among HIV-infected persons who enroll into BHS with initial CD4>350 and while still ART-naive. The underlying rationale for this comparison is the assessment of the immunologic and virologic implications of expanded/early ART. The primary endpoints for this analysis will be the change in CD4 count over time, and the proportion of participants with HIV-1 RNA < 400 copies/mL by the final visit, by randomized arm.

• 13<sup>th</sup> Secondary objective: To assess the accuracy and feasibility of point-of-care viral load testing in comparison to standard viral load platforms.

Sensitivity and specificity of the POC viral load testing against BHHRL standard procedure using the threshold of viral load at 10,000 copies/ml will be evaluated.

The POC and BHHRL measurements will be compared using Bablok and Passing regression analysis (Bablok and Passing 1985), which includes evaluation of the systematic and proportional errors, as well as correlation. For each phase, the difference of the POC value and the BHHRL standard procedure on the same sample will be plotted against the mean of the two measurements (Bland-Altman plot) to assess the comparability of the POC method with the BHHRL standard procedure, and estimate the mean bias (with 95% confidence interval) (Bland and Altman 1986).

Statistics and qualitative reports on operational characteristics of the POC procedures will be reported.

• 14<sup>th</sup> Secondary objective: To understand (through qualitative interviews) barriers to and facilitators of linkage to care and ART initiation among BHS participants.

Qualitative data related to linkage to care and initiation of ART will be gathered through focus group discussions (FGDs) and in-depth interviews (IDIs). Data will be collected in the CPCs from members of the BHS field team, the MOH nurse prescribers as well as from a subset of HIV-infected BHS participants who are eligible for ART. FGDs and IDIs will be semi-structured and based on a standardized guide. All FGDs and IDIs will be audio-recorded, transcribed and translated (when not in English). Investigators will read the transcripts and develop and agree on a codebook. An iterative process will be used to read transcripts, apply codes, compare and revise codes until consensus is reached about salient motivators and barriers for linking to care and initiating ART.

• 15<sup>th</sup> Secondary objective: To use BCPP data in analyses of the rates of and risk factors for major AIDS and non-AIDS illnesses/injuries/mortality among persons living with and without HIV in Botswana.

Measurements and survey responses from participants in the BHS, AHS, and ESS will be utilized to estimate the distribution of risk factors and frequency of health events in Botswana. The combined cohort (BHS, AHS, ESS) will also serve as a source for controls in case-control analyses and an estimate of population exposures in standardized incidence/morbidity/mortality analyses. Cases will be obtained from other sources, such as national registries, publicly available data, or other studies, with separate IRB approval where needed. Case-control and standardized incidence/mortality/morbidity analyses do not require release or sharing identifiable information outside of BCPP.

# 11. ETHICAL CONSIDERATIONS

#### 11.1. Ethical Review

The protocol, informed consent/assent forms, research participant education and recruitment materials, and other requested documents — and any subsequent modifications — will be reviewed and approved by the ethical review bodies responsible for oversight of research conducted at the study sites. Subsequent to initial review and approval, the responsible Institutional Review Boards/Ethical Committees (IRBs/ECs) will review the protocol at least annually.

#### 11.2. Informed Consent

Please see Table 12 below for a summary of the various approaches to informed consent for this protocol.

Potential participants will be given the opportunity to ask questions about the study. It will be emphasized that participation in any component of the research is completely voluntary. The informed consent process will occur in the language most comfortable for participants (usually in

Setswana). Consent materials will be translated into the local language and back-translated to ensure accuracy. Staff will obtain informed consent who have been designated this responsibility in study staff signature logs. Usually staff obtaining informed consent during household surveys and research blood draws will be healthcare auxiliaries and research assistants.

- BHS/AHS, HIC and ESS Household Representatives Verbal Consent for Household Representative: Consent will be obtained from the household representative to obtain the household structure. Informed consent for this aspect of study participation will be obtained from research volunteers aged 18 or older, without documenting the process in writing. A waiver of documentation of informed consent will be requested from IRBs and the informed consent script approved prior to use. The consent script (Household Script) will describe the purpose of the research activity, procedures to be followed, and the risks and benefits of participation. Only participants who verbally agree to participate will be asked to provide the requested data for this part of the study. A copy of the informed consent script will be offered to the participant. The reading level of the script has been estimated using Flesch-Kincaid and is below 6.0.
- BHS/AHS, HIC, ESS Citizen/Spouse of Citizen Participants in Household Surveys and Cohort, and individuals consenting to research blood draws or qualitative interviews: Written informed consent will be obtained from each eligible individual before completion of individual questionnaires and/or blood draws for study purposes. Residents aged 16-17 years old, if eligible, will be asked to provide written assent with a guardian's written permission. The informed consent/assent form will be given to the participant to read (for literate participants), or read by a trained study staff member (for illiterate participants). Required steps in the process will be driven electronically in household visits to ensure quality, consistency and completeness. Consent/assent will be documented by having the participant sign the informed consent/assent form or make a mark if the participant is illiterate; the latter will be witnessed by a third party. A copy of the informed consent/assent form will be offered to the participant, and if applicable, parent or legal guardian giving permission for a minor to participate. Staff will ensure that the participant takes a copy of a study contact card that contains study information and telephone numbers if the participant does not wish to take a copy of the consent. The reading levels of each consent/assent form have been estimated using Flesch-Kincaid and are below 6.0.
- **ESS Non-Citizen Adult Participants in ESS:** A waiver of the requirement to obtain a signed consent/assent form is requested from IRBs for non-citizen participants in the ESS. The request for this waiver is based on the U.S. Code of Federal Regulations Title 45 Part 46.117(c)(1). All data and specimens will be collected anonymously from these participants. Therefore, the only record linking the subject and the research would be the consent document and the principal risk would be potential harm resulting from a breach of confidentiality. A written statement regarding the ESS will be IRB-approved and provided to non-citizen participants prior to conducting survey procedures, but it will not bear the participant's name or signatures. The written statement will be given to the participant to read (for literate participants), or read by a trained study staff member (for illiterate participants in the presence of a witness). Parental permission will be sought with assent from any non-citizen participants 16-17 years old, but signatures will not be obtained per the waiver. Required steps in the process will be recorded with a checklist.

# Special Populations

*Minors*: Minors (participants ages 16-17) will only be enrolled in research activities if they can provide informed assent and with the written permission of a parent/legal guardian.

- ✓ Under circumstances where study staff suspect, or there is a reported incident of sexual abuse of a person under age 18, the study staff member must inform the relevant authorities; this is stated in the informed consent/assent forms.
- ✓ Referrals will be made to youth services if needed.

Institutionalized populations: Persons residing in institutions such as prisons will not be included in the study as they will not be available for household and community surveys. An enrolled participant who becomes imprisoned or involuntarily confined in a medical facility (e.g. for psychiatric illness) during the study will not undergo any study procedures during confinement. Visits missed due to absence will be recorded. Study procedures would only resume if the participant is released from confinement during the study period and is available and willing to complete any remaining study visits.

Non-citizens: Non-citizens who are not married to Botswana citizens are eligible to participate in the ESS, a one-time household survey at the end of the study. Increased likelihood of experiencing problems with securing housing, travel, exploitation in employment, and access to healthcare make non-citizens a potentially vulnerable population. Anonymous participation in the ESS will be offered to ensure protection for non-citizen participants. In particular, the sociodemographic information collected from non-citizens will be limited, including only age (year of birth, but not date of birth), gender, immigration status, place of primary residence (at the community level, not a physical address), for example. No names or personal identifiers will be collected from participants who are non-citizens. Referrals will be made to services that are available to non-citizens.

Table 12: Summary of Approach to Consent, Various Components of the Study

| Project<br>component | Targeted subjects | Activity | Consent<br>Type/Waiver<br>Requested | Consent<br>Material to be<br>Used | Provision for<br>Parental<br>Permission with<br>Assent? | Timing of<br>Obtaining<br>Consent |
|---|---|---|---|---|---|---|
| Household<br>structure | Head of household/representative in 20% households | Questionnaire regarding household structure and socioeconomic indicators | Verbal/Waiver requested for documentation of consent | Household<br>Script | No | внѕ то |
| BHS | Age-eligible members of 20% households, including HIV-infected persons and HIV-uninfected persons | Baseline and follow-up questionnaires Repeat HTC if not documented HIV-positive Research blood draws, if applicable Repeat CD4/VL, if applicable POC VL, if applicable | Written | BHS/HIC<br>Consent | Yes | BHS TO New participants may consent at T1 New participants at T2 will sign ESS consent |
| HIC | Age-eligible HIV-uninfected members of 20% households who meet HIC eligibility criteria (a subset of BHS participants) | Baseline and follow-up questionnaires Repeat HTC Research blood draws, CD4/VL/POC VL if applicable (i.e. for seroconverters) | Written | BHS/HIC<br>Consent | Yes | BHS TO, New<br>participants<br>may consent at<br>T1 |
| Blood draw for<br>research<br>purposes | <ul> <li>All HIV-infected persons in<br/>Combination Prevention<br/>communities</li> <li>BHS residents who decline<br/>survey participation but are<br/>willing to give a blood sample</li> </ul> | Blood for HIV-1 RNA, stored sample for HIV genotyping/resistance testing and incidence assay | Written | Research Blood<br>Draw Consent | Yes | Upon referral<br>to or<br>recruitment by<br>research staff |
| End of study<br>survey | All eligible residents (new enrollees from 20% BHS/HIC householdsand ~80% of remaining community members will be newly enrolled to ESS in 3 pairs of selected communities) | ESS questionnaire<br>Research blood draw, if<br>applicable<br>CD4/VL/POC VL if applicable | Written for<br>Citizens/Spouses<br>of Citizens; Waiver<br>requested for<br>non-citizens | ESS Consent | Yes for<br>Citizens/Spouses<br>of Citizens<br>No for Non-<br>Citizens | T2/ESS |
| Supplemental<br>Economic<br>Assessment for<br>Low CD4/OI | Residents with low CD4 or OIs seeking care (out- or inpatient) | Questionnaire regarding economic activity and quality of life | Written | Economics<br>Consent | No | Upon referral to research staff |

| Barriers to and | HIV-infected BHS participants | Focus group discussions | Written | ART Start | No | At T1 or later |
|---|---|---|---|---|---|---|
| facilitators of | BHS Research Assistants and Nurse | Individual in-depth interviews | | Interview | | |
| LTC and ART | Prescribers | | | Consent; ART | | |
| initiation | | | | Start Focus | | |
| | | | | Group Consent | | |
| | | | | for BHS; ART | | |
| | | | | Start Focus | | |
| | | | | Group Consent | | |
| | | | | for Staff | | |

#### 11.3. Risks

The risks, discomforts, and inconveniences that could be posed to subjects participating in this study include the following:

#### Survey Participants in the BHS, HIC, research blood draw after HTC, and ESS:

- Blood drawing may cause pain and bruising, and rarely, infection at the site where blood is drawn. Study participants may feel lightheaded or faint as a result.
- Repeated HIV testing and counseling in the HIC participants may cause stress, anxiety, or embarrassment. Participants are likely to become distressed if they learn they are HIV positive.
- Participants may become embarrassed, worried, or anxious when discussing their sexual practices, HIV risk factors, ways to protect their partner(s) against HIV, and/or ways to prevent acquiring HIV infection.
- Participants may experience discrimination as a result of being perceived by others to be HIVinfected or at high risk for HIV infection.
- Participants may have difficulty or conflict in their relationships if they choose to participate couples HIV testing, particularly if this results in perceived or disclosed infidelity.

#### 11.4. Benefits of Research Participation

#### Survey Participants in the BHS, HIC, research blood draw after HTC, and ESS:

Potential health benefits for 20% household residents include: earlier HTC delivered to their place of residence, earlier diagnosis of HIV-infection (and access to point-of-care CD4 result if ART-naive) with subsequent earlier enrollment in care and treatment or PMTCT, and earlier awareness of the importance of annual HTC and risk reduction practices for adults who test HIV-negative. HIV-infected individuals who consent to participate in the household surveys will also have access to a pre-ART viral load result at BHS enrollment and then repeat CD4 and viral load if ART-naïve at enrollment or at the study visit when HIV-positive status is recorded.

Those who participate in research blood draws independently of the household surveys may also benefit from a pre-ART viral load result; however, the test may not be run in real-time.

# 11.5. Confidentiality

No identifiable study data will be released to any unauthorized third party, without prior written approval of the participant, except as necessary for monitoring by the IRBs, the study sponsor, external monitors, OHRP, or the Botswana Ministry of Health.

#### During BHS, HIC, research blood draw after HTC, and ESS study procedures:

Project staff visiting households for study visits will identify an appropriately private space to counsel participants, perform HIV tests, and collect individual data. If private space is not available, or the participant does not wish to carry out study activities in the home, an appointment will be made to visit one of the study clinics instead. All study documents will be stored in a secure location and electronic data will be password protected. Full Drive Encryption will be implemented at the hardware layer of all devices storing protected health information. Only designated study staff will have access to study records.
#### De-identified data:

When de-identified datasets are created the following variables will be excluded: name, national identity number, phone numbers, address (other than community of residence), GPS coordinates, and all elements of dates (except year) for events related to the individual (birth, death, hospitalizations, clinic visits, etc.). BCPP does not collect data on persons >89 years, nor any biometric data or other identifiers.

# 11.6. Compensation and Incentives

- Baseline Household Survey (BHS) and HIV Incidence Cohort (HIC): Each participating resident will
  receive 20 Pula (about \$3) worth of air time as compensation for time dedicated to the study at
  each attended scheduled study visit.
- End of Study Survey (ESS): Each participating resident will receive 20 Pula (about \$3) worth of air time as compensation for time dedicated to the study at the End of Study Survey.

# 11.7. Protocol Compliance and Compliance with UN Convention on the Rights of the Child

Study staff will adhere to the ethical principles that have their origin in the Declaration of Helsinki (e.g., ICH E6, 45 CFR 46). The study will be conducted in accordance with the regulations of Botswana and the sponsor.

The US government is a signatory on the UN Convention on the Rights of the Child (defined as anyone under the age of 18) which requires that any research study or program activity which includes children that are identified as engaged in sex work, trafficked or victims of violence make special provisions for referral of these individuals to services. BCPP will report suspected cases to service providers (local police or social workers) as outlined in the Botswana National Guidelines for reporting child abuse or neglect. Contact information for the local police and social workers, and procedures for reporting suspected cases of child abuse or neglect are described in the study-specific SOP in the BCPP Study Manual. Local police and social workers will be contacted prior to the initiation of study activities in the community to ensure they are aware of the study activities in the community and the porcedures that will be followed should BCPP staff encounter suspected cases of abuse or neglect. As per national guidelines, reports of suspected abuse or neglect will be made to local authorities within 24 hours. Study personnel who may come in contact with these study participants will receive training on the appropriate procedures for handling these cases if they arise during the course of the study and training on the SOP documented in the regulatory files. The study will retain documentation of all reports that includes date of report, age of participant, and the name and type of service provider. No identified information will be retained in the documentation; documentation will be retained by the study for 2 years after study close-out. The informed consents for the study contain language that makes clear to the participant what is required to be reported to authorities and the impact on confidentiality.

# 11.8. Future Use of Stored Samples

Study participants will be asked to provide written informed consent for their specimens to be stored after the end of the study for possible future research testing. Any residual specimens of participants

who do not consent to long-term storage and additional testing will be destroyed at the end of the study after all protocol-required and quality assurance testing has been completed.

# 12. STUDY SAFETY AND MONITORING PLAN

# 12.1. Reporting Adverse Events

The Evaluation Protocol does not involve the administration of any study products.

The study team will report in real-time, to IRB's and to sponsors, any serious adverse events (SAEs) experienced by a participant or other individual, that in the opinion of the investigator are **BOTH unexpected and at least possibly related** to the research procedures. An SAE is defined as any untoward occurrence that:

- Results in death
- Is life-threatening (grade 4)
- Requires hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect, or
- Is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above.

This level of reporting is chosen for this observational aspect of the BCPP to avoid real-time reporting of all events (e.g. deaths, hospitalizations etc.) occurring in study communities that are definitely not related to study procedures (but to remain compliant with reportable new information generally required by IRBs).

# Timing of reporting:

Reportable events will be reported in accordance with institutional, sponsor, and study specific guidelines delineated in standard operating procedures for the study.

# **AE** reporting period:

The AE reporting period for this study is from the time of enrollment to the end of study follow-up for a participant.

# AE reporting process

Reportable events will be documented by the in-country study team who will then notify the IRBs, MoH, CDC-Atlanta, and Harvard teams. The incident will be discussed and a written action plan will be devised and implemented within 1 week of the initial report, if needed. Written documentation of all reportable events and event resolution will be retained in the study file. Reporting of events to IRBs and the study sponsor will follow institutional and IRB policies. If necessary, a formal report will be sent to the appropriate IRBs using the CDC's Incident Report Form 1254.

# 12.2. DSMB

DSMB review will take place prior to the start of the study and annually thereafter. Details of recommended interim analyses by the DSMB are provided in Section 5.4.

#### 12.3. Protocol Violations

The study will be conducted in full compliance with the protocol. The research team will ensure that volunteers are informed of and understand the risks of their participation in research. Protocol violations and cases of social harm will be documented using the appropriate study forms and reported to IRBs and sponsors in accordance with the institutional policies. Minor protocol violations that do not pose a threat to the health of participants will be compiled and reported to the IRBs at the time of annual IRB review. Incident reporting is the responsibility of the Principal Investigators of this study. Emergency departures from protocol that eliminate an apparent immediate hazard to a participant and are deemed crucial for the safety and well-being of that participant may be instituted for that participant only. In that case the Investigator will contact the IRBs and sponsor as soon as possible to document the reasons for violation and ensuing events.

# 12.4. Study Monitoring Plan

A complete monitoring plan will be developed and the site will complete a site activation checklist prior to study initiation. Internal (sponsor) and external monitors will travel to the study site according to a pre-determined monitoring schedule specified in the monitoring plan to conduct general monitoring. The study site will maintain a monitoring log to document all monitoring visits. Investigators and staff will grant access to the monitors to allow inspection and review study documents (e.g., consent forms, data collection forms, other source documents) and pertinent clinic records for confirmation of the study data. Study monitors will also inspect study facilities and documentation and may observe the performance of study procedures.

# 13. ADMINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION

# 13.1. Study Records and Document Retention

Complete, accurate, and current study records will be maintained and stored in a secure manner throughout the duration of the study and additionally for five years after study close-out. Study records include administrative documentation—including all reports and correspondence relating to the study—as well as documentation related to each participant screened and/or enrolled in the study, including informed consent forms, locator forms, case report forms, notations of all contacts with the participant, and all other source documents. Necessary documents to be maintained by the site before, during and after the study will be in accordance with GCP regulations and guidance. A complete list of needed documentation will be provided prior to initiation of the study and will appear in the study manual.

#### 13.2. Information Dissemination and Publication Plan

Study findings will be disseminated through presentations, reports and publication in peer-reviewed journals and other publications. In-country data and country specific information will be made available to national policy-makers, organizational, and implementing partners. A detailed publication and communication plan will be developed that describes the number and types of reports and manuscripts planned for the study and criteria for authorship. Formal presentations at conferences and scientific publications will follow CDC, Harvard, and MOH guidelines. A data sharing plan will also be developed that details the requirements and process for requesting access to stored data and samples for sub-studies and future analysis.

# 14. REFERENCES

- Ades, A. E., K. Claxton, et al. (2006). "Evidence synthesis, parameter correlation and probabilistic sensitivity analysis." Health Econ 15(4): 373-381.
- Alam, S., R. Meyer, et al. (2009). A model for HIV spread in a South African village, Lecture Notes in Computer Science. 5269: 33-45.
- Alkema, L., A. E. Raftery, et al. (2008). "Bayesian melding for estimating uncertainty in national HIV prevalence estimates." Sex Transm Infect 84 Suppl 1: i11-i16.
- Anglaret, X. and S. Eholié. (2012). "Early antiretroviral treatment and/or early isoniazid prophylaxis against tuberculosis in HIV-infected adults (ANRS 12136 TEMPRANO)." from <a href="http://clinicaltrials.gov/ct2/show/NCT00495651">http://clinicaltrials.gov/ct2/show/NCT00495651</a>.
- Attia, S., M. Egger, et al. (2009). "Sexual transmission of HIV according to viral load and antiretroviral therapy: systematic review and meta-analysis." <u>AIDS</u> 23(11): 1397-1404.
- Auvert, B., D. Taljaard, et al. (2005). "Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial." PLoS Med 2(11): e298.
- Bablok, W. and H. Passing (1985). "Application of statistical procedures in analytical instrument testing." <u>J</u>

  <u>Automat Chem</u> 7(2): 74-79.
- Bailey, R. C., S. Moses, et al. (2007). "Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial." <u>Lancet</u> 369(9562): 643-656.
- Barth, R. E., J. T. van der Meer, et al. (2008). "Effectiveness of highly active antiretroviral therapy administered by general practitioners in rural South Africa." <u>Eur J Clin Microbiol Infect Dis</u> 27(10): 977-984.
- Bendavid, E., M. L. Brandeau, et al. (2010). "Comparative effectiveness of HIV testing and treatment in highly endemic regions." <u>Arch Intern Med</u> 170(15): 1347-1354.
- Bennett, D. E., R. J. Camacho, et al. (2009). "Drug resistance mutations for surveillance of transmitted HIV-1 drug-resistance: 2009 update." <u>PLoS One</u> 4(3): e4724.
- Bershteyn, A., D. J. Klein, et al. (2012). "Description of the EMOD-HIV Model v0. 7." <u>arXiv preprint</u> <u>arXiv:1206.3720</u>.

- Bierman, W. F., M. A. van Agtmael, et al. (2009). "HIV monotherapy with ritonavir-boosted protease inhibitors: a systematic review." <u>AIDS</u> 23(3): 279-291.
- Bland, J. M. and D. G. Altman (1986). "Statistical methods for assessing agreement between two methods of clinical measurement." Lancet 1(8476): 307-310.
- Blitzstein, J. and P. Diaconis (2006). "A sequential importance sampling algorithm for generating random graphs with prescribed degrees. Available at: <a href="http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf">http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf</a>."
- Bouckaert, R., J. Heled, et al. (2014). "BEAST 2: a software platform for Bayesian evolutionary analysis." <u>PLoS</u>

  Comput Biol 10(4): e1003537.
- Boulle, A., G. Van Cutsem, et al. (2008). "Outcomes of nevirapine- and efavirenz-based antiretroviral therapy when coadministered with rifampicin-based antitubercular therapy." JAMA 300(5): 530-539.
- Braunstein, S. L., D. Nash, et al. (2011). "Dual testing algorithm of BED-CEIA and AxSYM Avidity Index assays performs best in identifying recent HIV infection in a sample of Rwandan sex workers." <u>PLoS One</u> 6(4): e18402.
- Brazier, J., J. Roberts, et al. (2002). "The estimation of a preference-based measure of health from the SF-36."

  J Health Econ 21(2): 271-292.
- Brazier, J., T. Usherwood, et al. (1998). "Deriving a preference-based single index from the UK SF-36 Health Survey." J Clin Epidemiol 51(11): 1115-1128.
- Briggs, A. H., M. C. Weinstein, et al. (2012). "Model parameter estimation and uncertainty analysis: a report of the ISPOR-SMDM Modeling Good Research Practices Task Force Working Group-6." Med Decis Making 32(5): 722-732.
- Central Statistics Office (2009). Botswana AIDS Impact Survey III (BAIS III), 2008. C. Kebonyethebe Johane. Gaborone, Botswana.
- Central Statistics Office (2009). Botswana Demographic Survey 2006. Gaborone, Central Statistics Office.
- Central Statistics Office (2009). Project Document: 2011 Population and Housing Census. Available at: <a href="http://unstats.un.org/unsd/censuskb20/Attachment453.aspx">http://unstats.un.org/unsd/censuskb20/Attachment453.aspx</a>. Gaborone, Central Statistics Office.
- Charalambous, S., C. Innes, et al. (2007). "Evaluation of a workplace HIV treatment programme in South Africa." <u>AIDS</u> 21 Suppl 3: S73-78.
- Coetzee, D., K. Hildebrand, et al. (2004). "Outcomes after two years of providing antiretroviral treatment in Khayelitsha, South Africa." AIDS 18(6): 887-895.
- Cohen, M. S., Y. Q. Chen, et al. (2011). "Prevention of HIV-1 infection with early antiretroviral therapy." N Engl J Med 365(6): 493-505.

- Cole, S. R., M. A. Hernan, et al. (2003). "Effect of highly active antiretroviral therapy on time to acquired immunodeficiency syndrome or death using marginal structural models." <u>Am J Epidemiol</u> 158(7): 687-694.
- Cornell, M., M. Schomaker, et al. (2012). "Gender differences in survival among adult patients starting antiretroviral therapy in South Africa: a multicentre cohort study." <u>PLoS Med</u> 9(9): e1001304.
- Curran, K., E. Njeuhmeli, et al. (2011). "Voluntary medical male circumcision: strategies for meeting the human resource needs of scale-up in southern and eastern Africa." <u>PLoS Med</u> 8(11): e1001129.
- Danel, C., R. Moh, et al. (2015). "A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa." N
  Engl J Med 373(9): 808-822.
- DART Virology Group and Trial Team (2006). "Virological response to a triple nucleoside/nucleotide analogue regimen over 48 weeks in HIV-1-infected adults in Africa." AIDS 20(10): 1391-1399.
- Delfraissy, J. F., P. Flandre, et al. (2008). "Lopinavir/ritonavir monotherapy or plus zidovudine and lamivudine in antiretroviral-naive HIV-infected patients." <u>AIDS</u> 22(3): 385-393.
- Drummond, M., R. Brown, et al. (2003). "Use of pharmacoeconomics information--report of the ISPOR Task Force on use of pharmacoeconomic/health economic information in health-care decision making."

  <u>Value Health</u> 6(4): 407-416.
- Duong, Y. T., R. Kassanjee, et al. (2015). "Recalibration of the limiting antigen avidity EIA to determine mean duration of recent infection in divergent HIV-1 subtypes." PLoS One 10(2): e0114947.
- Duong, Y. T., M. Qiu, et al. (2012). "Detection of Recent HIV-1 Infection Using a New Limiting-Antigen Avidity Assay: Potential for HIV-1 Incidence Estimates and Avidity Maturation Studies." <u>PLoS One</u> 7(3): e33328.
- Eaton, J. W., T. B. Hallett, et al. (2011). "Concurrent sexual partnerships and primary HIV infection: a critical interaction." <u>AIDS Behav</u> 15(4): 687-692.
- Enns, E. A. and M. L. Brandeau (2011). "Inferring model parameters in network-based disease simulation."

  Health Care Manag Sci 14(2): 174-188.
- EuroQol Group (1990). "EuroQol--a new facility for the measurement of health-related quality of life. The EuroQol Group." <u>Health Policy</u> 16(3): 199-208.
- Fauci, A. S. and G. K. Folkers (2012). "Toward an AIDS-free generation." JAMA 308(4): 343-344.
- Felsenstein, J. (1985). "Confidence Limits on Phylogenies: An Approach Using the Bootstrap." <u>Evolution</u> 39(4): 783-791.
- Felsenstein, J. (2004). Inferring Phylogenies. Sunderland, MA, Sinauer Associates.
- Finkelstein, D. M. (1986). "A proportional hazards model for interval-censored failure time data." <u>Biometrics</u> 42(4): 845-854.

- Fox, M. P., P. Ive, et al. (2010). "High rates of survival, immune reconstitution, and virologic suppression on second-line antiretroviral therapy in South Africa." <u>J Acquir Immune Defic Syndr</u> 53(4): 500-506.
- Fox, M. P. and S. Rosen (2010). "Patient retention in antiretroviral therapy programs up to three years on treatment in sub-Saharan Africa, 2007-2009: systematic review." Trop Med Int Health 15 Suppl 1: 1-15.
- Gail, M. H., D. P. Byar, et al. (1992). "Aspects of statistical design for the Community Intervention Trial for Smoking Cessation (COMMIT)." <u>Control Clin Trials</u> 13(1): 6-21.
- Gandhi, N. R., A. P. Moll, et al. (2009). "Successful integration of tuberculosis and HIV treatment in rural South Africa: the Sizonq'oba study." <u>J Acquir Immune Defic Syndr</u> 50(1): 37-43.
- Gardner, E. M., M. P. McLees, et al. (2011). "The spectrum of engagement in HIV care and its relevance to testand-treat strategies for prevention of HIV infection." Clin Infect Dis 52(6): 793-800.
- Gold, M. R., J. E. Siegel, et al., Eds. (1996). <u>Cost effectiveness in health and medicine</u>. New York, Oxford University Press.
- Gray, R. H., G. Kigozi, et al. (2007). "Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial." <u>Lancet</u> 369(9562): 657-666.
- Gray, R. T., M. H. Ghaus, et al. (2011). "Expected epidemiological impact of the introduction of a partially effective HIV vaccine among men who have sex with men in Australia." Vaccine 29(36): 6125-6129.
- Grinsztejn, B. and P. Mugyenyi. (2012). "Management using the latest technologies in resource-limited settings to optimize combination therapy after viral failure (MULTI-OCTAVE)." from <a href="http://clinicaltrials.gov/ct2/show/record/NCT01641367">http://clinicaltrials.gov/ct2/show/record/NCT01641367</a>.
- Habicht, J. P., C. G. Victora, et al. (1999). "Evaluation designs for adequacy, plausibility and probability of public health programme performance and impact." <a href="Int J Epidemiol">Int J Epidemiol</a> 28(1): 10-18.
- Hallett, T. B., J. M. Baeten, et al. (2011). "Optimal uses of antiretrovirals for prevention in HIV-1 serodiscordant heterosexual couples in South Africa: a modelling study." <u>PLoS Med</u> 8(11): e1001123.
- Halperin, D. T. (2009). "Combination HIV prevention must be based on evidence." Lancet 373(9663): 544-545.
- Hammond, R. and T. C. Harry (2008). "Efficacy of antiretroviral therapy in Africa: effect on immunological and virological outcome measures -- a meta-analysis." <a href="Int J STD AIDS">Int J STD AIDS</a> 19(5): 291-296.
- Handcock, M. S., D. R. Hunter, et al. (2003). "Software tools for the Statistical Modeling of Network Data. available at: <a href="http://statnet.org.">http://statnet.org.</a>"
- Hayes, R., F. Mosha, et al. (1995). "A community trial of the impact of improved sexually transmitted disease treatment on the HIV epidemic in rural Tanzania: 1. Design." <u>AIDS</u> 9(8): 919-926.
- Hayes, R. and L. H. Moulton (2009). Cluster Randomized Trials. Boca Raton, CRC Press.

- Helleringer, S. and H. P. Kohler (2007). "Sexual network structure and the spread of HIV in Africa: evidence from Likoma Island, Malawi." <u>AIDS</u> 21(17): 2323-2332.
- Holmes, C. B., R. Wood, et al. (2006). "CD4 decline and incidence of opportunistic infections in Cape Town, South Africa: implications for prophylaxis and treatment." <u>J Acquir Immune Defic Syndr</u> 42(4): 464-469.
- Hussey, M. A. and J. P. Hughes (2007). "Design and analysis of stepped wedge cluster randomized trials."

  <u>Contemp Clin Trials</u> 28(2): 182-191.
- Isogai, P. K., S. Rueda, et al. (2012). "Prediction of health preference values from CD4 counts in individuals with HIV." Med Decis Making: Epub 8 Aug 2012.
- Jani, I. V., N. E. Sitoe, et al. (2011). "Accurate CD4 T-cell enumeration and antiretroviral drug toxicity monitoring in primary healthcare clinics using point-of-care testing." AIDS 25(6): 807-812.
- Jelsma, J., E. Maclean, et al. (2005). "An investigation into the health-related quality of life of individuals living with HIV who are receiving HAART." <u>AIDS Care</u> 17(5): 579-588.
- Johnson, L. F., L. Alkema, et al. (2010). "A Bayesian approach to uncertainty analysis of sexually transmitted infection models." <u>Sex Transm Infect</u> 86(3): 169-174.
- Johnson, V. A., V. Calvez, et al. (2011). "2011 update of the drug resistance mutations in HIV-1." <u>Top Antivir</u> Med 19(4): 156-164.
- Joint United Nations Programme on HIV/AIDS (UNAIDS) (2010). Report on the Global AIDS Epidemic: HIV Estimates with Uncertainty Bounds. Geneva, UNAIDS.
- Jones, J. H. and M. S. Handcock (2003). "An assessment of preferential attachment as a mechanism for human sexual network formation." Proc Biol Sci 270(1520): 1123-1128.
- Kim, A. A., T. Hallett, et al. (2011). "Estimating HIV Incidence among Adults in Kenya and Uganda: A Systematic Comparison of Multiple Methods." <u>PLoS One</u> 6(3): e17535.
- Kreke, J. E., A. J. Schaefer, et al. (2004). "Simulation and critical care modeling." <u>Curr Opin Crit Care</u> 10(5): 395-398.
- Laeyendecker, O., R. Brookmeyer, et al. (2012). "Specificity of four laboratory approaches for cross-sectional HIV incidence determination: Analysis of samples from adults with known non-recent HIV infection from five African countries." <u>AIDS Res Hum Retroviruses</u>.
- Lancet (2010). "Evaluation: the top priority for global health." Lancet 375(9714): 526.
- Lara, A. M., B. N. Wakholi, et al. (2008). "Utility assessment of HIV/AIDS-related health states in HIV-infected Ugandans." <u>AIDS</u> 22 Suppl 1: S123-130.
- Leclerc, P. M., A. P. Matthews, et al. (2009). "Fitting the HIV epidemic in Zambia: a two-sex micro-simulation model." <u>PLoS One</u> 4(5): e5439.

- Little, R. J. and D. B. Rubin (2002). Statistical Analysis with Missing Data. New York, John Wiley and Sons.
- Losina, E., X. Anglaret, et al. (2006). "Impact of opportunistic diseases on chronic mortality in HIV-infected adults in Côte d'Ivoire." S Afr Med J 96(6): 526-529.
- Losina, E., Y. Chang, et al. (2008). Immunologic benefits of complete vs partial virologic suppression in patients initiating ART in Gugulethu, South Africa. Abstract 823. <u>15th Conference on Retroviruses and Opportunistic Infections</u>. Boston, MA.
- Losina, E., Y. Yazdanpanah, et al. (2007). "The independent effect of highly active antiretroviral therapy on severe opportunistic disease incidence and mortality in HIV-infected adults in Cote d'Ivoire." <u>Antivir Ther</u> 12(4): 543-551.
- Louwagie, G. M., M. O. Bachmann, et al. (2007). "Highly active antiretroviral treatment and health related quality of life in South African adults with human immunodeficiency virus infection: A cross-sectional analytical study." <a href="Mailto:BMC Public Health">BMC Public Health</a> 7: 244.
- Lundgren, J. D., A. G. Babiker, et al. (2015). "Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection." N Engl J Med 373(9): 795-807.
- Merson, M., N. Padian, et al. (2008). "Combination HIV prevention." Lancet 372(9652): 1805-1806.
- Meyer-Rath, G. and M. Over (2012). "HIV treatment as prevention: modelling the cost of antiretroviral treatment--state of the art and future directions." PLoS Med 9(7): e1001247.
- Modjarrad, K., E. Chamot, et al. (2008). "Impact of small reductions in plasma HIV RNA levels on the risk of heterosexual transmission and disease progression." <u>AIDS</u> 22(16): 2179-2185.
- Montaner, J. S., V. D. Lima, et al. (2010). "Association of highly active antiretroviral therapy coverage, population viral load, and yearly new HIV diagnoses in British Columbia, Canada: a population-based study." <u>Lancet</u> 376(9740): 532-539.
- Mtapuri-Zinyowera, S., M. Chideme, et al. (2010). "Evaluation of the PIMA point-of-care CD4 analyzer in VCT clinics in Zimbabwe." J Acquir Immune Defic Syndr 55(1): 1-7.
- Nachega, J. B., D. M. Stein, et al. (2004). "Adherence to antiretroviral therapy in HIV-infected adults in Soweto, South Africa." <u>AIDS Res Hum Retroviruses</u> 20(10): 1053-1056.
- Nei, M. and S. Kumar (2000). Molecular Evolution and Phylogenetics. New York, NY, Oxford University Press.
- Novitsky, V., H. Bussmann, et al. (2013). "Phylogenetic relatedness of circulating HIV-1C variants in Mochudi, Botswana." PLoS One 8(12): e80589.
- Novitsky, V., D. Kuhnert, et al. (2015). "Phylodynamic analysis of HIV sub-epidemics in Mochudi, Botswana." <u>Epidemics</u> 13: 44-55.
- Novitsky, V., S. Lagakos, et al. (2009). "Evolution of proviral gp120 over the first year of HIV-1 subtype C infection. NIHMSID # 79286." <u>Virology</u> 383(1): 47-59.

- Novitsky, V., S. Moyo, et al. (2014). "Impact of sampling density on the extent of HIV clustering." <u>AIDS Res</u> Hum Retroviruses 30(12): 1226-1235.
- Novitsky, V., S. Moyo, et al. (2015). "Importance of Viral Sequence Length and Number of Variable and Informative Sites in Analysis of HIV Clustering." <u>AIDS Res Hum Retroviruses</u> 31(5): 531-542.
- Novitsky, V., T. Ndung'u, et al. (2011). "Extended high viremics: a substantial fraction of individuals maintain high plasma viral RNA levels after acute HIV-1 subtype C infection." <u>AIDS</u> 25(12): 1515-1522.
- Novitsky, V., R. Wang, et al. (2011). "Evolutionary gamut of in vivo Gag substitutions during early HIV-1 subtype C infection." <u>Virology</u> 421(2): 119-128.
- Novitsky, V., R. Wang, et al. (2010). "HIV-1 subtype C-infected individuals maintaining high viral load as potential targets for the "test-and-treat" approach to reduce HIV transmission." <u>PLoS One</u> 5(4): e10148.
- Novitsky, V., R. Wang, et al. (2009). "Timing constraints of in vivo gag mutations during primary HIV-1 subtype C infection." PLoS One 4(11): e7727.
- Novitsky, V., R. Wang, et al. (2010). "Dynamics and timing of in vivo mutations at Gag residue 242 during primary HIV-1 subtype C infection." <u>Virology</u> 403(1): 37-46.
- Novitsky, V., M. Zahralban-Steele, et al. (2015). "Long-Range HIV Genotyping Using Viral RNA and Proviral DNA for Analysis of HIV Drug Resistance and HIV Clustering." J Clin Microbiol 53(8): 2581-2592.
- Padian, N. S., S. I. McCoy, et al. (2011). "Evaluation of large-scale combination HIV prevention programs: essential issues." <u>J Acquir Immune Defic Syndr</u> 58(2): e23-28.
- Paltiel, A. (2001). "Model-based drug evaluation in chronic disease: promise, pitfalls, and positioning." <u>Drug</u> Information Journal 35: 131-139.
- Phillips, A. N., D. Pillay, et al. (2011). "Effect on transmission of HIV-1 resistance of timing of implementation of viral load monitoring to determine switches from first to second-line antiretroviral regimens in resource-limited settings." <u>AIDS</u> 25(6): 843-850.
- Pitter, C., J. G. Kahn, et al. (2007). "Cost-effectiveness of cotrimoxazole prophylaxis among persons with HIV in Uganda." J Acquir Immune Defic Syndr 44(3): 336-343.
- Poole, D. and A. E. Raftery (2000). "Inference for deterministic simulation models: The Bayesian melding approach." J Am Stat Assoc 95(452): 1244-1255.
- Posada, D. (2008). "jModelTest: phylogenetic model averaging." Mol Biol Evol 25(7): 1253-1256.
- Prabhu, V. S., P. G. Farnham, et al. (2011). "Cost-effectiveness of HIV screening in STD clinics, emergency departments, and inpatient units: a model-based analysis." <u>PLoS One</u> 6(5): e19936.
- Pujades-Rodriguez, M., D. O'Brien, et al. (2008). "Second-line antiretroviral therapy in resource-limited settings: the experience of Medecins Sans Frontieres." <u>AIDS</u> 22(11): 1305-1312.

- Rajeev, K. H., B. Y. Yuvaraj, et al. (2012). "Impact of HIV/AIDS on quality of life of people living with HIV/AIDS in Chitradurga district, Karnataka." <u>Indian J Public Health</u> 56(2): 116-121.
- Rehle, T., L. Johnson, et al. (2015). "A Comparison of South African National HIV Incidence Estimates: A Critical Appraisal of Different Methods." <u>PLoS One</u> 10(7): e0133255.
- Robberstad, B. and J. A. Olsen (2010). "The health related quality of life of people living with HIV/AIDS in sub-Saharan Africa - a literature review and focus group study." <u>Cost Eff Resour Alloc</u> 8: 5.
- Rosen, S. and M. P. Fox (2011). "Retention in HIV Care between Testing and Treatment in Sub-Saharan Africa:

  A Systematic Review." <u>PLoS Med</u> 8(7): e1001056.
- Salichos, L. and A. Rokas (2013). "Inferring ancient divergences requires genes with strong phylogenetic signals." Nature 497(7449): 327-331.
- Salichos, L., A. Stamatakis, et al. (2014). "Novel information theory-based measures for quantifying incongruence among phylogenetic trees." <u>Mol Biol Evol</u> 31(5): 1261-1271.
- Saravanan, S., V. Madhavan, et al. (2012). "Darunavir Is a Good Third-Line Antiretroviral Agent for HIV Type 1Infected Patients Failing Second-Line Protease Inhibitor-Based Regimens in South India." <u>AIDS Res</u>
  Hum Retroviruses.
- Schneider, K., T. Puthanakit, et al. (2011). "Economic evaluation of monitoring virologic responses to antiretroviral therapy in HIV-infected children in resource-limited settings." AIDS 25(9): 1143-1151.
- Seyler, C., C. Adje-Toure, et al. (2007). "Impact of genotypic drug resistance mutations on clinical and immunological outcomes in HIV-infected adults on HAART in West Africa." <u>AIDS</u> 21(9): 1157-1164.
- Shapiro, R. L., M. D. Hughes, et al. (2010). "Antiretroviral regimens in pregnancy and breast-feeding in Botswana." N Engl J Med 362(24): 2282-2294.
- Simpson, K. N., M. P. Luo, et al. (2004). "Cost-effectiveness of lopinavir/ritonavir versus nelfinavir as the first-line highly active antiretroviral therapy regimen for HIV infection." <u>HIV Clin Trials</u> 5(5): 294-304.
- Society for Medical Decision Making and International Society for Pharmacoeconomics and Outcomes

  Research. "Joint modeling good research practices task force." Retrieved December 30, 2012, from <a href="http://www.ispor.org/taskforces/GRPModelingTf.asp">http://www.ispor.org/taskforces/GRPModelingTf.asp</a>.
- Stamatakis, A. (2006). "RAxML-VI-HPC: maximum likelihood-based phylogenetic analyses with thousands of taxa and mixed models." <u>Bioinformatics</u> 22(21): 2688-2690.
- Stamatakis, A. (2014). "RAxML version 8: a tool for phylogenetic analysis and post-analysis of large phylogenies." Bioinformatics 30(9): 1312-1313.
- Stover, J., L. Bollinger, et al. (2011). "Estimating the Impact and Cost of the WHO 2010 Recommendations for Antiretroviral Therapy." AIDS Res Treat 2011: 738271.

- Stover, J., B. Fidzani, et al. (2008). "Estimated HIV trends and program effects in Botswana." <u>PLoS One</u> 3(11): e3729.
- Stover, J., E. L. Korenromp, et al. (2011). "Long-term costs and health impact of continued global fund support for antiretroviral therapy." <u>PLoS One</u> 6(6): e21048.
- Sullivan, P. W., W. F. Lawrence, et al. (2005). "A national catalog of preference-based scores for chronic conditions in the United States." <u>Med Care</u> 43(7): 736-749.
- Tanser, F., T. Bärnighausen, et al. (2013). "High coverage of ART associated with decline in risk of HIV acquisition in rural KwaZulu-Natal, South Africa." <u>Science</u> 339(6122): 966-971.
- Tengs, T. O. and T. H. Lin (2002). "A meta-analysis of utility estimates for HIV/AIDS." Med Decis Making 22(6): 475-481.
- Tran, B. X., A. Ohinmaa, et al. (2012). "Quality of life profile and psychometric properties of the EQ-5D-5L in HIV/AIDS patients." Health Qual Life Outcomes 10(1): 132.
- Tsiatis, A. A. (2006). Semiparametric Theory and Missing Data. New York, Springer.
- Uhler, L. M., N. Kumarasamy, et al. (2010). "Cost-effectiveness of HIV testing referral strategies among tuberculosis patients in India." PLoS One 5(9).
- UNAIDS (2010). "Global Report: UNAIDS Report on the Global AIDS Epidemic. Available at: <a href="http://www.unaids.org/globalreport/global\_report.htm">http://www.unaids.org/globalreport/global\_report.htm</a>. Accessed February 2012.".
- UNAIDS. (2011). "Manual for costing HIV facilities and services." Retrieved December 14, 2012, from <a href="http://www.unaids.org/en/media/unaids/contentassets/documents/document/2011/20110523\_ma">http://www.unaids.org/en/media/unaids/contentassets/documents/document/2011/20110523\_ma</a> <a href="mailto:nual-costing-HIV">nual-costing-HIV facilities\_en.pdf</a>.
- UNAIDS (2013). WHO/UNAIDS Technical Update on HIV Incidence Assays for Surveillance and Epidemic Monitoring. Geneva, Joint United Nations Programme on HIV/AIDS: 6 pages.
- UNAIDS (2014). 90-90-90: An ambitious treatment target to help end the AIDS epidemic. Geneva.
- Ventelou, B., Y. Arrighi, et al. (2012). "The macroeconomic consequences of renouncing to universal access to antiretroviral treatment for HIV in Africa: a micro-simulation model." <u>PLoS One</u> 7(4): e34101.
- Walensky, R. P., E. L. Ross, et al. (2012). The cost-effectiveness of treatment as prevention: analysis of the HPTN 052 trial. Abstract FRLBC01. XIX International AIDS Conference. Washington DC, USA.
- Walensky, R. P., R. Wood, et al. (2008). "Scaling up antiretroviral therapy in South Africa: the impact of speed on survival." <u>J Infect Dis</u> 197(9): 1324-1332.
- Wallis, C. L., M. A. Papathanasopoulos, et al. (2010). "Affordable in-house antiretroviral drug resistance assay with good performance in non-subtype B HIV-1." <u>J Virol Methods</u> 163(2): 505-508.
- Wandeler, G., O. Keiser, et al. (2012). "Tenofovir in second-line ART in Zambia and South Africa: collaborative analysis of cohort studies." <u>J Acquir Immune Defic Syndr</u> 61(1): 41-48.

- Wang, B., N. Kumarasamy, et al. (2006). <u>Incidence of opportunistic infections (OIs) within specific CD4 strata in HIV-infected patients in Southern India. Abstract WEPE0279</u>. XVI International AIDS Conference, Toronto, Canada.
- Weinstein, M. C., B. O'Brien, et al. (2003). "Principles of good practice for decision analytic modeling in health-care evaluation: report of the ISPOR Task Force on Good Research Practices--Modeling Studies." <u>Value</u>
  Health 6(1): 9-17.
- Weinstein, M. C., J. E. Siegel, et al. (1996). "Recommendations of the Panel on Cost-effectiveness in Health and Medicine." <u>JAMA</u> 276(15): 1253-1258.
- World Health Organization (2011). When and how to use assays for recent infection to estimate HIV incidence at a population level. UNAIDS/WHO Working Group on Global HIV/AIDS and STI Surveillance. Geneva, World Health Organization: 48 pages.
- World Health Organization (2015). Guideline on When to Start Antiretroviral Therapy and on Pre-exposure Prophylaxis for HIV. Geneva, Switzerland.
- World Health Organization Division of Mental Health and Prevention of Substance Abuse (1997). WHOQOL: Measuring Quality of Life. Geneva, Switzerland.
- Wouters, E., W. Van Damme, et al. (2008). "Impact of baseline health and community support on antiretroviral treatment outcomes in HIV patients in South Africa." <u>AIDS</u> 22(18): 2545-2548.
- Zhang, Z., L. Sun, et al. (2007). "Regression analysis of failure time data with informative interval censoring."

  <u>Stat Med</u> 26(12): 2533-2546.
- Zhou, Z., N. Wagar, et al. (2011). "Optimization of a low cost and broadly sensitive genotyping assay for HIV-1 drug resistance surveillance and monitoring in resource-limited settings." PLoS One 6(11): e28184.
- Zimpel, R. R. and M. P. Fleck (2007). "Quality of life in HIV-positive Brazilians: application and validation of the WHOQOL-HIV, Brazilian version." <u>AIDS Care</u> 19(7): 923-930.

# Botswana Combination Prevention Project (BCPP) Intervention Protocol (Protocol #3)

# Implementation, Monitoring, and Evaluation of a Combination of HIV Prevention Interventions in Rural and Peri-Urban Communities in Botswana

# Version 6.0

**September 22, 2017** 

# **Collaborating Institutions:**

Botswana Ministry of Health (MOH)
Harvard T. H. Chan School of Public Health (Harvard Chan School)
U.S. Centers for Disease Control and Prevention (CDC)

# Funded by:

The United States President's Emergency Plan for AIDS Relief (PEPFAR) through United States Centers for Disease Control and Prevention (CDC)

#### PRINCIPAL INVESTIGATORS:

# Janet Moore, PhD

Branch Chief, HIV Prevention Branch

Division of Global HIV/AIDS (DGHA), Center for Global Health (CGH)

United States Centers for Disease Control and Prevention (CDC)

Address: 1600 Clifton Road, Atlanta, GA, 30333, U.S.A

Email: jym3@cdc.gov Office Phone: 404.639.8954

# Refeletswe Lebelonyane, MD

Combination Prevention Coordinator, MOH Ministry of Health, Botswana Government Enclave Plot No. 54609 Gaborone, Botswana

Email: rlebelonyane@gov.bw

# Shenaaz El Halabi, (PS) MPH

Permanent Secretary Botswana Ministry of Health

Address: Private Bag 0038, Gaborone, Botswana

Email: sel-halabi@gov.bw Office Phone: +267-363-2069

# Pamela Bachanas, PhD

Behavioral Scientist, HIV Prevention Branch

Division of Global HIV/AIDS (DGHA), Center for Global Health (CGH) United States Centers for Disease Control and Prevention (CDC)

Address: 1600 Clifton Road, Atlanta, GA, 30333, U.S.A

Email: ddt6@cdc.gov Office Phone: 404.639.8110

# **ROLES OF INSTITUTIONS AND PRINCIPAL INVESTIGATORS**

**Institutions**: Close coordination between MOH, CDC, HSPH, BHP, and other implementing partners is needed to ensure seamless implementation of research and program activities. MOH and CDC will lead and ultimately be responsible the Intervention Protocol and HSPH and BHP will lead the Evaluation Protocol.

**Principal Investigators:** 

**Janet Moore/ Pamela Bachanas:** CDC (PIs) responsible for preparation and design of the study protocol, monitoring of study progress, creation and monitoring of research budgets, and preparation of monthly progress reports.

**Refeletswe Lebelonyane/ Shenaaz El Halabi:** MOH Co-Principal Investigator (Co-PI) responsible for protocol review and in-country implementation oversight.

# **CO-INVESTIGATOR LISTS BY INSTITUTION**

# Botswana Ministry of Health (MOH), Gaborone, Botswana

| Name | Role | Contact Email |
|---|---|---|
| Ms. Dinah Ramaabya (Nursing) | ARV Program | dramaabya@gov.bw |
| Ms. Chipo Phetlo (Nursing) | PMTCT | cphetlo@gov.bw |
| Mr. S. Makathaye, Dip Health Educ. | BCIC | smalathaye@gov.bw |
| Mr. C. Ntsuape, BEd (Nursing Educ) | SMC | ontsuape@gov.bw |
| Ms. Nokuthula Manjingo (Nursing) | HIV Testing & Counselling | mmajingo@gov.bw |
| Dr. Joe Theu ((Medical Officer) | Clinical Care | jtheu@gov.bw_ |

# Centers for Disease Control and Prevention (CDC), Atlanta, GA, USA, and Gaborone, Botswana

| Name | Role | Contact Email |
|---|---|---|
| Elliot Raizes, MD | Clinical Consultant | gwq0@cdc.gov |
| Ebi Bile, BSc. MA, DU | In-country Lab Oversight | efb6@bw.cdc.gov |
| Peter Fonjungo, PhD | HQ Lab Oversight | pdf4@cdc.gov |
| Sherri Pals, PhD | Statistics | sfv3@cdc.gov |
| Chunfu Yang, PhD | Laboratory | cxy0@cdc.gov |
| Mary Grace Alwano | In Country HTC/ LTC Project Coordinator | mea9@bw.cdc.gov |
| Stephanie Behel, MPH | HTC and LTC | zmd7@cdc.gov |
| Naomi Bock, MD | Voluntary Medical MC | neb2@cdc.gov |
| Stephanie Davis, MD, MPH | Voluntary Medical MC | vic6@cdc.gov |
| Lisa Block, MS | Project Manager | kwk5@cdc.gov |
| Lisa Mills, MD | Co-investigator | loj7@cdc.gov |
| William Abrams | <b>Program Administration</b> | hvf8@cdc.gov |
| Arielle Lasry PhD | HTC Costing | ftn9@cdc.gov |

# Harvard T. H. Chan School of Public Health, Boston, MA, USA

| Name | Role | Contact Email |
|---|---|---|
| Myron Essex, DVM, PhD | Co-Investigator | messex@hsph.harvard.edu |
| Eric Tchetgen, PhD | Statistics and Epidemiology | etchetge@hsph.harvard.edu |
| Scott Dryden-Peterson, MD | Treatment and PMTCT | $scott\_peters on @post.harvard.edu$ |
| Shahin Lockman, MD, MSc | Treatment and PMTCT | slockman@hsph.harvard.edu |
| Rebeca Plank, MD | SMC | rplank@partners.org |
| Molly Pretorius Holme, MSc | Research operations | mpretori@hsph.harvard.edu |
| Roger Shapiro, MD, MPH | Treatment and PMTCT | rshapiro@hsph.harvard.edu |
| Kate Powis, MD, MPH | Research Operations, | kpowis@mgh.harvard.edu |
| Rate I Owis, IVID, IVII II | Treatment and PMTCT | kpowis@ingil.narvara.eau |

# Botswana-Harvard AIDS Institute Partnership (BHP), Gaborone, Botswana

| Role | Contact Email |
|---|---|
| Treatment and PMTCT, | tgaolathe@bhp.org.bw |
| Field research operations | |
| BHP research operations | jmakhema@bhp.org.bw |
| Lab | smoyo@bhp.org.bw |
| Community mobilization and | mmmalane@bhp.org.bw |
| research operations | minimalane@bilp.org.bw |
| Research data systems | ewidenfelt@bhp.org.bw |
| | Treatment and PMTCT, Field research operations BHP research operations Lab Community mobilization and research operations |

# TABLE OF CONTENTS

| Principal Investigators2 |
|---|
| List of Co-Investigators3 |
| Table of Contents |
| List of Tables and Figures |
| List of Acronyms and Appreviations |
| Intervention Protocol Synopisis10 |
| 1.0 INTRODUCTION |
| 1.1 Epidemic in Botswana |
| 1.2 Combination Prevention Interventions |
| 1.3 Antiretroviral Treatment as a Component of the Combination Prevention Package |
| 1.4 Proposed Combination Prevention (CP) Package |
| 1.5 Relationship Between Intervention Study Design and Impact Evaluation |
| 2.0 STUDY OBJECTIVES |
| 3.0 OVERVIEW OF STUDY METHODS16 |
| 4.0 STUDY POPULATIONS |
| 4.1 Selection of Study Communities |
| 4.2 Matching of Study Communities |
| 4.3 Eligibility of Community Members |
| 4.4 Enhancement of Services in all Study Communities |
| 4.5 Eligibility Criteria for Inclusion in Interventions in CP Communities |
| 4.6 Rationale for Exclusion in Interventions in CP Communities |
| 5.0 SAMPLE SIZE AND SAMPLE SELECTION METHODS21 |
| 6.0 INTERVENTION PROCEDURES22 |
| 6.1 Overview of Intervention Strategy |
| 6.2 Stakeholder Involvement, Community Engagement, and Community Mobilization |
| 6.3 HIV Testing and Counseling (HTC) |
| 6.4 Linkage to HIV Care and Treatment |
| 6.5 Male Circumcision (MC) |
| 6.6 Identification, Linkage, and Treatment of HIV+ Pregnant Women |
| 6.7 HIV Care and Treatment |
| 7.0 LABORATORY METHODS32 |
| 7.1 Overview of Laboratory Methods |
| 7.2 Training of Laboratory Personnel |
| 7.3 Specimen Collection, Transport, and Processing |

| 7.4 Laboratory Testing for HTC Campaigns |
|---|
| 7.5 Laboratory Testing for IDCC Patients |
| 7.6 Quality Assurance |
| 7.7 Biosafety and Waste Management |
| 7.8 Specimen Storage and Shipment |
| 8.0 DATA SYSTEMS AND MANAGEMENT35 |
| 8.1 Data Collection, Capture, and Flow |
| 8.2 Data Security |
| 8.3 Data Quality |
| 8.4 Confidentiality of data |
| 9.0 DATA AND ANALYSIS PLANS4 |
| 9.1 HIV Testing and Counseling and Linkage to Care |
| 9.2 Care and Treatment |
| 9.3 PMTCT Services |
| 9.4 Male Circumcision |
| 9.5 Analysis Plans |
| 10.0 ETHICAL CONSIDERATIONS |
| 10.1 Ethical Review |
| 10.2 Informed Consent |
| 10.3 Risks |
| 10.4 Benefits of Research Participation |
| 10.5 Confidentiality |
| 10.6 Protocol Compliance and Compliance with UN Convention on the Rights of the Child |
| 10.7 Future Use of Stored Samples |
| 11.0 STUDY SAFETY AND MONITORING PLAN49 |
| 11.1 Reporting Adverse Events |
| 11.2 Data Safety and Monitoring Board (DSMB) |
| 11.3 Protocol Violations |
| 11.4 Monitoring Plan |
| 12.0 ADMINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION |
| 12.1 Study Records and Document Retention |
| 12.2 Information Dissemination and Publication Plan |
| 13 O REFERENCES |

# **APPENDICES:**

# **Cross-Protocol Appendices:**

Appendix C2 A. List of Study Communities and Matching Criteria for Community Pairs

B. Back-up Communities in Selected 30 Communities Decline, unavailable or

deemed unsuitable for study inclusion

Figure A: Map of Study Communities in Three Regions

Figure B: Map of Study Communities in the Southern Region Figure C: Map of Study Communities in the Central Region Figure D: Map of Study Communities in the Northern Region

Appendix C3 Size of Study Populations
Appendix C4 Data Safety Monitoring Plan

Protocol 3 Appendix:

Appendix P1 Summary of Variables to be Collected for Ya Tsie Protocol 3

\_\_\_\_\_\_

# **LIST OF TABLES AND FIGURES**

Figure 1: Data Flow for Combination Prevention Communities

**Table 1:** Precision for 95% confidence intervals for uptake of CP interventions in CP communities

Table 2: BCPP Key Indicators

 Table 3: Summary of approach to consent for various components of the study

# **ACRONYMS AND ABBREVIATIONS**

AE adverse event

AIDS acquired immunodeficiency syndrome

AHS annual household surveys (follow-up visits of the BHS and HIC)

ANC antenatal clinic (or care)

ART antiretroviral treatment (or therapy)

ARV antiretroviral (drug)

BCPP Botswana Combination Prevention Project
BHHRL Botswana—Harvard HIV Reference Laboratory
BHP Botswana—Harvard AIDS Institute Partnership

BHS baseline household survey

CDC Centers for Disease Control and Prevention

CI confidence interval CP combination prevention

CPC combination prevention community

CRT community-randomized trial
DSMB Data Safety Monitoring Board
ECC enhanced care communities

ELISA enzyme-linked immunosorbent assay

ESS end of study survey

ETC expanded treatment cohort

HIC HIV incidence cohort

HIV-1 RNA human immunodeficiency virus
HIV-1 RNA load in plasma, viral load

HIVDR HIV drug resistance

HTC HIV testing and counseling

HVL high viral load

IAS International AIDS Society
IDCC infectious disease care clinic

IPMS integrated patient management system

IRB institutional review board

LFT liver function test
LTC linkage-to-care
MC male circumcision

M&E monitoring and evaluation

MOH Ministry of Health

MTCT mother-to-child (HIV) transmission
OHRP Office for Human Research Protections

OI opportunistic infection

Option B+ indefinite continuation of ART for women who start ART for PMTCT

PEP post-exposure prophylaxis

PEPFAR President's Emergency Plan for AIDS Relief

PII personally identifiable information

PIMS patient information management system

PMTCT prevention of mother-to-child (HIV) transmission

PLHIV people living with HIV

POC point-of-care

POB pregnant/pregnancy or breastfeeding

QA quality assurance

QC quality control
RHT Routine HIV testing
SAE serious adverse event
SD standard deviation

SMC safe male circumcision (Botswana government initiative)

SMS short message service
SOC standard of care
SoE schedule of events

SOP standard operating procedure

study arm a group of 15 communities that is randomized to receive either standard of care or

study interventions with respect to HIV prevention measures

TB tuberculosis
UN United Nations

UNAIDS Joint United Nations Program on HIV/AIDS

UTT Universal Test and Treat

VDC village development committee

VF virologic failure VL viral load

VPN virtual private network WHO World Health Organization

# **BCPP Intervention Protocol (#3)**

# **Protocol Synopsis**

**Overview:** The BCPP study is composed of 2 active interlocking protocols, the Evaluation Protocol (1) and the Intervention Protocol (3). The Closed Clinical Cohort Protocol (Protocol 2) was withdrawn in 2015. An overview of the overarching BCPP study is provided in the BCPP Overall Schema located in the Evaluation Protocol.

# **Primary Objective of Protocol 3**

1) To implement the combination prevention (CP) intervention package in combination prevention communities (CPC) and describe uptake of these interventions in CPCs (expanded HIV Testing and Counseling (HTC), strengthened Male Circumcision (MC), expanded HIV Care and Treatment, and strengthened PMTCT services).

# **Secondary Objectives of Protocol 3**

- 1) To describe retention in the clinical cascade of care from HIV diagnosis to viral suppression among all HIV-infected persons.
- 2) To describe uptake of expanded antiretroviral treatment (ART) and clinical outcomes including viral suppression among HIV-positive persons receiving expanded ART.
- 3) To examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions.
- 4) To examine demographic factors, including community of residence, that affect access to health care services.

# **Study Design:**

The BCPP study is a pair-matched community-randomized trial. This protocol describes the programmatic interventions, including expanded ART, and program monitoring activities that will be conducted as part of the larger BCPP project.

# **Study Population:**

Thirty community clusters were selected from three geographic regions in Botswana. Prerandomization, community pairs were matched on community characteristics thought to be associated with the outcome of interest of the BCPP (HIV incidence) to improve balance between arms and statistical efficiency. The average total population size of each of the targeted communities is 6,000 (range 2,400 - 12,000), giving a total population across all 30 communities of about 180,800, of whom about 105,000 are adults aged 16-64.

# **Study Procedures:**

Matched community pairs (15 communities per arm) were randomized 1:1 to Enhanced Care (ECC; Comparison) or Combination Prevention (CPC; Intervention) arms prior to the baseline household survey (BHS) that is conducted as part of the BCPP Evaluation Protocol. Initiation of intervention activities in the CPCs begin immediately following completion of enrollment in the BHS and continue for the duration of the study. CPCs receive the combination prevention intervention package, which includes strengthened HTC, MC linkage, PMTCT services, and expanded HIV care and treatment for HIV-infected persons 16-64 years. In addition, expanded ART for existing HIV-infected community clinic

patients will be offered in the CPCs. Routinely collected clinical data will be used to assess the clinical outcomes for all HIV positive patients.

**Study Duration:** All study activities will occur over a period of approximately 60 months.

# 1.0 INTRODUCTION AND BACKGROUND

# 1.1 Epidemic in Botswana

Thirty years into the global HIV pandemic, HIV prevalence and incidence remain high in sub-Saharan Africa. Although this region represents only 12% of the world's population, it accounts for approximately 67% of the world's 34 million HIV-infected persons, and annually, about 70% of the world's 2.7 million new infections occur in this region (UNAIDS 2010). Despite substantial progress in providing HIV treatment and prevention of mother-to-child transmission services (PMTCT) to its citizens, an estimated 25% of adult residents of Botswana are HIV-infected, the second highest adult HIV prevalence in the world, and about 14,000 persons are newly infected with HIV annually, the third highest national HIV incidence rate globally (UNAIDS 2010).

# 1.2 Combination Prevention Interventions

In the past five years several HIV prevention interventions have proven to be highly effective at reducing transmission of HIV and have offered hope for containing and possibly reversing epidemics in sub-Saharan Africa. For HIV-negative men, MC has been shown to significantly reduce HIV acquisition from HIV-infected female partners. Three randomized controlled trials of circumcision, involving more than 10,000 men in sub-Saharan Africa, demonstrated a 60% reduction in HIV acquisition risk (Auvert, Taljaard et al. 2005, Bailey, Moses et al. 2007, Gray, Kigozi et al. 2007). Additionally, antiretroviral treatment (ART) of HIV-infected persons has been shown to reduce viral load (VL) and consequently the risk of HIV transmission to uninfected partners in sero-discordant couples by as much as 96% (Cohen, Chen et al. 2011). Similarly, the use of antiretrovirals to prevent transmission of HIV from infected mothers to their infants during pregnancy, birth, and breastfeeding can reduce transmission to below 5% (Mahy, Stover et al. 2010; Shapiro, Hughs et al. 2013).

Despite considerable success in scaling up these interventions in many sub-Saharan African countries, especially those supported by the U.S. President's Emergency Plan for AIDS Relief (PEPFAR), adult HIV incidence has remained high (>1%) in many regions in Southern Africa (Botswana, Swaziland, Lesotho, Kwa-Zulu Natal in South Africa, and Southern Mozambique). Multiple factors may account for high HIV incidence in this part of the world. Firstly, viral characteristics of HIV-1 subtype C, endemic in Southern Africa, may make it more infectious than other viral subtypes (Novitsky, Wang et al. 2010, Novitsky, Ndung'u et al. 2011). For example, recent evidence suggests that about one third of persons infected with HIV-1 sub-type C, maintain very high viral loads (VL>50,000 copies/ml) for more than 6 months after sero-conversion. In contrast, viral load following HIV-1 subtype B infection (the prevalent subtype in the United States and Europe) resolves to a steady-state viral set point below 50,000 copies/ml in almost all individuals within four to six months (Daar, Moudgil et al. 1991, Mellors, Munoz et al. 1997, Kaufmann, Cunningham et al. 1998, Little, McLean et al. 1999).

Secondly, the scale and quality of the HIV prevention interventions may have been insufficient to reduce HIV incidence among adults in Southern Africa to levels observed in other parts of the world. For example, the main mechanism by which scale-up of HTC and antiretroviral therapy reduces HIV transmission risk in the community, is by reducing viral load in resident HIV-infected persons, ideally to undetectable levels (VL<400 copies/ml). Studies have suggested that every 0.5 log reduction in an individual's HIV-1 viral load is equivalent to a 40% reduction in individual HIV transmission risk

(Modjarrad, Chamot et al. 2008), and once the viral load is fully suppressed (VL <400 copies/ml) individual HIV transmission risk is virtually zero (Attia, Egger et al. 2009). Despite considerable scale-up of access to HTC and ART, poor retention of HIV-infected persons in the HIV care and treatment cascade from diagnosis to ART follow-up (Rosen and Fox 2011), has mitigated the ability of HTC and HIV care and treatment programs in Southern Africa to reduce the prevalence of HIV-infected persons with detectable viral loads (VL>400 copies/ml). In a meta-analysis of pre-ART retention in Africa, Rosen et al. reported that only 59% of newly diagnosed adults are successfully linked to HIV care and treatment services, only 46% are retained from initial registration and staging at the facility to ARTeligibility, and only 68% are retained from ART eligibility to ART initiation (Rosen and Fox 2011). Of those adults who initiate ART, ~30% are no longer on therapy by 3 years of follow-up, with most of those no longer in care considered lost to follow-up (Fox and Rosen 2010). Therefore, even if 50% of HIV-infected adults in Botswana know their HIV status (BAIS 2008), a considerably lower proportion have a suppressed viral load (Gardner, McLees et al. 2011). The remaining HIV-infected adults with unsuppressed viral load are still infectious and spreading virus in the community. Achieving high coverage of MC among HIV-negative males has also been challenging with most countries, including Botswana, unable to meet ambitious 80% coverage targets to date (Curran, Njeuhmeli et al. 2011).

In summary, despite having the tools to end the HIV epidemic (Fauci and Folkers 2012), insufficient scale, quality, and coordination of prevention interventions have significantly limited southern Africa's ability to sufficiently curb the HIV epidemic. This has led public health experts to call for a "combination prevention" strategy that involves implementing multiple prevention interventions with known efficacy in a geographic area at a scale, quality, and intensity to impact the epidemic (Merson, Padian et al. 2008, Piot, Bartos et al. 2008). Although most experts agree that synchronized implementation of a combination of prevention interventions is needed, there remains considerable debate about what components should be included in the essential combination prevention package (Merson, Padian et al. 2008, Halperin 2009). Four evidence-based interventions (HTC, ART, MC and PMTCT) are recommended for scale-up by almost all prevention experts and will form the cornerstone of the combination prevention package proposed as part of this project (see Section 1.4 below).

# 1.3 ART as a Component of the Combination Prevention Package

Data show that higher levels of HIV-1 RNA (viral load) are independently associated with both higher rates of HIV transmission and more rapid HIV clinical disease progression and CD4 decline. This study therefore originally included the use of a modified "treatment as prevention" approach that targeted not only those adults who need ART for their own health, but also those adults who are most likely to perpetuate HIV transmission within the community (those with viral load  $\geq$ 10,000 copies/ml). At the time of designing the BCPP in 2012 there was strong experimental evidence supporting initiation of ART at CD4 $\leq$ 350 cells/µL, or WHO Stage III/IV, but conclusive experimental evidence supporting patient benefit of ART initiation at higher CD4 counts, especially CD4 >500 cells/µL was lacking.

The 2013 WHO guidelines recommended initiation of ART in all HIV-infected adults with CD4 $\leq$ 500 cells/µL regardless of clinical stage. In an attempt to provide programmatic data for an anticipated change in CD4 threshold for ART initiation in Botswana and to enhance the power of the study to answer its primary objective, the threshold for ART initiation in the Combination Prevention arm was modified in early 2015 (from CD4 $\leq$ 350 to CD4 $\leq$ 500 regardless of viral load, in addition to offering expanded ART to persons with CD4>500 and viral load  $\geq$ 10,000).

Shortly thereafter, in July 2015, the WHO announced that it would revise ART guidelines to recommend universal treatment (regardless of CD4 count or HIV disease severity). The WHO's plans were informed by results from two clinical ART trials. One, the START trial, reported that early drug treatment of people with HIV cut their risk of serious illness or death by 57% (Lundgren, Babiker et al. 2015). Another, the TEMPRANO study, released findings that early ART significantly decreased morbidity overall and when restricted to patients with baseline CD4>500 cells/µL (Danel, Moh et al. 2015). WHO published an early release guideline on when to start ART and on pre-exposure prophylaxis for HIV in September 2015 (World Health Organization 2015). The BCPP study team, with the support of the DSMB and funder, is revising the intervention treatment initiation criteria once more to take these new results and WHO guidelines into account. Universal Test and Treat (UTT) is therefore included in the combination prevention package with version 4.0 of the protocols.

In June 2016, Botswana treatment guidelines changed to UTT. All PLHIV living within the Enhanced Care communities (ECC) are now eligible to receive ART according to these updated Botswana national guidelines. Residents in the Combination Prevention communities will also continue to receive universal treatment as prevention.

Through additional modeling, the study team has adjusted effect size and power calculations to reflect a move to UTT in both the Combination Prevention and Enhanced Care arms, using a range of roll-out timelines. This revised modeling also uses estimates of coverage (by HTC, LTC, ART, MC) that are consistent with what has been observed in BCPP thus far, rather than using the higher coverage "targets". Model-based estimates suggest that the impact of a change in treatment policy on the power to detect a difference in cumulative incidence (the primary objective of BCPP) may still yield at least 70% power (Protocol 1, v4.0, section 5.1.1), but the impact depends on the exact nature and timing of the implementation of changes in policy as well as other prevailing conditions. The retention of this level of power even with Enhanced Care communities moving to expanded access to ART is at least in part attributable to the fact that BCPP is implementing multiple HIV prevention interventions (including higher HTC coverage, linkage to HIV care/treatment, etc.).

# 1.4. Proposed Combination Prevention (CP) Package

In version 4.0 of this protocol, the combination package includes universal treatment of all PLHIV along with a package of interventions that are designed to: 1) Identify all HIV-infected adults in CP communities, 2) reduce barriers to ART initiation, 3) support adherence and retention on ART, 4) increase capacity of clinics to support aggressive ART scale-up, and 5) enhance the use of both individual and clinic-level data to ensure maintenance of quality of HIV care and treatment.

The revised combination prevention package for this project includes:

- Rapid scale-up of HTC services, with a target of ensuring ≥90% of HIV-infected adults aged 16-64 have documentation of their HIV-infected status.
- Rapid scale-up of universal ART for all HIV-infected adults, with a target of ensuring that <u>></u>93% of adults diagnosed with HIV infection are receiving ART.
- Rapid scale-up of retention in care and adherence interventions, with a target of ensuring that >95% of HIV-infected adults receiving ART are virally suppressed with HIV-1 RNA < 400 copies per ML.

- Scale-up of linkage to MC services, with a target of ensuring <u>></u>60% of HIV-negative men (aged 16–49) are circumcised.
- Rapid strengthening of PMTCT services, with a target of ensuring >90% of women initiated on indefinite ART (Option B+) during pregnancy remain in care and on treatment post-delivery.

The targets for intervention communities in this version of the Protocol have been revised from the targets in Protocol 3, version 3.0. Targets for ART initiation and viral load suppression have been raised based on the higher than expected baseline levels of ART initiation and viral load suppression coverage as measured in BCPP BHS and HTC campaign. The MC target has been lowered from 80% to 60%. This change is in accordance with the DSMB's 2013 recommendation based on concerns that the 80% target might not be realistic; results to date support these expectations.

To reach stated scale-up targets (cumulative over 3 years) several service uptake initiatives will be implemented, including (1) community mobilization to encourage HTC and MC uptake, (2) targeted HIV testing to include hard-to- reach populations, (3) strengthening linkage to care, treatment and/or PMTCT services for known HIV-infected adults not in care and newly diagnosed HIV-infected adults, (4) strengthening linkage to MC services for HIV-negative or HIV-unknown status males identified at HTC services, (5) strengthening retention in care and adherence to ART services at clinics (6) expansion and strengthening of HTC, ART, PMTCT services, and MC services through recruitment of additional health care personnel and counselors, and (7) strengthened monitoring and evaluation of prevention, care and treatment programs to ensure stated targets are reached.

Adults aged 16-64 will be targeted for service uptake because recent, nationally representative surveys of HIV prevalence and incidence (BAIS 2008) suggest that HIV incidence remains high (>1%) throughout this age group. Modeling exercises suggest that meeting scale-up targets by the end of two years of program implementation, and maintaining treatment coverage thereafter, could result in community HIV incidence reductions of 40% by the end of three years of implementation.

# 1.5. Relationship Between Intervention Study Design and Impact Evaluation

A separate protocol (BCPP Evaluation, Protocol #1) describes in detail the proposed plans for evaluating the impact of the combination prevention (CP) package on adult population level HIV incidence. In brief, a randomized design was proposed to provide experimental evidence of CP package impact and because population-level HIV incidence is the outcome of interest, a community (rather than individual) randomized trial is proposed. Thirty study communities have been selected and matched into pairs. Pair-matching is done to improve balance between study arms and statistical efficiency (Hayes and Moulton 2009). Communities within pairs were randomized to Combination Prevention Community and Enhanced Care Community (CPC and ECC) arms. Following community matching, a baseline 20% household survey (BHS) was implemented to recruit an HIV Incidence Cohort (HIC) of eligible, consenting, and HIV-negative adults aged 16-64. The HIC will be followed annually during Annual Household Survey (AHS) visits to assess cumulative HIV incidence over 30 months. Study participants who are not eligible for the HIC will also be followed annually in the AHS, to assess, in both study arms, uptake of HTC, ART, MC services and PMTCT services in each arm and to describe major health outcomes (such as death). Cumulative incidence will be compared between study arms to assess CP package impact.

Combination prevention package coverage in the community will be estimated at baseline (in the 20% BHS) and through a large end of study survey (ESS). In addition, during study conduct, progress in reaching target coverage levels will be captured from monitoring data collected as part of routine programmatic activities.

#### 2.0 STUDY OBJECTIVES

# **Primary Objective**

1) To implement the combination prevention (CP) intervention package in CPCs and describe uptake of these interventions (expanded HTC, strengthened MC, expanded HIV Care and Treatment, and strengthened PMTCT services).

# **Secondary Objectives**

- 1) To describe retention in the clinical cascade of care from HIV diagnosis to viral suppression for HIV-infected persons.
- 2) To describe uptake of expanded ART and clinical outcomes including viral suppression among HIV-positive persons receiving ART (UTT).
- 3) To examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions.
- 4) To examine demographic factors, including community of residence, that affect access to health care services.

# 3.0 OVERVIEW OF STUDY METHODS

As described in the introduction, the over-arching design is a pair-matched community-randomized trial (CRT). The full details of the CRT, including how communities were selected, how they were matched, community randomization, the BHS, enrollment of the HIV incidence cohorts (HIC), and the end of study survey (ESS), are described in the BCPP Evaluation Protocol. This protocol describes the interventions implemented in 15 communities randomly selected from the 30 study communities (*Appendix C2*), monitoring and evaluation (M&E) plans, and the program data systems.

#### **4.0 STUDY POPULATIONS**

# 4.1 Selection of Study Communities

Thirty communities (*Appendix C2*) in three geographic areas in Botswana: (1) around Gaborone in the south east, (2) around Francistown in the north east, and (3) in the region around Mahalapye, Serowe, and Palapye in the central eastern region, are included in the study. These communities were selected based on two criteria: (1) communities needed to be of sufficient size to meet sample size requirements for the HIV Incidence Cohort (described in BCPP Evaluation Protocol), and (2) implementation of the proposed combination prevention package needed to be feasible. Feasibility requirements are listed below:

# • Community Criteria

All communities must:

- Have a health center from which HIV care and treatment, PMTCT, or HTC can be provided.
- Be reachable by road via a <8 hour drive from Gaborone or Francistown. (CDC and the Ministry
  of Health have permanent, well-staffed offices in Gaborone and Francistown, while the Harvard</li>

- Chan School has a permanent office in Gaborone. This distance parameter makes the study easier to implement and monitor for quality control purposes).
- Have a clear geographic boundary such that it is reasonably easy to identify a household as either being part of, or outside of, the study community.

These inclusion criteria resulted in the exclusion of urban areas from the study. Approximately 61% of Batswana (plural noun for Botswana citizens) live in urban areas with a rate of urbanization of about 2.3% per year (annual rate of migration from rural or peri-urban regions into urban areas). Restricting the study to rural and peri-urban areas, besides being necessary for study feasibility, should not limit the generalizability of study findings to urban areas. If the combination prevention package is shown to be effective at reducing adult HIV incidence, the principle of scaling up combination prevention package coverage for prevention effectiveness should be applicable to urban settings.

The 30 study communities selected meet the criteria described above. The average total population size of each of the targeted communities is 5,855. Assuming an average community size of 5,855, we estimate a total population in all 30 study communities of about 175,664 people; 87,832 persons in the CPC arm of which ~58% of community residents are aged 16-64 (*Appendix C2/C3*). HIV prevalence among residents aged 16-64 is estimated at 25%, resulting in an estimated 25,471 HIV-infected residents aged 16-64 (12,736 per study arm).

# 4.2 Matching of Study Communities

Due to the small number of communities that can be enrolled in a community randomized trial for cost and feasibility reasons, the likelihood of imbalance of potential confounders between study arms is increased. A restricted randomization, matching, and stratification were considered as strategies to ensure balance between arms. A pair-matched design was chosen because:

- This approach is more likely than stratification to achieve balance between study arms;
- Matching has the added advantage of improving statistical efficiency compared with restricted randomization, and;
- Chosen matching covariates (see below) are quite closely correlated with the outcome of interest (adult HIV incidence), making a matched design of similar or increased statistical efficiency compared with a stratified design, even though a matched design entails greater loss of degrees of freedom.

Possible disadvantages of a pair-matched design include:

- Loss of both communities in a pair if one community drops out.
- It is not possible to assess whether the intervention effect varies between matched pairs, whereas, in a stratified design, opportunity to assess effect modification across strata would be possible.

The following matching criteria were chosen:

- Community size: Although community size in Botswana may not be associated with the outcome
  of interest (HIV incidence), achieving sample size balance between arms improves statistical
  efficiency.
- Baseline Access to Health Services including ART: Access to ART is associated with HIV incidence (Montaner, Lima et al. 2010, Tanser, Bärnighausen et al. 2012). Although some communities within matched pairs have access to primary care clinics and others have access to primary care hospitals,

in Botswana this does not appear to represent a significantly different level of access to health services.

- Age structure: Adult HIV prevalence and incidence are correlated with adult age (Central Statistics Office 2009). Age structures are very similar within the study community pairs. If we use the proportion of adults (16-64) who are in the highest risk for HIV infection (25-34) as an indicator of age structure, the median difference in this proportion is 2% (range 0-7%). [Note: we do not have age structure data for Gumare, Shakawe, Mandunyane, or Mmadinare, but based on the age structure of the other 26 selected communities, do not expect any significant differences in age structure within the matched pairs].
- Geographic location as measured by proximity to major urban centers (Hayes, Mosha et al. 1995).
   Geographic locations of communities within pairs, as estimated by average distance to the nearest large towns, are quite similar. For example, across 30 communities, the range of average distances to nearby urban centers ranges from 18-380 kilometers. However, following matching, the median difference in distance to an urban center between communities in a matched pair is 20 kilometers (range 3-150).

Access to community-specific measures of HIV prevalence [e.g., HIV prevalence measured from antenatal care (ANC) clinics] were not available prior to community selection/randomization. Previous successful pair-matched CRTs (Hayes, Mosha et al. 1995) where HIV incidence was the outcome of interest have also addressed the problem of absent baseline HIV prevalence estimates by using geographic location and other proxies of HIV prevalence as matching criteria.

- **4.3 Eligibility of Community Members** The following definitions of the study community will be used in the protocol:
- <u>Botswana Citizen:</u> A Botswana citizen is anyone who can produce proof of Botswana citizenship. (Usually this is the Omang number or Omang application receipt). The Omang number is needed in Botswana to access routine government services. It is anticipated, based on a community survey in Mochudi, and the 2011 census (Census 2011), that less than 3% of residents will be non-citizens.
- <u>Spouse of Botswana citizen</u>: A spouse of a Botswana citizen is a person who can produce evidence
  of being married to a Botswana citizen, usually a marriage certificate, and is therefore eligible to
  receive free medical services in Botswana.
- <u>Permanent study community resident:</u> An individual who reports spending on average ≥14 nights/month each month in that community for the past 12 months or an individual who recently moved into the community and reports spending on average ≥14 nights each month since arriving.
- <u>Part-time study community resident:</u> An individual who reports spending 3—13 nights (on average) each month in that community for the past 12 months or an individual who recently moved into the community and reports spending on average 3-13 nights each month since arriving.

• <u>Non-residents:</u> An individual who reports living outside of the community but is receiving treatment in the CP community clinic as well as those individuals with an unknown community of residence who are receiving treatment in the CP community clinic.

# 4.4 Enhancement of services in all study communities

One of the goals of BCPP is to provide enhancement of HIV prevention, care and treatment services in non-intervention (ECC) communities as well as expansion and strengthening of these services in the combination prevention communities. This goal is primarily motivated by two factors:

- 1) A commitment to offering the enhanced care communities tangible benefits from participating in this community randomized trial, and
- 2) The imperative to bring the standard of practice in all study community clinics close to the standard of care, so that the BCPP study is assessing the effect of the combination prevention interventions on HIV incidence.

For the purposes of BCPP, the term 'enhanced' will be used to signify activities done in all study communities (including Enhanced Care Communities) for the purposes delineated above, whereas the terms 'strengthened' and 'expanded' will be used to signify activities done in Combination Prevention Communities only, as part of the study's combination prevention intervention package. 'Strengthened' will signify that activities are already part of national policy and practice, whereas 'expanded' will signify that activities are beyond current national policy and practice (for example, 'expanded' antiretroviral therapy in the CPCs).

The following enhancements will be provided in all 30 study communities, including the ECCs:

- a) Baseline and Annual Household Surveys (Evaluation Protocol): As part of the BHS that occurs in all 30 communities (in both study arms), ~20% of adults are offered home-based HIV testing, point-of-care CD4 count if treatment-naïve, viral load testing, and referral for HIV care and treatment, PMTCT services, MC, and other health services as appropriate (TB screening, for example). HIV-infected persons who were ART naïve at entry to BHS or who seroconvert between study visits and are ART-naïve will also have annual point of care CD4 and viral load tests, and these results will be shared with participants/clinics respectively. HTC is also offered to household residents who do not wish to take part in the BHS/AHS, either by the BHS study team, the HTC campaign team, or by referral to local clinics where HIV testing is available.
- b) Clinical care quality assessment and quality improvement: BCPP and/or CDC Botswana will work through the Ministry of Health to support clinical quality care assessment and improvement. Existing or new Ministry of Health and CDC tools and quality improvement documents will be used or expanded in this effort.
- c) Clinical data system support: BCPP will provide technical assistance to the Ministry of Health to support improved implementation and utilization of clinical data systems (primarily PIMS2 and IPMS) in all 30 study communities.

d) Laboratory support: BCPP will provide technical assistance to Ministry of Health to help laboratories supporting clinics in all 30 study communities to perform at a level sufficient to meet the standard of care. Existing or new Ministry of Health and CDC tools and quality improvement documents may be used or expanded in this effort.

# 4.5 Eligibility Criteria for Inclusion in Interventions in CP Communities

This protocol provides the inclusion and exclusion criteria for access to the services provided as part of the Combination Prevention intervention package. Adults aged 16-64 will be targeted for service uptake because recent, nationally representative surveys of HIV prevalence and incidence (BAIS 2008) suggest that HIV incidence remains high (>1%) throughout this age group.

For clinical services, only those who are Botswana citizens or spouses of Botswana citizens can receive free services from Ministry of Health facilities. Non-citizen/non-spouse of citizen HIV-infected adults identified during testing will receive a referral to the health clinic in their community of residence, but will not be eligible for free services from Ministry of Health facilities, and thus will not be eligible for strengthened free services in intervention clinics.

Investigators propose that eligibility for interventions in the CPC arm be grouped into three categories (a) eligibility for expanded HTC services and (b) eligibility for strengthened linkage-to-MC services, and (c) eligibility for expanded treatment and follow-up.

# a) Eligibility for Expanded HTC

All adults ≥16 who wish to receive HTC services at health facilities, mobile testing units, or door-to-door programs in combination prevention communities (CPCs), are eligible to receive these HTC services. The rationale for proposing that non-residents of the CPC be able to access expanded HTC services is to improve community acceptance of the door-to-door and mobile HTC activities. Preliminary discussions with community leaders suggest that restricting access to a service like HTC which is being delivered to family homes and neighborhoods would be met with considerable resistance and community discontent.

Non-citizens of Botswana will also be provided HTC services in the CPC. Non-citizen/non-spouse of citizen HIV-infected adults identified during testing will receive a referral to the health clinic in their community of residence to connect them with available fee-based services including treatment.

# b) Eligibility for Strengthened Linkage-to-MC services

Noncitizens will continue to be eligible for enhanced linkage- to-MC services if they meet other eligibility criteria. Under the national MC programs, noncitizens who present directly to the MC tent requesting MC will be offered free services. Thus, all adult men 16 years or older who are HIV-negative or have unknown HIV status are eligible for strengthened linkage-to-MC services including men who decline HIV testing or have indeterminate results. Under current national guidelines, boys 13-15 years old will not be actively mobilized or included in linkage-to-MC though they can continue to receive free MC services at national locations if they present with parental permission.

# c) Eligibility for Universal Treatment

Universal treatment will be offered to all HIV-infected adults aged 16-64 who are Botswana citizens or spouses of Botswana citizens. HIV-infected persons referred through the study via BHS/AHS, HTC or

routine HIV testing (RHT) as well as existing patients already enrolled in care at the CPC clinics will be offered expanded treatment. The Infectious Disease Care Clinics (IDCC) treat all Botswana citizens and spouses of Botswana citizens regardless of the community in which they reside. Therefore, both residents and non-residents of the community will be included.

# 4.6 Rationale for Exclusion from Interventions in CP Communities

• Rationale Surrounding Need for Botswana Citizenship or for Being Spouse of Botswana Citizen: Although the Botswana Government provides free HTC services to non-citizens, free access to health services, including ART and PMTCT is restricted to a) persons who can produce valid documentation of Botswana citizenship or b) spouses of Botswana citizens. Combination prevention interventions will therefore not be available to non-citizens of Botswana unless married to a citizen, except in the case of HTC and MC services. The exception for MC will be made to bring study goals closer to aligning with WHO goals for protection of communities through MC provided to 60% of HIV-uninfected men - regardless of citizenship status - as noncitizens living in the community may share the same sexual networks with citizens.

Additionally, men who decline HIV testing may actually be those at greatest risk for HIV acquisition and thus could benefit most from MC. If such men were not offered MC and were later found to be positive at end of study they would have represented a missed opportunity for prevention.

• Rationale for Age Limits: Persons <16 years of age will be excluded from study participation because our intervention is targeting adults, and relevant study outcomes will be measured among adults. In Botswana, adults are considered those aged 16 or older. For example, all persons aged ≥16 can access medical services, including HTC, without guardian consent. Although individuals aged 16-17 can access medical services without guardian permission, participation in research still requires guardian permission, because the age of consent for research in Botswana is 18. Therefore, eligible 16-17 year-olds will be asked for assent to participate in research activities only after permission has been provided by the guardian.</p>

#### 5.0 SAMPLE SIZE AND SAMPLE SELECTION METHODS

The primary objective for the intervention protocol is to implement and describe uptake of CP interventions in CP communities. Combined (BHS and HTC) data for 7 intervention communities was used to derive average denominator sizes for the estimates of interest. These community-average sample sizes were multiplied by 15 to yield an estimate of the total denominator (see Table 1). For the estimate of uptake of HTC, we used the number of participants interviewed to be conservative, although estimates of HTC coverage will be extrapolated to persons not interviewed.

Table 1 presents confidence limits for all of the indicators of uptake of CP interventions for protocol 3, using targets presented earlier in the protocol. Sample size calculations were done using a simple binomial method to obtain standard errors and then multiplying standard errors by the square root of the variance inflation factor (VIF), which is [1+(m-1)\*ICC], where m is the average number of members of each group (here, participants within community), and ICC is the intraclass correlation coefficient,

reflecting the magnitude of the correlation within communities for the outcome measure of interest. No published ICCs were available for these outcomes, so we used one small and one large value, based on prior publications reporting ICCs for behavioral variables in HIV and STD studies (Zhang et al., 2013 and Pals et al., 2003).

Table 1. Precision for 95% confidence intervals for uptake of CP interventions in CP communities

| Outcome | Denominator<br>(per community) | Denominator<br>(Total across CP<br>communities) | ICC | Coverage | 95%<br>Confidence<br>Interval | CI<br>Width |
|---|---|---|---|---|---|---|
| HTC | 2469 | 37035 | .02 | 90% | 87.8, 92.2 | 2.2 |
| | 2469 | 37035 | .05 | 90% | 86.5 <i>,</i> 93.5 | 3.5 |
| PMTCT | 50 | 750 | .02 | 90% | 87.0, 93.0 | 3.0 |
| | 50 | 750 | .05 | 90% | 86.0, 94.0 | 4.0 |
| MC | 794 | 11910 | .02 | 60% | 56.4, 63.6 | 3.6 |
| | 794 | 11910 | .05 | 60% | 54.4, 65.6 | 5.6 |
| ART | 528 | 7920 | .02 | 93% | 91.1, 94.9 | 1.9 |
| | 528 | 7920 | .05 | 93% | 90.0, 96.0 | 3.0 |

Table 1 shows that where sample sizes are large and we expect rates of uptake closer to 100% (HTC and ART), precision is excellent. Where sample sizes are small (PMTCT) or rates expected closer to 50% (MC), we have less precision for estimates, but confidence interval widths are still less than ±6%. As the rate of the outcome variable of interest moves away from 50%, standard errors and confidence interval width will decrease. With a larger ICC, the variance inflation factor increases and confidence intervals will widen.

#### 6.0 INTERVENTION PROCEDURES

# **6.1** Overview of Intervention Strategy

Interventions described below are intended to: 1) be consistent with new WHO guidelines on treatment of HIV infection (World Health Organization, 2015), 2) streamline clinic procedures to accommodate expansion of treatment to all PLHIV, and 3) incorporate lessons learned during the first year of BCPP. Targeted strategies will be implemented to meet UNAIDS goals of 90% of PLHIV know their status, 90% of PLHIV who know their status are on treatment, and 90% of PLHIV on treatment are virally suppressed. Through reaching the UNAIDS goals, it is anticipated that there will be a reduction in HIV incidence in the CP communities as assessed in Protocol 1. The proposed BCPP interventions will demonstrate UTT and introduce a streamlined approach to finding, testing, and starting PLHIV on immediate treatment and retaining them on effective treatment over time. Specific engagement activities as well as the specific interventions being deployed are outlined in detail below.

# 6.2 Stakeholder Involvement, Community Engagement, and Community Mobilization

To enhance communities' acceptance and effectiveness of the combination prevention package, local government and community stakeholders will be highly engaged. Program implementers, including MOH at central-, district-, and facility-level, and NGOs supporting the MOH's public health mission in

study districts, have been engaged in the planning and continue to be involved in implementing all combination prevention interventions. These governing bodies include:

- National Government: MOH, CDC and Harvard Chan School investigators and program planners have presented project plans to (1) the Parliamentary Sub-committee on Health, (2) the Parliamentary Sub-committee on HIV/AIDS, and, (3) the House of Chiefs (a body of traditional leadership made of representatives of all communities in the country).
- District Government: Study communities are distributed across 13 of 29 districts in Botswana.
   Meetings and consultations have been held with the District AIDS Coordinator, District Multi-Sectoral AIDS Committee, and the District Health Management Teams.
- Community Government: At the community level, village political leadership has been consulted, including the traditional leadership of *Dikgosi* and *Dikgosana* (Chiefs and sub-chiefs), the Village Development Committees (VDCs), church leaders, and sporting clubs. Project plans were shared and discussed prior to initial implementation and ongoing support for the project is sought.

Investigators meet regularly with members of study Community Advisory Boards (CAB) to discuss community perceptions of the project. Minutes of these meeting are documented and shared with the study principals. Specific issues raised during CAB meetings are addressed as needed. There are four CABs located in the following regions: *South, Central, North, and Northwest.* The CABS have representatives from the study communities in that region.

Community mobilization activities are conducted in all communities; however, the scope and duration of the activities are greater in the CPCs. Activities focus primarily on increasing uptake of HTC and MC so that HIV-infected adults can access treatment and/or PMTCT and HIV-negative adults can access MC. Some of the methods to improve uptake of services include:

- o Public announcements from vehicles with loudspeakers (very common in Botswana),
- Community (kgotla) meetings, civic society activities, schools, and clinics as a platform to inform the community.
- Door-to-door canvassing of the community informing community members of the services that are available in the community, location and duration.
- Specific mobile activities (e.g., location of an HTC caravan near work and sporting locations or in residential areas after business hours (e.g., after 5 pm) targeting hard to reach populations like men.

# 6.3 HIV Testing and Counseling (HTC)

- a) Target: 90% of PLHIV know their status.
- b) Strategy: Based on the first round of HTC in BCPP, the HTC strategy is being modified for years 2 and 3. During the first year of HIV testing, approximately 70-% of HIV+ persons in the community were identified through concentrated testing efforts lasting 6-8 weeks. During the 2<sup>nd</sup> year of the study, HTC activities will be provided through continuous availability of services in the community and will focus on 1) finding incident cases of HIV infection by retesting persons found to be
negative during the 1<sup>st</sup> year; 2) finding the 25-30% of community members missed by the 1<sup>st</sup> year of testing in BCPP; and 3) identifying HIV+ persons who are new arrivals to the community.

The activities to fulfill the first objective of finding incident HIV cases include 1) repeating door-to-door HIV testing during year 2 in all homesteads from year 1; 2) monthly mobile testing at targeted community locations; and 3) strengthening routine HIV testing (RHT) in health facilities with a focus on antenatal clinics, outpatient departments and IDCC. To fulfill the 2<sup>nd</sup> objective, targeted testing activities will be used to find community members missed in the first year of testing in BCPP. Based on data collected in year 1 of BCPP, approximately 50% of men and 30% of women are missed through home-based testing. Targeted testing strategies to locate those missing in year 1 will include workplace testing, home-based testing on holidays and weekends, mobile testing at venues frequented by men and large-scale community activities that attract the majority of community members. To fulfill the 3<sup>rd</sup> objective, new arrivals to the community who are HIV+ will be found through re-enumeration of households and HIV testing while going door-to-door. New arrivals will also be identified during community mobile testing and large-scale community events that offer HIV testing. The HTC strategy for year 3 of BCPP will be based on findings from year 2 of the study, but is likely to focus on targeting populations missed in year 2.

In order to reach the target of the 90% of PLHIV knowing their status, cost-effective community-based HIV testing strategies are needed to find unidentified HIV-positive persons who are not accessing health care facilities, such as young women and men. An understanding of the incremental costs between strategies is key to determine the optimal mix of strategies to implement. Therefore, a cost analysis of different HTC models implemented through BCPP will be undertaken.

# c) Specific HIV Testing and Counseling Services:

- 1) Home-Based HTC: HTC counselors will go door-to-door and request verbal consent to: (1) map household GPS location, (2) record numbers of persons in each household, their age, and sex by interviewing the head of household or, if the head of household is absent, a household member 18 years of age or older (Household Enumeration Form), and (3) offer HTC services (HTC Intake Form). The following individuals will not be offered HTC:
  - a. Adults who have documentation of an HIV-positive status
  - Adults who have documentation of HIV-negative results obtained within the last 3
    months of the HTC encounter. (Documentation of HIV test results are recorded on the
    HTC Intake Form)
  - c. Persons <16 years old

If a household member is absent, the team conducting the home-based HTC activities will ask about an appropriate time to return to the household (*Household Enumeration Form*). Up to 3 repeat visits will be scheduled.

- 2) *Mobile HTC*: Mobile HTC caravans and tents will be placed in prominent locations of the community [e.g., at kgotlas (community meeting locations), or shopping centers]. Community mobilizers will engage the community via door-to-door 'mobilization' visits and in high traffic areas in the community such as shopping and transport areas and invite residents to get tested in the mobile units and tents. Lay counselors and support staff will be stationed in mobile venues consisting of a waiting area, private HTC area and a phlebotomy area. HTC will be offered to all individuals (residents and non-residents, citizens and non-citizens) who are not known to be HIV-infected according to national guidelines (i.e., adults who do not have an HIV test result card indicating HIV-positive status). Persons who tested will be asked to keep the card with their results safely for any future contact, e.g., during subsequent household visits (below).
- 3) Routine Facility-Based HTC: Routine HTC activities at health facilities will be strengthened by training facility-based counselors to offer RHT as part of integrated routine services in outpatient, IDCC, and antenatal (ANC) clinics. Facility-based counselors will be encouraged to provide testing to all adults receiving health care services at the clinic and to offer testing to all friends, family members, relatives, visitors, etc. (so-called non-patients) accompanying the patient to the clinic. In addition, the study will assist MOH ANC staff with strengthening of 3<sup>rd</sup> trimester re-testing among pregnant woman (see section 6.6). Routine HIV testing data will be extracted from PIMS2/IPMS to monitor coverage of testing in health facilities.
- 4) **Targeted Testing:** HTC for groups that are difficult to access through home-based, clinic-based, or other routine services will be targeted by providing services where these groups work or congregate and by offering HTC services at large, well-attended community events such as barbecues, health fairs, concerts, etc.
- 5) Additional Services for Persons Testing HIV-Positive: All HIV positive adults not on treatment are eligible for ART under current national guidelines so will not need to consent for treatment in the UTT intervention. HTC counselors are trained to integrate treatment preparation, adherence and readiness messages into their post-test counseling for HIV-positive persons to begin preparing participants for initiating ART at their first clinic visit. In addition, they will be counseled to expect a confirmation test for HIV positive results before initiating ART which will be conducted at the IDCC. All participants of HTC will be tested using the MOH rapid testing algorithm along with pre-test and post-test counseling that is recommended in the national guidelines.
- 6) Additional Services for Persons Testing HIV-Negative: The following services will be offered to newly identified or known HIV-negative adults:
  - Screening of all adults for TB, with a simple screening question, and referral of TB suspects to the nearest clinic for TB testing. TB suspects will be prioritized for evaluation at the clinic. In Zimbabwe and Zambia, this has been shown to reduce community prevalence of infectious TB and was well-accepted by the community (Corbett, Bandason et al. 2010).
  - Encourage MC uptake by HIV-negative males through linkage-to-MC services. These services also are offered to men with unknown HIV status. Further details of the linkage-to-MC service are provided in Section 6.5 below.

- HIV-negative pregnant women will be encouraged to enroll in ANC care and be retested in their 3<sup>rd</sup> trimester.

# 6.4 Linkage to HIV Care and Treatment

- a) Targets: 80% of adults identified as newly diagnosed or not currently in care are registered at the local study IDCC or are documented in care at another IDCC within 90 days of BCPP interview and 90% within 180 days of BCPP interview
- b) Strategy: To ensure that 90% of persons identified as HIV-infected initiate ART, persons newly identified as HIV-infected or PLHIV not connected to care and treatment must be linked to an IDCC. Data from the first year of BCPP suggest that about half of PLHIV link to care with very little prompting or follow-up. Another 50%, however, require additional supports. The linkage intervention package for BCPP includes: 1) counseling after diagnosis on the importance of immediate treatment and appointments made for PLHIV not already in care; 2) appointment reminders; and 3) tracking and tracing of persons who miss appointments at the IDCC. In addition, to enhance linkage rates, patients wishing to receive care/ART outside of their community will be able to link to any MOH IDCC.

# c) Specific Activities:

- 1) Counseling After Diagnosis and Scheduling Appointments at IDCC: Counselors will be available to: (1) provide immediate psychosocial support to help clients cope with their HIV-positive test result, (2) counsel participants on the importance of early entry into HIV care or PMTCT services and prepare them for treatment initiation and adherence at first clinic visit, and (3) help clients establish and achieve plans to enter care by identifying and troubleshooting real and perceived barriers to care (Gardner, Metsch et al. 2005, Gardner, Marks et al. 2007, Craw, Gardner et al. 2008, Gardner, Marks et al. 2009). Appointments at IDCCs in intervention communities will be scheduled as soon as possible for newly diagnosed individuals or PLHIV who are not enrolled in care and treatment. Some PLHIV may prefer to obtain care and treatment services at a clinic outside their community for privacy, proximity to job, or other reasons. For those PLHIV who choose to obtain care outside the study community, verification of enrollment in care will be obtained from the MOH data systems.
- 2) **Appointment Reminders:** PLHIV will be sent short message service (SMS) reminders about their upcoming appointments.
- 3) Tracking and Tracing: A record of all patients referred to care by BHS, HTC and RHT will be submitted to Site Coordinator at the local IDCC. The Site Coordinator at the IDCC will access names of those referred and will track them to ensure they keep their first appointment. Names and contact information of those who don't keep their appointments will be turned over to the community counselor for tracing and case management. The intensified participant tracing program includes telephone calls and home visits for persons who missed a scheduled appointment up to 180 days after either diagnosis or BCPP interview for known HIV positive persons (Participant Tracing Log).
- 4) Counseling, Appointments and Tracing for PLHIV Identified who are already on ART

- Patients who are on ART, enrolled in care at the study IDCC, are not late for an appointment, and have a future appointment scheduled will be encouraged to remain adherent to ART and appointments.
- Patients who have initiated ART and are enrolled in care at the IDCC and are late for their next appointment or who do not have a future appointment scheduled will be (1) counseled on the importance of adherence and appointment keeping, (2) given a new appointment at the clinic, and (3) have phone number and residential address information obtained to facilitate follow-up (retention tracing of participants already in care and late for their scheduled appointments is described in section 6.7 below).
- Patients who are on ART and not enrolled in care at the study clinic will be counseled to remain adherent to ART and in care; they will also be informed of expanded and strengthened services available at the study clinic and will be given an appointment to the study clinic. Follow-up for these patients will be limited to only an SMS reminder for their appointment. Verification of the patients' enrollment at another clinic outside the study community and ART status will be obtained from MOH data systems.
- 5) Retrospective Tracking and Tracing of PLHIV who Did Not Link to Care: Given the change in the 2016 Botswana national treatment guidelines, HIV-positive participants not on ART who did not link to care from Round 1 (October 2013 February 2016) will be retrospectively contacted by the Ministry of Health clinic staff or a community counselor and informed that all HIV-positive persons are now eligible for ART, regardless of CD4 count or condition. Participants from Round 1 and Round 2 (June 2016 present) who previously did not give permission for follow-up may also be contacted, as the new guidelines recommend tracking all HIV-positive persons identified to care and treatment sites. Specifically,
  - Contact with the participant will be attempted by a Ministry of Health clinic staff member or a community counselor to inform the participant that the national guidelines have changed and all persons that are HIV-positive are now eligible for ART. They will also be informed that it is critical for their health and the health of their partners and children to get on ART as early as possible, and that the clinic offers services to help community members get into care and on treatment. Staff will use the updated talking points from the Linkage to Care SOP revised (see Appendix XX, Section 3.8).
  - Participants will be given an appointment at the clinic with a health care provider and will be encouraged to keep it.
  - If there is no current phone number for the participant, a home visit will be conducted by a clinic staff member or a community counselor. Up to 3 attempts to contact the participant will be made through alternating phone and home visits.
  - Participants from Round 1 who have not linked to care will be contacted beyond the follow-up period specified in the protocol (e.g., 180 days) in order to ensure the new guidelines are being implemented with all participants. Paricipants from Round 2 who were enrolled during the time between the introduction of the new guidelines and field implementation (November 2016) may also be followed beyond the 180 day window.

A note to file will be documented at each of the 15 intervention sites noting the procedural changes and follow-up provided to those individuals who previously did not link and declined follow-up.

#### 6.5 Male Circumcision

- a) Target: 60% of HIV-negative 16-49-year-old males are circumcised
- b) Strategy: BCPP's SMC intervention in the second year will be streamlined from the full-service campaign model used in the first year to a program that mobilizes and links interested men to existing services in nearby locations. MC services are expected to be provided in five of the 15 CPC sites using PEPFAR programmatic support. In all other districts, nearby services funded by Global Fund or MOH will be used, though distances to these services from CPCs is likely to vary. All CPCs are expected to have at least one service option available. Therefore, BCPP funding will not be used to support direct service delivery but to mobilize and link men in BCPP communities to existing MC services. Modified SMC services are expected to begin when the second round of BCPP interventions are implemented, approximately February 2016.

# c) Specific Activities:

- 1) Mobilization: In the first round of BCPP activities, SMC depended heavily on community-based mobilizers and referrals from the BCPP HTC Campaign and BHS to generate client demand. A basic level of this ongoing mobilization will continue. HTC and BHS will refer men to community mobilizers by passing contact information with consent; the mobilizers will then follow up with these men and link them to nearby services. Mobilizers will also work directly with communities to mobilize men for services. Incentives for mobilizers through a performance-based contract may be utilized to improve mobilization efforts. In addition to encouraging potential clients to obtain MC, mobilizers will disseminate service information about linkage sites, transport schedules, and assist with coordinating transportation.
- **2)** Coordination: A small number of full-time coordinators will oversee all the CPCs. Their responsibilities will include identifying and liaising with locally-available SMC services to confirm their schedules and notify them of expected clientele numbers on transportation days; supervising mobilizers; coordinating transportation; and follow-up with service sites to collect the necessary data. A senior BCPP staff member will keep the MOH SMC coordinator up to date on these activities.
- **3) Transportation:** In each CPC, transportation will be offered at least monthly to nearby SMC services, on days of the week determined to be optimal. Transportation will also be provided for day-2 and day-7 follow-up visits, and will remain available for adverse event emergencies.
- **4) Data collection:** Individual-level data will not be collected at SMC service provision sites by BCPP, but aggregate data will be requested from these sites. Specifically, at these sites, the coordinator will make attempts at least quarterly via physical visits and register reviews to ascertain how many HIV-negative/unknown men 16-49 years of age from the CPC were served. The coordinator will also collect aggregate data from the transfer logs to gather numbers of men transported to SMC services. Finally, the coordinator will collect aggregate data on number of men referred and mobilized from demand creation records completed by HTS and BHS staff as well as SMC mobilizers (*Male Circumcision Tracking Sheet*).

## 6.6 Identification, Linkage, and Treatment of HIV+ Pregnant Women

- a) Target: 90% of women initiated on indefinite ART (Option B+) during pregnancy remain in care and on treatment post-delivery.
- b) Strategy: Strengthening PMTCT activities is important to ensure that HIV-infected pregnant women are identified, linked to care, and remain on ART post-delivery. Currently, Option B+ is the national standard of prevention of mother-to-child transmission in Botswana. Therefore, BCPP intervention and control communities will provide Option B+ interventions for all HIV+ pregnant women. The BCPP program for pregnant women will focus on strengthening three activities in PMTCT settings in intervention communities: 1) strengthening of third trimester retesting within the ANC; 2) linkage to HIV treatment for all HIV-infected pregnant and post-partum women; and 3) retention on ART post-delivery.

## c) Specific Activities:

- 1) Strengthening third trimester retesting: BCPP staff work with MOH clinic staff to strengthen capacity to identify women who are due for third trimester retesting. MOH clinic staff will use client contact information from the ANC register to make phone calls and schedule appointments with all HIV-negative pregnant women who have not completed third trimester retesting. MOH clinic staff will keep a record of clients called for third trimester retesting. Third trimester retesting will be monitored through PIMS/IPMS by the IDCC clinic.
- 2) Linkage and Retention for HIV-infected Women: Ensuring HIV-positive pregnant women receive ART and remain on ART following delivery is a key priority. All HIV positive pregnant women identified through the BHS and HTC campaigns are referred to the IDCC for HIV care and treatment. In addition, HIV+ post-partum women are referred to the IDCC to continue ART indefinitely (Option B+). Those who do not keep IDCC appointments will be tracked by the IDCC Site Coordinator and followed by community counselors to ensure they link or re-link to the IDCC post-delivery. Similarly, retention activities will track women who have begun Option B+ to ensure that they stay in care and on ART indefinitely. Those who are 14 or more days late for an appointment or pharmacy pick up will be contacted by MOH clinic staff and/or the IDCC Site Coordinator (*Linkage, Retention and Adherence Tracing Verbal Consent Script*) and community counselors will provide supportive counseling and new appointments through phone and home visits (*Participant Tracing Log*) as outlined in section 6.4.

#### **6.7 HIV Care and Treatment**

## a) Targets:

- 1) 93% of PLHIV aged 16–64 who know their status are receiving ART
- 2) 95% of PLHIV aged 16-64 who are on ART are virally suppressed
- b) Strategy: Prior versions of BCPP Protocol 3 introduced anti-retroviral treatment outside Botswana national guidelines (CD4 < 350, WHO stage III or IV). With the revised WHO recommendations to treat all HIV-infected persons, Version 4.0 of Protocol 3 proposes to start all HIV+ adults in CPCs on immediate treatment and retain them on treatment (UTT). To demonstrate methods for

implementation of UTT for later adoption by the Botswana MOH, BCPP will embed UTT treatment interventions within the national ART program (MASA). The package of interventions described below are designed to 1) reduce barriers to ART initiation by simplifying procedures and making services easily available 2) increase capacity of IDCCs to support aggressive ART scale-up, and 3) enhance the use of both individual and clinic-level data to monitor uptake of HIV care and treatment.

# c) Specific HIV Care and Treatment Activities:

- 1) Confirmation of HIV status: All HIV+ referrals into the clinic as well as existing pre-ART patients will be confirmed with an HIV test administered by IDCC staff as recommended by WHO before initiating ART (World Health Organization, July 2015).
- **2)** Same day ART initiation: Patients who are not on ART will be offered initiation (or re-initiation) of ART on the day of their first clinic visit if blood draws are possible that day. Adherence counseling, screening for opportunistic infections, and blood draw for baseline pre-ART safety labs will occur on the day of ART initiation. Patients who decline ART initiation (or re-initiation) will be given a 1 month follow-up appointment for re-consideration of ART initiation.
- **3)** Frequency of clinic follow-up visits: Patients on ART who are stable (e.g., virally suppressed, no opportunistic infections, keeping appointments, etc.) will be offered a reduced frequency of scheduled visits as compared to the current MASA standards. Patients will be followed according to national program standards for the first year. For stable patients on ART for longer than 12 months, visits with a clinician every 6 months will be implemented. IDCC patients already on ART will follow the streamlined schedule according to their time on ART.
- **4)** Frequency of visits for laboratory testing: Routine laboratory testing will be offered to patients according to the national guidelines with the exception of CD4 counts which will only be measured at baseline, after 12 months on ART, and at the discretion of the clinician. Also, wherever possible, patients will have their blood drawn at the time of routine clinic visits rather than on separate days to further reduce the frequency of clinic visits and clinic congestion. All laboratory results will be reviewed by the clinic staff within 4 weeks of blood draws, and patients will be contacted by clinic staff for review of any abnormal lab results.
- **5)** Frequency of dispensing visits: Patients who are stable after 12 months of ART (e.g., virally suppressed, no opportunistic infections, keeping appointments, etc.) will be dispensed up to 3 months of ARVs if there is adequate stock in the clinic at the time of dispensing rather than being required to return after only 1 month for a dispensing visit. The pharmacy will update a patient's next refill appointment in PIMS2/IPMS if more than one month is dispensed. Stable patients will have monthly, bi-monthly or quarterly refill appointments, which may coincide with the semi-annual clinician visits.
- **6) Retention Intervention:** Resources will be available in CP communities to ensure that all PLHIV are retained in care. The retention intervention will focus efforts on those who have missed treatment appointments and/or pharmacy pick-ups. Persons eligible for retention tracing will be identified by the IDCC staff using their electronic data system.

Existing IDCC patients who have missed appointments or pharmacy pick-ups are contacted by MOH clinic staff by phone or home visits and are asked if they agree to have a community counselor contact them to provide retention support activities. Patients who do not consent to retention support intervention activities are reminded about the importance of staying in care/linking back into care, and thanked for their time (*Linkage, Retention and Adherence Tracing Verbal Consent Script; Retention Tracing Contact Log*).

Patients who consent to intervention activities receive retention support services by clinic staff and community counselors including SMS reminders of appointments, rescheduling of missed appointments, and tracing and supportive counseling through home visits and telephone calls for defaulters (>14 days late for appointment or pharmacy pick-up) and Lost to Follow Up (LTFU; > 90 days late for an appointment). Clinic data systems are monitored to determine if these patients have relinked to the IDCC (*Retention Tracking Log, Participant Tracing Form*).

7) Adherence Intervention: IDCCs typically use self-reports, pill counts, pharmacy refill data and viral loads to monitor adherence. These adherence monitoring strategies are promoted in all study sites. All PLHIV on ART in CPCs are offered an increased level of adherence counseling and support above and beyond what is routinely offered within the setting of government clinics. Eligible persons who would benefit from increased adherence support are identified by the clinic staff.

Eligible patients are contacted by MOH clinic staff by phone or home visit (*Retention and Adherence Outreach Script* and are asked if they agree to have a community counselor contact them to provide adherence support activities (*Linkage, Retention and Adherence Tracing Verbal Consent Script*). Patients who do not consent to adherence support intervention activities are reminded about the importance of taking ART as prescribed, and thanked for their time.

Patients who consent to intervention activities (*Adherence Intervention Verbal Consent/Assent Script*) receive adherence intervention services including an assessment (*Adherence Assessment Tool*), assignment of case manager, and additional counseling to assess and resolve individual adherence challenges. In addition, the following services may also be delivered depending upon the person's circumstances and assessment: referral to social worker; SMS reminders; home visits; pill box issuance; depression screening; support with HIV disclosure; alcohol assessment; treatment buddy/mopati; VL repeat; assignment of earlier appointment; and change in ART regimen (for those in whom side effects/medication acceptability might be mitigated through substitution). All adherence interventions will be documented as will the outcome of the efforts, on the *Adherence Intervention Tracing Log*.

## **Patient CARE in Other Study Clinics or Non-Study Clinics**

Finding solutions so that as many BCPP patients as possible can receive expanded ART initiation is important for reaching ART saturation in CP communities, however the study is constrained and cannot easily perform study activities or install study staff at sites which are not CP community clinics. As a solution, the following options will be offered to patients, if during counseling it is determined that they face challenges to participation in study activities at the IDCC in their own community:

1) BCPP activities at <u>any</u> CP community clinic: Initiation and receipt of ART will be allowed at <u>any</u> CP community clinic at which a participant would be able to receive services. Note that the

study will not be able to provide transport or any additional compensation for these individuals. Follow-up data from PIMS2 or IPMS will be obtained on these individuals for study purposes from the CPC clinic the participant chooses.

2) ART initiation activities at <u>own</u> community clinic, followed by transfer to <u>any</u> MOH clinic: Services including ART initiation will be provided at the participant's own CPC, followed by facilitated transfer to any MOH HIV care and treatment facility (including those not in study communities) for continued ART. Follow-up data on these individuals will be obtained from routine medical information sources such as PIMS2 or the national HIV data warehouse.

# **Identifying Patients for UTT**

To find all eligible PLHIV not currently on ART and initiate them on treatment, BCPP priorities will include approaching the Expanded Treatment Cohort (described in BCPP Protocol 3 version 3.0) in early 2016

to offer ART initiation for those not on ART. Another strategy to identify eligible PLHIV not currently on ART will include data mining of the MOH electronic patient systems to seek PLHIV categorized as "pre-ART" to approach them about immediate ART initiation (*Script for Outreach Pre-ART Clinic Patients*). These two mechanisms in combination with expanded HTC activities outlined earlier will yield the scale-up of ART initiation necessary to meet both treatment and viral suppression targets.

## 7.0 LABORATORY METHODS

Detailed laboratory procedures are described in Standard Operating Procedures (SOPs) that are maintained at each laboratory supporting the study. The BCPP Laboratory Manual provides an overview of routine testing that is conducted at Ministry of Health laboratories and more detailed study specific procedures for testing conducted at CDC, Harvard Chan School, BHP laboratories. In addition, all study staff has received a Field Operations Procedures Manual which serves as a procedural guide during actual specimen and data collection.

## 7.1 Overview of Laboratory Methods

An overview of the types of laboratory tests, sample types, and the location of the testing is provided below. The intervention component of the project uses the following laboratories and locations:

- 1. BHHRL: MOH regional HIV Reference Lab (Gaborone). BHHRL is a hybrid institution with management shared by Harvard and MOH.
- 2. NHHRL: MOH regional HIV Reference Lab (Francistown)
- 3. MOH District and primary Labs (Botswana-multi-sites)
- 4. MOH clinics in CPC communities
- 5. Field sites: households and community venues conducting surveys and HTC campaigns
- 6. CDC: International Laboratory Branch at Centers for Disease Control and Prevention (Atlanta) and CDC Laboratories (Gaborone and Francistown)
- 7. BHP (Botswana Harvard Partnership Laboratory)
- 8. Harvard T. H. Chan School of Public Health (Boston)

A minimum laboratory enhancement package has been implemented in laboratories supporting study sites. Each study-associated laboratory adheres to site and study specific SOPs for proper processing, labelling, transport, testing and storage of specimens as outlined in the BCPP Laboratory Manual. The laboratory study team provides guidance and technical support to the laboratories to implement and

maintain a quality management system which includes continuous quality improvement, adherence to biosafety, enrollment in EQA programs, review and maintenance of standard operating procedures for laboratory testing, timely procurement and forecasting reagent and supply needs, and documentation of training for all laboratory personnel. Adherence to these standards is routinely monitored by the laboratory study team.

# 7.2 Training of Laboratory Personnel

All laboratory personnel participate in study-specific training prior to study initiation. Training includes an overview of the BCPP study design and study-specific laboratory methodologies (with assessment for competency) in addition to Research Ethics and good clinical laboratory practices including QA/QC (quality assurance/quality control) and laboratory record keeping procedures. Study staff responsible for providing HTC complete the required training curriculum recognized by the Ministry of Health. Study staff members who collect blood samples and conduct laboratory analyses receive training in universal precautions, sample collection, and testing of study samples. Additional refresher trainings are scheduled during the study to ensure consistency and address training needs as they arise.

# 7.3 Specimen Collection, Transport, and Processing

Specimens are collected from participants at study field sites and samples transported to designated laboratories for processing, testing, and storage. Testing may also occur at study field sites.

# **Sample Types and Sources**

- a) <u>Capillary blood samples</u>: Finger prick samples are collected in a microtube using a blade lancet by trained staff at study field sites according to BCPP finger prick SOP and used for the HIV rapid tests.
- b) <u>Venous blood samples</u>: Several types of venous blood draws occur at the IDCC during routine management of patients, and will be done following MOH procedures for phlebotomy, (including appropriate blood volumes and processing). At the IDCC, venous blood samples will be collected for drug resistance testing per national guidelines.

# 7.4 Laboratory testing for HTC campaigns (returned to participant and/or participant file with exception of viral load test)

a) HIV Diagnostic Testing: HIV diagnostic testing will be conducted in the study communities and clinics per national HIV testing guidelines using Botswana government-approved serial rapid tests as outlined in the 2016 testing algorithm in the national treatment guidelines. Other testing algorithms may be substituted if in alignment with national guidelines. Verification will be conducted on all newly diagnosed and known HIV-positive persons before initiating ART according to WHO recommendations (World Health Organization, July 2015). All HIV tests will be conducted according to the manufacturer's guidelines and BCPP SOPs. If results of the initial serial rapid tests are discordant, then per national guidelines two rapid tests will again be performed in parallel. If the second pair of tests is discordant, the participant will be referred to the clinic for re-testing in 2-4 weeks with a referral recommending ELISA testing. A 3 ml venous blood specimen will be taken at the visit and sent to a reference laboratory for further testing using ELISA (Murex HIV 1.2.0 test, Genetic Systems HIV 1.2 plus O, BioRad HIV-1/HIV-2 plus O EIA,) and/or Western blot). The results from the EIA and/or Western Blot will supersede the discordant and/or indeterminate results obtained in the field. The IDCC Site Coordinator reviews the HTC register at the clinic in PIMS2 or IPMS to determine if HTC campaign participants with indeterminate results received confirmatory testing. HTC participants with indeterminate rapid test results, and who do not have a documented retest at the clinic are referred to a community counselor for tracing and follow-up services.

# 7.5 Laboratory Testing for IDCC patients

Clinical laboratory testing is performed in MOH labs in accordance with the National Guidelines. Testing procedures follow approved standard operating procedures for each laboratory where testing is conducted.

# a) Hematology and Clinical Chemistry

Basic blood work is used to assess participant health status for initiation and monitoring ARV treatment in HIV-infected individuals; however, ART initiation will occur before all lab results are available. The following tests may be conducted per MOH guidelines:

- Hematology: Full Blood Count (FBC) to include hemoglobin, hematocrit, red blood cell count (RBC), mean corpuscular volume (MCV), white blood cell count (WBC), differential WBC, absolute neutrophil count (ANC), and platelets.
- Clinical Chemistry:
  - o Liver Function Tests (LFT): Total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase.
  - Glucose (fasting or non-fasting)
  - Electrolytes: sodium and chloride
  - o Renal Function Tests (RFT): Urea and Creatinine: An estimated creatinine clearance
  - CrCl in cc/minute can be estimated from formulas using patient sex, age, weight, and serum creatinine (in um/L):

Males:  $1.22 \times [(140 - age in yrs) \times wt (kg)]/[serum Cr]$ 

Females:  $1.037 \times [(140 - age in yrs) \times wt (kg)]/[serum Cr]$ 

- b) <u>Syphilis testing (RPR and VDRL</u>): As per Botswana guidelines, non-treponemal tests for syphilis (rapid plasma reagin or Venereal Disease Research Laboratory tests) will be performed according to the manufacturer's instructions.
- c) <u>CD4:</u> Point of care and flow-based CD4 methods are used dependent upon availability of CD4 instruments. Testing follows manufacturer's instructions and national guidelines for use.
- d) <u>HIV-1 RNA Viral Load:</u> HIV-1 plasma RNA viral load is quantified for monitoring of ART-naïve HIV-infected individuals and monitoring of viral suppression in HIV-infected individuals receiving ART (at 3 and 6 months after ART initiation and every 6 month thereafter according to current national ART guidelines or per Adherence Intervention Procedures).
- e) <u>HIV drug resistance testing</u>: Drug resistance testing is offered per national guidelines and under circumstances described in section 6.11.
- f) Pap smear: Pap smears are performed and findings managed according to national guidelines.
- g) <u>Pregnancy Testing</u>: If pregnancy is suspected but not confirmed by LMP (last menstrual period) or exam, a urine pregnancy test is performed for confirmation of pregnancy as per MOH procedure.

## 7.6 Quality Assurance

Standard operating procedures (SOPs) are used for all tests as well as quality assurance/quality control (QA/QC) procedures. Laboratory staff conducting testing participate in a proficiency testing and 5% of all tests (or as indicated by laboratory specific SOP) are subjected to internal quality control processes. The QA/QC plan includes periodic monthly reviews of EQA performance, collaboration with the CDC laboratories, enrollment in appropriate EQA schemes, and inter-laboratory comparisons. External quality assurance and proficiency testing programs includes: CD4 count, HIV-1 RNA load, Hematology (FBC), and clinical chemistry analytes. Laboratories are monitored throughout the study by the study team and external monitors as requested by the study sponsor. QA for HTC conducted in the communities and through RHT in the clinics include weekly QC exercises for counselors in the field, participation in proficiency testing programs, monitoring and site visits from lab personnel, and biweekly monitoring of the concordance rates of HIV serial tests conducted in the field. A small sample of HIV-positive tests may be retested in the lab for QA purposes.

# 7.7 Biosafety and Waste Management

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate blood and secretion precautions are employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the United States Centers for Disease Control and Prevention. All infectious specimens are transported in accordance with the IATA guidelines using designated courier services.

# 7.8 Specimen Storage and Shipment

The IDCC Site Coordinator coordinates shipment of specimens as required. Selected samples may be transferred to the CDC (Atlanta) or Harvard Chan School (Boston) laboratories for external quality assurance, viral load, and drug resistance/level testing. Specimens are stored until all protocol-related and quality assurance testing have been completed.

## **8.0 DATA SYSTEMS AND MANAGEMENT**

The overall system to capture data, record outcomes and analyze results is an integration of multiple data collection sources for all BCPP interventions into a single research data base or data warehouse. Each BCPP activity has underlying systems of data capture and management which serve as the "system of record" containing the source records for all study data captured within the scope of that activity. A variety of data capture methodologies are used across the BCPP activities including online reference data retrieval (e.g., community maps), paperless point of service/survey capture, and paper and electronic chart/registry abstraction. Process, study participant status, and calculated data are also generated by the data systems of the BCPP activities and exchanged between systems and stored in the research database.

Each system must also interface with other activity data systems to exchange data as required to successfully implement the study. This includes maintaining participant registries, referrals, and key eligibility and status data, as well as underlying denominators within study arms and components. In

this section, we provide an overview of the data management for BCPP including data capture, data flow, security, confidentiality, access and quality.

# 8.1 Data collection, Capture and Flow

HTC data forms (*Household Enumeration Form, HTC Intake Form*) are collected with the OpenDataKit (ODK) software using handheld tablets running the Android operating system. HTC counselors are trained in the use of these handheld tablets for electronic data entry at the point of HTC, which includes door-to-door home visits and mobile HTC sites.

Community counselors also record their tracing activities for linkage and retention on the *Participant Tracing Log* using these handheld mobile devices.

HTC and Linkage to Care forms are synced to the clinic-level study database at least daily. Completed forms are deleted from the tablets following the sync.

Clinic Site Coordinators manage screening, adherence and retention activities using both the hand-held data devices and OpenClinica.

The MOH has an electronic data system known as the Patient Information Management System 2 or PIMS2. PIMS2 is a SQL-based, client-server application which runs on a local clinic network and has been implemented in BCPP community clinics. PIMS2 captures data for a variety of programs, including: facility-based routine HTC, MC, ANC, maternity, and post-natal care. HIV care and treatment data are regularly extracted from PIMS into the clinic-level study database via a secured Virtual LAN (VLAN) connection between the local clinic network on which PIMS2 operates and the BCPP network.

Some larger BCPP community clinics have migrated to a web-based system to record patient-level data which runs on the Botswana Government's data network. This Integrated Patient Management System or IPMS captures program data that are similar to PIMS and includes an integrated laboratory information system. IPMS data will be regularly extracted from the IPMS central data repository onto the BCPP central data server.

The MOH strongly encourages the use of PIMS or IPMS where available. Therefore, nurse prescribers, physicians, midwives, lay counselors and other clinic staff within the 30 BCPP communities record patient registration and appointments, and enter consultation, laboratory and pharmacy data into PIMS or IPMS. *Appendix P1* outlines the selected data elements transferred from MOH systems to the BCPP central data server.

MC staff members responsible for the coordinating linkage of eligible men to MC will distill aggregate data on numbers of total and eligible men transported to MC from the transportation logs and will also engage with service delivery providers to obtain numbers of eligible men served on non-transport days. This data will be entered into an electronic or paper-based custom data collection form monthly.

On a daily basis during the BHS/AHS surveys in all 30 communities, BHS/AHS referral and locator data files are transferred from BHP's electronic data capture system to the clinic via secure copy on the BCPP network in the clinic and processed into the clinic-level study database. At CPCs, BHS referrals are combined with HTC referrals. In all community clinics, referral data is used to produce operational

reports for use in the clinic. In CPCs, an encrypted flash drive is used to retrieve updated referral files from the clinic's study database and to transfer updated data from the MC client tracking tool to the clinic-level study database.

On a nightly basis, data from all clinic-level study databases is copied to the BCPP central data server in Gaborone over the secure BCPP VPN. As needed, the BCPP senior data manager in Gaborone will work with IDCC Site Coordinators or other clinic level staff to reconcile data issues.

The Research Database is designed in PostgreSQL and housed on the BCPP central data server at the CDC-Botswana Gaborone office. It is populated with data pulled up from all the clinic level study databases as well as data from IPMS, PIMS, CD4 data from PIMAs, and baseline, annual and end of study survey data transferred from BHP's EDC via secure copy.

The diagram in Figure 1 offers a schematic representation of the data flows from all sources described above to the central BCPP data warehouse for the intervention communities (CPCs). For all PLHIV in the study communities we obtain clinical data from the existing MOH's electronic patient data systems (PIMS or IPMS).

Figure 1: Data Flow diagram for CPCs



## 8.2 Data Security

The CDC Data Manager is responsible the security of BCPP data collected for the Intervention protocol. The Botswana MOH is responsible for the security of data collected through routine MOH systems, including PIMS and IPMS. All BCPP-specific systems supporting clinic data reside within the clinic network where a firewall, encryption keys, user logins, and physical security and access, and routine data back-up measures have been put into place to ensure data security and integrity.

Laptops and tablets used for data capture and processing are encrypted and require user logins to prevent unauthorized users from accessing data. Laptops, tablets and all study related paper-based forms and logs are stored in locked cabinets or locked trunks when not in active use. The clinic laptops which serve as the local clinic-level study databases are locked in secure cabinets. Daily data transfers from tablets and the MC Epi Info system minimize the risk of data loss should the device be lost or corrupted. Clinic-level study databases are backed up on to the local encrypted hard drive and the backup files are transferred to the BCPP central data server in Gaborone using secure copy. The

backups from all of the clinic-level study databases and the central data server will be backed up to tape daily. The BCPP central data server at the CDC-Botswana Gaborone office is located in a locked, climate controlled server room managed by CDC IT staff in compliance with CDC IT policies.

A virtual private network (VPN) connects each clinic-level study database to the BCPP data center. The VPN provides a secure network over which data can be transmitted and through which data managers and IT staff can access clinic systems. VPN accounts are provided to study staff as needed and CDC DM lead approval is required for access to study data systems managed by CDC. Within the BCPP network, access to devices, databases, and directories are managed based on user roles. Data in transit over the BCPP network is encrypted, password protected and transmitted through secure connections using secure-shell (SSH) protocols; encrypted, password protected memory sticks are used for data transfer when direct network connections are not available.

The Botswana MOH is responsible for the security of PIMS and IPMS data. PIMS resides on secure local networks at each clinic and IPMS runs on the secure Government Data Network (GDN). Both the local network and the GDN use PIMS are regularly backed up via secure memory sticks. IPMS backups are managed through the IPMS central data store in compliance with Botswana MOH IT policies. CDC DM and IT will work with MOH counterparts to strengthen data security policies and practices.

# 8.3 Data quality

ODK Surveys on the tablets and Epilnfo have built-in validation tools to minimize data entry errors. These include range restrictions for numeric data, pre-defined values (code sets) for categorical data, and logic checks. Valid responses are required for key fields to ensure completeness and skip patterns will be used to prevent extraneous data entry and encourage proper form completion. Error messages and caution notices will be used to alert staff when they enter faulty data so that they are aware and can correct the problem.

HTC and linkage to care staff receive training on both the contents of the tools and use of the tablets and ODK software. Supervisors review the data forms for completeness and supervise corrections prior to synching of the tablets. SMC staff will receive training on proper completion of MOH tools and use of the Epi Info client tracker. Data managers will monitor system performance throughout implementation.

## 8.4 Confidentiality of data

CDC DM is responsible for protecting the privacy of all study participants and ensuring the proper handling of all personal health information and contact information collected for BCPP under Protocol 3. All components of the distributed data systems implement both electronic and physical security procedures for "data in use" within secure networks and devices. Encryption is implemented to render electronically stored subject identity and personal health information unusable, unreadable, or indecipherable to unauthorized individuals for "data in motion" and "data at rest". Encrypted personally identifiable information (PII) will be transmitted within the BCPP system by way of the secured VPN only.

PII, including name, national identity card number (Omang) and locator data (address, phone numbers), is collected as part of HTC to facilitate referral and linkage of clients with services (e.g. IDCC, ANC, SMC). BHS collects similar information and includes necessary PII in the transfer of referral and

locator data to the clinic. PII is collected as a part of patient registration in both PIMS and IPMS as required by MOH to ensure patients are eligible to receive services.

PII maintained in the clinic study databases are not transferred to the central database on the BCPP server; Omang is encrypted with a one-way hash prior to transfer to the BCPP server for the purpose of linking data across data systems. Where there is consent from the client to access medical records or a waiver of consent to extract identified data from the clinic systems (PIMS and IPMS), clinic data can be linked with BHS referrals and HTC data using the hashed Omang.

All study staff are trained on data confidentiality. Site staff access to PII and locator data is limited to health care providing staff which are required to reliably identify a participant, and staff engaged in linking patients consenting for contact with services. A minimal number of staff have access to the study databases where PII is stored and the operational reports which present PII to site staff; DM can access these data when required for system maintenance or to provide user support.

#### 9.0 DATA AND ANALYSIS PLANS

The primary objective of the Intervention Protocol is to implement and describe uptake of Combination Prevention interventions in CPCs. Secondary objectives will describe retention in the clinical cascade of care from HIV diagnosis to viral suppression among all HIV-infected persons. The key indicators for analyzing results of BCPP objectives are outlined in Table 2.

•

**Table 2. BCPP Key Indicators** 

| Indicator Name | | Coverage vs. Numerator BCPP Performance | | Denominator |
|---|---|---|---|---|
| 1. | % of HIV+ Adults* who Know their Status | Coverage | # of HIV+ Adults estimated to know<br>their HIV status | # of Adults estimated to<br>be HIV+ |
| 2. | % of HIV+ Adults in<br>Care | Coverage | # of HIV+ Adults in Care | # of HIV+ Adults<br>estimated to know their<br>HIV status |
| 3. | % of HIV+ Adults on<br>ART | Coverage | #of HIV+ Adults on ART | # of HIV+ Adults<br>estimated to know their<br>HIV status |
| 4. | % of HIV+ Adults with<br>Viral Suppression | Coverage | # of HIV+ Adults with VL<1000Copies/ML | #of HIV+ Adults on ART |
| 5. | % of HIV+ Adults Identified through BCPP who know their status | BCPP<br>Performance | # of HIV+ Adults Identified (new & known) through BCPP who know their status | # of Adults estimated to<br>be HIV+ |
| 6. | % of PLHIV Newly<br>Diagnosed through<br>BCPP | BCPP<br>Performance | # of Adults Identified as Newly<br>Diagnosed HIV+ through BCPP | # of HIV+ Adults Identified (new & known) through BCPP who know their status |
| 7. | % of PLHIV Linked to<br>Care | BCPP<br>Performance | # of HIV+ Adults Identified as Newly Diagnosed or Not Currently in Care at IDCC who were seen at IDCC within 90 and 180 days of Interview | # HIV+ Adults Identified<br>as Newly Diagnosed or<br>Currently Not in Care at<br>IDCC |
| 8. | % of PLHIV Initiating (or re-starting) ART | BCPP<br>Performance | # of Eligible HIV+ Adults Identified Not<br>on ART who Start or Re-Start ART | # of HIV+ Adults<br>Identified not on ART |
| 9. | % of PLHIV Retained<br>on ART (12 months<br>Post ART Start or<br>Restart) | BCPP<br>Performance | # of HIV+ Adults Identified Not on ART<br>who Start or Re-Start ART and Remain<br>on ART after 12 Months | # of Eligible HIV+ Adults<br>Identified Not on ART<br>who Start or Re-Start ART |
| 10. | % of PLHIV on ART with Viral Suppression (12 Months post ART Initiation or Restart) | BCPP<br>Performance | # of HIV+ Adults Identified Not on ART who Start or Re-Start ART and have VL<1000Copies/ML after 12 Months | # of Eligible HIV+ Adults<br>Identified Not on ART<br>who Start or Re-Start ART |

In the section below, data and the data sources for the outcomes of interest are identified for each intervention within the combination prevention package of services (HTC and Linkage to care, HIV care and treatment, MC and PMTCT services). In addition, the data analysis plans are provided for the study objectives.

# 9.1 HIV Testing and Counseling and Linkage to Care

The HTC services aim to maximize the number of PLHIV who know their status within the community. Predictors of HTC uptake will be examined including demographics, prior testing history, partner status, etc. Participants reached through mobile vs home-based testing will be described including age

and gender. Characteristics of HIV-positive persons identified will be described, including but not limited to demographics, testing history, new or previous HIV diagnosis, history of HIV care, CD4 count, and ART status. Data sources will include the *Household Enumeration Form, HTC Intake Form, and BHS* collected during the HTC activities. In addition, facility-based testing will be monitored in CPCs through RHT data in PIMS2 or IPMS.

All HIV-positive participants given appointments at the HIV care and treatment clinic in the study communities are tracked to ensure they link to care. Those who keep appointments at the study clinic within 90 and up to 180 days of the BCPP interview as recorded in PIMS2 or IPMS are considered "linked" to care. Those participants who report they are receiving care at another clinic outside the study community will be verified by PIMS2 or IPMS and will be considered linked to care if that have an IDCC appointment within 90 and up to 180 days of their BCPP interview date. In addition, at one year from the interview data, electronic data systems will be checked to determine if participants who did not link or register within 90 days have registered in care.

Predictors of linkage to care will be examined including but not limited to, demographics, new or previous diagnosis, CD4 count, and time to first appointment from interview. In addition, rates of linkage to care will be compared among participants who received interventions services and those who did not.

Data sources include referrals from HTC and BHS (*HTC Intake*, *BHS*), PIMS2 and IPMS for details of registration into care and treatment, and the *Participant Tracing Log* where all linkage to care follow-up activities are recorded. In addition, the Ministry of Health's Central Data Warehouse will be queried to identify (or confirm self-reported enrollment) of community residents who register for HIV care and treatment outside of the local study community.

Further, estimations of the operational costs associated with the expanded HTC and linkage to care interventions paired with the total cost by intervention with their corresponding BCPP performance indicator will be used to estimate the average costs per person. The financial costing approach is described below, in the cost analysis plan.

#### 9.2 Care and Treatment

For HIV care and treatment objectives, the overall number of PLHIV enrolled in the IDCC and on ART including community residents getting care at clinics outside the community will be described. Specific focus will be given to examination of patterns of health care utilization by residents and non-residents of the community. The key outcomes for analysis are ART initiation, adherence, retention and virologic suppression. We will also describe the laboratory results showing toxicity, and adverse events among the clinic population on ART. ART initiation will be measured by start date of ART among all HIV-positive patients initiated on ART as recorded in the electronic patient management system. Length of time from BCPP interview or encounter to date of initiation on ART will be recorded and monitored. ART coverage will be measured by the number of HIV-positive community residents receiving ART out of the estimated number of HIV-positive community residents.

Adherence levels will be assessed through self-reports, pill counts and pharmacy refill data from the electronic data systems and also from the adherence intervention tools. Based on the self-reports, pill counts and pharmacy refill data, an aggregate measure of adherence will be calculated (e.g., good,

limited or poor). Adherence levels at a community clinic will be measured by the percentage of clinic patients with an adherence assessment of good, limited and poor adherence. Retention of HIV-positive persons in care and on treatment will be measured during a defined period of time (e.g. 12 and 24 months). The number of HIV-positive clinic patients who are community residents and who remain in care (had a clinic visit within 6 months) and on treatment (pharmacy pick up and clinic visit within 3 months) during a defined period among all patients from the community who were registered at the clinic during that time will be considered retained in care or on treatment. The number of patients who missed clinic visits, defaulted from care and were lost to follow up will also be recorded from the electronic patient management system during a defined period. Virologic suppression will be assessed from the electronic data systems and will be defined as those HIV-positive patients on ART with a viral load of less than or equal to 400 copies/ml among all patients on ART.

Predictors of retention, ART initiation, adherence and virologic suppression will be examined. As the inverse of retention, predictors of loss to follow will be examined. For those on ART, predictors of defaulting on ART will be examined.

All clinic patients will have data captured in the existing MOH electronic patient management systems. Clinical outcomes, including but not limited to ART eligibility and initiation, WHO stage, lab results, death, adherence, retention, viral suppression, and adverse events, will be assessed using routinely collected clinical data that is captured in the electronic medical record (see Appendix P1). In addition, the Ministry of Health's Central Data Warehouse or other sources of routine medical information will be queried to identify clinic participation, ART eligibility, ART initiation and virologic suppression among community residents receiving services outside of the local study community clinic. Secondary descriptive analyses for key clinical indicators will be conducted on these data. In the CPCs, retention intervention data will be recorded on the *Participant Tracing Log*, and adherence intervention data will be recorded on the *Adherence Assessment Tool* and the *Adherence Intervention Tracing Form*.

## **9.3 PMTCT Services**

Rates of 3<sup>rd</sup> trimester retesting among pregnant women will be assessed using the MOH Antenatal Care and Maternity registers and the MOH patient management systems. Among HIV-negative pregnant women enrolled in ANC care, the percent who were retested for HIV between 32-36 weeks will be recorded and monitored over the course of the study.

Rates of linkage to care among HIV-positive post-partum women will be reported. Once discharged from ANC care, HIV-positive post-partum women will be given appointments at the local IDCC. Those who kept the appointments and registered at the clinic as recorded in the electronic patient management system will be "linked" to care. Those who were previously registered patients in the IDCC who re-link to care will be considered re-linked. Predictors of linkage to care among HIV-positive post-partum women will be examined including but not limited to, demographics, time since diagnosis, CD4 count, viral load, and time since delivery. In addition, rates of linkage to care will be compared among participants who received intervention services and those who did not. Retention in care among post-partum women will be measured the same as among all HIV-positive patients in the IDCCs (see above) and recorded in the electronic patient management system. Rates of retention on ART in post-partum women at one year post-delivery will be described. In addition, predictors of post-partum

women who default from ART will be examined including demographics, time since diagnosis, time since delivery, CD4 count, and viral load.

Tracing activities with HIV-positive post-partum women referred to the HIV care and treatment clinic will be recorded on the *Participant Tracing Log*. The MOH patient management system will be used to verify registration of post-partum women in the IDCC. In addition, the Ministry of Health's Central Data Warehouse will be queried to identify women who temporarily access care and treatment services outside of the local study community during their period of postpartum confinement.

## 9.4 Male Circumcision

Through linkage to MC services, the MC program aims to maximize coverage of circumcision among males, which is defined as the percentage of HIV-uninfected men (aged 16-49) residing in CPC communities who are circumcised. Community-level MC uptake among all and eligible men will be reported. **BHS** and **ESS** surveys will be used to obtain cross-sectional true estimates of MC coverage, based on self-report. These surveys are described in the BCPP Evaluation Protocol (Protocol 1). Further, MC coverage will be estimated using records of MCs performed as well as the baseline MC prevalence reported by the HTC and BHS campaigns. MC coverage will be evaluated based on the most recent census estimates of the study community population as well as on the enumerated study population.

#### 9.5 ANALYSIS PLANS

For the primary outcomes, uptake of the CP interventions, we will estimate the percentage of participants eligible for and receiving the intervention using BHS and HTC data to identify those eligible, and BHS, HTC and clinic data to identify those receiving interventions. Confidence limits for each outcome will be estimated using robust standard errors to account for within-community clustering.

The first secondary objective is to examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions. We will fit Generalized Estimating Equations (GEE) models with robust standard errors to account for the clustering within communities. Independent variables for these models will be chosen based on prior literature and hypotheses about how various demographic, clinical and social/behavioral factors impact uptake of HTC, PMTCT, ART and MC. For MC, this type of analysis will only be possible for year 1 interventions because individual-level data on men obtaining MC will not be collected in subsequent years. Variables will be chosen a priori based on theoretical justification rather than statistical results and all chosen variables retained in the model to adjust for confounding.

To compare clinical outcomes, including viral suppression, among HIV-positive persons in CPCs who initiate expanded ART to those who initiate ART according to national guidelines, we will use tests appropriate to clustered data and the distribution of the outcomes of interest. For example, for viral suppression, we will use GEE models to account for the clustering within communities and test for a difference between groups (those initiating expanded ART vs. those who initiate according to guidelines). Since each community will contain both of these groups of participants, clustering has less impact on statistical tests, but still should be taken into account in the analysis to provide appropriate effect estimates and confidence limits.

To estimate the percentage of participants retained on ART among HIV-positive pregnant or breastfeeding women who initiate Option B+ (indefinite ART post-delivery), we will determine the number of HIV-positive pregnant women who initiate Option B+ during the study using BHS, HTC and clinic data, and determine the number retained on ART using clinic data. Confidence limits will be estimated using robust standard errors as for the primary outcome. Three costing studies of HTC and LTC services are planned. First, estimates of costs of home-based testing and mobile testing during the community-based HTC campaigns, including the cost per person and per new HIV case identified will be compared. Second, incremental costs and outcomes of strengthening facility-based routine testing relative to the standard of care will be estimated. Lastly, to assess the impact of the expanded linkage activities, estimates of the costs and outcomes of these tracking & tracing services will be calculated. Outcomes are defined as the number of new or previously diagnosed HIV-infected persons not in care, who register at an IDCC without engaging tracking and tracing services, and who register at an IDCC within 90 and 180 days of their HTC encounter.

A mixed top-down and micro-costing approach will be used to estimate costs. All relevant direct medical costs such as labor and materials, and direct non-medical costs such as program support and administrative overhead will be considered.

Analyses will be conducted from the perspective of the health care system indicating that the costs included would be those typically associated with the providers and payers of care, and would exclude the costs and productivity losses incurred by patients and their informal caregivers. The most significant cost component is expected to be labor, for which the main categories include: HTC lay counselors and supervisors, LTC Coordinators, drivers, and community mobilizers.

Labor time will be estimated by analyzing data records on clients seen, then confirmed through communication with staff and managers, and, as needed, through observation. Other cost items will be estimated through a combination of resource utilization and expenditure records. Any research related expenses will be removed in order for the resulting cost analyses to be useful for the projection of operational program costs. Costs of tests conducted through the baseline and annual household surveys administered by the Botswana Harvard Partnership will not be considered.

Cost and outcome data will be collected, retrospectively, from routine monitoring program data stored in the central study database and from actual program expenditures incurred over the period corresponding to the HTC and LTC programmatic efforts from all BCPP communities. The analytic horizon will begin in November 2013 and correspond to the period during which the HTC campaign and LTC program are delivered in a community. Unit costs (e.g. Cost per tested, Cost per new diagnosis, Cost per person linked) will estimated by dividing total costs by the relevant BCPP performance indicator. Where applicable any future costs will be discounted to their present value at a standard rate of 3%. As needed, costs will be converted from Botswana Pula to US dollars. Costs will be presented in 2015 US dollars. We will conduct univariate sensitivity analysis to identify the inputs which most impact the results and gauge the robustness of the conclusions. Data analysis will be conducted using Microsoft Excel and SAS.

# **10.0 ETHICAL CONSIDERATIONS**

## 10.1 Ethical Review

The protocol, informed consent/parental permission forms/assent forms, research participant education and recruitment materials, and other requested documents — and any subsequent modifications — will be reviewed and approved by the ethical review bodies responsible for oversight of research conducted at the study sites. The Institutional Review Boards/Ethical Committees (IRBs/ECs) for CDC and the Health Research & Development Committee, Botswana Ministry of Health will review the protocol at least annually.

## **10.2 Informed Consent**

# a) Interventions and strengthened programs:

HTC: National guidelines for obtaining verbal consent prior to receiving HTC services, for adults aged 16 or older, will be followed. Linkage-to-care interventions now fall under the Ministry of Health's 2016 national treatment guidelines which recommend that all HIV-positive persons identified be referred and tracked to the HIV care and treatment clinic. Therefore, all linkage to care follow up tracking will now be considered standard of care and will not require permission. However, participants who do not link to care and receive tracking and tracing follow up services will have the option to discontinue those services at any time they request. Similarly, active retention tracing of participants late for appointments has been implemented in several ART clinics in Botswana with plans to expand the scope of this program. For Retention Tracing, clinic patient contact information (name, phone number, address), OMANG (patient medical ID number) and appointment history are abstracted from MOH register and PIMS2 database for retention tracing of clinic patients who have missed scheduled clinic appointments These patients will be contacted by an MOH staff member and permission will be obtained to send BCPP counselors out for tracing and follow up services.

<u>Adherence Intervention</u>: Clinic patients identified as being non-adherent will be asked to consent for the adherence intervention (*Linkage, Retention & Adherence Intervention Verbal Consent*) which requests permission to administer the Adherence Assessment Form.

The informed consent process will occur in the language most comfortable for participants (usually in Setswana) at 8.0 reading level or below. Permission/assent will be documented by having the participant sign the permission/assent form or make a mark if the participant is illiterate; the latter will be witnessed by a third party. A copy of the informed consent/assent form will be offered to the participant, and if applicable, parent or legal guardian giving permission for a minor to participate. Staff will ensure that the participant takes a copy of a study contact card that contains study information and telephone numbers if the participant does not wish to take a copy of the permission/assent form.

## b) Special Populations

*Minors:* Minors (participants ages 16-17) are only enrolled with the written permission of a parent/legal guardian and if they provide informed assent.

- ✓ Under circumstances where clinical or study staff suspect, or there is a reported incident of sexual abuse of a person under age 18, the study staff member must inform the relevant authorities; this is stated in the permission/assent forms.
- ✓ Referrals will be made to youth services if needed.

- c) Use of Routine Programmatic Data: A waiver of informed consent was previously granted for the following activities:
  - 1) Medical record use in accordance with 45CFR 46.116 (d) to extract a limited, preselected dataset (Appendix P1) from MOH clinical data systems in the clinic population in Enhanced Care and Combination Prevention Communities. This is done by linking BHS and HTC data with clinic data to monitor the care and treatment cascade from HIV testing and referral through clinic enrollment, ART initiation and adherence, and retention in care. Procedures for extracting, matching between sources, and de-identification of this data are described in Section 8. Limitation of data-to-data elements based on consent/waiver-of-consent will be applied during the transfer of data from the clinics into the study database. Although not all data elements are part of the matching algorithm, data are matched using date of birth and Omang number. Once match is assigned, the data retained for analysis is de-identified in accordance with the consent/waiver-of-consent and the stipulations of the study protocols.
  - 2) A waiver of informed consent was previously granted for the following: a) data from the HTC Intake questionnaire that is collected as part of HTC programmatic services in households and tent venues in the Combination Prevention Communities, and b) abstraction of aggregate program data from MC and HTC facilities.

The waiver is appropriate because (1) the analysis involves no more than minimal risk to human subjects, and personal identifiers are encrypted for data handlers and analysts; (2) the evaluation does not adversely affect the rights and welfare of the subjects; (3) the evaluation cannot practicably be carried out without the waiver because it is not possible to obtain consent from all service recipients without infringing on the ability to carry out the program in an efficient manner; and (4) if consent for routine data use from all participants was requested, this might reasonably constitute an unnecessary waste of an individual's time. The types of consents being requested for activities in this study are described in Table 3.

Table 3: Summary of approach to consent for various components of the study

| Project | Targeted subjects | Activity | Consent | Comment |
|---|---|---|---|---|
| component | | | | |
| HTC | Persons not documented to be HIV-infected | Routine HIV counseling and testing | Verbal consent | |
| Programmatic<br>Interventions | Eligible residents of study communities | Use of testing (rapid test) and intake data from HTC, linkage to HIV care, TB screening, retention support and PMTCT services | Waiver of consent/assent granted | 45 CFR<br>46.116 (d) |
| Use of routine-<br>clinical data | Clinic population, all communities | Use of routinely-collected, program data-see Appendix P1 | Waiver of consent/assent granted | 45 CFR<br>46.116 (d) |
| Clinic Patient<br>Retention and<br>Adherence | IDCC patient population in CPCs | Data collection and permission to follow-up | Linkage, Retention &<br>Adherence Tracing<br>Verbal Consent Script | |

#### 10.3 Risks

The risks, discomforts, and inconveniences that could be posed to subjects participating in this project include the following:

## • HTC Participants:

- O Blood drawing may cause pain and bruising, and rarely, infection at the site where blood is drawn. Study participants may feel lightheaded or faint as a result.
- Repeated HTC may cause stress, anxiety, or embarrassment. Participants are likely to become distressed if they learn they are HIV positive.
- Participants may become embarrassed, worried, or anxious when discussing their sexual practices, HIV risk factors, ways to protect their partner(s) against HIV, and/or ways to prevent acquiring HIV infection.
- Participants may experience discrimination as a result of being perceived by others to be HIVinfected.

# • Other Strengthened Program Interventions:

- Other strengthened interventions, including linkage for HIV care, ANC, TB screening, and retention support all carry very minimal risk to participants.
- Persons starting ART: In addition to the risks described above for survey participants, risks for patients initiating ART include:

Adults starting ART are at risk of ART-related adverse events (e.g., hepatitis, severe skin rash, renal dysfunction, drug resistance, need for regimen change, etc.).

## 10.4 Benefits of Research Participation

- **HTC:** Potential health benefits include: earlier HTC delivered to their place of residence, earlier diagnosis of HIV-infection with subsequent earlier enrollment in care and treatment or PMTCT, earlier awareness of the importance of annual HTC and risk reduction practices for adults who test HIV-negative, and earlier awareness of the benefits of MC for HIV negative males.
- Other Strengthened Program Interventions: Evidence for health benefits of linkage-to-care and adherence/ retention interventions are described in Section 6.
- UTT: The benefits of earlier initiation of ART might include improved survival and reduction in incidence of adverse events [such as serious non-AIDS events like myocardial infarction, or AIDSrelated morbidity (e.g., a new WHO stage III/IV condition)] as well as decreased likelihood of transmitting HIV to others.

## **10.5 Confidentiality**

No information concerning the study or the data will be released to any unauthorized third party, without prior written approval of the participant, except as necessary for monitoring by the IRBs, the study sponsor, OHRP, or the Botswana Ministry of Health. No data with subject identifiers will be released.

# • HTC, linkage to care, and HIV care and treatment following HIV diagnosis:

Project staff visiting households for study visits will identify an appropriately private space to counsel participants, perform HIV tests, and collect individual data. If private space is not available, or the participant does not wish to carry out study activities in the home, an appointment will be made to visit one of the mobile units or study clinics instead. All study documents, including any papers or files containing personal contact information (such as telephone numbers and addresses), will be stored in a secure location and electronic data will be password protected. Full Drive Encryption will be implemented at the hardware layer of all devices storing protected health information. Only designated study staff will have access to study records.

# Linkage to MC and MC

MC mobilization will be conducted according to national standards for mobilization. These standards include protections for transport registers and mobilization registers with PII.

#### **IDCC Care and Treatment:**

Care at the clinic will be provided in adherence with MOH confidentiality guidelines. Consultations between patients and clinic/research staff will occur in a private location. All consent forms kept by investigators are stored in locked steel cabinets at the clinic or on password-protected electronic devices (e.g., tablets). All paper forms are stored in locked steel cabinets and transported in sealed boxes to Gaborone. All data collected via MOH data systems or entered from paper questionnaires are kept securely on password-protected log-in screens.

## 10.6 Protocol Compliance and Compliance with UN Convention on the Rights of the Child

Study staff will adhere to the ethical principles that are reflected in the Declaration of Helsinki (e.g., ICH E6, 45 CFR 46). The study will be conducted in accordance with the Botswana and Sponsor regulations.

The US government is a signatory on the UN Convention on the Rights of the Child (defined as anyone under the age of 18) which requires that any research study or program activity which includes children that are identified as engaged in sex work, trafficked or victims of violence make special provisions for referral of these individuals to services. BCPP will report suspected cases to designated service providers (local police or social workers) as outlined in the Botswana National Guidelines for reporting child abuse or neglect. Contact information for the local police and social workers, and procedures for reporting suspected cases of child abuse or neglect are described in study specific SOP in the BCPP Study Manual. Local police and social workers will be contacted prior to the initiation of study activities in the community to ensure they are aware of the study activities in the community and the procedures that will be followed should BCPP staff encounter suspected cases of abuse or neglect. As per national guidelines, reports of suspected abuse or neglect will be made to local authorities within 24 hours. Study personnel who may come in contact with these study participants will receive training on the appropriate procedures for handling these cases if they arise during the course of the study and training on the SOP documented in the regulatory files. The study will retain documentation of all reports that includes date of report, age of participant, and the name and type of service provider. No identified information will be retained in the documentation; documentation will be retained by the study for 2 years after study close-out. The informed consents for the study contain

language that makes clear to the participant what is required to be reported to authorities and the impact on confidentiality.

#### 11.0 STUDY SAFETY AND MONITORING PLAN

## **11.1** Reporting Adverse Events

# Expedited Adverse Event (EAE) Reporting Requirements for this Study:

The study team will report in real-time, to overseeing IRB's and to sponsors, any AE following any exposure to the study interventions that is BOTH possibly related to study intervention and unexpected, and which is a Serious Adverse Event (SAE). An SAE is defined as any untoward occurrence that:

- Results in death
- Is life-threatening (grade 4)
- Requires hospitalization or prolongation of hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect

This level of reporting is chosen to avoid real-time EAE reporting of all deaths, hospitalizations, etc. occurring in study communities that are definitely not related to study procedures.

Study interventions are defined as:

- 1. Antiretroviral therapy implemented as per BCPP protocol
- 2. HIV testing as part of the HTC campaigns
- 3. Any other study-related activity in which harm (including social harm) could occur.

With regard to ART intervention, EAE reporting will be restricted to SAEs that are possibly related to initiating ART beyond national guidelines.

## Timing of EAE reporting:

EAEs will be reported to CDC and HRDC within 2 business days of the study investigators becoming aware of the event.

## Grading Severity of Events:

The most current Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) dated November 2014 will be used (or more current version, if applicable), and is available on the RSC website (<a href="http://rsc.tech-res.com/">http://rsc.tech-res.com/</a>).

## Non-EAE Adverse Event and Incident Reporting:

The risk of adverse events related to the use of ART has been established and there is no indication that enrollees, with intact immune systems, who are receiving ART, are likely to have a higher risk of adverse events.

SAEs that do not meet the criteria for EAEs (i.e. an SAE that is NOT related to the study intervention) will be submitted quarterly to the IRB. A table listing all unrelated SAEs that occurred in the specified quarter will be submitted to the IRB along with a brief narrative of each event. Per discussions with the CDC IRB, SAEs that are unrelated to the study intervention will NOT be reported using the official CDC forms (.1254/.1254S).

# **Adverse Event Reporting Period:**

The expedited AE reporting period for this study is from the time of initial study contact to the last study contact for a participant.

## AE reporting process

Reportable events will be documented by the in-country study team who will then notify the IRBs, MOH, CDC-Atlanta, and Harvard Chan School teams. The incident will be discussed and a written action plan will be devised and implemented within 1 week of the initial report, if needed. Written documentation of all events and event resolution will be retained in the study file. Reporting of EAEs, SAEs and AEs to IRBs and the study sponsor will follow institutional and IRB policies. If applicable, a formal report will be sent to the appropriate IRBs using the CDC's Incident Report Form 1254.

## 11.2 **DSMB**

Proposed Schedule of DSMB Reviews and Interim Data Analysis

The BCPP is divided into three interlocking protocols (two active protocols, after Protocol 2 was terminated in 2015), and the investigators expect that DSMB review will require information regarding interim study results and study conduct from all three. The combination prevention package under study includes the following interventions that are outside of current SOC in Botswana: provision of ART for all HIV-infected adults regardless of WHO Stage or CD4 count and streamlined ART delivery. Hence, the reports will provide information needed to evaluate the adverse and favorable effects of such interventions on individually treated patients as well as on the communities in which they reside. The study will require at least 6 reviews, DSMB 1-6, proposed to take place at baseline and at the end of years 1, 2, 3, 4, and 5. DSMB 3 and 4 will evaluate intervention rollout and safety. At DSMB 5, the DSMB can recommend stopping for efficacy or extending the study by 1 year should there be low intervention coverage or a lower than expected incidence rate in the Enhanced Care arm. To demonstrate that the study has reasonable power to answer the study questions given information up to the time of each review, investigators will provide the DSMB with assessments of the adequacy of coverage of proposed interventions; estimated conditional power given available incidence information will be provided at DSMB 4 and all subsequent reviews. While there will be separate reports for each of the protocols, each report will make use of the data available from all protocols. Details of the DSMB review plan for each protocol are provided in that protocol, and the full detailed plan is provided in **Appendix C4**.

# 11.3 Protocol Violations

The study will be conducted in full compliance with the protocol. The research team will ensure that volunteers are informed of and understand the risks of their participation in research. Protocol violations and cases of social harm will be documented using the appropriate study forms and reported to IRBs and sponsors in accordance with the institutional policies. Minor protocol violations that do not pose a threat to the health or welfare of participants will be compiled and reported to the IRBs at the time of annual IRB review. Incident reporting is the responsibility of the Principal Investigators of

this study. Emergency departures from protocol that eliminate an apparent immediate hazard to participants and are deemed crucial for the safety and well-being of that participant may be instituted for that participant only. In that case the Investigator will contact the IRBs and sponsor as soon as possible to document the reasons for violation and ensuing events.

## 11.4 Monitoring Plan

A complete monitoring plan has been developed and the site will complete a study site activation checklist prior to study initiation. Internal (sponsor) and external monitors will travel to the study site according to a pre-determined monitoring schedule specified in the monitoring plan to conduct general monitoring. The study site will maintain a monitoring log to document all monitoring visits. Investigators and staff will grant access to the monitors to allow inspection and review study documents (e.g., consent forms, data collection forms, other source documents) and pertinent clinic records for confirmation of the study data. Study monitors will also inspect study facilities and documentation and may observe the performance of study procedures.

## 12.0 ADMINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION

# 12.1 Study Records and Document Retention

Complete, accurate, and current study records will be maintained and stored in a secure manner throughout the duration of the study and additionally for five years after study close-out. Study records include administrative documentation— including all reports and correspondence relating to the study— as well as documentation related to each participant screened and/or enrolled in the study, including informed consent forms, locator forms, case report forms, notations of all contacts with the participant, and all other source documents. Necessary documents to be maintained by the site before, during and after the study will be in accordance with GCP regulations and guidance. A complete list of needed documentation will be provided prior to initiation of the study and will appear in the study manual.

## 12.2 Information Dissemination and Publication Plan

Study findings will be disseminated through presentations, reports and publication in peer-reviewed journals and other publications. In-country data and country specific information will be made available to national policy-makers, organizational, and implementing partners. A detailed publication and communication plan will be developed that describes the number and types of reports and manuscripts planned for the study and criteria for authorship. Formal presentations at conferences and scientific publications will follow CDC, Harvard Chan School, and MOH guidelines. A data sharing plan will also be developed that details the requirements and process for requesting access to stored data and a samples for sub-studies and future analysis.

#### 13.0 REFERENCES

Ananworanich, J., Gayet-Ageron, A., Le Braz, M., Prasithsirikul, W., Chetchotisakd, P., Kiertiburanakul, S., et al. (2006). CD4-guided scheduled treatment interruptions compared with continuous therapy for patients infected with HIV-1: results of the Staccato randomised trial. Lancet, 368(9534), 459–465. doi:10.1016/S0140-6736(06)69153-8.

Attia, S., M. Egger, M. Muller, M. Zwahlen and N. Low (2009). "Sexual transmission of HIV according to viral load and antiretroviral therapy: systematic review and meta-analysis." <u>AIDS</u> 23(11): 1397-1404.

Auld, A. F., N. Wambua, J. Onyango, B. Marston, G. Namulanda, M. Ackers, T. Oluoch, A. Karisa, A. Hightower, R. W. Shiraishi, A. Nakashima and J. Sitienei (2010). "Piloting the use of personal digital assistants for tuberculosis and human immunodeficiency virus surveillance, Kenya, 2007." <a href="Int J Tuberc Lung Dis">Int J Tuberc Lung Dis</a> 14(9): 1140-1146.

Auvert, B., D. Taljaard, E. Lagarde, J. Sobngwi-Tambekou, R. Sitta and A. Puren (2005). "Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial." <u>PLoS Med</u> 2(11): e298.

Bailey, R. C., S. Moses, C. B. Parker, K. Agot, I. Maclean, J. N. Krieger, C. F. Williams, R. T. Campbell and J. O. Ndinya-Achola (2007). "Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial." <u>Lancet</u> 369(9562): 643-656.

BAIS (2008). "The Botswana HIV/AIDS Impact Survey III Results. Available: http://www.gov.bw/Global/NACA%20Ministry/wana/BAIS%20III Stats%20Press.pdf."

BAIS (2012). Botswana National AIDS Coordinating Agency. The Fourth Botswana HIV/AIDS Impact Survey IV-2012. Accessed 17 July 2014 at <a href="http://www.naca.gov.bw/sites/default/files/BAIS%20IV%20Protocol.pdf">http://www.naca.gov.bw/sites/default/files/BAIS%20IV%20Protocol.pdf</a>

Binik, A., C. Weijer, A. D. McRae, J. M. Grimshaw, R. Boruch, J. C. Brehaut, A. Donner, M. P. Eccles, R. Saginur, M. Taljaard and M. Zwarenstein (2011). "Does clinical equipoise apply to cluster randomized trials in health research?" <u>Trials</u> 12: 118.

Blitzstein, J. and P. Diaconis (2006). "A sequential importance sampling algorithm for generating random graphs with prescribed degrees. Available at: <a href="http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf">http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf</a>."

Census (2011). "Project Document: 2011 Population and Housing Census. Available at: http://unstats.un.org/unsd/censuskb20/Attachment453.aspx."

Central Statistics Office (2009). Botswana AIDS Impact Survey III (BAIS III), 2008. C. Kebonyethebe Johane. Gaborone, Botswana.

Ciaranello AL, Perez F, Engelsmann B, Walensky RP, Mushavi A, Rusibamayila A, et al. Cost-effectiveness of World Health Organization 2010 guidelines for prevention of mother-to-child HIV transmission in Zimbabwe. *Clin Infect Dis* 2013,56:430-446.

Cohen, M. S., Y. Q. Chen, M. McCauley, T. Gamble, M. C. Hosseinipour, N. Kumarasamy, J. G. Hakim, J. Kumwenda, B. Grinsztejn, J. H. Pilotto, S. V. Godbole, S. Mehendale, S. Chariyalertsak, B. R. Santos, K. H. Mayer, I. F. Hoffman, S. H. Eshleman, E. Piwowar-Manning, L. Wang, J. Makhema, L. A. Mills, G. de Bruyn, I. Sanne, J. Eron, J. Gallant, D. Havlir, S. Swindells, H. Ribaudo, V. Elharrar, D. Burns, T. E. Taha, K. Nielsen-Saines, D. Celentano, M. Essex and T. R. Fleming (2011). "Prevention of HIV-1 infection with early antiretroviral therapy." N Engl J Med 365(6): 493-505.

Corbett, E. L., T. Bandason, T. Duong, E. Dauya, B. Makamure, G. J. Churchyard, B. G. Williams, S. S. Munyati, A. E. Butterworth, P. R. Mason, S. Mungofa and R. J. Hayes (2010). "Comparison of two active case-finding strategies for community-based diagnosis of symptomatic smear-positive tuberculosis and control of infectious tuberculosis in Harare, Zimbabwe (DETECTB): a cluster-randomised trial." <u>Lancet</u> 376(9748): 1244-1253.

Craw, J. A., L. I. Gardner, G. Marks, R. C. Rapp, J. Bosshart, W. A. Duffus, A. Rossman, S. L. Coughlin, D. Gruber, L. A. Safford, J. Overton and K. Schmitt (2008). "Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II." <u>J Acquir Immune Defic Syndr</u> 47(5): 597-606.

Curran, K., E. Njeuhmeli, A. Mirelman, K. Dickson, T. Adamu, P. Cherutich, H. Mahler, B. Fimbo, T. K. Mavuso, J. Albertini, L. Fitzgerald, N. Bock, J. Reed, D. Castor and D. Stanton (2011). "Voluntary medical male circumcision: strategies for meeting the human resource needs of scale-up in southern and eastern Africa." <u>PLoS Med</u> 8(11): e1001129.

Daar, E. S., T. Moudgil, R. D. Meyer and D. D. Ho (1991). "Transient high levels of viremia in patients with primary human immunodeficiency virus type 1 infection." N Engl J Med 324(14): 961-964.

Ding, M., P. Tarwater, M. Rodriguez, R. Chatterjee, D. Ratner, Y. Yamamura, P. Roy, J. Mellors, D. Neogi, Y. Chen and P. Gupta (2009). "Estimation of the predictive role of plasma viral load on CD4 decline in HIV-1 subtype C-

Donnell, D., J. M. Baeten, J. Kiarie, K. K. Thomas, W. Stevens, C. R. Cohen, J. McIntyre, J. R. Lingappa, C. Celum and H. S. V. H. I. V. T. S. T. Partners in Prevention (2010). "Heterosexual HIV-1 transmission after initiation of antiretroviral therapy: a prospective cohort analysis." Lancet 375(9731): 2092-2098.

infected subjects in India." J Acquir Immune Defic Syndr 50(2): 119-125.

Eaton, J. W., T. B. Hallett and G. P. Garnett (2011). "Concurrent sexual partnerships and primary HIV infection: a critical interaction." <u>AIDS Behav</u> 15(4): 687-692.

Faal, M., N. Naidoo, D. K. Glencross, W. D. Venter and R. Osih (2011). "Providing immediate CD4 count results at HIV testing improves ART initiation." <u>J Acquir Immune Defic Syndr</u> 58(3): e54-59. Fauci, A. S. and G. K. Folkers (2012). "Toward an AIDS-free generation." <u>JAMA</u> 308(4): 343-344.

Fasawe O, Avila C, Shaffer N, Schouten E, Chimbwandira F, Hoos D, et al. Cost-Effectiveness Analysis of Option B+ for HIV Prevention and Treatment of Mothers and Children in Malawi. *PLoS One* 2013,8:e57778.

Fox, M. P. and S. Rosen (2010). "Patient retention in antiretroviral therapy programs up to three years on treatment in sub-Saharan Africa, 2007-2009: systematic review." Trop Med Int Health 15 Suppl 1: 1-15.

Gardner, E. M., M. P. McLees, J. F. Steiner, C. Del Rio and W. J. Burman (2011). "The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection." <u>Clin Infect Dis</u> 52(6): 793-800.

Gardner, L. I., G. Marks, J. Craw, L. Metsch, S. Strathdee, P. Anderson-Mahoney, C. del Rio and G. Antiretroviral Treatment Access Study (2009). "Demographic, psychological, and behavioral modifiers of the Antiretroviral Treatment Access Study (ARTAS) intervention." <u>AIDS Patient Care STDS</u> 23(9): 735-742.

Gardner, L. I., G. Marks, L. R. Metsch, A. M. Loughlin, C. O'Daniels, C. del Rio, P. Anderson-Mahoney, J. D. Wilkinson and A. S. Group (2007). "Psychological and behavioral correlates of entering care for HIV infection: the Antiretroviral Treatment Access Study (ARTAS)." <u>AIDS Patient Care STDS</u> 21(6): 418-425.

Gardner, L. I., L. R. Metsch, P. Anderson-Mahoney, A. M. Loughlin, C. del Rio, S. Strathdee, S. L. Sansom, H. A. Siegal, A. E. Greenberg, S. D. Holmberg, T. Antiretroviral and G. Access Study Study (2005). "Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care." <u>AIDS</u> 19(4): 423-431. Geng, E. H., D. Nash, A. Kambugu, Y. Zhang, P. Braitstein, K. A. Christopoulos, W. Muyindike, M. B. Bwana, C. T. Yiannoutsos, M. L. Petersen and J. N. Martin (2010). "Retention in care among HIV-infected patients in resource-limited settings: emerging insights and new directions." <u>Curr HIV/AIDS Rep</u> 7(4): 234-244.

Granich, R. M., C. F. Gilks, C. Dye, K. M. De Cock and B. G. Williams (2009). "Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model." Lancet 373(9657): 48-57.

Gray, R. H., G. Kigozi, D. Serwadda, F. Makumbi, S. Watya, F. Nalugoda, N. Kiwanuka, L. H. Moulton, M. A. Chaudhary, M. Z. Chen, N. K. Sewankambo, F. Wabwire-Mangen, M. C. Bacon, C. F. Williams, P. Opendi, S. J. Reynolds, O. Laeyendecker, T. C. Quinn and M. J. Wawer (2007). "Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial." <u>Lancet</u> 369(9562): 657-666.

Habicht, J. P., C. G. Victora and J. P. Vaughan (1999). "Evaluation designs for adequacy, plausibility and probability of public health programme performance and impact." <u>Int J Epidemiol</u> 28(1): 10-18.

Halperin, D. T. (2009). "Combination HIV prevention must be based on evidence." <u>Lancet</u> 373(9663): 544-545. Handcock, M. S., D. R. Hunter, C. T. Butts, S. M. Goodreau and M. Morris (2003). "Software tools for the Statistical Modeling of Network Data. available at: <a href="http://statnet.org.">http://statnet.org.</a>"

Hayes, R., F. Mosha, A. Nicoll, H. Grosskurth, J. Newell, J. Todd, J. Killewo, J. Rugemalila and D. Mabey (1995). "A community trial of the impact of improved sexually transmitted disease treatment on the HIV epidemic in rural Tanzania: 1. Design." <u>AIDS</u> 9(8): 919-926.

Hayes, R. and L. H. Moulton (2009). <u>Cluster Randomized Trials</u>. Boca Raton, CRC Press. Helleringer, S. and H. P. Kohler (2007). "Sexual network structure and the spread of HIV in Africa: evidence from Likoma Island, Malawi." <u>AIDS</u> 21(17): 2323-2332.

HHS (2011). "Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents. Avaiable at: http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf."

HHS (2012). "Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Available at: http://infosida.nih.gov/contentfiles/lvguidelines/adultandadolescentglsp.pdf. Accessed 19 August 2012.".

Hussey, M. A. and J. P. Hughes (2007). "Design and analysis of stepped wedge cluster randomized trials." <u>Contemp Clin Trials</u> 28(2): 182-191.

Jani, I. V., N. E. Sitoe, P. L. Chongo, E. R. Alfai, J. I. Quevedo, O. Tobaiwa, J. D. Lehe and T. F. Peter (2011). "Accurate CD4 T-cell enumeration and antiretroviral drug toxicity monitoring in primary healthcare clinics using point-of-care testing." <u>AIDS</u> 25(6): 807-812.

Jones, J. H. and M. S. Handcock (2003). "An assessment of preferential attachment as a mechanism for human sexual network formation." <u>Proc Biol Sci</u> 270(1520): 1123-1128.

Kaufmann, G. R., P. Cunningham, A. D. Kelleher, J. Zaunders, A. Carr, J. Vizzard, M. Law and D. A. Cooper (1998). "Patterns of viral dynamics during primary human immunodeficiency virus type 1 infection. The Sydney Primary HIV Infection Study Group." <u>J Infect Dis</u> 178(6): 1812-1815.

Kim, A. A., T. Hallett, J. Stover, E. Gouws, J. Musinguzi, P. K. Mureithi, R. Bunnell, J. Hargrove, J. Mermin, R. K. Kaiser, A. Barsigo and P. D. Ghys (2011). "Estimating HIV Incidence among Adults in Kenya and Uganda: A Systematic Comparison of Multiple Methods." <u>PLoS One</u> 6(3): e17535.

Kitahata, M. M., S. J. Gange, A. G. Abraham, B. Merriman, M. S. Saag, A. C. Justice, R. S. Hogg, S. G. Deeks, J. J. Eron, J. T. Brooks, S. B. Rourke, M. J. Gill, R. J. Bosch, J. N. Martin, M. B. Klein, L. P. Jacobson, B. Rodriguez, T. R. Sterling, G. D. Kirk, S. Napravnik, A. R. Rachlis, L. M. Calzavara, M. A. Horberg, M. J. Silverberg, K. A. Gebo, J. J. Goedert, C. A. Benson, A. C. Collier, S. E. Van Rompaey, H. M. Crane, R. G. McKaig, B. Lau, A. M. Freeman, R. D. Moore and N.-A. Investigators (2009). "Effect of early versus deferred antiretroviral therapy for HIV on survival." N Engl J Med 360(18): 1815-1826.

Lawn, S. D., A. D. Harries, B. G. Williams, R. E. Chaisson, E. Losina, K. M. De Cock and R. Wood (2011). "Antiretroviral therapy and the control of HIV-associated tuberculosis. Will ART do it?" <a href="Int J Tuberc Lung Dis">Int J Tuberc Lung Dis</a> 15(5): 571-581.

Lester, R. T., P. Ritvo, E. J. Mills, A. Kariri, S. Karanja, M. H. Chung, W. Jack, J. Habyarimana, M. Sadatsafavi, M. Najafzadeh, C. A. Marra, B. Estambale, E. Ngugi, T. B. Ball, L. Thabane, L. J. Gelmon, J. Kimani, M. Ackers and F. A. Plummer (2010). "Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial." <u>Lancet</u> 376(9755): 1838-1845.

Lingappa, J. R., J. P. Hughes, R. S. Wang, J. M. Baeten, C. Celum, G. E. Gray, W. S. Stevens, D. Donnell, M. S. Campbell, C. Farquhar, M. Essex, J. I. Mullins, R. W. Coombs, H. Rees, L. Corey, A. Wald and H. S. V. H. I. V. T. S. T. Partners in Prevention (2010). "Estimating the impact of plasma HIV-1 RNA reductions on heterosexual HIV-1 transmission risk." <u>PLoS One</u> 5(9): e12598.

Little, S. J., A. R. McLean, C. A. Spina, D. D. Richman and D. V. Havlir (1999). "Viral dynamics of acute HIV-1 infection." <u>J Exp Med</u> 190(6): 841-850.

Lyles, R. H., C. Chu, J. W. Mellors, J. B. Margolick, R. Detels, J. V. Giorgi, Q. Al-Shboul and J. P. Phair (1999). "Prognostic value of plasma HIV RNA in the natural history of Pneumocystis carinii pneumonia, cytomegalovirus and Mycobacterium avium complex. Multicenter AIDS Cohort Study." <u>AIDS</u> 13(3): 341-349

Mahy, M., J. Stover, K. Kiragu, C. Hayashi, P. Akwara, C. Luo, K. Stanecki, R. Ekpini and N. Shaffer (2010). "What will it take to achieve virtual elimination of mother-to-child transmission of HIV? An assessment of current progress and future needs." <u>Sex Transm Infect</u> 86 Suppl 2: ii48-55.

Mellors, J. W., J. B. Margolick, J. P. Phair, C. R. Rinaldo, R. Detels, L. P. Jacobson and A. Munoz (2007). "Prognostic value of HIV-1 RNA, CD4 cell count, and CD4 Cell count slope for progression to AIDS and death in untreated HIV-1 infection." <u>JAMA</u> 297(21): 2349-2350.

Mellors, J. W., A. Munoz, J. V. Giorgi, J. B. Margolick, C. J. Tassoni, P. Gupta, L. A. Kingsley, J. A. Todd, A. J. Saah, R. Detels, J. P. Phair and C. R. Rinaldo, Jr. (1997). "Plasma viral load and CD4+ lymphocytes as prognostic markers of HIV-1 infection." <u>Ann Intern Med</u> 126(12): 946-954.

Mellors, J. W., C. R. Rinaldo, Jr., P. Gupta, R. M. White, J. A. Todd and L. A. Kingsley (1996). "Prognosis in HIV-1 infection predicted by the quantity of virus in plasma." Science 272(5265): 1167-1170.

Merson, M., N. Padian, T. J. Coates, G. R. Gupta, S. M. Bertozzi, P. Piot, P. Mane, M. Bartos and H. I. V. P. S. A. Lancet (2008). "Combination HIV prevention." <u>Lancet</u> 372(9652): 1805-1806.

Microsoft (2011). "HIV/AIDS Information System Taps Existing Cell Phone Texting Capabilities. Available at: <a href="http://research.microsoft.com/en-us/collaboration/papers/botswana.pdf">http://research.microsoft.com/en-us/collaboration/papers/botswana.pdf</a>."

MMWR. Impact of an Innovative Approach to Prevent Mother-to-Child Transmission of HIV — Malawi, July 2011–September 2012. March 1, 2013 / 62(08);148-151.

Modjarrad, K., E. Chamot and S. H. Vermund (2008). "Impact of small reductions in plasma HIV RNA levels on the risk of heterosexual transmission and disease progression." <u>AIDS</u> 22(16): 2179-2185.

Montaner, J. S., V. D. Lima, R. Barrios, B. Yip, E. Wood, T. Kerr, K. Shannon, P. R. Harrigan, R. S. Hogg, P. Daly and P. Kendall (2010). "Association of highly active antiretroviral therapy coverage, population viral load, and yearly new HIV diagnoses in British Columbia, Canada: a population-based study." <u>Lancet</u> 376(9740): 532-539. Mtapuri-Zinyowera, S., M. Chideme, D. Mangwanya, O. Mugurungi, S. Gudukeya, K. Hatzold, A. Mangwiro, G. Bhattacharya, J. Lehe and T. Peter (2010). "Evaluation of the PIMA point-of-care CD4 analyzer in VCT clinics in Zimbabwe." J Acquir Immune Defic Syndr 55(1): 1-7.

Novitsky, V., T. Ndung'u, R. Wang, H. Bussmann, F. Chonco, J. Makhema, V. De Gruttola, B. D. Walker and M. Essex (2011). "Extended high viremics: a substantial fraction of individuals maintain high plasma viral RNA levels after acute HIV-1 subtype C infection." <u>AIDS</u> 25(12): 1515-1522.

Novitsky, V., R. Wang, H. Bussmann, S. Lockman, M. Baum, R. Shapiro, I. Thior, C. Wester, C. W. Wester, A. Ogwu, A. Asmelash, R. Musonda, A. Campa, S. Moyo, E. van Widenfelt, M. Mine, C. Moffat, M. Mmalane, J. Makhema, R. Marlink, P. Gilbert, G. R. Seage, 3rd, V. DeGruttola and M. Essex (2010). "HIV-1 subtype C-infected individuals maintaining high viral load as potential targets for the "test-and-treat" approach to reduce HIV transmission." PLoS One 5(4): e10148.

Padian, N. S., S. I. McCoy, S. Manian, D. Wilson, B. Schwartlander and S. M. Bertozzi (2011). "Evaluation of large-scale combination HIV prevention programs: essential issues." <u>J Acquir Immune Defic Syndr</u> 58(2): e23-28.

PEPFAR (2009). "Celebrating Life: The U.S. President's Emergency Plan for AIDS Relief 2009 Annual Report to Congress – Highlights. Accessed 3 September 2011 at: http://www.pepfar.gov/documents/organization/113878.pdf."

Piot, P., M. Bartos, H. Larson, D. Zewdie and P. Mane (2008). "Coming to terms with complexity: a call to action for HIV prevention." Lancet 372(9641): 845-859.

Rosen, S. and M. P. Fox (2011). "Retention in HIV Care between Testing and Treatment in Sub-Saharan Africa: A Systematic Review." <u>PLoS Med</u> 8(7): e1001056.

Severe, P., M. A. Juste, A. Ambroise, L. Eliacin, C. Marchand, S. Apollon, A. Edwards, H. Bang, J. Nicotera, C. Godfrey, R. M. Gulick, W. D. Johnson, Jr., J. W. Pape and D. W. Fitzgerald (2010). "Early versus standard antiretroviral therapy for HIV-infected adults in Haiti." N Engl J Med 363(3): 257-265.

Shapiro RL, Kitch D, Ogwu A, Hughes M, Lockman S, Powis K, Souda S, Moffat C, Moyo S, McIntosh K, Widenfelt E, Zwerski S, Mazhani L, Makhema J, Essex M. HIV transmission and 24-month survival in a randomized trial of HAART to prevent MTCT during pregnancy and breastfeeding in Botswana (The Mma Bana Study). AIDS. 2013 (in press).

Stover, J., L. Bollinger and C. Avila (2011). "Estimating the Impact and Cost of the WHO 2010 Recommendations for Antiretroviral Therapy." <u>AIDS Res Treat</u> 2011: 738271

Stover, J., B. Fidzani, B. C. Molomo, T. Moeti and G. Musuka (2008). "Estimated HIV trends and program effects in Botswana." PLoS One 3(11): e3729.

Stover, J., E. L. Korenromp, M. Blakley, R. Komatsu, K. Viisainen, L. Bollinger and R. Atun (2011). "Long-term costs and health impact of continued global fund support for antiretroviral therapy." <u>PLoS One</u> 6(6): e21048. Tanser, F., T. Bärnighausen, E. Grapsa and M.-L. Newell (2012). "Effect of ART Coverage on Rate of New HIV Infections in a Hyper-endemic, Rural Population: South Africa." <u>19th Conference on Retroviruses and Opportunistic Infections; March 5-8; Seattle, USA. Available: http://www.retroconference.org/2012b/Abstracts/45379.htm. Accessed 4 July 2012.</u>

Tanser, F., T. Bärnighausen, E. Grapsa, J. Zaidi and M. L. Newell (2013). "High Coverage of ART Associated with Decline in Risk of HIV Acquisition in Rural KwaZulu-Natal, South Africa." <u>Science</u> 339(966).

UNAIDS (2010). "Global Report: UNAIDS Report on the Global AIDS Epidemic. Available at: <a href="http://www.unaids.org/globalreport/globalreport.htm">http://www.unaids.org/globalreport/global report.htm</a>. Accessed February 2012.".

Van Rooyen, H., R. V. Barnabas, Z. Phakathi, P. Joseph, M. Krows, T. Hong, J. Baeten and C. Celum (2012). "HIV testing uptake and linkages to HIV treatment through home-based HIV counseling and testing and facilitated referral in Kwa-Zulu Natal, South Africa." <u>CROI 2012</u>.

Walensky, R. P., L. L. Wolf, R. Wood, M. O. Fofana, K. A. Freedberg, N. A. Martinson, A. D. Paltiel, X. Anglaret, M. C. Weinstein and E. Losina (2009). "When to start antiretroviral therapy in resource-limited settings." <u>Ann Intern Med</u> 151(3): 157-166.

WHO (2003). "World health Organization. WHO Guide to Cost-Effectiveness Analysis - 2003." Geneva, Switzerland: WHO; 2003. Accessed August 11, 2010: http://www.who.int/choice/publications/p 2003 generalised cea.pdf.

WHO (2010). World Health Organization. Towards universal access: Scaling up priority HIV/AIDS interventions in the health sector - Progress report 2010. Geneva, Switzerland: WHO; 2010. . Avaliable: http://wwwwhoint/hiv/pub/2010progressreport/full report enpdf. Accessed 29 September 2010.

WHO (2011). "Global HIV./AIDS Response. Epidemic update and health sector progress towards Universal Access. Available:

http://www.unaids.org/en/media/unaids/contentassets/documents/unaidspublication/2011/20111130\_UA\_Report\_en.pdf. Accessed 24 August 2012."

WHO (2013) "Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV infection" Available: http://apps.who.int/iris/bitstream/10665/85321/1/9789241505727\_eng.pdf Accessed 5 December 2013

World Health Organization. Use of Antiretroviral Drugs for Treating Pregnant Women and Preventing HIV Infection in Infants. Programmatic Update. April, 2012. http://www.who.int/hiv/pub/mtct/programmatic\_update2012/en/.

World health Organization. Consolidated Guidelines on HIV Testing Services. July, 2015. <a href="http://www.who.int/hiv/pub/guidelines/hiv-testing-services/en/">http://www.who.int/hiv/pub/guidelines/hiv-testing-services/en/</a>

World Health Organization. Guideline on When to Start Antiretrovoral Therapy and on Pre-Exposure Prophylaxis for HIV. September, 2015.

Writing Committee for the, C. C. (2011). "Timing of HAART initiation and clinical outcomes in human immunodeficiency virus type 1 seroconverters." <u>Arch Intern Med</u> 171(17): 1560-1569.
# Botswana Combination Prevention Project (BCPP) Intervention Protocol (Protocol #3)

## Implementation, Monitoring, and Evaluation of a Combination of HIV Prevention Interventions in Rural and Peri-Urban Communities in Botswana

#### Version 6.0

**September 22, 2017** 

#### **Collaborating Institutions:**

Botswana Ministry of Health (MOH)
Harvard T. H. Chan School of Public Health (Harvard Chan School)
U.S. Centers for Disease Control and Prevention (CDC)

#### Funded by:

The United States President's Emergency Plan for AIDS Relief (PEPFAR) through United States Centers for Disease Control and Prevention (CDC)

#### PRINCIPAL INVESTIGATORS:

#### Janet Moore, PhD

Branch Chief, HIV Prevention Branch

Division of Global HIV/AIDS (DGHA), Center for Global Health (CGH)

United States Centers for Disease Control and Prevention (CDC)

Address: 1600 Clifton Road, Atlanta, GA, 30333, U.S.A

Email: jym3@cdc.gov Office Phone: 404.639.8954

#### Refeletswe Lebelonyane, MD

Combination Prevention Coordinator, MOH Ministry of Health, Botswana Government Enclave Plot No. 54609 Gaborone, Botswana

Email: rlebelonyane@gov.bw

#### Shenaaz El Halabi, (PS) MPH

Permanent Secretary Botswana Ministry of Health

Address: Private Bag 0038, Gaborone, Botswana

Email: sel-halabi@gov.bw Office Phone: +267-363-2069

#### Pamela Bachanas, PhD

Behavioral Scientist, HIV Prevention Branch

Division of Global HIV/AIDS (DGHA), Center for Global Health (CGH) United States Centers for Disease Control and Prevention (CDC)

Address: 1600 Clifton Road, Atlanta, GA, 30333, U.S.A

Email: ddt6@cdc.gov Office Phone: 404.639.8110

#### **ROLES OF INSTITUTIONS AND PRINCIPAL INVESTIGATORS**

**Institutions**: Close coordination between MOH, CDC, HSPH, BHP, and other implementing partners is needed to ensure seamless implementation of research and program activities. MOH and CDC will lead and ultimately be responsible the Intervention Protocol and HSPH and BHP will lead the Evaluation Protocol.

**Principal Investigators:** 

**Janet Moore/ Pamela Bachanas:** CDC (PIs) responsible for preparation and design of the study protocol, monitoring of study progress, creation and monitoring of research budgets, and preparation of monthly progress reports.

**Refeletswe Lebelonyane/ Shenaaz El Halabi:** MOH Co-Principal Investigator (Co-PI) responsible for protocol review and in-country implementation oversight.

#### **CO-INVESTIGATOR LISTS BY INSTITUTION**

#### Botswana Ministry of Health (MOH), Gaborone, Botswana

| Name | Role | Contact Email |
|---|---|---|
| Ms. Dinah Ramaabya (Nursing) | ARV Program | dramaabya@gov.bw |
| Ms. Chipo Phetlo (Nursing) | PMTCT | cphetlo@gov.bw |
| Mr. S. Makathaye, Dip Health Educ. | BCIC | smalathaye@gov.bw |
| Mr. C. Ntsuape, BEd (Nursing Educ) | SMC | ontsuape@gov.bw |
| Ms. Nokuthula Manjingo (Nursing) | HIV Testing & Counselling | mmajingo@gov.bw |
| Dr. Joe Theu ((Medical Officer) | Clinical Care | jtheu@gov.bw_ |

#### Centers for Disease Control and Prevention (CDC), Atlanta, GA, USA, and Gaborone, Botswana

| Name | Role | Contact Email |
|---|---|---|
| Elliot Raizes, MD | Clinical Consultant | gwq0@cdc.gov |
| Ebi Bile, BSc. MA, DU | In-country Lab Oversight | efb6@bw.cdc.gov |
| Peter Fonjungo, PhD | HQ Lab Oversight | pdf4@cdc.gov |
| Sherri Pals, PhD | Statistics | sfv3@cdc.gov |
| Chunfu Yang, PhD | Laboratory | cxy0@cdc.gov |
| Mary Grace Alwano | In Country HTC/ LTC Project Coordinator | mea9@bw.cdc.gov |
| Stephanie Behel, MPH | HTC and LTC | zmd7@cdc.gov |
| Naomi Bock, MD | Voluntary Medical MC | neb2@cdc.gov |
| Stephanie Davis, MD, MPH | Voluntary Medical MC | vic6@cdc.gov |
| Lisa Block, MS | Project Manager | kwk5@cdc.gov |
| Lisa Mills, MD | Co-investigator | loj7@cdc.gov |
| William Abrams | <b>Program Administration</b> | hvf8@cdc.gov |
| Arielle Lasry PhD | HTC Costing | ftn9@cdc.gov |

#### Harvard T. H. Chan School of Public Health, Boston, MA, USA

| Name | Role | Contact Email |
|---|---|---|
| Myron Essex, DVM, PhD | Co-Investigator | messex@hsph.harvard.edu |
| Eric Tchetgen, PhD | Statistics and Epidemiology | etchetge@hsph.harvard.edu |
| Scott Dryden-Peterson, MD | Treatment and PMTCT | $scott\_peters on @post.harvard.edu$ |
| Shahin Lockman, MD, MSc | Treatment and PMTCT | slockman@hsph.harvard.edu |
| Rebeca Plank, MD | SMC | rplank@partners.org |
| Molly Pretorius Holme, MSc | Research operations | mpretori@hsph.harvard.edu |
| Roger Shapiro, MD, MPH | Treatment and PMTCT | rshapiro@hsph.harvard.edu |
| Kate Powis, MD, MPH | Research Operations, | kpowis@mgh.harvard.edu |
| Rate I Owis, IVID, IVII II | Treatment and PMTCT | kpowis@ingil.narvara.eau |

#### Botswana-Harvard AIDS Institute Partnership (BHP), Gaborone, Botswana

| Role | Contact Email |
|---|---|
| Treatment and PMTCT, | tgaolathe@bhp.org.bw |
| Field research operations | |
| BHP research operations | jmakhema@bhp.org.bw |
| Lab | smoyo@bhp.org.bw |
| Community mobilization and | mmmalane@bhp.org.bw |
| research operations | minimalane@bilp.org.bw |
| Research data systems | ewidenfelt@bhp.org.bw |
| | Treatment and PMTCT, Field research operations BHP research operations Lab Community mobilization and research operations |

#### TABLE OF CONTENTS

| Principal Investigators2 |
|---|
| List of Co-Investigators3 |
| Table of Contents |
| List of Tables and Figures |
| List of Acronyms and Appreviations |
| Intervention Protocol Synopisis10 |
| 1.0 INTRODUCTION |
| 1.1 Epidemic in Botswana |
| 1.2 Combination Prevention Interventions |
| 1.3 Antiretroviral Treatment as a Component of the Combination Prevention Package |
| 1.4 Proposed Combination Prevention (CP) Package |
| 1.5 Relationship Between Intervention Study Design and Impact Evaluation |
| 2.0 STUDY OBJECTIVES |
| 3.0 OVERVIEW OF STUDY METHODS16 |
| 4.0 STUDY POPULATIONS |
| 4.1 Selection of Study Communities |
| 4.2 Matching of Study Communities |
| 4.3 Eligibility of Community Members |
| 4.4 Enhancement of Services in all Study Communities |
| 4.5 Eligibility Criteria for Inclusion in Interventions in CP Communities |
| 4.6 Rationale for Exclusion in Interventions in CP Communities |
| 5.0 SAMPLE SIZE AND SAMPLE SELECTION METHODS21 |
| 6.0 INTERVENTION PROCEDURES22 |
| 6.1 Overview of Intervention Strategy |
| 6.2 Stakeholder Involvement, Community Engagement, and Community Mobilization |
| 6.3 HIV Testing and Counseling (HTC) |
| 6.4 Linkage to HIV Care and Treatment |
| 6.5 Male Circumcision (MC) |
| 6.6 Identification, Linkage, and Treatment of HIV+ Pregnant Women |
| 6.7 HIV Care and Treatment |
| 7.0 LABORATORY METHODS32 |
| 7.1 Overview of Laboratory Methods |
| 7.2 Training of Laboratory Personnel |
| 7.3 Specimen Collection, Transport, and Processing |

| 7.4 Laboratory Testing for HTC Campaigns |
|---|
| 7.5 Laboratory Testing for IDCC Patients |
| 7.6 Quality Assurance |
| 7.7 Biosafety and Waste Management |
| 7.8 Specimen Storage and Shipment |
| 8.0 DATA SYSTEMS AND MANAGEMENT35 |
| 8.1 Data Collection, Capture, and Flow |
| 8.2 Data Security |
| 8.3 Data Quality |
| 8.4 Confidentiality of data |
| 9.0 DATA AND ANALYSIS PLANS4 |
| 9.1 HIV Testing and Counseling and Linkage to Care |
| 9.2 Care and Treatment |
| 9.3 PMTCT Services |
| 9.4 Male Circumcision |
| 9.5 Analysis Plans |
| 10.0 ETHICAL CONSIDERATIONS |
| 10.1 Ethical Review |
| 10.2 Informed Consent |
| 10.3 Risks |
| 10.4 Benefits of Research Participation |
| 10.5 Confidentiality |
| 10.6 Protocol Compliance and Compliance with UN Convention on the Rights of the Child |
| 10.7 Future Use of Stored Samples |
| 11.0 STUDY SAFETY AND MONITORING PLAN49 |
| 11.1 Reporting Adverse Events |
| 11.2 Data Safety and Monitoring Board (DSMB) |
| 11.3 Protocol Violations |
| 11.4 Monitoring Plan |
| 12.0 ADMINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION |
| 12.1 Study Records and Document Retention |
| 12.2 Information Dissemination and Publication Plan |
| 13 O REFERENCES |

#### **APPENDICES:**

#### **Cross-Protocol Appendices:**

Appendix C2 A. List of Study Communities and Matching Criteria for Community Pairs

B. Back-up Communities in Selected 30 Communities Decline, unavailable or

deemed unsuitable for study inclusion

Figure A: Map of Study Communities in Three Regions

Figure B: Map of Study Communities in the Southern Region Figure C: Map of Study Communities in the Central Region Figure D: Map of Study Communities in the Northern Region

Appendix C3 Size of Study Populations
Appendix C4 Data Safety Monitoring Plan

Protocol 3 Appendix:

Appendix P1 Summary of Variables to be Collected for Ya Tsie Protocol 3

\_\_\_\_\_\_

#### **LIST OF TABLES AND FIGURES**

Figure 1: Data Flow for Combination Prevention Communities

**Table 1:** Precision for 95% confidence intervals for uptake of CP interventions in CP communities

Table 2: BCPP Key Indicators

 Table 3: Summary of approach to consent for various components of the study

#### **ACRONYMS AND ABBREVIATIONS**

AE adverse event

AIDS acquired immunodeficiency syndrome

AHS annual household surveys (follow-up visits of the BHS and HIC)

ANC antenatal clinic (or care)

ART antiretroviral treatment (or therapy)

ARV antiretroviral (drug)

BCPP Botswana Combination Prevention Project
BHHRL Botswana—Harvard HIV Reference Laboratory
BHP Botswana—Harvard AIDS Institute Partnership

BHS baseline household survey

CDC Centers for Disease Control and Prevention

CI confidence interval CP combination prevention

CPC combination prevention community

CRT community-randomized trial
DSMB Data Safety Monitoring Board
ECC enhanced care communities

ELISA enzyme-linked immunosorbent assay

ESS end of study survey

ETC expanded treatment cohort

HIC HIV incidence cohort

HIV-1 RNA human immunodeficiency virus
HIV-1 RNA load in plasma, viral load

HIVDR HIV drug resistance

HTC HIV testing and counseling

HVL high viral load

IAS International AIDS Society
IDCC infectious disease care clinic

IPMS integrated patient management system

IRB institutional review board

LFT liver function test
LTC linkage-to-care
MC male circumcision

M&E monitoring and evaluation

MOH Ministry of Health

MTCT mother-to-child (HIV) transmission
OHRP Office for Human Research Protections

OI opportunistic infection

Option B+ indefinite continuation of ART for women who start ART for PMTCT

PEP post-exposure prophylaxis

PEPFAR President's Emergency Plan for AIDS Relief

PII personally identifiable information

PIMS patient information management system

PMTCT prevention of mother-to-child (HIV) transmission

PLHIV people living with HIV

POC point-of-care

POB pregnant/pregnancy or breastfeeding

QA quality assurance

QC quality control
RHT Routine HIV testing
SAE serious adverse event
SD standard deviation

SMC safe male circumcision (Botswana government initiative)

SMS short message service
SOC standard of care
SoE schedule of events

SOP standard operating procedure

study arm a group of 15 communities that is randomized to receive either standard of care or

study interventions with respect to HIV prevention measures

TB tuberculosis
UN United Nations

UNAIDS Joint United Nations Program on HIV/AIDS

UTT Universal Test and Treat

VDC village development committee

VF virologic failure VL viral load

VPN virtual private network WHO World Health Organization

#### **BCPP Intervention Protocol (#3)**

#### **Protocol Synopsis**

**Overview:** The BCPP study is composed of 2 active interlocking protocols, the Evaluation Protocol (1) and the Intervention Protocol (3). The Closed Clinical Cohort Protocol (Protocol 2) was withdrawn in 2015. An overview of the overarching BCPP study is provided in the BCPP Overall Schema located in the Evaluation Protocol.

#### **Primary Objective of Protocol 3**

1) To implement the combination prevention (CP) intervention package in combination prevention communities (CPC) and describe uptake of these interventions in CPCs (expanded HIV Testing and Counseling (HTC), strengthened Male Circumcision (MC), expanded HIV Care and Treatment, and strengthened PMTCT services).

#### **Secondary Objectives of Protocol 3**

- 1) To describe retention in the clinical cascade of care from HIV diagnosis to viral suppression among all HIV-infected persons.
- 2) To describe uptake of expanded antiretroviral treatment (ART) and clinical outcomes including viral suppression among HIV-positive persons receiving expanded ART.
- 3) To examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions.
- 4) To examine demographic factors, including community of residence, that affect access to health care services.

#### **Study Design:**

The BCPP study is a pair-matched community-randomized trial. This protocol describes the programmatic interventions, including expanded ART, and program monitoring activities that will be conducted as part of the larger BCPP project.

#### **Study Population:**

Thirty community clusters were selected from three geographic regions in Botswana. Prerandomization, community pairs were matched on community characteristics thought to be associated with the outcome of interest of the BCPP (HIV incidence) to improve balance between arms and statistical efficiency. The average total population size of each of the targeted communities is 6,000 (range 2,400 - 12,000), giving a total population across all 30 communities of about 180,800, of whom about 105,000 are adults aged 16-64.

#### **Study Procedures:**

Matched community pairs (15 communities per arm) were randomized 1:1 to Enhanced Care (ECC; Comparison) or Combination Prevention (CPC; Intervention) arms prior to the baseline household survey (BHS) that is conducted as part of the BCPP Evaluation Protocol. Initiation of intervention activities in the CPCs begin immediately following completion of enrollment in the BHS and continue for the duration of the study. CPCs receive the combination prevention intervention package, which includes strengthened HTC, MC linkage, PMTCT services, and expanded HIV care and treatment for HIV-infected persons 16-64 years. In addition, expanded ART for existing HIV-infected community clinic

patients will be offered in the CPCs. Routinely collected clinical data will be used to assess the clinical outcomes for all HIV positive patients.

**Study Duration:** All study activities will occur over a period of approximately 60 months.

#### 1.0 INTRODUCTION AND BACKGROUND

#### 1.1 Epidemic in Botswana

Thirty years into the global HIV pandemic, HIV prevalence and incidence remain high in sub-Saharan Africa. Although this region represents only 12% of the world's population, it accounts for approximately 67% of the world's 34 million HIV-infected persons, and annually, about 70% of the world's 2.7 million new infections occur in this region (UNAIDS 2010). Despite substantial progress in providing HIV treatment and prevention of mother-to-child transmission services (PMTCT) to its citizens, an estimated 25% of adult residents of Botswana are HIV-infected, the second highest adult HIV prevalence in the world, and about 14,000 persons are newly infected with HIV annually, the third highest national HIV incidence rate globally (UNAIDS 2010).

#### 1.2 Combination Prevention Interventions

In the past five years several HIV prevention interventions have proven to be highly effective at reducing transmission of HIV and have offered hope for containing and possibly reversing epidemics in sub-Saharan Africa. For HIV-negative men, MC has been shown to significantly reduce HIV acquisition from HIV-infected female partners. Three randomized controlled trials of circumcision, involving more than 10,000 men in sub-Saharan Africa, demonstrated a 60% reduction in HIV acquisition risk (Auvert, Taljaard et al. 2005, Bailey, Moses et al. 2007, Gray, Kigozi et al. 2007). Additionally, antiretroviral treatment (ART) of HIV-infected persons has been shown to reduce viral load (VL) and consequently the risk of HIV transmission to uninfected partners in sero-discordant couples by as much as 96% (Cohen, Chen et al. 2011). Similarly, the use of antiretrovirals to prevent transmission of HIV from infected mothers to their infants during pregnancy, birth, and breastfeeding can reduce transmission to below 5% (Mahy, Stover et al. 2010; Shapiro, Hughs et al. 2013).

Despite considerable success in scaling up these interventions in many sub-Saharan African countries, especially those supported by the U.S. President's Emergency Plan for AIDS Relief (PEPFAR), adult HIV incidence has remained high (>1%) in many regions in Southern Africa (Botswana, Swaziland, Lesotho, Kwa-Zulu Natal in South Africa, and Southern Mozambique). Multiple factors may account for high HIV incidence in this part of the world. Firstly, viral characteristics of HIV-1 subtype C, endemic in Southern Africa, may make it more infectious than other viral subtypes (Novitsky, Wang et al. 2010, Novitsky, Ndung'u et al. 2011). For example, recent evidence suggests that about one third of persons infected with HIV-1 sub-type C, maintain very high viral loads (VL>50,000 copies/ml) for more than 6 months after sero-conversion. In contrast, viral load following HIV-1 subtype B infection (the prevalent subtype in the United States and Europe) resolves to a steady-state viral set point below 50,000 copies/ml in almost all individuals within four to six months (Daar, Moudgil et al. 1991, Mellors, Munoz et al. 1997, Kaufmann, Cunningham et al. 1998, Little, McLean et al. 1999).

Secondly, the scale and quality of the HIV prevention interventions may have been insufficient to reduce HIV incidence among adults in Southern Africa to levels observed in other parts of the world. For example, the main mechanism by which scale-up of HTC and antiretroviral therapy reduces HIV transmission risk in the community, is by reducing viral load in resident HIV-infected persons, ideally to undetectable levels (VL<400 copies/ml). Studies have suggested that every 0.5 log reduction in an individual's HIV-1 viral load is equivalent to a 40% reduction in individual HIV transmission risk

(Modjarrad, Chamot et al. 2008), and once the viral load is fully suppressed (VL <400 copies/ml) individual HIV transmission risk is virtually zero (Attia, Egger et al. 2009). Despite considerable scale-up of access to HTC and ART, poor retention of HIV-infected persons in the HIV care and treatment cascade from diagnosis to ART follow-up (Rosen and Fox 2011), has mitigated the ability of HTC and HIV care and treatment programs in Southern Africa to reduce the prevalence of HIV-infected persons with detectable viral loads (VL>400 copies/ml). In a meta-analysis of pre-ART retention in Africa, Rosen et al. reported that only 59% of newly diagnosed adults are successfully linked to HIV care and treatment services, only 46% are retained from initial registration and staging at the facility to ARTeligibility, and only 68% are retained from ART eligibility to ART initiation (Rosen and Fox 2011). Of those adults who initiate ART, ~30% are no longer on therapy by 3 years of follow-up, with most of those no longer in care considered lost to follow-up (Fox and Rosen 2010). Therefore, even if 50% of HIV-infected adults in Botswana know their HIV status (BAIS 2008), a considerably lower proportion have a suppressed viral load (Gardner, McLees et al. 2011). The remaining HIV-infected adults with unsuppressed viral load are still infectious and spreading virus in the community. Achieving high coverage of MC among HIV-negative males has also been challenging with most countries, including Botswana, unable to meet ambitious 80% coverage targets to date (Curran, Njeuhmeli et al. 2011).

In summary, despite having the tools to end the HIV epidemic (Fauci and Folkers 2012), insufficient scale, quality, and coordination of prevention interventions have significantly limited southern Africa's ability to sufficiently curb the HIV epidemic. This has led public health experts to call for a "combination prevention" strategy that involves implementing multiple prevention interventions with known efficacy in a geographic area at a scale, quality, and intensity to impact the epidemic (Merson, Padian et al. 2008, Piot, Bartos et al. 2008). Although most experts agree that synchronized implementation of a combination of prevention interventions is needed, there remains considerable debate about what components should be included in the essential combination prevention package (Merson, Padian et al. 2008, Halperin 2009). Four evidence-based interventions (HTC, ART, MC and PMTCT) are recommended for scale-up by almost all prevention experts and will form the cornerstone of the combination prevention package proposed as part of this project (see Section 1.4 below).

#### 1.3 ART as a Component of the Combination Prevention Package

Data show that higher levels of HIV-1 RNA (viral load) are independently associated with both higher rates of HIV transmission and more rapid HIV clinical disease progression and CD4 decline. This study therefore originally included the use of a modified "treatment as prevention" approach that targeted not only those adults who need ART for their own health, but also those adults who are most likely to perpetuate HIV transmission within the community (those with viral load  $\geq$ 10,000 copies/ml). At the time of designing the BCPP in 2012 there was strong experimental evidence supporting initiation of ART at CD4 $\leq$ 350 cells/µL, or WHO Stage III/IV, but conclusive experimental evidence supporting patient benefit of ART initiation at higher CD4 counts, especially CD4 >500 cells/µL was lacking.

The 2013 WHO guidelines recommended initiation of ART in all HIV-infected adults with CD4 $\leq$ 500 cells/µL regardless of clinical stage. In an attempt to provide programmatic data for an anticipated change in CD4 threshold for ART initiation in Botswana and to enhance the power of the study to answer its primary objective, the threshold for ART initiation in the Combination Prevention arm was modified in early 2015 (from CD4 $\leq$ 350 to CD4 $\leq$ 500 regardless of viral load, in addition to offering expanded ART to persons with CD4>500 and viral load  $\geq$ 10,000).

Shortly thereafter, in July 2015, the WHO announced that it would revise ART guidelines to recommend universal treatment (regardless of CD4 count or HIV disease severity). The WHO's plans were informed by results from two clinical ART trials. One, the START trial, reported that early drug treatment of people with HIV cut their risk of serious illness or death by 57% (Lundgren, Babiker et al. 2015). Another, the TEMPRANO study, released findings that early ART significantly decreased morbidity overall and when restricted to patients with baseline CD4>500 cells/µL (Danel, Moh et al. 2015). WHO published an early release guideline on when to start ART and on pre-exposure prophylaxis for HIV in September 2015 (World Health Organization 2015). The BCPP study team, with the support of the DSMB and funder, is revising the intervention treatment initiation criteria once more to take these new results and WHO guidelines into account. Universal Test and Treat (UTT) is therefore included in the combination prevention package with version 4.0 of the protocols.

In June 2016, Botswana treatment guidelines changed to UTT. All PLHIV living within the Enhanced Care communities (ECC) are now eligible to receive ART according to these updated Botswana national guidelines. Residents in the Combination Prevention communities will also continue to receive universal treatment as prevention.

Through additional modeling, the study team has adjusted effect size and power calculations to reflect a move to UTT in both the Combination Prevention and Enhanced Care arms, using a range of roll-out timelines. This revised modeling also uses estimates of coverage (by HTC, LTC, ART, MC) that are consistent with what has been observed in BCPP thus far, rather than using the higher coverage "targets". Model-based estimates suggest that the impact of a change in treatment policy on the power to detect a difference in cumulative incidence (the primary objective of BCPP) may still yield at least 70% power (Protocol 1, v4.0, section 5.1.1), but the impact depends on the exact nature and timing of the implementation of changes in policy as well as other prevailing conditions. The retention of this level of power even with Enhanced Care communities moving to expanded access to ART is at least in part attributable to the fact that BCPP is implementing multiple HIV prevention interventions (including higher HTC coverage, linkage to HIV care/treatment, etc.).

#### 1.4. Proposed Combination Prevention (CP) Package

In version 4.0 of this protocol, the combination package includes universal treatment of all PLHIV along with a package of interventions that are designed to: 1) Identify all HIV-infected adults in CP communities, 2) reduce barriers to ART initiation, 3) support adherence and retention on ART, 4) increase capacity of clinics to support aggressive ART scale-up, and 5) enhance the use of both individual and clinic-level data to ensure maintenance of quality of HIV care and treatment.

The revised combination prevention package for this project includes:

- Rapid scale-up of HTC services, with a target of ensuring ≥90% of HIV-infected adults aged 16-64 have documentation of their HIV-infected status.
- Rapid scale-up of universal ART for all HIV-infected adults, with a target of ensuring that <u>></u>93% of adults diagnosed with HIV infection are receiving ART.
- Rapid scale-up of retention in care and adherence interventions, with a target of ensuring that >95% of HIV-infected adults receiving ART are virally suppressed with HIV-1 RNA < 400 copies per ML.

- Scale-up of linkage to MC services, with a target of ensuring <u>></u>60% of HIV-negative men (aged 16–49) are circumcised.
- Rapid strengthening of PMTCT services, with a target of ensuring >90% of women initiated on indefinite ART (Option B+) during pregnancy remain in care and on treatment post-delivery.

The targets for intervention communities in this version of the Protocol have been revised from the targets in Protocol 3, version 3.0. Targets for ART initiation and viral load suppression have been raised based on the higher than expected baseline levels of ART initiation and viral load suppression coverage as measured in BCPP BHS and HTC campaign. The MC target has been lowered from 80% to 60%. This change is in accordance with the DSMB's 2013 recommendation based on concerns that the 80% target might not be realistic; results to date support these expectations.

To reach stated scale-up targets (cumulative over 3 years) several service uptake initiatives will be implemented, including (1) community mobilization to encourage HTC and MC uptake, (2) targeted HIV testing to include hard-to- reach populations, (3) strengthening linkage to care, treatment and/or PMTCT services for known HIV-infected adults not in care and newly diagnosed HIV-infected adults, (4) strengthening linkage to MC services for HIV-negative or HIV-unknown status males identified at HTC services, (5) strengthening retention in care and adherence to ART services at clinics (6) expansion and strengthening of HTC, ART, PMTCT services, and MC services through recruitment of additional health care personnel and counselors, and (7) strengthened monitoring and evaluation of prevention, care and treatment programs to ensure stated targets are reached.

Adults aged 16-64 will be targeted for service uptake because recent, nationally representative surveys of HIV prevalence and incidence (BAIS 2008) suggest that HIV incidence remains high (>1%) throughout this age group. Modeling exercises suggest that meeting scale-up targets by the end of two years of program implementation, and maintaining treatment coverage thereafter, could result in community HIV incidence reductions of 40% by the end of three years of implementation.

#### 1.5. Relationship Between Intervention Study Design and Impact Evaluation

A separate protocol (BCPP Evaluation, Protocol #1) describes in detail the proposed plans for evaluating the impact of the combination prevention (CP) package on adult population level HIV incidence. In brief, a randomized design was proposed to provide experimental evidence of CP package impact and because population-level HIV incidence is the outcome of interest, a community (rather than individual) randomized trial is proposed. Thirty study communities have been selected and matched into pairs. Pair-matching is done to improve balance between study arms and statistical efficiency (Hayes and Moulton 2009). Communities within pairs were randomized to Combination Prevention Community and Enhanced Care Community (CPC and ECC) arms. Following community matching, a baseline 20% household survey (BHS) was implemented to recruit an HIV Incidence Cohort (HIC) of eligible, consenting, and HIV-negative adults aged 16-64. The HIC will be followed annually during Annual Household Survey (AHS) visits to assess cumulative HIV incidence over 30 months. Study participants who are not eligible for the HIC will also be followed annually in the AHS, to assess, in both study arms, uptake of HTC, ART, MC services and PMTCT services in each arm and to describe major health outcomes (such as death). Cumulative incidence will be compared between study arms to assess CP package impact.

Combination prevention package coverage in the community will be estimated at baseline (in the 20% BHS) and through a large end of study survey (ESS). In addition, during study conduct, progress in reaching target coverage levels will be captured from monitoring data collected as part of routine programmatic activities.

#### 2.0 STUDY OBJECTIVES

#### **Primary Objective**

1) To implement the combination prevention (CP) intervention package in CPCs and describe uptake of these interventions (expanded HTC, strengthened MC, expanded HIV Care and Treatment, and strengthened PMTCT services).

#### **Secondary Objectives**

- 1) To describe retention in the clinical cascade of care from HIV diagnosis to viral suppression for HIV-infected persons.
- 2) To describe uptake of expanded ART and clinical outcomes including viral suppression among HIV-positive persons receiving ART (UTT).
- 3) To examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions.
- 4) To examine demographic factors, including community of residence, that affect access to health care services.

#### 3.0 OVERVIEW OF STUDY METHODS

As described in the introduction, the over-arching design is a pair-matched community-randomized trial (CRT). The full details of the CRT, including how communities were selected, how they were matched, community randomization, the BHS, enrollment of the HIV incidence cohorts (HIC), and the end of study survey (ESS), are described in the BCPP Evaluation Protocol. This protocol describes the interventions implemented in 15 communities randomly selected from the 30 study communities (*Appendix C2*), monitoring and evaluation (M&E) plans, and the program data systems.

#### **4.0 STUDY POPULATIONS**

#### 4.1 Selection of Study Communities

Thirty communities (*Appendix C2*) in three geographic areas in Botswana: (1) around Gaborone in the south east, (2) around Francistown in the north east, and (3) in the region around Mahalapye, Serowe, and Palapye in the central eastern region, are included in the study. These communities were selected based on two criteria: (1) communities needed to be of sufficient size to meet sample size requirements for the HIV Incidence Cohort (described in BCPP Evaluation Protocol), and (2) implementation of the proposed combination prevention package needed to be feasible. Feasibility requirements are listed below:

#### • Community Criteria

All communities must:

- Have a health center from which HIV care and treatment, PMTCT, or HTC can be provided.
- Be reachable by road via a <8 hour drive from Gaborone or Francistown. (CDC and the Ministry
  of Health have permanent, well-staffed offices in Gaborone and Francistown, while the Harvard</li>

- Chan School has a permanent office in Gaborone. This distance parameter makes the study easier to implement and monitor for quality control purposes).
- Have a clear geographic boundary such that it is reasonably easy to identify a household as either being part of, or outside of, the study community.

These inclusion criteria resulted in the exclusion of urban areas from the study. Approximately 61% of Batswana (plural noun for Botswana citizens) live in urban areas with a rate of urbanization of about 2.3% per year (annual rate of migration from rural or peri-urban regions into urban areas). Restricting the study to rural and peri-urban areas, besides being necessary for study feasibility, should not limit the generalizability of study findings to urban areas. If the combination prevention package is shown to be effective at reducing adult HIV incidence, the principle of scaling up combination prevention package coverage for prevention effectiveness should be applicable to urban settings.

The 30 study communities selected meet the criteria described above. The average total population size of each of the targeted communities is 5,855. Assuming an average community size of 5,855, we estimate a total population in all 30 study communities of about 175,664 people; 87,832 persons in the CPC arm of which ~58% of community residents are aged 16-64 (*Appendix C2/C3*). HIV prevalence among residents aged 16-64 is estimated at 25%, resulting in an estimated 25,471 HIV-infected residents aged 16-64 (12,736 per study arm).

#### 4.2 Matching of Study Communities

Due to the small number of communities that can be enrolled in a community randomized trial for cost and feasibility reasons, the likelihood of imbalance of potential confounders between study arms is increased. A restricted randomization, matching, and stratification were considered as strategies to ensure balance between arms. A pair-matched design was chosen because:

- This approach is more likely than stratification to achieve balance between study arms;
- Matching has the added advantage of improving statistical efficiency compared with restricted randomization, and;
- Chosen matching covariates (see below) are quite closely correlated with the outcome of interest (adult HIV incidence), making a matched design of similar or increased statistical efficiency compared with a stratified design, even though a matched design entails greater loss of degrees of freedom.

Possible disadvantages of a pair-matched design include:

- Loss of both communities in a pair if one community drops out.
- It is not possible to assess whether the intervention effect varies between matched pairs, whereas, in a stratified design, opportunity to assess effect modification across strata would be possible.

The following matching criteria were chosen:

- Community size: Although community size in Botswana may not be associated with the outcome
  of interest (HIV incidence), achieving sample size balance between arms improves statistical
  efficiency.
- Baseline Access to Health Services including ART: Access to ART is associated with HIV incidence (Montaner, Lima et al. 2010, Tanser, Bärnighausen et al. 2012). Although some communities within matched pairs have access to primary care clinics and others have access to primary care hospitals,

in Botswana this does not appear to represent a significantly different level of access to health services.

- Age structure: Adult HIV prevalence and incidence are correlated with adult age (Central Statistics Office 2009). Age structures are very similar within the study community pairs. If we use the proportion of adults (16-64) who are in the highest risk for HIV infection (25-34) as an indicator of age structure, the median difference in this proportion is 2% (range 0-7%). [Note: we do not have age structure data for Gumare, Shakawe, Mandunyane, or Mmadinare, but based on the age structure of the other 26 selected communities, do not expect any significant differences in age structure within the matched pairs].
- Geographic location as measured by proximity to major urban centers (Hayes, Mosha et al. 1995).
   Geographic locations of communities within pairs, as estimated by average distance to the nearest large towns, are quite similar. For example, across 30 communities, the range of average distances to nearby urban centers ranges from 18-380 kilometers. However, following matching, the median difference in distance to an urban center between communities in a matched pair is 20 kilometers (range 3-150).

Access to community-specific measures of HIV prevalence [e.g., HIV prevalence measured from antenatal care (ANC) clinics] were not available prior to community selection/randomization. Previous successful pair-matched CRTs (Hayes, Mosha et al. 1995) where HIV incidence was the outcome of interest have also addressed the problem of absent baseline HIV prevalence estimates by using geographic location and other proxies of HIV prevalence as matching criteria.

- **4.3 Eligibility of Community Members** The following definitions of the study community will be used in the protocol:
- <u>Botswana Citizen:</u> A Botswana citizen is anyone who can produce proof of Botswana citizenship. (Usually this is the Omang number or Omang application receipt). The Omang number is needed in Botswana to access routine government services. It is anticipated, based on a community survey in Mochudi, and the 2011 census (Census 2011), that less than 3% of residents will be non-citizens.
- <u>Spouse of Botswana citizen</u>: A spouse of a Botswana citizen is a person who can produce evidence
  of being married to a Botswana citizen, usually a marriage certificate, and is therefore eligible to
  receive free medical services in Botswana.
- <u>Permanent study community resident:</u> An individual who reports spending on average ≥14 nights/month each month in that community for the past 12 months or an individual who recently moved into the community and reports spending on average ≥14 nights each month since arriving.
- <u>Part-time study community resident:</u> An individual who reports spending 3—13 nights (on average) each month in that community for the past 12 months or an individual who recently moved into the community and reports spending on average 3-13 nights each month since arriving.

• <u>Non-residents:</u> An individual who reports living outside of the community but is receiving treatment in the CP community clinic as well as those individuals with an unknown community of residence who are receiving treatment in the CP community clinic.

#### 4.4 Enhancement of services in all study communities

One of the goals of BCPP is to provide enhancement of HIV prevention, care and treatment services in non-intervention (ECC) communities as well as expansion and strengthening of these services in the combination prevention communities. This goal is primarily motivated by two factors:

- 1) A commitment to offering the enhanced care communities tangible benefits from participating in this community randomized trial, and
- 2) The imperative to bring the standard of practice in all study community clinics close to the standard of care, so that the BCPP study is assessing the effect of the combination prevention interventions on HIV incidence.

For the purposes of BCPP, the term 'enhanced' will be used to signify activities done in all study communities (including Enhanced Care Communities) for the purposes delineated above, whereas the terms 'strengthened' and 'expanded' will be used to signify activities done in Combination Prevention Communities only, as part of the study's combination prevention intervention package. 'Strengthened' will signify that activities are already part of national policy and practice, whereas 'expanded' will signify that activities are beyond current national policy and practice (for example, 'expanded' antiretroviral therapy in the CPCs).

The following enhancements will be provided in all 30 study communities, including the ECCs:

- a) Baseline and Annual Household Surveys (Evaluation Protocol): As part of the BHS that occurs in all 30 communities (in both study arms), ~20% of adults are offered home-based HIV testing, point-of-care CD4 count if treatment-naïve, viral load testing, and referral for HIV care and treatment, PMTCT services, MC, and other health services as appropriate (TB screening, for example). HIV-infected persons who were ART naïve at entry to BHS or who seroconvert between study visits and are ART-naïve will also have annual point of care CD4 and viral load tests, and these results will be shared with participants/clinics respectively. HTC is also offered to household residents who do not wish to take part in the BHS/AHS, either by the BHS study team, the HTC campaign team, or by referral to local clinics where HIV testing is available.
- b) Clinical care quality assessment and quality improvement: BCPP and/or CDC Botswana will work through the Ministry of Health to support clinical quality care assessment and improvement. Existing or new Ministry of Health and CDC tools and quality improvement documents will be used or expanded in this effort.
- c) Clinical data system support: BCPP will provide technical assistance to the Ministry of Health to support improved implementation and utilization of clinical data systems (primarily PIMS2 and IPMS) in all 30 study communities.

d) Laboratory support: BCPP will provide technical assistance to Ministry of Health to help laboratories supporting clinics in all 30 study communities to perform at a level sufficient to meet the standard of care. Existing or new Ministry of Health and CDC tools and quality improvement documents may be used or expanded in this effort.

#### 4.5 Eligibility Criteria for Inclusion in Interventions in CP Communities

This protocol provides the inclusion and exclusion criteria for access to the services provided as part of the Combination Prevention intervention package. Adults aged 16-64 will be targeted for service uptake because recent, nationally representative surveys of HIV prevalence and incidence (BAIS 2008) suggest that HIV incidence remains high (>1%) throughout this age group.

For clinical services, only those who are Botswana citizens or spouses of Botswana citizens can receive free services from Ministry of Health facilities. Non-citizen/non-spouse of citizen HIV-infected adults identified during testing will receive a referral to the health clinic in their community of residence, but will not be eligible for free services from Ministry of Health facilities, and thus will not be eligible for strengthened free services in intervention clinics.

Investigators propose that eligibility for interventions in the CPC arm be grouped into three categories (a) eligibility for expanded HTC services and (b) eligibility for strengthened linkage-to-MC services, and (c) eligibility for expanded treatment and follow-up.

#### a) Eligibility for Expanded HTC

All adults ≥16 who wish to receive HTC services at health facilities, mobile testing units, or door-to-door programs in combination prevention communities (CPCs), are eligible to receive these HTC services. The rationale for proposing that non-residents of the CPC be able to access expanded HTC services is to improve community acceptance of the door-to-door and mobile HTC activities. Preliminary discussions with community leaders suggest that restricting access to a service like HTC which is being delivered to family homes and neighborhoods would be met with considerable resistance and community discontent.

Non-citizens of Botswana will also be provided HTC services in the CPC. Non-citizen/non-spouse of citizen HIV-infected adults identified during testing will receive a referral to the health clinic in their community of residence to connect them with available fee-based services including treatment.

#### b) Eligibility for Strengthened Linkage-to-MC services

Noncitizens will continue to be eligible for enhanced linkage- to-MC services if they meet other eligibility criteria. Under the national MC programs, noncitizens who present directly to the MC tent requesting MC will be offered free services. Thus, all adult men 16 years or older who are HIV-negative or have unknown HIV status are eligible for strengthened linkage-to-MC services including men who decline HIV testing or have indeterminate results. Under current national guidelines, boys 13-15 years old will not be actively mobilized or included in linkage-to-MC though they can continue to receive free MC services at national locations if they present with parental permission.

#### c) Eligibility for Universal Treatment

Universal treatment will be offered to all HIV-infected adults aged 16-64 who are Botswana citizens or spouses of Botswana citizens. HIV-infected persons referred through the study via BHS/AHS, HTC or

routine HIV testing (RHT) as well as existing patients already enrolled in care at the CPC clinics will be offered expanded treatment. The Infectious Disease Care Clinics (IDCC) treat all Botswana citizens and spouses of Botswana citizens regardless of the community in which they reside. Therefore, both residents and non-residents of the community will be included.

#### 4.6 Rationale for Exclusion from Interventions in CP Communities

• Rationale Surrounding Need for Botswana Citizenship or for Being Spouse of Botswana Citizen: Although the Botswana Government provides free HTC services to non-citizens, free access to health services, including ART and PMTCT is restricted to a) persons who can produce valid documentation of Botswana citizenship or b) spouses of Botswana citizens. Combination prevention interventions will therefore not be available to non-citizens of Botswana unless married to a citizen, except in the case of HTC and MC services. The exception for MC will be made to bring study goals closer to aligning with WHO goals for protection of communities through MC provided to 60% of HIV-uninfected men - regardless of citizenship status - as noncitizens living in the community may share the same sexual networks with citizens.

Additionally, men who decline HIV testing may actually be those at greatest risk for HIV acquisition and thus could benefit most from MC. If such men were not offered MC and were later found to be positive at end of study they would have represented a missed opportunity for prevention.

• Rationale for Age Limits: Persons <16 years of age will be excluded from study participation because our intervention is targeting adults, and relevant study outcomes will be measured among adults. In Botswana, adults are considered those aged 16 or older. For example, all persons aged ≥16 can access medical services, including HTC, without guardian consent. Although individuals aged 16-17 can access medical services without guardian permission, participation in research still requires guardian permission, because the age of consent for research in Botswana is 18. Therefore, eligible 16-17 year-olds will be asked for assent to participate in research activities only after permission has been provided by the guardian.</p>

#### 5.0 SAMPLE SIZE AND SAMPLE SELECTION METHODS

The primary objective for the intervention protocol is to implement and describe uptake of CP interventions in CP communities. Combined (BHS and HTC) data for 7 intervention communities was used to derive average denominator sizes for the estimates of interest. These community-average sample sizes were multiplied by 15 to yield an estimate of the total denominator (see Table 1). For the estimate of uptake of HTC, we used the number of participants interviewed to be conservative, although estimates of HTC coverage will be extrapolated to persons not interviewed.

Table 1 presents confidence limits for all of the indicators of uptake of CP interventions for protocol 3, using targets presented earlier in the protocol. Sample size calculations were done using a simple binomial method to obtain standard errors and then multiplying standard errors by the square root of the variance inflation factor (VIF), which is [1+(m-1)\*ICC], where m is the average number of members of each group (here, participants within community), and ICC is the intraclass correlation coefficient,

reflecting the magnitude of the correlation within communities for the outcome measure of interest. No published ICCs were available for these outcomes, so we used one small and one large value, based on prior publications reporting ICCs for behavioral variables in HIV and STD studies (Zhang et al., 2013 and Pals et al., 2003).

Table 1. Precision for 95% confidence intervals for uptake of CP interventions in CP communities

| Outcome | Denominator<br>(per community) | Denominator<br>(Total across CP<br>communities) | ICC | Coverage | 95%<br>Confidence<br>Interval | CI<br>Width |
|---|---|---|---|---|---|---|
| HTC | 2469 | 37035 | .02 | 90% | 87.8, 92.2 | 2.2 |
| | 2469 | 37035 | .05 | 90% | 86.5 <i>,</i> 93.5 | 3.5 |
| PMTCT | 50 | 750 | .02 | 90% | 87.0, 93.0 | 3.0 |
| | 50 | 750 | .05 | 90% | 86.0, 94.0 | 4.0 |
| MC | 794 | 11910 | .02 | 60% | 56.4, 63.6 | 3.6 |
| | 794 | 11910 | .05 | 60% | 54.4, 65.6 | 5.6 |
| ART | 528 | 7920 | .02 | 93% | 91.1, 94.9 | 1.9 |
| | 528 | 7920 | .05 | 93% | 90.0, 96.0 | 3.0 |

Table 1 shows that where sample sizes are large and we expect rates of uptake closer to 100% (HTC and ART), precision is excellent. Where sample sizes are small (PMTCT) or rates expected closer to 50% (MC), we have less precision for estimates, but confidence interval widths are still less than ±6%. As the rate of the outcome variable of interest moves away from 50%, standard errors and confidence interval width will decrease. With a larger ICC, the variance inflation factor increases and confidence intervals will widen.

#### 6.0 INTERVENTION PROCEDURES

#### **6.1** Overview of Intervention Strategy

Interventions described below are intended to: 1) be consistent with new WHO guidelines on treatment of HIV infection (World Health Organization, 2015), 2) streamline clinic procedures to accommodate expansion of treatment to all PLHIV, and 3) incorporate lessons learned during the first year of BCPP. Targeted strategies will be implemented to meet UNAIDS goals of 90% of PLHIV know their status, 90% of PLHIV who know their status are on treatment, and 90% of PLHIV on treatment are virally suppressed. Through reaching the UNAIDS goals, it is anticipated that there will be a reduction in HIV incidence in the CP communities as assessed in Protocol 1. The proposed BCPP interventions will demonstrate UTT and introduce a streamlined approach to finding, testing, and starting PLHIV on immediate treatment and retaining them on effective treatment over time. Specific engagement activities as well as the specific interventions being deployed are outlined in detail below.

#### 6.2 Stakeholder Involvement, Community Engagement, and Community Mobilization

To enhance communities' acceptance and effectiveness of the combination prevention package, local government and community stakeholders will be highly engaged. Program implementers, including MOH at central-, district-, and facility-level, and NGOs supporting the MOH's public health mission in

study districts, have been engaged in the planning and continue to be involved in implementing all combination prevention interventions. These governing bodies include:

- National Government: MOH, CDC and Harvard Chan School investigators and program planners have presented project plans to (1) the Parliamentary Sub-committee on Health, (2) the Parliamentary Sub-committee on HIV/AIDS, and, (3) the House of Chiefs (a body of traditional leadership made of representatives of all communities in the country).
- District Government: Study communities are distributed across 13 of 29 districts in Botswana.
   Meetings and consultations have been held with the District AIDS Coordinator, District Multi-Sectoral AIDS Committee, and the District Health Management Teams.
- Community Government: At the community level, village political leadership has been consulted, including the traditional leadership of *Dikgosi* and *Dikgosana* (Chiefs and sub-chiefs), the Village Development Committees (VDCs), church leaders, and sporting clubs. Project plans were shared and discussed prior to initial implementation and ongoing support for the project is sought.

Investigators meet regularly with members of study Community Advisory Boards (CAB) to discuss community perceptions of the project. Minutes of these meeting are documented and shared with the study principals. Specific issues raised during CAB meetings are addressed as needed. There are four CABs located in the following regions: *South, Central, North, and Northwest.* The CABS have representatives from the study communities in that region.

Community mobilization activities are conducted in all communities; however, the scope and duration of the activities are greater in the CPCs. Activities focus primarily on increasing uptake of HTC and MC so that HIV-infected adults can access treatment and/or PMTCT and HIV-negative adults can access MC. Some of the methods to improve uptake of services include:

- o Public announcements from vehicles with loudspeakers (very common in Botswana),
- Community (kgotla) meetings, civic society activities, schools, and clinics as a platform to inform the community.
- Door-to-door canvassing of the community informing community members of the services that are available in the community, location and duration.
- Specific mobile activities (e.g., location of an HTC caravan near work and sporting locations or in residential areas after business hours (e.g., after 5 pm) targeting hard to reach populations like men.

#### 6.3 HIV Testing and Counseling (HTC)

- a) Target: 90% of PLHIV know their status.
- b) Strategy: Based on the first round of HTC in BCPP, the HTC strategy is being modified for years 2 and 3. During the first year of HIV testing, approximately 70-% of HIV+ persons in the community were identified through concentrated testing efforts lasting 6-8 weeks. During the 2<sup>nd</sup> year of the study, HTC activities will be provided through continuous availability of services in the community and will focus on 1) finding incident cases of HIV infection by retesting persons found to be

negative during the 1<sup>st</sup> year; 2) finding the 25-30% of community members missed by the 1<sup>st</sup> year of testing in BCPP; and 3) identifying HIV+ persons who are new arrivals to the community.

The activities to fulfill the first objective of finding incident HIV cases include 1) repeating door-to-door HIV testing during year 2 in all homesteads from year 1; 2) monthly mobile testing at targeted community locations; and 3) strengthening routine HIV testing (RHT) in health facilities with a focus on antenatal clinics, outpatient departments and IDCC. To fulfill the 2<sup>nd</sup> objective, targeted testing activities will be used to find community members missed in the first year of testing in BCPP. Based on data collected in year 1 of BCPP, approximately 50% of men and 30% of women are missed through home-based testing. Targeted testing strategies to locate those missing in year 1 will include workplace testing, home-based testing on holidays and weekends, mobile testing at venues frequented by men and large-scale community activities that attract the majority of community members. To fulfill the 3<sup>rd</sup> objective, new arrivals to the community who are HIV+ will be found through re-enumeration of households and HIV testing while going door-to-door. New arrivals will also be identified during community mobile testing and large-scale community events that offer HIV testing. The HTC strategy for year 3 of BCPP will be based on findings from year 2 of the study, but is likely to focus on targeting populations missed in year 2.

In order to reach the target of the 90% of PLHIV knowing their status, cost-effective community-based HIV testing strategies are needed to find unidentified HIV-positive persons who are not accessing health care facilities, such as young women and men. An understanding of the incremental costs between strategies is key to determine the optimal mix of strategies to implement. Therefore, a cost analysis of different HTC models implemented through BCPP will be undertaken.

#### c) Specific HIV Testing and Counseling Services:

- 1) Home-Based HTC: HTC counselors will go door-to-door and request verbal consent to: (1) map household GPS location, (2) record numbers of persons in each household, their age, and sex by interviewing the head of household or, if the head of household is absent, a household member 18 years of age or older (Household Enumeration Form), and (3) offer HTC services (HTC Intake Form). The following individuals will not be offered HTC:
  - a. Adults who have documentation of an HIV-positive status
  - Adults who have documentation of HIV-negative results obtained within the last 3
    months of the HTC encounter. (Documentation of HIV test results are recorded on the
    HTC Intake Form)
  - c. Persons <16 years old

If a household member is absent, the team conducting the home-based HTC activities will ask about an appropriate time to return to the household (*Household Enumeration Form*). Up to 3 repeat visits will be scheduled.

- 2) *Mobile HTC*: Mobile HTC caravans and tents will be placed in prominent locations of the community [e.g., at kgotlas (community meeting locations), or shopping centers]. Community mobilizers will engage the community via door-to-door 'mobilization' visits and in high traffic areas in the community such as shopping and transport areas and invite residents to get tested in the mobile units and tents. Lay counselors and support staff will be stationed in mobile venues consisting of a waiting area, private HTC area and a phlebotomy area. HTC will be offered to all individuals (residents and non-residents, citizens and non-citizens) who are not known to be HIV-infected according to national guidelines (i.e., adults who do not have an HIV test result card indicating HIV-positive status). Persons who tested will be asked to keep the card with their results safely for any future contact, e.g., during subsequent household visits (below).
- 3) Routine Facility-Based HTC: Routine HTC activities at health facilities will be strengthened by training facility-based counselors to offer RHT as part of integrated routine services in outpatient, IDCC, and antenatal (ANC) clinics. Facility-based counselors will be encouraged to provide testing to all adults receiving health care services at the clinic and to offer testing to all friends, family members, relatives, visitors, etc. (so-called non-patients) accompanying the patient to the clinic. In addition, the study will assist MOH ANC staff with strengthening of 3<sup>rd</sup> trimester re-testing among pregnant woman (see section 6.6). Routine HIV testing data will be extracted from PIMS2/IPMS to monitor coverage of testing in health facilities.
- 4) **Targeted Testing:** HTC for groups that are difficult to access through home-based, clinic-based, or other routine services will be targeted by providing services where these groups work or congregate and by offering HTC services at large, well-attended community events such as barbecues, health fairs, concerts, etc.
- 5) Additional Services for Persons Testing HIV-Positive: All HIV positive adults not on treatment are eligible for ART under current national guidelines so will not need to consent for treatment in the UTT intervention. HTC counselors are trained to integrate treatment preparation, adherence and readiness messages into their post-test counseling for HIV-positive persons to begin preparing participants for initiating ART at their first clinic visit. In addition, they will be counseled to expect a confirmation test for HIV positive results before initiating ART which will be conducted at the IDCC. All participants of HTC will be tested using the MOH rapid testing algorithm along with pre-test and post-test counseling that is recommended in the national guidelines.
- 6) Additional Services for Persons Testing HIV-Negative: The following services will be offered to newly identified or known HIV-negative adults:
  - Screening of all adults for TB, with a simple screening question, and referral of TB suspects to the nearest clinic for TB testing. TB suspects will be prioritized for evaluation at the clinic. In Zimbabwe and Zambia, this has been shown to reduce community prevalence of infectious TB and was well-accepted by the community (Corbett, Bandason et al. 2010).
  - Encourage MC uptake by HIV-negative males through linkage-to-MC services. These services also are offered to men with unknown HIV status. Further details of the linkage-to-MC service are provided in Section 6.5 below.

- HIV-negative pregnant women will be encouraged to enroll in ANC care and be retested in their 3<sup>rd</sup> trimester.

#### 6.4 Linkage to HIV Care and Treatment

- a) Targets: 80% of adults identified as newly diagnosed or not currently in care are registered at the local study IDCC or are documented in care at another IDCC within 90 days of BCPP interview and 90% within 180 days of BCPP interview
- b) Strategy: To ensure that 90% of persons identified as HIV-infected initiate ART, persons newly identified as HIV-infected or PLHIV not connected to care and treatment must be linked to an IDCC. Data from the first year of BCPP suggest that about half of PLHIV link to care with very little prompting or follow-up. Another 50%, however, require additional supports. The linkage intervention package for BCPP includes: 1) counseling after diagnosis on the importance of immediate treatment and appointments made for PLHIV not already in care; 2) appointment reminders; and 3) tracking and tracing of persons who miss appointments at the IDCC. In addition, to enhance linkage rates, patients wishing to receive care/ART outside of their community will be able to link to any MOH IDCC.

#### c) Specific Activities:

- 1) Counseling After Diagnosis and Scheduling Appointments at IDCC: Counselors will be available to: (1) provide immediate psychosocial support to help clients cope with their HIV-positive test result, (2) counsel participants on the importance of early entry into HIV care or PMTCT services and prepare them for treatment initiation and adherence at first clinic visit, and (3) help clients establish and achieve plans to enter care by identifying and troubleshooting real and perceived barriers to care (Gardner, Metsch et al. 2005, Gardner, Marks et al. 2007, Craw, Gardner et al. 2008, Gardner, Marks et al. 2009). Appointments at IDCCs in intervention communities will be scheduled as soon as possible for newly diagnosed individuals or PLHIV who are not enrolled in care and treatment. Some PLHIV may prefer to obtain care and treatment services at a clinic outside their community for privacy, proximity to job, or other reasons. For those PLHIV who choose to obtain care outside the study community, verification of enrollment in care will be obtained from the MOH data systems.
- 2) **Appointment Reminders:** PLHIV will be sent short message service (SMS) reminders about their upcoming appointments.
- 3) Tracking and Tracing: A record of all patients referred to care by BHS, HTC and RHT will be submitted to Site Coordinator at the local IDCC. The Site Coordinator at the IDCC will access names of those referred and will track them to ensure they keep their first appointment. Names and contact information of those who don't keep their appointments will be turned over to the community counselor for tracing and case management. The intensified participant tracing program includes telephone calls and home visits for persons who missed a scheduled appointment up to 180 days after either diagnosis or BCPP interview for known HIV positive persons (Participant Tracing Log).
- 4) Counseling, Appointments and Tracing for PLHIV Identified who are already on ART

- Patients who are on ART, enrolled in care at the study IDCC, are not late for an appointment, and have a future appointment scheduled will be encouraged to remain adherent to ART and appointments.
- Patients who have initiated ART and are enrolled in care at the IDCC and are late for their next appointment or who do not have a future appointment scheduled will be (1) counseled on the importance of adherence and appointment keeping, (2) given a new appointment at the clinic, and (3) have phone number and residential address information obtained to facilitate follow-up (retention tracing of participants already in care and late for their scheduled appointments is described in section 6.7 below).
- Patients who are on ART and not enrolled in care at the study clinic will be counseled to remain adherent to ART and in care; they will also be informed of expanded and strengthened services available at the study clinic and will be given an appointment to the study clinic. Follow-up for these patients will be limited to only an SMS reminder for their appointment. Verification of the patients' enrollment at another clinic outside the study community and ART status will be obtained from MOH data systems.
- 5) Retrospective Tracking and Tracing of PLHIV who Did Not Link to Care: Given the change in the 2016 Botswana national treatment guidelines, HIV-positive participants not on ART who did not link to care from Round 1 (October 2013 February 2016) will be retrospectively contacted by the Ministry of Health clinic staff or a community counselor and informed that all HIV-positive persons are now eligible for ART, regardless of CD4 count or condition. Participants from Round 1 and Round 2 (June 2016 present) who previously did not give permission for follow-up may also be contacted, as the new guidelines recommend tracking all HIV-positive persons identified to care and treatment sites. Specifically,
  - Contact with the participant will be attempted by a Ministry of Health clinic staff member or a community counselor to inform the participant that the national guidelines have changed and all persons that are HIV-positive are now eligible for ART. They will also be informed that it is critical for their health and the health of their partners and children to get on ART as early as possible, and that the clinic offers services to help community members get into care and on treatment. Staff will use the updated talking points from the Linkage to Care SOP revised (see Appendix XX, Section 3.8).
  - Participants will be given an appointment at the clinic with a health care provider and will be encouraged to keep it.
  - If there is no current phone number for the participant, a home visit will be conducted by a clinic staff member or a community counselor. Up to 3 attempts to contact the participant will be made through alternating phone and home visits.
  - Participants from Round 1 who have not linked to care will be contacted beyond the follow-up period specified in the protocol (e.g., 180 days) in order to ensure the new guidelines are being implemented with all participants. Paricipants from Round 2 who were enrolled during the time between the introduction of the new guidelines and field implementation (November 2016) may also be followed beyond the 180 day window.

A note to file will be documented at each of the 15 intervention sites noting the procedural changes and follow-up provided to those individuals who previously did not link and declined follow-up.

#### 6.5 Male Circumcision

- a) Target: 60% of HIV-negative 16-49-year-old males are circumcised
- b) Strategy: BCPP's SMC intervention in the second year will be streamlined from the full-service campaign model used in the first year to a program that mobilizes and links interested men to existing services in nearby locations. MC services are expected to be provided in five of the 15 CPC sites using PEPFAR programmatic support. In all other districts, nearby services funded by Global Fund or MOH will be used, though distances to these services from CPCs is likely to vary. All CPCs are expected to have at least one service option available. Therefore, BCPP funding will not be used to support direct service delivery but to mobilize and link men in BCPP communities to existing MC services. Modified SMC services are expected to begin when the second round of BCPP interventions are implemented, approximately February 2016.

#### c) Specific Activities:

- 1) Mobilization: In the first round of BCPP activities, SMC depended heavily on community-based mobilizers and referrals from the BCPP HTC Campaign and BHS to generate client demand. A basic level of this ongoing mobilization will continue. HTC and BHS will refer men to community mobilizers by passing contact information with consent; the mobilizers will then follow up with these men and link them to nearby services. Mobilizers will also work directly with communities to mobilize men for services. Incentives for mobilizers through a performance-based contract may be utilized to improve mobilization efforts. In addition to encouraging potential clients to obtain MC, mobilizers will disseminate service information about linkage sites, transport schedules, and assist with coordinating transportation.
- **2)** Coordination: A small number of full-time coordinators will oversee all the CPCs. Their responsibilities will include identifying and liaising with locally-available SMC services to confirm their schedules and notify them of expected clientele numbers on transportation days; supervising mobilizers; coordinating transportation; and follow-up with service sites to collect the necessary data. A senior BCPP staff member will keep the MOH SMC coordinator up to date on these activities.
- **3) Transportation:** In each CPC, transportation will be offered at least monthly to nearby SMC services, on days of the week determined to be optimal. Transportation will also be provided for day-2 and day-7 follow-up visits, and will remain available for adverse event emergencies.
- **4) Data collection:** Individual-level data will not be collected at SMC service provision sites by BCPP, but aggregate data will be requested from these sites. Specifically, at these sites, the coordinator will make attempts at least quarterly via physical visits and register reviews to ascertain how many HIV-negative/unknown men 16-49 years of age from the CPC were served. The coordinator will also collect aggregate data from the transfer logs to gather numbers of men transported to SMC services. Finally, the coordinator will collect aggregate data on number of men referred and mobilized from demand creation records completed by HTS and BHS staff as well as SMC mobilizers (*Male Circumcision Tracking Sheet*).

#### 6.6 Identification, Linkage, and Treatment of HIV+ Pregnant Women

- a) Target: 90% of women initiated on indefinite ART (Option B+) during pregnancy remain in care and on treatment post-delivery.
- b) Strategy: Strengthening PMTCT activities is important to ensure that HIV-infected pregnant women are identified, linked to care, and remain on ART post-delivery. Currently, Option B+ is the national standard of prevention of mother-to-child transmission in Botswana. Therefore, BCPP intervention and control communities will provide Option B+ interventions for all HIV+ pregnant women. The BCPP program for pregnant women will focus on strengthening three activities in PMTCT settings in intervention communities: 1) strengthening of third trimester retesting within the ANC; 2) linkage to HIV treatment for all HIV-infected pregnant and post-partum women; and 3) retention on ART post-delivery.

#### c) Specific Activities:

- 1) Strengthening third trimester retesting: BCPP staff work with MOH clinic staff to strengthen capacity to identify women who are due for third trimester retesting. MOH clinic staff will use client contact information from the ANC register to make phone calls and schedule appointments with all HIV-negative pregnant women who have not completed third trimester retesting. MOH clinic staff will keep a record of clients called for third trimester retesting. Third trimester retesting will be monitored through PIMS/IPMS by the IDCC clinic.
- 2) Linkage and Retention for HIV-infected Women: Ensuring HIV-positive pregnant women receive ART and remain on ART following delivery is a key priority. All HIV positive pregnant women identified through the BHS and HTC campaigns are referred to the IDCC for HIV care and treatment. In addition, HIV+ post-partum women are referred to the IDCC to continue ART indefinitely (Option B+). Those who do not keep IDCC appointments will be tracked by the IDCC Site Coordinator and followed by community counselors to ensure they link or re-link to the IDCC post-delivery. Similarly, retention activities will track women who have begun Option B+ to ensure that they stay in care and on ART indefinitely. Those who are 14 or more days late for an appointment or pharmacy pick up will be contacted by MOH clinic staff and/or the IDCC Site Coordinator (*Linkage, Retention and Adherence Tracing Verbal Consent Script*) and community counselors will provide supportive counseling and new appointments through phone and home visits (*Participant Tracing Log*) as outlined in section 6.4.

#### **6.7 HIV Care and Treatment**

#### a) Targets:

- 1) 93% of PLHIV aged 16–64 who know their status are receiving ART
- 2) 95% of PLHIV aged 16-64 who are on ART are virally suppressed
- b) Strategy: Prior versions of BCPP Protocol 3 introduced anti-retroviral treatment outside Botswana national guidelines (CD4 < 350, WHO stage III or IV). With the revised WHO recommendations to treat all HIV-infected persons, Version 4.0 of Protocol 3 proposes to start all HIV+ adults in CPCs on immediate treatment and retain them on treatment (UTT). To demonstrate methods for

implementation of UTT for later adoption by the Botswana MOH, BCPP will embed UTT treatment interventions within the national ART program (MASA). The package of interventions described below are designed to 1) reduce barriers to ART initiation by simplifying procedures and making services easily available 2) increase capacity of IDCCs to support aggressive ART scale-up, and 3) enhance the use of both individual and clinic-level data to monitor uptake of HIV care and treatment.

#### c) Specific HIV Care and Treatment Activities:

- 1) Confirmation of HIV status: All HIV+ referrals into the clinic as well as existing pre-ART patients will be confirmed with an HIV test administered by IDCC staff as recommended by WHO before initiating ART (World Health Organization, July 2015).
- **2)** Same day ART initiation: Patients who are not on ART will be offered initiation (or re-initiation) of ART on the day of their first clinic visit if blood draws are possible that day. Adherence counseling, screening for opportunistic infections, and blood draw for baseline pre-ART safety labs will occur on the day of ART initiation. Patients who decline ART initiation (or re-initiation) will be given a 1 month follow-up appointment for re-consideration of ART initiation.
- **3)** Frequency of clinic follow-up visits: Patients on ART who are stable (e.g., virally suppressed, no opportunistic infections, keeping appointments, etc.) will be offered a reduced frequency of scheduled visits as compared to the current MASA standards. Patients will be followed according to national program standards for the first year. For stable patients on ART for longer than 12 months, visits with a clinician every 6 months will be implemented. IDCC patients already on ART will follow the streamlined schedule according to their time on ART.
- **4)** Frequency of visits for laboratory testing: Routine laboratory testing will be offered to patients according to the national guidelines with the exception of CD4 counts which will only be measured at baseline, after 12 months on ART, and at the discretion of the clinician. Also, wherever possible, patients will have their blood drawn at the time of routine clinic visits rather than on separate days to further reduce the frequency of clinic visits and clinic congestion. All laboratory results will be reviewed by the clinic staff within 4 weeks of blood draws, and patients will be contacted by clinic staff for review of any abnormal lab results.
- **5)** Frequency of dispensing visits: Patients who are stable after 12 months of ART (e.g., virally suppressed, no opportunistic infections, keeping appointments, etc.) will be dispensed up to 3 months of ARVs if there is adequate stock in the clinic at the time of dispensing rather than being required to return after only 1 month for a dispensing visit. The pharmacy will update a patient's next refill appointment in PIMS2/IPMS if more than one month is dispensed. Stable patients will have monthly, bi-monthly or quarterly refill appointments, which may coincide with the semi-annual clinician visits.
- **6) Retention Intervention:** Resources will be available in CP communities to ensure that all PLHIV are retained in care. The retention intervention will focus efforts on those who have missed treatment appointments and/or pharmacy pick-ups. Persons eligible for retention tracing will be identified by the IDCC staff using their electronic data system.

Existing IDCC patients who have missed appointments or pharmacy pick-ups are contacted by MOH clinic staff by phone or home visits and are asked if they agree to have a community counselor contact them to provide retention support activities. Patients who do not consent to retention support intervention activities are reminded about the importance of staying in care/linking back into care, and thanked for their time (*Linkage, Retention and Adherence Tracing Verbal Consent Script; Retention Tracing Contact Log*).

Patients who consent to intervention activities receive retention support services by clinic staff and community counselors including SMS reminders of appointments, rescheduling of missed appointments, and tracing and supportive counseling through home visits and telephone calls for defaulters (>14 days late for appointment or pharmacy pick-up) and Lost to Follow Up (LTFU; > 90 days late for an appointment). Clinic data systems are monitored to determine if these patients have relinked to the IDCC (*Retention Tracking Log, Participant Tracing Form*).

7) Adherence Intervention: IDCCs typically use self-reports, pill counts, pharmacy refill data and viral loads to monitor adherence. These adherence monitoring strategies are promoted in all study sites. All PLHIV on ART in CPCs are offered an increased level of adherence counseling and support above and beyond what is routinely offered within the setting of government clinics. Eligible persons who would benefit from increased adherence support are identified by the clinic staff.

Eligible patients are contacted by MOH clinic staff by phone or home visit (*Retention and Adherence Outreach Script* and are asked if they agree to have a community counselor contact them to provide adherence support activities (*Linkage, Retention and Adherence Tracing Verbal Consent Script*). Patients who do not consent to adherence support intervention activities are reminded about the importance of taking ART as prescribed, and thanked for their time.

Patients who consent to intervention activities (*Adherence Intervention Verbal Consent/Assent Script*) receive adherence intervention services including an assessment (*Adherence Assessment Tool*), assignment of case manager, and additional counseling to assess and resolve individual adherence challenges. In addition, the following services may also be delivered depending upon the person's circumstances and assessment: referral to social worker; SMS reminders; home visits; pill box issuance; depression screening; support with HIV disclosure; alcohol assessment; treatment buddy/mopati; VL repeat; assignment of earlier appointment; and change in ART regimen (for those in whom side effects/medication acceptability might be mitigated through substitution). All adherence interventions will be documented as will the outcome of the efforts, on the *Adherence Intervention Tracing Log*.

#### **Patient CARE in Other Study Clinics or Non-Study Clinics**

Finding solutions so that as many BCPP patients as possible can receive expanded ART initiation is important for reaching ART saturation in CP communities, however the study is constrained and cannot easily perform study activities or install study staff at sites which are not CP community clinics. As a solution, the following options will be offered to patients, if during counseling it is determined that they face challenges to participation in study activities at the IDCC in their own community:

1) BCPP activities at <u>any</u> CP community clinic: Initiation and receipt of ART will be allowed at <u>any</u> CP community clinic at which a participant would be able to receive services. Note that the

study will not be able to provide transport or any additional compensation for these individuals. Follow-up data from PIMS2 or IPMS will be obtained on these individuals for study purposes from the CPC clinic the participant chooses.

2) ART initiation activities at <u>own</u> community clinic, followed by transfer to <u>any</u> MOH clinic: Services including ART initiation will be provided at the participant's own CPC, followed by facilitated transfer to any MOH HIV care and treatment facility (including those not in study communities) for continued ART. Follow-up data on these individuals will be obtained from routine medical information sources such as PIMS2 or the national HIV data warehouse.

#### **Identifying Patients for UTT**

To find all eligible PLHIV not currently on ART and initiate them on treatment, BCPP priorities will include approaching the Expanded Treatment Cohort (described in BCPP Protocol 3 version 3.0) in early 2016

to offer ART initiation for those not on ART. Another strategy to identify eligible PLHIV not currently on ART will include data mining of the MOH electronic patient systems to seek PLHIV categorized as "pre-ART" to approach them about immediate ART initiation (*Script for Outreach Pre-ART Clinic Patients*). These two mechanisms in combination with expanded HTC activities outlined earlier will yield the scale-up of ART initiation necessary to meet both treatment and viral suppression targets.

#### 7.0 LABORATORY METHODS

Detailed laboratory procedures are described in Standard Operating Procedures (SOPs) that are maintained at each laboratory supporting the study. The BCPP Laboratory Manual provides an overview of routine testing that is conducted at Ministry of Health laboratories and more detailed study specific procedures for testing conducted at CDC, Harvard Chan School, BHP laboratories. In addition, all study staff has received a Field Operations Procedures Manual which serves as a procedural guide during actual specimen and data collection.

#### 7.1 Overview of Laboratory Methods

An overview of the types of laboratory tests, sample types, and the location of the testing is provided below. The intervention component of the project uses the following laboratories and locations:

- 1. BHHRL: MOH regional HIV Reference Lab (Gaborone). BHHRL is a hybrid institution with management shared by Harvard and MOH.
- 2. NHHRL: MOH regional HIV Reference Lab (Francistown)
- 3. MOH District and primary Labs (Botswana-multi-sites)
- 4. MOH clinics in CPC communities
- 5. Field sites: households and community venues conducting surveys and HTC campaigns
- 6. CDC: International Laboratory Branch at Centers for Disease Control and Prevention (Atlanta) and CDC Laboratories (Gaborone and Francistown)
- 7. BHP (Botswana Harvard Partnership Laboratory)
- 8. Harvard T. H. Chan School of Public Health (Boston)

A minimum laboratory enhancement package has been implemented in laboratories supporting study sites. Each study-associated laboratory adheres to site and study specific SOPs for proper processing, labelling, transport, testing and storage of specimens as outlined in the BCPP Laboratory Manual. The laboratory study team provides guidance and technical support to the laboratories to implement and

maintain a quality management system which includes continuous quality improvement, adherence to biosafety, enrollment in EQA programs, review and maintenance of standard operating procedures for laboratory testing, timely procurement and forecasting reagent and supply needs, and documentation of training for all laboratory personnel. Adherence to these standards is routinely monitored by the laboratory study team.

#### 7.2 Training of Laboratory Personnel

All laboratory personnel participate in study-specific training prior to study initiation. Training includes an overview of the BCPP study design and study-specific laboratory methodologies (with assessment for competency) in addition to Research Ethics and good clinical laboratory practices including QA/QC (quality assurance/quality control) and laboratory record keeping procedures. Study staff responsible for providing HTC complete the required training curriculum recognized by the Ministry of Health. Study staff members who collect blood samples and conduct laboratory analyses receive training in universal precautions, sample collection, and testing of study samples. Additional refresher trainings are scheduled during the study to ensure consistency and address training needs as they arise.

#### 7.3 Specimen Collection, Transport, and Processing

Specimens are collected from participants at study field sites and samples transported to designated laboratories for processing, testing, and storage. Testing may also occur at study field sites.

#### **Sample Types and Sources**

- a) <u>Capillary blood samples</u>: Finger prick samples are collected in a microtube using a blade lancet by trained staff at study field sites according to BCPP finger prick SOP and used for the HIV rapid tests.
- b) <u>Venous blood samples</u>: Several types of venous blood draws occur at the IDCC during routine management of patients, and will be done following MOH procedures for phlebotomy, (including appropriate blood volumes and processing). At the IDCC, venous blood samples will be collected for drug resistance testing per national guidelines.

### 7.4 Laboratory testing for HTC campaigns (returned to participant and/or participant file with exception of viral load test)

a) HIV Diagnostic Testing: HIV diagnostic testing will be conducted in the study communities and clinics per national HIV testing guidelines using Botswana government-approved serial rapid tests as outlined in the 2016 testing algorithm in the national treatment guidelines. Other testing algorithms may be substituted if in alignment with national guidelines. Verification will be conducted on all newly diagnosed and known HIV-positive persons before initiating ART according to WHO recommendations (World Health Organization, July 2015). All HIV tests will be conducted according to the manufacturer's guidelines and BCPP SOPs. If results of the initial serial rapid tests are discordant, then per national guidelines two rapid tests will again be performed in parallel. If the second pair of tests is discordant, the participant will be referred to the clinic for re-testing in 2-4 weeks with a referral recommending ELISA testing. A 3 ml venous blood specimen will be taken at the visit and sent to a reference laboratory for further testing using ELISA (Murex HIV 1.2.0 test, Genetic Systems HIV 1.2 plus O, BioRad HIV-1/HIV-2 plus O EIA,) and/or Western blot). The results from the EIA and/or Western Blot will supersede the discordant and/or indeterminate results obtained in the field. The IDCC Site Coordinator reviews the HTC register at the clinic in PIMS2 or IPMS to determine if HTC campaign participants with indeterminate results received confirmatory testing. HTC participants with indeterminate rapid test results, and who do not have a documented retest at the clinic are referred to a community counselor for tracing and follow-up services.

#### 7.5 Laboratory Testing for IDCC patients

Clinical laboratory testing is performed in MOH labs in accordance with the National Guidelines. Testing procedures follow approved standard operating procedures for each laboratory where testing is conducted.

#### a) Hematology and Clinical Chemistry

Basic blood work is used to assess participant health status for initiation and monitoring ARV treatment in HIV-infected individuals; however, ART initiation will occur before all lab results are available. The following tests may be conducted per MOH guidelines:

- Hematology: Full Blood Count (FBC) to include hemoglobin, hematocrit, red blood cell count (RBC), mean corpuscular volume (MCV), white blood cell count (WBC), differential WBC, absolute neutrophil count (ANC), and platelets.
- Clinical Chemistry:
  - o Liver Function Tests (LFT): Total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase.
  - Glucose (fasting or non-fasting)
  - Electrolytes: sodium and chloride
  - o Renal Function Tests (RFT): Urea and Creatinine: An estimated creatinine clearance
  - CrCl in cc/minute can be estimated from formulas using patient sex, age, weight, and serum creatinine (in um/L):

Males:  $1.22 \times [(140 - age in yrs) \times wt (kg)]/[serum Cr]$ 

Females:  $1.037 \times [(140 - age in yrs) \times wt (kg)]/[serum Cr]$ 

- b) <u>Syphilis testing (RPR and VDRL</u>): As per Botswana guidelines, non-treponemal tests for syphilis (rapid plasma reagin or Venereal Disease Research Laboratory tests) will be performed according to the manufacturer's instructions.
- c) <u>CD4:</u> Point of care and flow-based CD4 methods are used dependent upon availability of CD4 instruments. Testing follows manufacturer's instructions and national guidelines for use.
- d) <u>HIV-1 RNA Viral Load:</u> HIV-1 plasma RNA viral load is quantified for monitoring of ART-naïve HIV-infected individuals and monitoring of viral suppression in HIV-infected individuals receiving ART (at 3 and 6 months after ART initiation and every 6 month thereafter according to current national ART guidelines or per Adherence Intervention Procedures).
- e) <u>HIV drug resistance testing</u>: Drug resistance testing is offered per national guidelines and under circumstances described in section 6.11.
- f) Pap smear: Pap smears are performed and findings managed according to national guidelines.
- g) <u>Pregnancy Testing</u>: If pregnancy is suspected but not confirmed by LMP (last menstrual period) or exam, a urine pregnancy test is performed for confirmation of pregnancy as per MOH procedure.

#### 7.6 Quality Assurance

Standard operating procedures (SOPs) are used for all tests as well as quality assurance/quality control (QA/QC) procedures. Laboratory staff conducting testing participate in a proficiency testing and 5% of all tests (or as indicated by laboratory specific SOP) are subjected to internal quality control processes. The QA/QC plan includes periodic monthly reviews of EQA performance, collaboration with the CDC laboratories, enrollment in appropriate EQA schemes, and inter-laboratory comparisons. External quality assurance and proficiency testing programs includes: CD4 count, HIV-1 RNA load, Hematology (FBC), and clinical chemistry analytes. Laboratories are monitored throughout the study by the study team and external monitors as requested by the study sponsor. QA for HTC conducted in the communities and through RHT in the clinics include weekly QC exercises for counselors in the field, participation in proficiency testing programs, monitoring and site visits from lab personnel, and biweekly monitoring of the concordance rates of HIV serial tests conducted in the field. A small sample of HIV-positive tests may be retested in the lab for QA purposes.

#### 7.7 Biosafety and Waste Management

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate blood and secretion precautions are employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the United States Centers for Disease Control and Prevention. All infectious specimens are transported in accordance with the IATA guidelines using designated courier services.

#### 7.8 Specimen Storage and Shipment

The IDCC Site Coordinator coordinates shipment of specimens as required. Selected samples may be transferred to the CDC (Atlanta) or Harvard Chan School (Boston) laboratories for external quality assurance, viral load, and drug resistance/level testing. Specimens are stored until all protocol-related and quality assurance testing have been completed.

#### **8.0 DATA SYSTEMS AND MANAGEMENT**

The overall system to capture data, record outcomes and analyze results is an integration of multiple data collection sources for all BCPP interventions into a single research data base or data warehouse. Each BCPP activity has underlying systems of data capture and management which serve as the "system of record" containing the source records for all study data captured within the scope of that activity. A variety of data capture methodologies are used across the BCPP activities including online reference data retrieval (e.g., community maps), paperless point of service/survey capture, and paper and electronic chart/registry abstraction. Process, study participant status, and calculated data are also generated by the data systems of the BCPP activities and exchanged between systems and stored in the research database.

Each system must also interface with other activity data systems to exchange data as required to successfully implement the study. This includes maintaining participant registries, referrals, and key eligibility and status data, as well as underlying denominators within study arms and components. In

this section, we provide an overview of the data management for BCPP including data capture, data flow, security, confidentiality, access and quality.

#### 8.1 Data collection, Capture and Flow

HTC data forms (*Household Enumeration Form, HTC Intake Form*) are collected with the OpenDataKit (ODK) software using handheld tablets running the Android operating system. HTC counselors are trained in the use of these handheld tablets for electronic data entry at the point of HTC, which includes door-to-door home visits and mobile HTC sites.

Community counselors also record their tracing activities for linkage and retention on the *Participant Tracing Log* using these handheld mobile devices.

HTC and Linkage to Care forms are synced to the clinic-level study database at least daily. Completed forms are deleted from the tablets following the sync.

Clinic Site Coordinators manage screening, adherence and retention activities using both the hand-held data devices and OpenClinica.

The MOH has an electronic data system known as the Patient Information Management System 2 or PIMS2. PIMS2 is a SQL-based, client-server application which runs on a local clinic network and has been implemented in BCPP community clinics. PIMS2 captures data for a variety of programs, including: facility-based routine HTC, MC, ANC, maternity, and post-natal care. HIV care and treatment data are regularly extracted from PIMS into the clinic-level study database via a secured Virtual LAN (VLAN) connection between the local clinic network on which PIMS2 operates and the BCPP network.

Some larger BCPP community clinics have migrated to a web-based system to record patient-level data which runs on the Botswana Government's data network. This Integrated Patient Management System or IPMS captures program data that are similar to PIMS and includes an integrated laboratory information system. IPMS data will be regularly extracted from the IPMS central data repository onto the BCPP central data server.

The MOH strongly encourages the use of PIMS or IPMS where available. Therefore, nurse prescribers, physicians, midwives, lay counselors and other clinic staff within the 30 BCPP communities record patient registration and appointments, and enter consultation, laboratory and pharmacy data into PIMS or IPMS. *Appendix P1* outlines the selected data elements transferred from MOH systems to the BCPP central data server.

MC staff members responsible for the coordinating linkage of eligible men to MC will distill aggregate data on numbers of total and eligible men transported to MC from the transportation logs and will also engage with service delivery providers to obtain numbers of eligible men served on non-transport days. This data will be entered into an electronic or paper-based custom data collection form monthly.

On a daily basis during the BHS/AHS surveys in all 30 communities, BHS/AHS referral and locator data files are transferred from BHP's electronic data capture system to the clinic via secure copy on the BCPP network in the clinic and processed into the clinic-level study database. At CPCs, BHS referrals are combined with HTC referrals. In all community clinics, referral data is used to produce operational
reports for use in the clinic. In CPCs, an encrypted flash drive is used to retrieve updated referral files from the clinic's study database and to transfer updated data from the MC client tracking tool to the clinic-level study database.

On a nightly basis, data from all clinic-level study databases is copied to the BCPP central data server in Gaborone over the secure BCPP VPN. As needed, the BCPP senior data manager in Gaborone will work with IDCC Site Coordinators or other clinic level staff to reconcile data issues.

The Research Database is designed in PostgreSQL and housed on the BCPP central data server at the CDC-Botswana Gaborone office. It is populated with data pulled up from all the clinic level study databases as well as data from IPMS, PIMS, CD4 data from PIMAs, and baseline, annual and end of study survey data transferred from BHP's EDC via secure copy.

The diagram in Figure 1 offers a schematic representation of the data flows from all sources described above to the central BCPP data warehouse for the intervention communities (CPCs). For all PLHIV in the study communities we obtain clinical data from the existing MOH's electronic patient data systems (PIMS or IPMS).

Figure 1: Data Flow diagram for CPCs



### 8.2 Data Security

The CDC Data Manager is responsible the security of BCPP data collected for the Intervention protocol. The Botswana MOH is responsible for the security of data collected through routine MOH systems, including PIMS and IPMS. All BCPP-specific systems supporting clinic data reside within the clinic network where a firewall, encryption keys, user logins, and physical security and access, and routine data back-up measures have been put into place to ensure data security and integrity.

Laptops and tablets used for data capture and processing are encrypted and require user logins to prevent unauthorized users from accessing data. Laptops, tablets and all study related paper-based forms and logs are stored in locked cabinets or locked trunks when not in active use. The clinic laptops which serve as the local clinic-level study databases are locked in secure cabinets. Daily data transfers from tablets and the MC Epi Info system minimize the risk of data loss should the device be lost or corrupted. Clinic-level study databases are backed up on to the local encrypted hard drive and the backup files are transferred to the BCPP central data server in Gaborone using secure copy. The

backups from all of the clinic-level study databases and the central data server will be backed up to tape daily. The BCPP central data server at the CDC-Botswana Gaborone office is located in a locked, climate controlled server room managed by CDC IT staff in compliance with CDC IT policies.

A virtual private network (VPN) connects each clinic-level study database to the BCPP data center. The VPN provides a secure network over which data can be transmitted and through which data managers and IT staff can access clinic systems. VPN accounts are provided to study staff as needed and CDC DM lead approval is required for access to study data systems managed by CDC. Within the BCPP network, access to devices, databases, and directories are managed based on user roles. Data in transit over the BCPP network is encrypted, password protected and transmitted through secure connections using secure-shell (SSH) protocols; encrypted, password protected memory sticks are used for data transfer when direct network connections are not available.

The Botswana MOH is responsible for the security of PIMS and IPMS data. PIMS resides on secure local networks at each clinic and IPMS runs on the secure Government Data Network (GDN). Both the local network and the GDN use PIMS are regularly backed up via secure memory sticks. IPMS backups are managed through the IPMS central data store in compliance with Botswana MOH IT policies. CDC DM and IT will work with MOH counterparts to strengthen data security policies and practices.

## 8.3 Data quality

ODK Surveys on the tablets and Epilnfo have built-in validation tools to minimize data entry errors. These include range restrictions for numeric data, pre-defined values (code sets) for categorical data, and logic checks. Valid responses are required for key fields to ensure completeness and skip patterns will be used to prevent extraneous data entry and encourage proper form completion. Error messages and caution notices will be used to alert staff when they enter faulty data so that they are aware and can correct the problem.

HTC and linkage to care staff receive training on both the contents of the tools and use of the tablets and ODK software. Supervisors review the data forms for completeness and supervise corrections prior to synching of the tablets. SMC staff will receive training on proper completion of MOH tools and use of the Epi Info client tracker. Data managers will monitor system performance throughout implementation.

### 8.4 Confidentiality of data

CDC DM is responsible for protecting the privacy of all study participants and ensuring the proper handling of all personal health information and contact information collected for BCPP under Protocol 3. All components of the distributed data systems implement both electronic and physical security procedures for "data in use" within secure networks and devices. Encryption is implemented to render electronically stored subject identity and personal health information unusable, unreadable, or indecipherable to unauthorized individuals for "data in motion" and "data at rest". Encrypted personally identifiable information (PII) will be transmitted within the BCPP system by way of the secured VPN only.

PII, including name, national identity card number (Omang) and locator data (address, phone numbers), is collected as part of HTC to facilitate referral and linkage of clients with services (e.g. IDCC, ANC, SMC). BHS collects similar information and includes necessary PII in the transfer of referral and

locator data to the clinic. PII is collected as a part of patient registration in both PIMS and IPMS as required by MOH to ensure patients are eligible to receive services.

PII maintained in the clinic study databases are not transferred to the central database on the BCPP server; Omang is encrypted with a one-way hash prior to transfer to the BCPP server for the purpose of linking data across data systems. Where there is consent from the client to access medical records or a waiver of consent to extract identified data from the clinic systems (PIMS and IPMS), clinic data can be linked with BHS referrals and HTC data using the hashed Omang.

All study staff are trained on data confidentiality. Site staff access to PII and locator data is limited to health care providing staff which are required to reliably identify a participant, and staff engaged in linking patients consenting for contact with services. A minimal number of staff have access to the study databases where PII is stored and the operational reports which present PII to site staff; DM can access these data when required for system maintenance or to provide user support.

#### 9.0 DATA AND ANALYSIS PLANS

The primary objective of the Intervention Protocol is to implement and describe uptake of Combination Prevention interventions in CPCs. Secondary objectives will describe retention in the clinical cascade of care from HIV diagnosis to viral suppression among all HIV-infected persons. The key indicators for analyzing results of BCPP objectives are outlined in Table 2.

•

**Table 2. BCPP Key Indicators** 

| Indicator Name | | Coverage vs. Numerator BCPP Performance | | Denominator |
|---|---|---|---|---|
| 1. | % of HIV+ Adults* who Know their Status | Coverage | # of HIV+ Adults estimated to know<br>their HIV status | # of Adults estimated to<br>be HIV+ |
| 2. | % of HIV+ Adults in<br>Care | Coverage | # of HIV+ Adults in Care | # of HIV+ Adults<br>estimated to know their<br>HIV status |
| 3. | % of HIV+ Adults on<br>ART | Coverage | #of HIV+ Adults on ART | # of HIV+ Adults<br>estimated to know their<br>HIV status |
| 4. | % of HIV+ Adults with<br>Viral Suppression | Coverage | # of HIV+ Adults with VL<1000Copies/ML | #of HIV+ Adults on ART |
| 5. | % of HIV+ Adults Identified through BCPP who know their status | BCPP<br>Performance | # of HIV+ Adults Identified (new & known) through BCPP who know their status | # of Adults estimated to<br>be HIV+ |
| 6. | % of PLHIV Newly<br>Diagnosed through<br>BCPP | BCPP<br>Performance | # of Adults Identified as Newly<br>Diagnosed HIV+ through BCPP | # of HIV+ Adults Identified (new & known) through BCPP who know their status |
| 7. | % of PLHIV Linked to<br>Care | BCPP<br>Performance | # of HIV+ Adults Identified as Newly Diagnosed or Not Currently in Care at IDCC who were seen at IDCC within 90 and 180 days of Interview | # HIV+ Adults Identified<br>as Newly Diagnosed or<br>Currently Not in Care at<br>IDCC |
| 8. | % of PLHIV Initiating (or re-starting) ART | BCPP<br>Performance | # of Eligible HIV+ Adults Identified Not<br>on ART who Start or Re-Start ART | # of HIV+ Adults<br>Identified not on ART |
| 9. | % of PLHIV Retained<br>on ART (12 months<br>Post ART Start or<br>Restart) | BCPP<br>Performance | # of HIV+ Adults Identified Not on ART<br>who Start or Re-Start ART and Remain<br>on ART after 12 Months | # of Eligible HIV+ Adults<br>Identified Not on ART<br>who Start or Re-Start ART |
| 10. | % of PLHIV on ART with Viral Suppression (12 Months post ART Initiation or Restart) | BCPP<br>Performance | # of HIV+ Adults Identified Not on ART who Start or Re-Start ART and have VL<1000Copies/ML after 12 Months | # of Eligible HIV+ Adults<br>Identified Not on ART<br>who Start or Re-Start ART |

In the section below, data and the data sources for the outcomes of interest are identified for each intervention within the combination prevention package of services (HTC and Linkage to care, HIV care and treatment, MC and PMTCT services). In addition, the data analysis plans are provided for the study objectives.

# 9.1 HIV Testing and Counseling and Linkage to Care

The HTC services aim to maximize the number of PLHIV who know their status within the community. Predictors of HTC uptake will be examined including demographics, prior testing history, partner status, etc. Participants reached through mobile vs home-based testing will be described including age

and gender. Characteristics of HIV-positive persons identified will be described, including but not limited to demographics, testing history, new or previous HIV diagnosis, history of HIV care, CD4 count, and ART status. Data sources will include the *Household Enumeration Form, HTC Intake Form, and BHS* collected during the HTC activities. In addition, facility-based testing will be monitored in CPCs through RHT data in PIMS2 or IPMS.

All HIV-positive participants given appointments at the HIV care and treatment clinic in the study communities are tracked to ensure they link to care. Those who keep appointments at the study clinic within 90 and up to 180 days of the BCPP interview as recorded in PIMS2 or IPMS are considered "linked" to care. Those participants who report they are receiving care at another clinic outside the study community will be verified by PIMS2 or IPMS and will be considered linked to care if that have an IDCC appointment within 90 and up to 180 days of their BCPP interview date. In addition, at one year from the interview data, electronic data systems will be checked to determine if participants who did not link or register within 90 days have registered in care.

Predictors of linkage to care will be examined including but not limited to, demographics, new or previous diagnosis, CD4 count, and time to first appointment from interview. In addition, rates of linkage to care will be compared among participants who received interventions services and those who did not.

Data sources include referrals from HTC and BHS (*HTC Intake*, *BHS*), PIMS2 and IPMS for details of registration into care and treatment, and the *Participant Tracing Log* where all linkage to care follow-up activities are recorded. In addition, the Ministry of Health's Central Data Warehouse will be queried to identify (or confirm self-reported enrollment) of community residents who register for HIV care and treatment outside of the local study community.

Further, estimations of the operational costs associated with the expanded HTC and linkage to care interventions paired with the total cost by intervention with their corresponding BCPP performance indicator will be used to estimate the average costs per person. The financial costing approach is described below, in the cost analysis plan.

#### 9.2 Care and Treatment

For HIV care and treatment objectives, the overall number of PLHIV enrolled in the IDCC and on ART including community residents getting care at clinics outside the community will be described. Specific focus will be given to examination of patterns of health care utilization by residents and non-residents of the community. The key outcomes for analysis are ART initiation, adherence, retention and virologic suppression. We will also describe the laboratory results showing toxicity, and adverse events among the clinic population on ART. ART initiation will be measured by start date of ART among all HIV-positive patients initiated on ART as recorded in the electronic patient management system. Length of time from BCPP interview or encounter to date of initiation on ART will be recorded and monitored. ART coverage will be measured by the number of HIV-positive community residents receiving ART out of the estimated number of HIV-positive community residents.

Adherence levels will be assessed through self-reports, pill counts and pharmacy refill data from the electronic data systems and also from the adherence intervention tools. Based on the self-reports, pill counts and pharmacy refill data, an aggregate measure of adherence will be calculated (e.g., good,

limited or poor). Adherence levels at a community clinic will be measured by the percentage of clinic patients with an adherence assessment of good, limited and poor adherence. Retention of HIV-positive persons in care and on treatment will be measured during a defined period of time (e.g. 12 and 24 months). The number of HIV-positive clinic patients who are community residents and who remain in care (had a clinic visit within 6 months) and on treatment (pharmacy pick up and clinic visit within 3 months) during a defined period among all patients from the community who were registered at the clinic during that time will be considered retained in care or on treatment. The number of patients who missed clinic visits, defaulted from care and were lost to follow up will also be recorded from the electronic patient management system during a defined period. Virologic suppression will be assessed from the electronic data systems and will be defined as those HIV-positive patients on ART with a viral load of less than or equal to 400 copies/ml among all patients on ART.

Predictors of retention, ART initiation, adherence and virologic suppression will be examined. As the inverse of retention, predictors of loss to follow will be examined. For those on ART, predictors of defaulting on ART will be examined.

All clinic patients will have data captured in the existing MOH electronic patient management systems. Clinical outcomes, including but not limited to ART eligibility and initiation, WHO stage, lab results, death, adherence, retention, viral suppression, and adverse events, will be assessed using routinely collected clinical data that is captured in the electronic medical record (see Appendix P1). In addition, the Ministry of Health's Central Data Warehouse or other sources of routine medical information will be queried to identify clinic participation, ART eligibility, ART initiation and virologic suppression among community residents receiving services outside of the local study community clinic. Secondary descriptive analyses for key clinical indicators will be conducted on these data. In the CPCs, retention intervention data will be recorded on the *Participant Tracing Log*, and adherence intervention data will be recorded on the *Adherence Assessment Tool* and the *Adherence Intervention Tracing Form*.

## **9.3 PMTCT Services**

Rates of 3<sup>rd</sup> trimester retesting among pregnant women will be assessed using the MOH Antenatal Care and Maternity registers and the MOH patient management systems. Among HIV-negative pregnant women enrolled in ANC care, the percent who were retested for HIV between 32-36 weeks will be recorded and monitored over the course of the study.

Rates of linkage to care among HIV-positive post-partum women will be reported. Once discharged from ANC care, HIV-positive post-partum women will be given appointments at the local IDCC. Those who kept the appointments and registered at the clinic as recorded in the electronic patient management system will be "linked" to care. Those who were previously registered patients in the IDCC who re-link to care will be considered re-linked. Predictors of linkage to care among HIV-positive post-partum women will be examined including but not limited to, demographics, time since diagnosis, CD4 count, viral load, and time since delivery. In addition, rates of linkage to care will be compared among participants who received intervention services and those who did not. Retention in care among post-partum women will be measured the same as among all HIV-positive patients in the IDCCs (see above) and recorded in the electronic patient management system. Rates of retention on ART in post-partum women at one year post-delivery will be described. In addition, predictors of post-partum

women who default from ART will be examined including demographics, time since diagnosis, time since delivery, CD4 count, and viral load.

Tracing activities with HIV-positive post-partum women referred to the HIV care and treatment clinic will be recorded on the *Participant Tracing Log*. The MOH patient management system will be used to verify registration of post-partum women in the IDCC. In addition, the Ministry of Health's Central Data Warehouse will be queried to identify women who temporarily access care and treatment services outside of the local study community during their period of postpartum confinement.

### 9.4 Male Circumcision

Through linkage to MC services, the MC program aims to maximize coverage of circumcision among males, which is defined as the percentage of HIV-uninfected men (aged 16-49) residing in CPC communities who are circumcised. Community-level MC uptake among all and eligible men will be reported. **BHS** and **ESS** surveys will be used to obtain cross-sectional true estimates of MC coverage, based on self-report. These surveys are described in the BCPP Evaluation Protocol (Protocol 1). Further, MC coverage will be estimated using records of MCs performed as well as the baseline MC prevalence reported by the HTC and BHS campaigns. MC coverage will be evaluated based on the most recent census estimates of the study community population as well as on the enumerated study population.

#### 9.5 ANALYSIS PLANS

For the primary outcomes, uptake of the CP interventions, we will estimate the percentage of participants eligible for and receiving the intervention using BHS and HTC data to identify those eligible, and BHS, HTC and clinic data to identify those receiving interventions. Confidence limits for each outcome will be estimated using robust standard errors to account for within-community clustering.

The first secondary objective is to examine demographic, clinical, and social/behavioral facilitators and barriers to uptake of CP interventions. We will fit Generalized Estimating Equations (GEE) models with robust standard errors to account for the clustering within communities. Independent variables for these models will be chosen based on prior literature and hypotheses about how various demographic, clinical and social/behavioral factors impact uptake of HTC, PMTCT, ART and MC. For MC, this type of analysis will only be possible for year 1 interventions because individual-level data on men obtaining MC will not be collected in subsequent years. Variables will be chosen a priori based on theoretical justification rather than statistical results and all chosen variables retained in the model to adjust for confounding.

To compare clinical outcomes, including viral suppression, among HIV-positive persons in CPCs who initiate expanded ART to those who initiate ART according to national guidelines, we will use tests appropriate to clustered data and the distribution of the outcomes of interest. For example, for viral suppression, we will use GEE models to account for the clustering within communities and test for a difference between groups (those initiating expanded ART vs. those who initiate according to guidelines). Since each community will contain both of these groups of participants, clustering has less impact on statistical tests, but still should be taken into account in the analysis to provide appropriate effect estimates and confidence limits.

To estimate the percentage of participants retained on ART among HIV-positive pregnant or breastfeeding women who initiate Option B+ (indefinite ART post-delivery), we will determine the number of HIV-positive pregnant women who initiate Option B+ during the study using BHS, HTC and clinic data, and determine the number retained on ART using clinic data. Confidence limits will be estimated using robust standard errors as for the primary outcome. Three costing studies of HTC and LTC services are planned. First, estimates of costs of home-based testing and mobile testing during the community-based HTC campaigns, including the cost per person and per new HIV case identified will be compared. Second, incremental costs and outcomes of strengthening facility-based routine testing relative to the standard of care will be estimated. Lastly, to assess the impact of the expanded linkage activities, estimates of the costs and outcomes of these tracking & tracing services will be calculated. Outcomes are defined as the number of new or previously diagnosed HIV-infected persons not in care, who register at an IDCC without engaging tracking and tracing services, and who register at an IDCC within 90 and 180 days of their HTC encounter.

A mixed top-down and micro-costing approach will be used to estimate costs. All relevant direct medical costs such as labor and materials, and direct non-medical costs such as program support and administrative overhead will be considered.

Analyses will be conducted from the perspective of the health care system indicating that the costs included would be those typically associated with the providers and payers of care, and would exclude the costs and productivity losses incurred by patients and their informal caregivers. The most significant cost component is expected to be labor, for which the main categories include: HTC lay counselors and supervisors, LTC Coordinators, drivers, and community mobilizers.

Labor time will be estimated by analyzing data records on clients seen, then confirmed through communication with staff and managers, and, as needed, through observation. Other cost items will be estimated through a combination of resource utilization and expenditure records. Any research related expenses will be removed in order for the resulting cost analyses to be useful for the projection of operational program costs. Costs of tests conducted through the baseline and annual household surveys administered by the Botswana Harvard Partnership will not be considered.

Cost and outcome data will be collected, retrospectively, from routine monitoring program data stored in the central study database and from actual program expenditures incurred over the period corresponding to the HTC and LTC programmatic efforts from all BCPP communities. The analytic horizon will begin in November 2013 and correspond to the period during which the HTC campaign and LTC program are delivered in a community. Unit costs (e.g. Cost per tested, Cost per new diagnosis, Cost per person linked) will estimated by dividing total costs by the relevant BCPP performance indicator. Where applicable any future costs will be discounted to their present value at a standard rate of 3%. As needed, costs will be converted from Botswana Pula to US dollars. Costs will be presented in 2015 US dollars. We will conduct univariate sensitivity analysis to identify the inputs which most impact the results and gauge the robustness of the conclusions. Data analysis will be conducted using Microsoft Excel and SAS.

# **10.0 ETHICAL CONSIDERATIONS**

### 10.1 Ethical Review

The protocol, informed consent/parental permission forms/assent forms, research participant education and recruitment materials, and other requested documents — and any subsequent modifications — will be reviewed and approved by the ethical review bodies responsible for oversight of research conducted at the study sites. The Institutional Review Boards/Ethical Committees (IRBs/ECs) for CDC and the Health Research & Development Committee, Botswana Ministry of Health will review the protocol at least annually.

### **10.2 Informed Consent**

# a) Interventions and strengthened programs:

HTC: National guidelines for obtaining verbal consent prior to receiving HTC services, for adults aged 16 or older, will be followed. Linkage-to-care interventions now fall under the Ministry of Health's 2016 national treatment guidelines which recommend that all HIV-positive persons identified be referred and tracked to the HIV care and treatment clinic. Therefore, all linkage to care follow up tracking will now be considered standard of care and will not require permission. However, participants who do not link to care and receive tracking and tracing follow up services will have the option to discontinue those services at any time they request. Similarly, active retention tracing of participants late for appointments has been implemented in several ART clinics in Botswana with plans to expand the scope of this program. For Retention Tracing, clinic patient contact information (name, phone number, address), OMANG (patient medical ID number) and appointment history are abstracted from MOH register and PIMS2 database for retention tracing of clinic patients who have missed scheduled clinic appointments These patients will be contacted by an MOH staff member and permission will be obtained to send BCPP counselors out for tracing and follow up services.

<u>Adherence Intervention</u>: Clinic patients identified as being non-adherent will be asked to consent for the adherence intervention (*Linkage, Retention & Adherence Intervention Verbal Consent*) which requests permission to administer the Adherence Assessment Form.

The informed consent process will occur in the language most comfortable for participants (usually in Setswana) at 8.0 reading level or below. Permission/assent will be documented by having the participant sign the permission/assent form or make a mark if the participant is illiterate; the latter will be witnessed by a third party. A copy of the informed consent/assent form will be offered to the participant, and if applicable, parent or legal guardian giving permission for a minor to participate. Staff will ensure that the participant takes a copy of a study contact card that contains study information and telephone numbers if the participant does not wish to take a copy of the permission/assent form.

## b) Special Populations

*Minors:* Minors (participants ages 16-17) are only enrolled with the written permission of a parent/legal guardian and if they provide informed assent.

- ✓ Under circumstances where clinical or study staff suspect, or there is a reported incident of sexual abuse of a person under age 18, the study staff member must inform the relevant authorities; this is stated in the permission/assent forms.
- ✓ Referrals will be made to youth services if needed.

- c) Use of Routine Programmatic Data: A waiver of informed consent was previously granted for the following activities:
  - 1) Medical record use in accordance with 45CFR 46.116 (d) to extract a limited, preselected dataset (Appendix P1) from MOH clinical data systems in the clinic population in Enhanced Care and Combination Prevention Communities. This is done by linking BHS and HTC data with clinic data to monitor the care and treatment cascade from HIV testing and referral through clinic enrollment, ART initiation and adherence, and retention in care. Procedures for extracting, matching between sources, and de-identification of this data are described in Section 8. Limitation of data-to-data elements based on consent/waiver-of-consent will be applied during the transfer of data from the clinics into the study database. Although not all data elements are part of the matching algorithm, data are matched using date of birth and Omang number. Once match is assigned, the data retained for analysis is de-identified in accordance with the consent/waiver-of-consent and the stipulations of the study protocols.
  - 2) A waiver of informed consent was previously granted for the following: a) data from the HTC Intake questionnaire that is collected as part of HTC programmatic services in households and tent venues in the Combination Prevention Communities, and b) abstraction of aggregate program data from MC and HTC facilities.

The waiver is appropriate because (1) the analysis involves no more than minimal risk to human subjects, and personal identifiers are encrypted for data handlers and analysts; (2) the evaluation does not adversely affect the rights and welfare of the subjects; (3) the evaluation cannot practicably be carried out without the waiver because it is not possible to obtain consent from all service recipients without infringing on the ability to carry out the program in an efficient manner; and (4) if consent for routine data use from all participants was requested, this might reasonably constitute an unnecessary waste of an individual's time. The types of consents being requested for activities in this study are described in Table 3.

Table 3: Summary of approach to consent for various components of the study

| Project | Targeted subjects | Activity | Consent | Comment |
|---|---|---|---|---|
| component | | | | |
| HTC | Persons not documented to be HIV-infected | Routine HIV counseling and testing | Verbal consent | |
| Programmatic<br>Interventions | Eligible residents of study communities | Use of testing (rapid test) and intake data from HTC, linkage to HIV care, TB screening, retention support and PMTCT services | Waiver of consent/assent granted | 45 CFR<br>46.116 (d) |
| Use of routine-<br>clinical data | Clinic population, all communities | Use of routinely-collected, program data-see Appendix P1 | Waiver of consent/assent granted | 45 CFR<br>46.116 (d) |
| Clinic Patient<br>Retention and<br>Adherence | IDCC patient population in CPCs | Data collection and permission to follow-up | Linkage, Retention &<br>Adherence Tracing<br>Verbal Consent Script | |

### 10.3 Risks

The risks, discomforts, and inconveniences that could be posed to subjects participating in this project include the following:

### HTC Participants:

- O Blood drawing may cause pain and bruising, and rarely, infection at the site where blood is drawn. Study participants may feel lightheaded or faint as a result.
- Repeated HTC may cause stress, anxiety, or embarrassment. Participants are likely to become distressed if they learn they are HIV positive.
- Participants may become embarrassed, worried, or anxious when discussing their sexual practices, HIV risk factors, ways to protect their partner(s) against HIV, and/or ways to prevent acquiring HIV infection.
- Participants may experience discrimination as a result of being perceived by others to be HIVinfected.

## Other Strengthened Program Interventions:

- Other strengthened interventions, including linkage for HIV care, ANC, TB screening, and retention support all carry very minimal risk to participants.
- Persons starting ART: In addition to the risks described above for survey participants, risks for patients initiating ART include:

Adults starting ART are at risk of ART-related adverse events (e.g., hepatitis, severe skin rash, renal dysfunction, drug resistance, need for regimen change, etc.).

### 10.4 Benefits of Research Participation

- **HTC:** Potential health benefits include: earlier HTC delivered to their place of residence, earlier diagnosis of HIV-infection with subsequent earlier enrollment in care and treatment or PMTCT, earlier awareness of the importance of annual HTC and risk reduction practices for adults who test HIV-negative, and earlier awareness of the benefits of MC for HIV negative males.
- Other Strengthened Program Interventions: Evidence for health benefits of linkage-to-care and adherence/ retention interventions are described in Section 6.
- UTT: The benefits of earlier initiation of ART might include improved survival and reduction in incidence of adverse events [such as serious non-AIDS events like myocardial infarction, or AIDSrelated morbidity (e.g., a new WHO stage III/IV condition)] as well as decreased likelihood of transmitting HIV to others.

### **10.5 Confidentiality**

No information concerning the study or the data will be released to any unauthorized third party, without prior written approval of the participant, except as necessary for monitoring by the IRBs, the study sponsor, OHRP, or the Botswana Ministry of Health. No data with subject identifiers will be released.

# • HTC, linkage to care, and HIV care and treatment following HIV diagnosis:

Project staff visiting households for study visits will identify an appropriately private space to counsel participants, perform HIV tests, and collect individual data. If private space is not available, or the participant does not wish to carry out study activities in the home, an appointment will be made to visit one of the mobile units or study clinics instead. All study documents, including any papers or files containing personal contact information (such as telephone numbers and addresses), will be stored in a secure location and electronic data will be password protected. Full Drive Encryption will be implemented at the hardware layer of all devices storing protected health information. Only designated study staff will have access to study records.

# Linkage to MC and MC

MC mobilization will be conducted according to national standards for mobilization. These standards include protections for transport registers and mobilization registers with PII.

#### **IDCC Care and Treatment:**

Care at the clinic will be provided in adherence with MOH confidentiality guidelines. Consultations between patients and clinic/research staff will occur in a private location. All consent forms kept by investigators are stored in locked steel cabinets at the clinic or on password-protected electronic devices (e.g., tablets). All paper forms are stored in locked steel cabinets and transported in sealed boxes to Gaborone. All data collected via MOH data systems or entered from paper questionnaires are kept securely on password-protected log-in screens.

## 10.6 Protocol Compliance and Compliance with UN Convention on the Rights of the Child

Study staff will adhere to the ethical principles that are reflected in the Declaration of Helsinki (e.g., ICH E6, 45 CFR 46). The study will be conducted in accordance with the Botswana and Sponsor regulations.

The US government is a signatory on the UN Convention on the Rights of the Child (defined as anyone under the age of 18) which requires that any research study or program activity which includes children that are identified as engaged in sex work, trafficked or victims of violence make special provisions for referral of these individuals to services. BCPP will report suspected cases to designated service providers (local police or social workers) as outlined in the Botswana National Guidelines for reporting child abuse or neglect. Contact information for the local police and social workers, and procedures for reporting suspected cases of child abuse or neglect are described in study specific SOP in the BCPP Study Manual. Local police and social workers will be contacted prior to the initiation of study activities in the community to ensure they are aware of the study activities in the community and the procedures that will be followed should BCPP staff encounter suspected cases of abuse or neglect. As per national guidelines, reports of suspected abuse or neglect will be made to local authorities within 24 hours. Study personnel who may come in contact with these study participants will receive training on the appropriate procedures for handling these cases if they arise during the course of the study and training on the SOP documented in the regulatory files. The study will retain documentation of all reports that includes date of report, age of participant, and the name and type of service provider. No identified information will be retained in the documentation; documentation will be retained by the study for 2 years after study close-out. The informed consents for the study contain

language that makes clear to the participant what is required to be reported to authorities and the impact on confidentiality.

#### 11.0 STUDY SAFETY AND MONITORING PLAN

## **11.1** Reporting Adverse Events

## Expedited Adverse Event (EAE) Reporting Requirements for this Study:

The study team will report in real-time, to overseeing IRB's and to sponsors, any AE following any exposure to the study interventions that is BOTH possibly related to study intervention and unexpected, and which is a Serious Adverse Event (SAE). An SAE is defined as any untoward occurrence that:

- Results in death
- Is life-threatening (grade 4)
- Requires hospitalization or prolongation of hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect

This level of reporting is chosen to avoid real-time EAE reporting of all deaths, hospitalizations, etc. occurring in study communities that are definitely not related to study procedures.

Study interventions are defined as:

- 1. Antiretroviral therapy implemented as per BCPP protocol
- 2. HIV testing as part of the HTC campaigns
- 3. Any other study-related activity in which harm (including social harm) could occur.

With regard to ART intervention, EAE reporting will be restricted to SAEs that are possibly related to initiating ART beyond national guidelines.

## Timing of EAE reporting:

EAEs will be reported to CDC and HRDC within 2 business days of the study investigators becoming aware of the event.

### Grading Severity of Events:

The most current Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) dated November 2014 will be used (or more current version, if applicable), and is available on the RSC website (<a href="http://rsc.tech-res.com/">http://rsc.tech-res.com/</a>).

## Non-EAE Adverse Event and Incident Reporting:

The risk of adverse events related to the use of ART has been established and there is no indication that enrollees, with intact immune systems, who are receiving ART, are likely to have a higher risk of adverse events.

SAEs that do not meet the criteria for EAEs (i.e. an SAE that is NOT related to the study intervention) will be submitted quarterly to the IRB. A table listing all unrelated SAEs that occurred in the specified quarter will be submitted to the IRB along with a brief narrative of each event. Per discussions with the CDC IRB, SAEs that are unrelated to the study intervention will NOT be reported using the official CDC forms (.1254/.1254S).

## **Adverse Event Reporting Period:**

The expedited AE reporting period for this study is from the time of initial study contact to the last study contact for a participant.

## AE reporting process

Reportable events will be documented by the in-country study team who will then notify the IRBs, MOH, CDC-Atlanta, and Harvard Chan School teams. The incident will be discussed and a written action plan will be devised and implemented within 1 week of the initial report, if needed. Written documentation of all events and event resolution will be retained in the study file. Reporting of EAEs, SAEs and AEs to IRBs and the study sponsor will follow institutional and IRB policies. If applicable, a formal report will be sent to the appropriate IRBs using the CDC's Incident Report Form 1254.

### 11.2 **DSMB**

Proposed Schedule of DSMB Reviews and Interim Data Analysis

The BCPP is divided into three interlocking protocols (two active protocols, after Protocol 2 was terminated in 2015), and the investigators expect that DSMB review will require information regarding interim study results and study conduct from all three. The combination prevention package under study includes the following interventions that are outside of current SOC in Botswana: provision of ART for all HIV-infected adults regardless of WHO Stage or CD4 count and streamlined ART delivery. Hence, the reports will provide information needed to evaluate the adverse and favorable effects of such interventions on individually treated patients as well as on the communities in which they reside. The study will require at least 6 reviews, DSMB 1-6, proposed to take place at baseline and at the end of years 1, 2, 3, 4, and 5. DSMB 3 and 4 will evaluate intervention rollout and safety. At DSMB 5, the DSMB can recommend stopping for efficacy or extending the study by 1 year should there be low intervention coverage or a lower than expected incidence rate in the Enhanced Care arm. To demonstrate that the study has reasonable power to answer the study questions given information up to the time of each review, investigators will provide the DSMB with assessments of the adequacy of coverage of proposed interventions; estimated conditional power given available incidence information will be provided at DSMB 4 and all subsequent reviews. While there will be separate reports for each of the protocols, each report will make use of the data available from all protocols. Details of the DSMB review plan for each protocol are provided in that protocol, and the full detailed plan is provided in **Appendix C4**.

# 11.3 Protocol Violations

The study will be conducted in full compliance with the protocol. The research team will ensure that volunteers are informed of and understand the risks of their participation in research. Protocol violations and cases of social harm will be documented using the appropriate study forms and reported to IRBs and sponsors in accordance with the institutional policies. Minor protocol violations that do not pose a threat to the health or welfare of participants will be compiled and reported to the IRBs at the time of annual IRB review. Incident reporting is the responsibility of the Principal Investigators of

this study. Emergency departures from protocol that eliminate an apparent immediate hazard to participants and are deemed crucial for the safety and well-being of that participant may be instituted for that participant only. In that case the Investigator will contact the IRBs and sponsor as soon as possible to document the reasons for violation and ensuing events.

## 11.4 Monitoring Plan

A complete monitoring plan has been developed and the site will complete a study site activation checklist prior to study initiation. Internal (sponsor) and external monitors will travel to the study site according to a pre-determined monitoring schedule specified in the monitoring plan to conduct general monitoring. The study site will maintain a monitoring log to document all monitoring visits. Investigators and staff will grant access to the monitors to allow inspection and review study documents (e.g., consent forms, data collection forms, other source documents) and pertinent clinic records for confirmation of the study data. Study monitors will also inspect study facilities and documentation and may observe the performance of study procedures.

### 12.0 ADMINISTRATIVE PROCEDURES AND INFORMATION DISSEMINATION

## 12.1 Study Records and Document Retention

Complete, accurate, and current study records will be maintained and stored in a secure manner throughout the duration of the study and additionally for five years after study close-out. Study records include administrative documentation— including all reports and correspondence relating to the study— as well as documentation related to each participant screened and/or enrolled in the study, including informed consent forms, locator forms, case report forms, notations of all contacts with the participant, and all other source documents. Necessary documents to be maintained by the site before, during and after the study will be in accordance with GCP regulations and guidance. A complete list of needed documentation will be provided prior to initiation of the study and will appear in the study manual.

### 12.2 Information Dissemination and Publication Plan

Study findings will be disseminated through presentations, reports and publication in peer-reviewed journals and other publications. In-country data and country specific information will be made available to national policy-makers, organizational, and implementing partners. A detailed publication and communication plan will be developed that describes the number and types of reports and manuscripts planned for the study and criteria for authorship. Formal presentations at conferences and scientific publications will follow CDC, Harvard Chan School, and MOH guidelines. A data sharing plan will also be developed that details the requirements and process for requesting access to stored data and a samples for sub-studies and future analysis.

#### 13.0 REFERENCES

Ananworanich, J., Gayet-Ageron, A., Le Braz, M., Prasithsirikul, W., Chetchotisakd, P., Kiertiburanakul, S., et al. (2006). CD4-guided scheduled treatment interruptions compared with continuous therapy for patients infected with HIV-1: results of the Staccato randomised trial. Lancet, 368(9534), 459–465. doi:10.1016/S0140-6736(06)69153-8.

Attia, S., M. Egger, M. Muller, M. Zwahlen and N. Low (2009). "Sexual transmission of HIV according to viral load and antiretroviral therapy: systematic review and meta-analysis." <u>AIDS</u> 23(11): 1397-1404.

Auld, A. F., N. Wambua, J. Onyango, B. Marston, G. Namulanda, M. Ackers, T. Oluoch, A. Karisa, A. Hightower, R. W. Shiraishi, A. Nakashima and J. Sitienei (2010). "Piloting the use of personal digital assistants for tuberculosis and human immunodeficiency virus surveillance, Kenya, 2007." <a href="Int J Tuberc Lung Dis">Int J Tuberc Lung Dis</a> 14(9): 1140-1146.

Auvert, B., D. Taljaard, E. Lagarde, J. Sobngwi-Tambekou, R. Sitta and A. Puren (2005). "Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial." <u>PLoS Med</u> 2(11): e298.

Bailey, R. C., S. Moses, C. B. Parker, K. Agot, I. Maclean, J. N. Krieger, C. F. Williams, R. T. Campbell and J. O. Ndinya-Achola (2007). "Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial." <u>Lancet</u> 369(9562): 643-656.

BAIS (2008). "The Botswana HIV/AIDS Impact Survey III Results. Available: http://www.gov.bw/Global/NACA%20Ministry/wana/BAIS%20III Stats%20Press.pdf."

BAIS (2012). Botswana National AIDS Coordinating Agency. The Fourth Botswana HIV/AIDS Impact Survey IV-2012. Accessed 17 July 2014 at <a href="http://www.naca.gov.bw/sites/default/files/BAIS%20IV%20Protocol.pdf">http://www.naca.gov.bw/sites/default/files/BAIS%20IV%20Protocol.pdf</a>

Binik, A., C. Weijer, A. D. McRae, J. M. Grimshaw, R. Boruch, J. C. Brehaut, A. Donner, M. P. Eccles, R. Saginur, M. Taljaard and M. Zwarenstein (2011). "Does clinical equipoise apply to cluster randomized trials in health research?" <u>Trials</u> 12: 118.

Blitzstein, J. and P. Diaconis (2006). "A sequential importance sampling algorithm for generating random graphs with prescribed degrees. Available at: <a href="http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf">http://www-stat.stanford.edu/~cgates/PERSI/papers/GraphAlgorithm.pdf</a>."

Census (2011). "Project Document: 2011 Population and Housing Census. Available at: http://unstats.un.org/unsd/censuskb20/Attachment453.aspx."

Central Statistics Office (2009). Botswana AIDS Impact Survey III (BAIS III), 2008. C. Kebonyethebe Johane. Gaborone, Botswana.

Ciaranello AL, Perez F, Engelsmann B, Walensky RP, Mushavi A, Rusibamayila A, et al. Cost-effectiveness of World Health Organization 2010 guidelines for prevention of mother-to-child HIV transmission in Zimbabwe. *Clin Infect Dis* 2013,56:430-446.

Cohen, M. S., Y. Q. Chen, M. McCauley, T. Gamble, M. C. Hosseinipour, N. Kumarasamy, J. G. Hakim, J. Kumwenda, B. Grinsztejn, J. H. Pilotto, S. V. Godbole, S. Mehendale, S. Chariyalertsak, B. R. Santos, K. H. Mayer, I. F. Hoffman, S. H. Eshleman, E. Piwowar-Manning, L. Wang, J. Makhema, L. A. Mills, G. de Bruyn, I. Sanne, J. Eron, J. Gallant, D. Havlir, S. Swindells, H. Ribaudo, V. Elharrar, D. Burns, T. E. Taha, K. Nielsen-Saines, D. Celentano, M. Essex and T. R. Fleming (2011). "Prevention of HIV-1 infection with early antiretroviral therapy." N Engl J Med 365(6): 493-505.

Corbett, E. L., T. Bandason, T. Duong, E. Dauya, B. Makamure, G. J. Churchyard, B. G. Williams, S. S. Munyati, A. E. Butterworth, P. R. Mason, S. Mungofa and R. J. Hayes (2010). "Comparison of two active case-finding strategies for community-based diagnosis of symptomatic smear-positive tuberculosis and control of infectious tuberculosis in Harare, Zimbabwe (DETECTB): a cluster-randomised trial." <u>Lancet</u> 376(9748): 1244-1253.

Craw, J. A., L. I. Gardner, G. Marks, R. C. Rapp, J. Bosshart, W. A. Duffus, A. Rossman, S. L. Coughlin, D. Gruber, L. A. Safford, J. Overton and K. Schmitt (2008). "Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II." <u>J Acquir Immune Defic Syndr</u> 47(5): 597-606.

Curran, K., E. Njeuhmeli, A. Mirelman, K. Dickson, T. Adamu, P. Cherutich, H. Mahler, B. Fimbo, T. K. Mavuso, J. Albertini, L. Fitzgerald, N. Bock, J. Reed, D. Castor and D. Stanton (2011). "Voluntary medical male circumcision: strategies for meeting the human resource needs of scale-up in southern and eastern Africa." <u>PLoS Med</u> 8(11): e1001129.

Daar, E. S., T. Moudgil, R. D. Meyer and D. D. Ho (1991). "Transient high levels of viremia in patients with primary human immunodeficiency virus type 1 infection." N Engl J Med 324(14): 961-964.

Ding, M., P. Tarwater, M. Rodriguez, R. Chatterjee, D. Ratner, Y. Yamamura, P. Roy, J. Mellors, D. Neogi, Y. Chen and P. Gupta (2009). "Estimation of the predictive role of plasma viral load on CD4 decline in HIV-1 subtype C-

Donnell, D., J. M. Baeten, J. Kiarie, K. K. Thomas, W. Stevens, C. R. Cohen, J. McIntyre, J. R. Lingappa, C. Celum and H. S. V. H. I. V. T. S. T. Partners in Prevention (2010). "Heterosexual HIV-1 transmission after initiation of antiretroviral therapy: a prospective cohort analysis." Lancet 375(9731): 2092-2098.

infected subjects in India." J Acquir Immune Defic Syndr 50(2): 119-125.

Eaton, J. W., T. B. Hallett and G. P. Garnett (2011). "Concurrent sexual partnerships and primary HIV infection: a critical interaction." <u>AIDS Behav</u> 15(4): 687-692.

Faal, M., N. Naidoo, D. K. Glencross, W. D. Venter and R. Osih (2011). "Providing immediate CD4 count results at HIV testing improves ART initiation." <u>J Acquir Immune Defic Syndr</u> 58(3): e54-59. Fauci, A. S. and G. K. Folkers (2012). "Toward an AIDS-free generation." <u>JAMA</u> 308(4): 343-344.

Fasawe O, Avila C, Shaffer N, Schouten E, Chimbwandira F, Hoos D, et al. Cost-Effectiveness Analysis of Option B+ for HIV Prevention and Treatment of Mothers and Children in Malawi. *PLoS One* 2013,8:e57778.

Fox, M. P. and S. Rosen (2010). "Patient retention in antiretroviral therapy programs up to three years on treatment in sub-Saharan Africa, 2007-2009: systematic review." Trop Med Int Health 15 Suppl 1: 1-15.

Gardner, E. M., M. P. McLees, J. F. Steiner, C. Del Rio and W. J. Burman (2011). "The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection." <u>Clin Infect Dis</u> 52(6): 793-800.

Gardner, L. I., G. Marks, J. Craw, L. Metsch, S. Strathdee, P. Anderson-Mahoney, C. del Rio and G. Antiretroviral Treatment Access Study (2009). "Demographic, psychological, and behavioral modifiers of the Antiretroviral Treatment Access Study (ARTAS) intervention." <u>AIDS Patient Care STDS</u> 23(9): 735-742.

Gardner, L. I., G. Marks, L. R. Metsch, A. M. Loughlin, C. O'Daniels, C. del Rio, P. Anderson-Mahoney, J. D. Wilkinson and A. S. Group (2007). "Psychological and behavioral correlates of entering care for HIV infection: the Antiretroviral Treatment Access Study (ARTAS)." <u>AIDS Patient Care STDS</u> 21(6): 418-425.

Gardner, L. I., L. R. Metsch, P. Anderson-Mahoney, A. M. Loughlin, C. del Rio, S. Strathdee, S. L. Sansom, H. A. Siegal, A. E. Greenberg, S. D. Holmberg, T. Antiretroviral and G. Access Study Study (2005). "Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care." <u>AIDS</u> 19(4): 423-431. Geng, E. H., D. Nash, A. Kambugu, Y. Zhang, P. Braitstein, K. A. Christopoulos, W. Muyindike, M. B. Bwana, C. T. Yiannoutsos, M. L. Petersen and J. N. Martin (2010). "Retention in care among HIV-infected patients in resource-limited settings: emerging insights and new directions." <u>Curr HIV/AIDS Rep</u> 7(4): 234-244.

Granich, R. M., C. F. Gilks, C. Dye, K. M. De Cock and B. G. Williams (2009). "Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model." Lancet 373(9657): 48-57.

Gray, R. H., G. Kigozi, D. Serwadda, F. Makumbi, S. Watya, F. Nalugoda, N. Kiwanuka, L. H. Moulton, M. A. Chaudhary, M. Z. Chen, N. K. Sewankambo, F. Wabwire-Mangen, M. C. Bacon, C. F. Williams, P. Opendi, S. J. Reynolds, O. Laeyendecker, T. C. Quinn and M. J. Wawer (2007). "Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial." <u>Lancet</u> 369(9562): 657-666.

Habicht, J. P., C. G. Victora and J. P. Vaughan (1999). "Evaluation designs for adequacy, plausibility and probability of public health programme performance and impact." <u>Int J Epidemiol</u> 28(1): 10-18.

Halperin, D. T. (2009). "Combination HIV prevention must be based on evidence." <u>Lancet</u> 373(9663): 544-545. Handcock, M. S., D. R. Hunter, C. T. Butts, S. M. Goodreau and M. Morris (2003). "Software tools for the Statistical Modeling of Network Data. available at: <a href="http://statnet.org.">http://statnet.org.</a>"

Hayes, R., F. Mosha, A. Nicoll, H. Grosskurth, J. Newell, J. Todd, J. Killewo, J. Rugemalila and D. Mabey (1995). "A community trial of the impact of improved sexually transmitted disease treatment on the HIV epidemic in rural Tanzania: 1. Design." <u>AIDS</u> 9(8): 919-926.

Hayes, R. and L. H. Moulton (2009). <u>Cluster Randomized Trials</u>. Boca Raton, CRC Press. Helleringer, S. and H. P. Kohler (2007). "Sexual network structure and the spread of HIV in Africa: evidence from Likoma Island, Malawi." <u>AIDS</u> 21(17): 2323-2332.

HHS (2011). "Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents. Avaiable at: http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf."

HHS (2012). "Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Available at: http://infosida.nih.gov/contentfiles/lvguidelines/adultandadolescentglsp.pdf. Accessed 19 August 2012.".

Hussey, M. A. and J. P. Hughes (2007). "Design and analysis of stepped wedge cluster randomized trials." <u>Contemp Clin Trials</u> 28(2): 182-191.

Jani, I. V., N. E. Sitoe, P. L. Chongo, E. R. Alfai, J. I. Quevedo, O. Tobaiwa, J. D. Lehe and T. F. Peter (2011). "Accurate CD4 T-cell enumeration and antiretroviral drug toxicity monitoring in primary healthcare clinics using point-of-care testing." <u>AIDS</u> 25(6): 807-812.

Jones, J. H. and M. S. Handcock (2003). "An assessment of preferential attachment as a mechanism for human sexual network formation." <u>Proc Biol Sci</u> 270(1520): 1123-1128.

Kaufmann, G. R., P. Cunningham, A. D. Kelleher, J. Zaunders, A. Carr, J. Vizzard, M. Law and D. A. Cooper (1998). "Patterns of viral dynamics during primary human immunodeficiency virus type 1 infection. The Sydney Primary HIV Infection Study Group." <u>J Infect Dis</u> 178(6): 1812-1815.

Kim, A. A., T. Hallett, J. Stover, E. Gouws, J. Musinguzi, P. K. Mureithi, R. Bunnell, J. Hargrove, J. Mermin, R. K. Kaiser, A. Barsigo and P. D. Ghys (2011). "Estimating HIV Incidence among Adults in Kenya and Uganda: A Systematic Comparison of Multiple Methods." <u>PLoS One</u> 6(3): e17535.

Kitahata, M. M., S. J. Gange, A. G. Abraham, B. Merriman, M. S. Saag, A. C. Justice, R. S. Hogg, S. G. Deeks, J. J. Eron, J. T. Brooks, S. B. Rourke, M. J. Gill, R. J. Bosch, J. N. Martin, M. B. Klein, L. P. Jacobson, B. Rodriguez, T. R. Sterling, G. D. Kirk, S. Napravnik, A. R. Rachlis, L. M. Calzavara, M. A. Horberg, M. J. Silverberg, K. A. Gebo, J. J. Goedert, C. A. Benson, A. C. Collier, S. E. Van Rompaey, H. M. Crane, R. G. McKaig, B. Lau, A. M. Freeman, R. D. Moore and N.-A. Investigators (2009). "Effect of early versus deferred antiretroviral therapy for HIV on survival." N Engl J Med 360(18): 1815-1826.

Lawn, S. D., A. D. Harries, B. G. Williams, R. E. Chaisson, E. Losina, K. M. De Cock and R. Wood (2011). "Antiretroviral therapy and the control of HIV-associated tuberculosis. Will ART do it?" <a href="Int J Tuberc Lung Dis">Int J Tuberc Lung Dis</a> 15(5): 571-581.

Lester, R. T., P. Ritvo, E. J. Mills, A. Kariri, S. Karanja, M. H. Chung, W. Jack, J. Habyarimana, M. Sadatsafavi, M. Najafzadeh, C. A. Marra, B. Estambale, E. Ngugi, T. B. Ball, L. Thabane, L. J. Gelmon, J. Kimani, M. Ackers and F. A. Plummer (2010). "Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial." <u>Lancet</u> 376(9755): 1838-1845.

Lingappa, J. R., J. P. Hughes, R. S. Wang, J. M. Baeten, C. Celum, G. E. Gray, W. S. Stevens, D. Donnell, M. S. Campbell, C. Farquhar, M. Essex, J. I. Mullins, R. W. Coombs, H. Rees, L. Corey, A. Wald and H. S. V. H. I. V. T. S. T. Partners in Prevention (2010). "Estimating the impact of plasma HIV-1 RNA reductions on heterosexual HIV-1 transmission risk." <u>PLoS One</u> 5(9): e12598.

Little, S. J., A. R. McLean, C. A. Spina, D. D. Richman and D. V. Havlir (1999). "Viral dynamics of acute HIV-1 infection." <u>J Exp Med</u> 190(6): 841-850.

Lyles, R. H., C. Chu, J. W. Mellors, J. B. Margolick, R. Detels, J. V. Giorgi, Q. Al-Shboul and J. P. Phair (1999). "Prognostic value of plasma HIV RNA in the natural history of Pneumocystis carinii pneumonia, cytomegalovirus and Mycobacterium avium complex. Multicenter AIDS Cohort Study." <u>AIDS</u> 13(3): 341-349

Mahy, M., J. Stover, K. Kiragu, C. Hayashi, P. Akwara, C. Luo, K. Stanecki, R. Ekpini and N. Shaffer (2010). "What will it take to achieve virtual elimination of mother-to-child transmission of HIV? An assessment of current progress and future needs." <u>Sex Transm Infect</u> 86 Suppl 2: ii48-55.

Mellors, J. W., J. B. Margolick, J. P. Phair, C. R. Rinaldo, R. Detels, L. P. Jacobson and A. Munoz (2007). "Prognostic value of HIV-1 RNA, CD4 cell count, and CD4 Cell count slope for progression to AIDS and death in untreated HIV-1 infection." <u>JAMA</u> 297(21): 2349-2350.

Mellors, J. W., A. Munoz, J. V. Giorgi, J. B. Margolick, C. J. Tassoni, P. Gupta, L. A. Kingsley, J. A. Todd, A. J. Saah, R. Detels, J. P. Phair and C. R. Rinaldo, Jr. (1997). "Plasma viral load and CD4+ lymphocytes as prognostic markers of HIV-1 infection." <u>Ann Intern Med</u> 126(12): 946-954.

Mellors, J. W., C. R. Rinaldo, Jr., P. Gupta, R. M. White, J. A. Todd and L. A. Kingsley (1996). "Prognosis in HIV-1 infection predicted by the quantity of virus in plasma." Science 272(5265): 1167-1170.

Merson, M., N. Padian, T. J. Coates, G. R. Gupta, S. M. Bertozzi, P. Piot, P. Mane, M. Bartos and H. I. V. P. S. A. Lancet (2008). "Combination HIV prevention." <u>Lancet</u> 372(9652): 1805-1806.

Microsoft (2011). "HIV/AIDS Information System Taps Existing Cell Phone Texting Capabilities. Available at: <a href="http://research.microsoft.com/en-us/collaboration/papers/botswana.pdf">http://research.microsoft.com/en-us/collaboration/papers/botswana.pdf</a>."

MMWR. Impact of an Innovative Approach to Prevent Mother-to-Child Transmission of HIV — Malawi, July 2011–September 2012. March 1, 2013 / 62(08);148-151.

Modjarrad, K., E. Chamot and S. H. Vermund (2008). "Impact of small reductions in plasma HIV RNA levels on the risk of heterosexual transmission and disease progression." <u>AIDS</u> 22(16): 2179-2185.

Montaner, J. S., V. D. Lima, R. Barrios, B. Yip, E. Wood, T. Kerr, K. Shannon, P. R. Harrigan, R. S. Hogg, P. Daly and P. Kendall (2010). "Association of highly active antiretroviral therapy coverage, population viral load, and yearly new HIV diagnoses in British Columbia, Canada: a population-based study." <u>Lancet</u> 376(9740): 532-539. Mtapuri-Zinyowera, S., M. Chideme, D. Mangwanya, O. Mugurungi, S. Gudukeya, K. Hatzold, A. Mangwiro, G. Bhattacharya, J. Lehe and T. Peter (2010). "Evaluation of the PIMA point-of-care CD4 analyzer in VCT clinics in Zimbabwe." J Acquir Immune Defic Syndr 55(1): 1-7.

Novitsky, V., T. Ndung'u, R. Wang, H. Bussmann, F. Chonco, J. Makhema, V. De Gruttola, B. D. Walker and M. Essex (2011). "Extended high viremics: a substantial fraction of individuals maintain high plasma viral RNA levels after acute HIV-1 subtype C infection." <u>AIDS</u> 25(12): 1515-1522.

Novitsky, V., R. Wang, H. Bussmann, S. Lockman, M. Baum, R. Shapiro, I. Thior, C. Wester, C. W. Wester, A. Ogwu, A. Asmelash, R. Musonda, A. Campa, S. Moyo, E. van Widenfelt, M. Mine, C. Moffat, M. Mmalane, J. Makhema, R. Marlink, P. Gilbert, G. R. Seage, 3rd, V. DeGruttola and M. Essex (2010). "HIV-1 subtype C-infected individuals maintaining high viral load as potential targets for the "test-and-treat" approach to reduce HIV transmission." PLoS One 5(4): e10148.

Padian, N. S., S. I. McCoy, S. Manian, D. Wilson, B. Schwartlander and S. M. Bertozzi (2011). "Evaluation of large-scale combination HIV prevention programs: essential issues." <u>J Acquir Immune Defic Syndr</u> 58(2): e23-28.

PEPFAR (2009). "Celebrating Life: The U.S. President's Emergency Plan for AIDS Relief 2009 Annual Report to Congress – Highlights. Accessed 3 September 2011 at: http://www.pepfar.gov/documents/organization/113878.pdf."

Piot, P., M. Bartos, H. Larson, D. Zewdie and P. Mane (2008). "Coming to terms with complexity: a call to action for HIV prevention." Lancet 372(9641): 845-859.

Rosen, S. and M. P. Fox (2011). "Retention in HIV Care between Testing and Treatment in Sub-Saharan Africa: A Systematic Review." <u>PLoS Med</u> 8(7): e1001056.

Severe, P., M. A. Juste, A. Ambroise, L. Eliacin, C. Marchand, S. Apollon, A. Edwards, H. Bang, J. Nicotera, C. Godfrey, R. M. Gulick, W. D. Johnson, Jr., J. W. Pape and D. W. Fitzgerald (2010). "Early versus standard antiretroviral therapy for HIV-infected adults in Haiti." N Engl J Med 363(3): 257-265.

Shapiro RL, Kitch D, Ogwu A, Hughes M, Lockman S, Powis K, Souda S, Moffat C, Moyo S, McIntosh K, Widenfelt E, Zwerski S, Mazhani L, Makhema J, Essex M. HIV transmission and 24-month survival in a randomized trial of HAART to prevent MTCT during pregnancy and breastfeeding in Botswana (The Mma Bana Study). AIDS. 2013 (in press).

Stover, J., L. Bollinger and C. Avila (2011). "Estimating the Impact and Cost of the WHO 2010 Recommendations for Antiretroviral Therapy." <u>AIDS Res Treat</u> 2011: 738271

Stover, J., B. Fidzani, B. C. Molomo, T. Moeti and G. Musuka (2008). "Estimated HIV trends and program effects in Botswana." PLoS One 3(11): e3729.

Stover, J., E. L. Korenromp, M. Blakley, R. Komatsu, K. Viisainen, L. Bollinger and R. Atun (2011). "Long-term costs and health impact of continued global fund support for antiretroviral therapy." <u>PLoS One</u> 6(6): e21048. Tanser, F., T. Bärnighausen, E. Grapsa and M.-L. Newell (2012). "Effect of ART Coverage on Rate of New HIV Infections in a Hyper-endemic, Rural Population: South Africa." <u>19th Conference on Retroviruses and Opportunistic Infections; March 5-8; Seattle, USA. Available: http://www.retroconference.org/2012b/Abstracts/45379.htm. Accessed 4 July 2012.</u>

Tanser, F., T. Bärnighausen, E. Grapsa, J. Zaidi and M. L. Newell (2013). "High Coverage of ART Associated with Decline in Risk of HIV Acquisition in Rural KwaZulu-Natal, South Africa." <u>Science</u> 339(966).

UNAIDS (2010). "Global Report: UNAIDS Report on the Global AIDS Epidemic. Available at: <a href="http://www.unaids.org/globalreport/globalreport.htm">http://www.unaids.org/globalreport/global report.htm</a>. Accessed February 2012.".

Van Rooyen, H., R. V. Barnabas, Z. Phakathi, P. Joseph, M. Krows, T. Hong, J. Baeten and C. Celum (2012). "HIV testing uptake and linkages to HIV treatment through home-based HIV counseling and testing and facilitated referral in Kwa-Zulu Natal, South Africa." <u>CROI 2012</u>.

Walensky, R. P., L. L. Wolf, R. Wood, M. O. Fofana, K. A. Freedberg, N. A. Martinson, A. D. Paltiel, X. Anglaret, M. C. Weinstein and E. Losina (2009). "When to start antiretroviral therapy in resource-limited settings." <u>Ann Intern Med</u> 151(3): 157-166.

WHO (2003). "World health Organization. WHO Guide to Cost-Effectiveness Analysis - 2003." Geneva, Switzerland: WHO; 2003. Accessed August 11, 2010: http://www.who.int/choice/publications/p 2003 generalised cea.pdf.

WHO (2010). World Health Organization. Towards universal access: Scaling up priority HIV/AIDS interventions in the health sector - Progress report 2010. Geneva, Switzerland: WHO; 2010. . Avaliable: http://wwwwhoint/hiv/pub/2010progressreport/full report enpdf. Accessed 29 September 2010.

WHO (2011). "Global HIV./AIDS Response. Epidemic update and health sector progress towards Universal Access. Available:

http://www.unaids.org/en/media/unaids/contentassets/documents/unaidspublication/2011/20111130\_UA\_Report\_en.pdf. Accessed 24 August 2012."

WHO (2013) "Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV infection" Available: http://apps.who.int/iris/bitstream/10665/85321/1/9789241505727\_eng.pdf Accessed 5 December 2013

World Health Organization. Use of Antiretroviral Drugs for Treating Pregnant Women and Preventing HIV Infection in Infants. Programmatic Update. April, 2012. http://www.who.int/hiv/pub/mtct/programmatic\_update2012/en/.

World health Organization. Consolidated Guidelines on HIV Testing Services. July, 2015. <a href="http://www.who.int/hiv/pub/guidelines/hiv-testing-services/en/">http://www.who.int/hiv/pub/guidelines/hiv-testing-services/en/</a>

World Health Organization. Guideline on When to Start Antiretrovoral Therapy and on Pre-Exposure Prophylaxis for HIV. September, 2015.

Writing Committee for the, C. C. (2011). "Timing of HAART initiation and clinical outcomes in human immunodeficiency virus type 1 seroconverters." <u>Arch Intern Med</u> 171(17): 1560-1569.